# Emulating the SUSTAIN-6 Cardiovascular Outcome Trial in Healthcare Claims Data

NCT06659744

30<sup>th</sup> July 2025

# 1. Title Page

| Title | Comparative effectiveness of semaglutide and tirzepatide in patients at elevated cardiovascular risk with type 2 diabetes and obesity: Emulating the SUSTAIN-6 |
|---|---|
| | Cardiovascular Outcome Trial in Healthcare Claims Data |
| Research question & Objectives | This study is part of a three-stage project evaluating the comparative |
| | effectiveness of semaglutide and tirzepatide in patients at elevated |
| | cardiovascular risk with type 2 diabetes and obesity: |
| | The SUSTAIN-6 evaluates the effect of injectable semaglutide versus placebo on |
| | the risk of major adverse cardiovascular event (MACE) among patients with type |
| | 2 diabetes and high cardiovascular risk. |
| Protocol version | Version 1 |
| Last update date | 30 <sup>th</sup> July 2025 |
| Contributors | Primary investigators contact information: |
| | Dr. Nils Krüger, nkruger1@bwh.harvard.edu |
| | Dr. Shirley Wang, swang1@bwh.harvard.edu |
| | Contributor names: |
| | Dr. Krüger implemented the study design in the Aetion Evidence Platform. He is |
| | responsible for the validity of the design and analytic choices. All implementation |
| | steps are recorded and the implementation history is archived in the platform. |
| Study registration | Site: clinicaltrials.gov |
| | Identifier: NCT06659744 |
| Sponsor | Organization: N/A |
| | Contact: N/A |
| Conflict of interest | Dr. Krüger has no conflict of interest. |
| | Dr. Wang has consulted for Cytel Incs, Exponent Inc, and MITRE an FFRDC for |
| | Centers for Medicare and Medicaid for unrelated work. |

# **Table of contents**

| . Title Page | 1 |
|---|---|
| 2. Abstract | 3 |
| 3. Amendments and updates | 4 |
| . Rationale and background | 4 |
| . Research question and objectives | 5 |
| Table 1 Primary and secondary research questions and objective | 5 |
| 5. Research methods | 7 |
| 6.1 Study design | 7 |
| 6.2 Study design diagram when following the eligibility criteria of the SUSTAIN-6 trial (Figure 1). | 8 |
| 6.3 Setting | 9 |
| 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population | 9 |
| 6.3.2 Context and rationale for study inclusion criteria: | 9 |
| 6.3.3 Context and rationale for study exclusion criteria | 9 |
| 6.4 Variables | 9 |
| 6.4.1 Context and rationale for exposure(s) of interest | 9 |
| 6.4.2 Context and rationale for outcome(s) of interest | 9 |
| 6.4.3 Context and rationale for follow up | 10 |
| Table 2. Operational Definitions of Follow Up | 10 |
| 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) | 11 |
| Table 3. Operational Definitions of Covariates | 11 |
| 6.5 Data analysis | 46 |
| 6.5.1 Context and rationale for analysis plan | 46 |
| Table 4. Primary, secondary, and subgroup analysis specification | 46 |
| Table 5. Sensitivity analyses – rationale, strengths and limitations | 48 |
| 6.5.2 Comparison of Results Between Database Studies and RCTs | 48 |
| 6.6 Data sources | 49 |
| 6.6.1 Context and rationale for data sources | 49 |
| Table 6. Metadata about data sources and software | 50 |
| 6.7 Data management | 50 |
| 6.8. Quality control | 52 |
| 6.9. Study size and feasibility | 52 |
| . Limitation of the methods | 52 |
| 8. Protection of human subjects | 53 |

| 9. I | References | 53 |
|---|---|---|
| 10. | . Appendices | 55 |
| | 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment | 55 |
| | 2 Code algorithms | 55 |
| | 3 Flowchart for cohort assembly | 55 |
| | 4 1st feasibility assessment | 55 |
| | 5 2nd feasibility assessment | 55 |
| | 6 Balance Assessment - PS Distribution and C-Statistic | 55 |
| | 7 Balance Assessment - Table 1 | 56 |

## 2. Abstract

This is a non-randomized, non-interventional study that is part of the *Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims:* Applying Techniques of Epidemiology (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as possible in healthcare insurance claims data, the SUSTAIN6 trial described below. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization cannot be emulated in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The SUSTAIN6 trial is a non-inferiority trial to evaluate the effect of injectable semaglutide, a glucagon-like peptide-1 receptor agonist (GLP-1-RA), versus placebo on time to first occurrence of any major adverse cardiovascular event (MACE), defined as cardiovascular death, myocardial infarction, or stroke among patients with type 2 diabetes mellitus (T2DM).

The database study designed to emulate SUSTAIN6 trial will be a new-user active comparative study, where we compare the effect of injectable semaglutide versus sitagliptin on MACE outcome among patients with T2DM. Sitagliptin was selected to act as an active-comparator proxy for placebo. Sitagliptin and the class of dipeptidyl peptidase-4 (DPP-4) inhibitors have been demonstrated not to have an effect on MACE in a series of RCTs, and they are used in similar stages of disease/line of therapy as semaglutide, as well as being of similar cost.

The study will use three data sources: Optum Clinformatics, Merative MarketScan, and Medicare.

Optum: Study period between January 1, 2018 to February 28, 2025.

MarketScan: Study period between January 1, 2018 to December 31, 2023.

Medicare: Study period between January 1, 2018 to December 31, 2020.

# 3. Amendments and updates

| Version date | Version number | Section of protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 24 <sup>th</sup> July 2025 | 1 | All sections | This version of the emulation of SUSTAIN-6 is part of a 3-stage study that aims to compare tirzepatide vs semaglutide in patients at cardiovascular risk with type 2 diabetes and obesity. This project builds on a protocol for emulating SUSTAIN6 that was developed for a different project with a different objective. The changes include: • Extending cohort entry and follow up to include data up to February 28, 2025 in Optum data • Adding additional secondary outcomes (including individual components of the primary endpoint) • Adding additional variables to the propensity score to address confounding for added outcomes • Changing assessment windows for various design elements (e.g., covariate assessment window, eligibility criteria) of the study | This project builds on a version of an emulation of SUSTAIN-6 that was conducted for different objectives than this study. This protocol includes updates to align the study design with other components of the 3-stage study. Differences in results between the versions of SUSTAIN emulations may occur due to the differences in objectives and design/implementation. |

# 4. Rationale and background

The purpose of this protocol is to describe the emulation of the SUSTAIN6 trial (NCT01720446). The trial enrolled 3,297 participants between February and December 2013. The trial design is event-driven to collect 122 events, which assumes an annual 1.98% event rate in both arms over 2.1 years, which would result in 90% power, to reject a 1.8 hazard ratio at a significance level of 0.05 to assess non-inferiority.<sup>1,2</sup>

Injectable semaglutide became available on December 5, 2017 under the brand name Ozempic.<sup>3</sup> On January 16, 2020, the approval was expanded to include cardiovascular risk reduction in adults with type 2 diabetes mellitus and known heart disease. On March 28, 2022, Novo Nordisk received FDA approval for a higher-dose semaglutide (2 mg) to provide improved glycemic control for adults with T2DM. Meanwhile, semaglutide received its first FDA approval for the treatment of obesity in adults under the brand name Wegovy on June 4, 2021. On December 23, 2022, the approval was extended to include teenagers aged 12 and older. Later, on March 8, 2024, Wegovy was additionally approved for cardiovascular risk reduction in people with overweight or obesity and established cardiovascular disease. Most recently, on January 28, 2025, Ozempic became the first and only GLP-1-RA approved to reduce the risk of worsening kidney disease and cardiovascular death in adults with Type 2 diabetes and chronic kidney disease.

Sitagliptin was specifically chosen as an active comparator that could proxy for placebo because a major randomized controlled trial on cardiovascular outcomes demonstrated that it does not affect the cardiovascular outcomes under investigation.<sup>4</sup> This contrasts with other DPP4i such as saxagliptin, which has raised concerns regarding potential increased risks of heart failure, <sup>5-8</sup> and linagliptin, which is commonly prescribed for patients with renal impairment because it does not require dose modifications based on kidney function, potentially leading to increased confounding compared to sitagliptin.<sup>9,10</sup> Sodium-glucose cotransporter-2 (SGLT2) inhibitors would not be a neutral comparator, as they significantly reduce clinically important kidney events, kidney failure, and cardiovascular events.<sup>11-14</sup> Sulfonylureas (SUs), though inexpensive and widely used, are a poor comparator in cardiovascular outcome studies due to their association with hypoglycemia, weight gain, and channeling bias, as they are often prescribed to elderly, lower socioeconomic status patients with higher baseline cardiovascular risk, making direct comparisons to GLP-1-RAs less reliable.<sup>15</sup>

# 5. Research question and objectives

#### Table 1 Primary and secondary research questions and objective

### A. Primary research question and objective

| Objective: | To evaluate the effect of injectable semaglutide versus sitagliptin on MACE outcomes (CV |
|---|---|
| | death, nonfatal MI, or nonfatal stroke) in patients with diabetes and established or subclinical |
| | CV disease. |

| Hypothesis: | We hypothesize that semaglutide will be superior to sitagliptin at preventing MACE. |
|---|---|
| Population (mention key inclusion-exclusion criteria): | Individuals with T2DM, who are either aged 50 years or above with an established cardiovascular disease, or aged 60 years or above with a subclinical cardiovascular disease. |
| Exposure: | Injectable Semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Major adverse cardiac event (MACE), including myocardial infarction, stroke, and all cause death. |
| Time (when follow up begins and ends): | One day after cohort entry date until the first of outcome, disenrollment, end of study period, 365 days after cohort entry date, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP1 agonists (including oral Semaglutide), Other DPP4 or Pramlintide, Nursing home admission. |
| Setting: | Patients may be treated in outpatient settings. The outcome will be measured from inpatient hospitalizations and/or death. |
| Main measure of effect: | Hazard ratio. |

# **B.** Secondary research questions and objectives

| Objective: | To evaluate the effect of injectable semaglutide versus sitagliptin on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients meeting the eligibility criteria of the SUSTAIN-6 trial. |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will be superior to sitagliptin at preventing all-cause mortality, myocardial infarction, or stroke. |
| Population (mention key inclusion-exclusion criteria): | Individuals with T2DM, who are either aged 50 years or above with an established cardiovascular disease, or aged 60 years or above with a subclinical cardiovascular disease. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | The individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, and stroke. |

| Time (when follow up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, death, 365 days after cohort entry date, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP1 agonists (including injectable semaglutide). |
|---|---|
| Setting: | The outcome will be measured from inpatient hospitalizations and death. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the effect of injectable semaglutide versus sitagliptin on negative control outcomes, including (1) hernia and (2) lumbar radiculopathy. |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will not have a different effect than sitagliptin. |
| Population (mention key inclusion-exclusion criteria): | Individuals with T2DM, who are either aged 50 years or above with an established cardiovascular disease, or aged 60 years or above with a subclinical cardiovascular disease. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Separate analyses were run for hernia and lumbar radiculopathy. |
| Time (when follow up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, death, 365 days after cohort entry date, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP1 agonists (including injectable semaglutide). |
| Setting: | Patients may be treated in outpatient settings. The outcome will be measured from outpatient procedure codes. |
| Main measure of effect: | Hazard ratio. |

# 6. Research methods

### 6.1 Study design

Research design (e.g. cohort, case-control, etc.): New user active comparator cohort study.

Rationale for study design choice: A new user active comparator cohort study is a powerful design that may be able to address confounding by indication. It accomplishes this, in large part, through judicious selection of an appropriate active-comparator group. While selection of an appropriate comparator in the design phase is crucial, cohort studies often require additional adjustment of measurable confounders. A common method for adjusting for confounding is via a propensity score (PS).

# **6.2 Study design diagram** when following the eligibility criteria of the SUSTAIN-6 trial (Figure 1).

Cohort Entry Date (CED, Day 0) [Dispensation of exposure group (Semaglutide)] OR [Dispensation of reference group (Sitagliptin)] INCL: Anti-diabetic drug naive OR treated with 1-2 oral antidiabetics OR NPH insulin OR long-acting insulin Days [-183, 0] INCL: Age at least 50 OR 60, male or female sex Days [0, 0] dCensoring criteria: · Occurrence of outcomes EXCL: T1DM, heart failure (NYHA IV), chronic dialysis, pregnancy, proliferative retinopathy/ maculopathy
Days [-365, 0] Death Disenrollment · End of study period 365 days after CED EXCL: Prior use of Pramlintide or other GLP-1-RA/ DPP4I, chronic/ acute pancreatitis, liver disease, drug dependence/ buse disorders, nursing home admission, missing age/ gender Days [-183, 0] Discontinuation (30 days grace window and risk-window) Use of other DPP4i/ Pramlintide/ GLP-1RA (including oral semaglutide) Nursing home admission EXCL: Insulin use (except short term), diabetic ketoacidosis, acute cerebrovascular event Days [-91, 0] EXCL: Concurrent use of both study drugs Days [0] Covariate Assessment Window: BMI Days [-730, 0] Covariate Assessment Window: Pre-exposure characteristics except age, sex, BMI
Days [-365, 0] PRIMARY OUTCOME: Covariate Assessment Window: Age, sex Days [0] Composite of all-cause mortality, myocardial infarction, and stroke Follow-up Window Days [1, Censor<sup>d</sup>] Day 0 Time

Figure 1. Exposure-based cohort entry where the cohort entry date is selected after application of exclusion criteria

#### 6.3 Setting

#### 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population

Time 0 in the database study was defined to emulate randomization to treatment with injectable semaglutide versus sitagliptin in the clinical trial design. See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

#### **6.3.2** Context and rationale for study inclusion criteria:

Study inclusion criteria were defined to emulate the inclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in Appendix 3.

## 6.3.3 Context and rationale for study exclusion criteria

Study exclusion criteria were defined to emulate the exclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in Appendix 3.

#### 6.4 Variables

#### **6.4.1** Context and rationale for exposure(s) of interest

The exposure and comparator were defined to emulate the agents compared for the trial, Injectable Semaglutide versus Sitagliptin. See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

## Algorithm to define duration of exposure effect:

Assuming the effect of pill lasts for 45 days after the days' supply, we allow 45 days gap between the dispensation (grace period) and also add 45 days at the end of days' supply of dispensation (exposure risk window).

#### 6.4.2 Context and rationale for outcome(s) of interest

The primary outcome for the database study was defined to emulate the primary outcome of the trial, i.e., MACE (composite of cardiovascular death, myocardial infarction, or stroke). Due to the inability to capture cause of death in our emulation, we modified the MACE outcome to capture all-cause mortality, myocardial infarction, or stroke. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. Optum includes death information from the inpatient discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. MarketScan includes information from the inpatient discharged dead status as well as social security death master file. Medicare includes information from the inpatient discharged dead status, NDI cause of death, and social security death master file. The positive predictive value for the myocardial infarction outcome algorithm using ICD-9 codes was observed to be 88.4% and 94% in validation studies. The PPV for the ischemic stroke outcome algorithm was 95% in a validation study using ICD9 codes. The ICD9 code algorithms were mapped to ICD10 codes and reviewed by a clinician, but the performance of the mapped codes was not further validated.

Secondary outcomes from the trial that will be evaluated include:

1. Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, and stroke.

Control outcomes of interest include:

- 1. Hernia (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for tirzepatide vs dulaglutide.
- 2. Lumbar radiculopathy (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for tirzepatide vs dulaglutide.

#### 6.4.3 Context and rationale for follow up

Both on-treatment (OT) and intention-to-treat (ITT) analyses will be conducted. Adherence in clinical practice databases is expected to be much worse than in the trial, therefore the OT analysis will be the primary analysis. The OT analysis targets the relative hazard of outcomes while on treatment and may more closely emulate the effect observed in highly adherent trial participants. Both OT and ITT analyses will be conducted with up to 1-year follow-up.

**Table 2. Operational Definitions of Follow Up** 

| Follow up start | Day 1 | |
|---|---|---|
| Follow up end <sup>1</sup> | Select all that apply | Specify |
| Date of outcome | Yes | |
| Date of death | Yes | Part of the outcome |
| End of observation in data | Yes | Date of disenrollment |
| <b>Day X following index date</b> (specify day) | Yes | Day 365 |
| <b>End of study period</b> (specify date) | Yes | Dates for different databases (Optum: February 28, 2025, Marketscan December 31, 2023, Medicare December 31, 2020) |
| End of exposure<br>(specify operational details,<br>e.g. stockpiling algorithm, grace period) | Yes | 45 days grace window and 45 days risk window |
| <b>Date of add to/switch from exposure</b> (specify algorithm) | Yes | Date of augmentation or switching from an exposure to a comparator and vice versa. |
| Other date (specify) | Yes | Censor upon starting any other GLP1 agonists, including oral semaglutide, other DPP4 inhibitors or pramlintide, nursing home admission |

# 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications)

We identified a series of covariates that were likely confounders due to being strong risk factors for the primary outcome that were associated with choice of treatment. These include demographics, disease severity related variables, comorbid conditions, comedications, frailty, healthcare utilization and markers of health seeking behaviour.

**Table 3. Operational Definitions of Covariates** 

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Demographics | | | | | | | | | |
| Age | Cohort entry<br>year – year of<br>birth, (last<br>observed<br>value in the<br>baseline) | Continuous | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| Gender | Male, Female<br>(last observed<br>value in the<br>baseline) | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| Race* | White, Black,<br>Other (Asian,<br>Hispanic),<br>Missing/Unkn<br>own (last | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |

<sup>&</sup>lt;sup>1</sup> Follow up ends at the first occurrence of any of the selected criteria that end follow up.


| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Concomitant use or initiation of insulin | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of sulfonylureas | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of SGLT2i | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of other glucose-lowering drugs | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of metformin | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of insulin | | | | | | | | | |
| Doct was of | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of sulfonylureas | | | | | | | | | |
| , (OOLTO) | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of SGLT2i | | | | | | | | | |
| Past use of other glucose-lowering drugs | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart failure medic | cations | | | | | | | | |
| ACEi / ARB | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide; | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| ARNI | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Thiazides | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Beta-blockers | | | | | | | | | |
| Calcium channel | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| blockers | | | | | | | | | |
| Digoxin / Digitoxin | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide; | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | |
| Loop diuretics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Other diuretics Intravenous diuretics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Nitrates | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Other medications | | | | | | | | | |

#### Other medications

| Characteristics | Details | Type of variable | Assessmen t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Anti ovelovitlomico | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anti-arrhythmics Statins | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| PCSK9 inhibitors<br>and other lipid-<br>lowering drugs | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antiplatelet agents | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Oral<br>anticoagulants | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| COPD/Asthma<br>medication | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| NCAID | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| NSAIDs Oral | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Osteoporosis agents (incl. bisphosphonates) | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Opioids | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Characteristics | Details | Type of variable | Assessmen t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anti-depressants | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antipsychotics | | | | | | | | | |
| Anxiolytics/hypnotics, | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| benzodiazepines | | | | | | | | | |
| Medication for | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| dementia | | | | | | | | | |
| Urinary tract infections antibiotics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Laxatives | | | | | | | | | |
| Healthcare utilizat | ion markers | | | | | | | | |
| Number of distinct<br>medications,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of office<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>endocrinologist<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>cardiologist visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Number of internal<br>medicine/family<br>medicine visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Electrocardiogram<br>s, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Echocardiograms,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pharmacy out-of-<br>pocket cost,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Unique brand<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Unique generic<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Ratio of unique<br>brand to generic<br>medications,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Healthy behavior n | narkers | | | | | | | | |
| Colonoscopy /<br>Sigmoidoscopy | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Flu vaccine /<br>Pneumococcal<br>vaccine | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pap smear test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide; | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | |
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| PSA test | | | | | | | | | |
| Fecal occult blood<br>test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Bone mineral<br>density tests | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Mammograms | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure: | n/a | Appendix, |
| Telemedicine | | a. y | [ 2 3 3, 3] | , | 3. 1,113. 33 | , | Injectable<br>Semaglutide; | 1.7,5 | Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | |
| Laboratory and dia | gnostic tests | | | | | | | | |
| Number of HbA1c<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of lipid<br>panels, median<br>(iqr), mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>creatinine tests,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>natriuretic peptide<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Number of urine<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Lab values | | · | | | | | | | |
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| HbA1c** | | | | | | | | | |
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Glucose** | | | | | | | | | |
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Creatinine** | | | | | | | | | |
| Systolic blood<br>pressure** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart rate** | | | | | | | | | |
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| BMI** | | | | | | | | | |
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| eGFR** | | | | | | | | | |
| LDL** (mg/dl; | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| mean, sd) | | | | | | | | | |
| HDL** (mg/dl;<br>mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Total cholesterol**<br>(mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Triglyceride** (mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Burden of comorbi | dities | | | • | | | | | |
| Combined comorbidity score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Gagne et al.,<br>Sun et al. <sup>20,21</sup> |
| Frailty score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Kim et al. <sup>22</sup> |
| Baseline hospitaliz | rations and bos | enital matrics | | | | | | | |
| Paseille Hospitaliz | ations and nos | ppirai ilieti ics | | | | | | | |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Number of any<br>hospitalization,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Any hospitalization<br>within prior 91<br>days; n (%) | | Binary | [-91, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Any hospitalization<br>within prior 92-<br>365 days; n (%) | | Binary | [-365, -92] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| 0, 1, >1<br>hospitalizations<br>(any) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Hospitalization for heart failure; n (%) | | Binary | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Emergency<br>department visits;<br>n (%) | | Binary | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Calendar year of co | ohort entry | | | | | | | | |
| | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2018 | | | | | | | | | |
| | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2019 | | | | | | | | | |
| | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2020 | | | | | | | | | |
| 2021 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| 2022 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2023 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2024 | | | | | | | | | |
| | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide;<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2025 | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup>IP = inpatient, OP = outpatient, ED = emergency department, OT = other, n/a = not applicable

<sup>&</sup>lt;sup>2</sup>See appendix for listing of clinical codes for each study parameter

<sup>&</sup>lt;sup>3</sup>Specify whether a diagnosis code is required to be in the primary position (main reason for encounter)

<sup>\*</sup>Available for Optum Clinformatics and Medicare

<sup>\*\*</sup>Not used in the PS model

<sup>\*\*\*</sup>Available for Medicare

### **6.5 Data analysis**

### **6.5.1** Context and rationale for analysis plan

The study will use a propensity score (PS) 1:1 nearest neighbor matching with a caliper of 0.01 on the propensity score scale. The PS will be estimated as the probability of initiating injectable semaglutide versus sitagliptin given the baseline patient characteristics using multivariable logistic regression models. As diagnostics for PS models, the study will evaluate distributional covariate balance using standardized differences and c-statistics post-matching. The study will estimate the hazard ratio for injectable semaglutide versus Sitagliptin inhibitor on MACE outcome in the matched population using a Cox proportional hazards model.

Table 4. Primary, secondary, and subgroup analysis specification

#### A. Primary analysis

| Hypothesis: | Injectable Semaglutide might decrease risk of MACE outcome compared to Sitagliptin in those with diabetes |
|---|---|
| | and established or subclinical CV disease. |
| Exposure contrast: | Injectable Semaglutide vs Sitagliptin. |
| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching |
| Comounting adjustment method | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | N/A. |

# **B.** Secondary Analyses

| Hypothesis: | Injectable semaglutide does not increase the risk of occurrence of the individual components of the primary |
|---|---|
| | endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients with diabetes and established or subclinical CV disease when following the eligibility criteria of the SUSTAIN-6 trial. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards for all-cause mortality, Aalen-Johansen estimator for myocardial |
| (provide details or code) | infarction and stroke to account for the competing risk of death. |
| | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Injectable semaglutide has no effect on risk of negative control outcomes compared to sitagliptin. Negative |
|---|---|
| | control outcomes include (1) hernia and (2) lumbar radiculopathy. |
| Exposure contrast: | njectable semaglutide vs sitagliptin. |
| Outcome: | Separate analyses were run for each negative control outcome, including (1) hernia and (2) lumbar radiculopathy |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | utcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |

| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
|---|---|
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | N/A. |

Table 5. Sensitivity analyses – rationale, strengths and limitations

| | What is being varied? How? | Why?<br>(What do you expect to<br>learn?) | Strengths of the sensitivity analysis compared to the primary | Limitations of the sensitivity analysis compared to the primary |
|---|---|---|---|---|
| Negative control outcomes, including hernia, lumbar radiculopathy | We evaluate negative control outcomes of hernia and lumbar radiculopathy, where no causal effect is expected from tirzepatide, or dulaglutide. | We will evaluate the potential impact of residual confounding on this outcome for which there is not expected to be a causal effect | The evaluates the robustness of the interpretation of the primary analysis by evaluating the potential magnitude of unmeasured confounding | This analysis assumes that the confounding structure is the same or similar for the negative control outcome as the outcome of interest |
| Effect estimation in individuals with HbA1c measurement. | The population will be restricted to individuals with a HbA1c measurement in the 120 days before cohort entry. | To assess the impact of restricting to individuals with HbA1c measurement and including HbA1c in the PS model. | Includes baseline glycemic information as captured in laboratory HbA1c measurements. | This approach highly restricts the number of eligible individuals under study and thereby the statistical power of the analysis. |
| As-started analyses (observational analogue to intention-to-treat) to address potential informative censoring. | To address potential informative censoring. | We will consider the first-<br>used medication for 365<br>days without considering<br>drug discontinuation or<br>switching, mimicking an<br>"intention-to-treat"<br>approach. | Reflects follow-up regimen of RCT. | Persistence of drug use is shorter in clinical practice whereas adherence is typically higher in RCTs. Therefore, we expect the estimated effects will be diluted toward the null, underestimating the true treatment effect had patients remained on therapy. |

#### **6.5.2 Comparison of Results Between Database Studies and RCTs**

We will attempt to benchmark the results of the secondary analysis from the database study against the composite end point of MACE observed in the SUSTAIN-6 trial. It is important to note that this end point had few outcomes in the trial. Consequently, failure to replicate the RCT findings is not necessarily indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons, nor does failure to replicate provide information about the validity of the trial result.<sup>23</sup> Assessment of concordance in results between the database study-trial pair will use the

metrics previously implemented in the RCT-DUPLICATE initiative, namely statistical significance agreement, estimate agreement, and standardized difference agreement. In this project, "full" statistical significance agreement was defined by estimates and confidence intervals on the same side of null; estimate agreement was defined by whether estimates for the trial emulation fell within the 95% CI for the trial results; standardized difference agreement between treatment effect estimates from trials and emulations was defined by standardized differences |Z| < 1.96 ( $Z = \frac{(\theta_{RCT} - \theta_{RWE})}{(\sqrt{q^2}_{RCT} - \theta^2_{RWE})}$  where are the treatment effect estimates and the  $\hat{\sigma}^2$  are associated variances). In addition, "partial" significance agreement was defined as meeting pre-specified non-inferiority criteria even though a more highly powered database study may have indicated superiority.<sup>23,24</sup>

#### 6.6 Data sources

#### 6.6.1 Context and rationale for data sources

Reason for selection: The study will be conducted in 3 US health care claims databases: Optum Clinformatics (2018-Feb 2024), Merative Marketscan (2018-2022) and Medicare (a sample that includes all patients with diabetes or heart failure diagnosis, 2018-2020)

Strengths of data source(s): Each data source contains deidentified, longitudinal, date-stamped information on patient enrollment, demographics, inpatient/outpatient diagnosis and procedures, admission and discharge dates, and medication dispensation. The death data is captured in the Optum database from inpatient discharge status, social security death master file, and deaths scraped from obituaries or other sources. The death data in MarketScan is captured from the social security death master file and inpatient discharge status. It is recognized that the social security death master file has high specificity and positive predictive value for deaths. While this data resource has under captured deaths since 2011, the capture of deaths is not expected to be differential between compared exposure groups. The death data is captured in the Medicare database from inpatient discharge status, and social security death master file.<sup>25–27</sup>

Limitations of data source(s): Patient healthcare encounters are only observable when they are enrolled in an insurance plan that contributes to the database. Patients may change insurance plans for multiple reasons. Both Optum Clinformatics and Merative MarketScan are primarily employer based insurance databases where patients may disenroll with job changes. Patients in Medicare may move in and out of fee-for-service plans. We are excluding person-time in health maintenance organization (HMO) plans due to concerns about the completeness of capture of diagnoses and procedures. This means that we require patients to be enrolled in Medicare parts AB and D during the baseline assessment window and censor patients if they switch to part C. In claims data, dispensing data for inpatient medication is unavailable. Diagnoses reflect billing practices, therefore algorithms (preferably validated) are needed for accurate phenotyping of patient conditions. Services that are not covered by insurance do not appear in the data. The trial evaluated cardiovascular deaths, however we will evaluate all cause death in the emulation because most deaths in this cohort of patients at high cardiovascular risk will be related to cardiovascular reasons, the cause of death is not recorded for databases not linked to NDI, and the performance of NDI at identifying cardiovascular causes of death may be suboptimal.<sup>27</sup>

Data source provenance/curation: Information about Optum Clinformatics and Merative MarketScan can be found in data dictionaries and user guides that are provided to clients. Information about Medicare data provenance and curation can be found on the ResDac website.<sup>28</sup>

Table 6. Metadata about data sources and software

| | Data 1 | Data 2 | Data 3 |
|---|---|---|---|
| Data Source(s): | Optum Clinformatics | Merative Marketscan | Medicare |
| Study Period: | 1 <sup>st</sup> Jan 2018-28 <sup>th</sup> Feb 2025 | 1 <sup>st</sup> Jan 2018-31 <sup>st</sup> Dec 2023 | 1 <sup>st</sup> Jan 2018-31 <sup>st</sup> Dec 2020 |
| Eligible Cohort Entry Period: | 1 <sup>st</sup> Jan 2018-28 <sup>th</sup> Feb 2025 | 1 <sup>st</sup> Jan 2018-31 <sup>st</sup> Dec 2023 | 1 <sup>st</sup> Jan 2018-31 <sup>st</sup> Dec 2020 |
| Data Version (or date of last update): | April 2025 | Mortality Cut Set A<br>Received 2025-05-01 | DUA 59286_Received 2023-10-17 |
| Data sampling/extraction criteria: | n/a | n/a | Patients with a diabetes or heart failure diagnosis |
| Type(s) of data: | Administrative healthcare claims | Administrative healthcare claims | Administrative healthcare claims |
| Data linkage: | n/a | n/a | Linkage to National Death<br>Index |
| Conversion to CDM*: | n/a | n/a | n/a |
| Software for data management: | Aetion Evidence Platform® (2025) | Aetion Evidence Platform® (2025) | Aetion Evidence Platform® (2025) |

<sup>\*</sup>CDM = Common Data Model

#### **6.7 Data management**

Tracking data: The Data Use Agreement (DUA) Custodian (Principal Investigator) and the Division Operations Manager (Winta Tekle) are responsible for receiving and creating a record of new data associated with the given request. The Operations Manager is responsible for all indexing and archiving of documents and electronic media related to data that the Division receives and will log data location, data contents, and associated DUA and Institutional Review Board (IRB) numbers in the Division's centralized tracking system.

Handling and storage: In-scope data will be stored utilizing Mass General Brigham approved information systems – i.e., Division servers and Mass General Brigham network storage.

Archiving: Data retention and any removal will be executed by the Division Operations Manager (Winta Tekle) and Data Manager (Todd MacGarvey). The Division follows Mass General Brigham enterprise record retention policies and follow the terms of the agreement through which the in-scope data was received.

Information security: The Division follows Mass General Brigham's Enterprise Information Security Program (EISP). The EISP helps by providing assurance that Mass General Brigham information and information systems are protected from unauthorized access, use, disclosure, duplication, modification, or destruction in order to maintain their confidentiality, integrity, and availability. To that end, the EISP policies, standards and procedures

create an information security framework that is aligned with the recommendations of the International Organization for Standardization's (ISO) publication 27001 and the National Institute of Standards and Technology's (NIST) publication 800-53 Family of Controls and MGB regulatory and legal requirements (as a HIPAA covered entity).

Mass General Brigham workforce members are required to complete new workforce privacy and information security training upon hire and annually thereafter. Refresh training is provided as appropriate. Mass General Brigham workforce members are required to review and sign a Confidentiality Agreement upon hire and annually thereafter. Additionally, we follow Enterprise Information Security and Privacy policies, including Managing Workforce Members Information Security Responsibilities Policy, which was developed to help assure that Mass General Brigham workforce members are competent and eligible to support the information security responsibilities associated with their role. Mass General Brigham workforce, including Division staff, are required to comply with Enterprise Information Security and Privacy Policies.

Facilities: The research team uses a highly secure, state-of-the-art, computing facility housed at Mass General Brigham's Corporate Data Centers in Needham and Marlborough, Massachusetts as well as Amazon Web Services (AWS). We maintain redundant storage for maximal data integrity and high-speed data access.

The Division uses Mass General Brigham corporate provisioned servers to analyze and store data in connection with this project. There are strict access controls enforced by technical means to ensure that only study staff who have been approved to conduct data analyses and contracted data engineers are able to access data (e.g., Mass General Brigham Authentication (Active Directory) utilized; auditing, logging, and monitoring enabled; firewalls enabled; etc.). All Division servers used in this study are accessible to only authorized staff only through the MGB network and utilizing VPN as appropriate (i.e., users must be on the network and logged into VPN to access). Mass General Brigham has a network information security monitoring team and in-scope servers are enrolled in enterprise security tools (e.g., vulnerability scanning service, antivirus, etc.).

The Division also uses AWS. In-scope AWS services / resources have undergone review and assessment by Mass General Brigham's Information Security Risk Assessment Team/ InfoSec Risk Management Team as required and in alignment with NIST 800-30: Guide for Conducting Risk Assessments. In-scope AWS servers are for our exclusive use (reserved instances), are covered under our organization's Business Associate Agreement with AWS. In-scope servers are housed in anonymous facilities that are not branded as AWS facilities. Physical access is strictly controlled both at the perimeter and at building ingress points by professional security staff utilizing video surveillance, intrusion detection systems, and other electronic means.

Security attributes and controls for the Division's use of in-scope AWS in connection with this project include: encryption at rest and in transit (industry standard AES-256 encryption, SSL/TSL), anti-malware, latest OS updates and patches as well as anti-virus; multi-factor authentication (MFA), Identity and Access Management, including SSO; auditing and logging; principle of least privilege, including for traffic and ports (e.g., deny all default configurations), use of VPC enabled Step functions, etc.; separation between environments; minimum necessary (out of the box AWS roles are not used as they can be overly permissive); all data would reside in the US domestic regions – use only US east HIPAA compliant region; performance monitoring enabled and reviewed as per internal processes; passwords compliant with enterprise password policy and, as appropriate, more protective password requirements; etc. Our Division's AWS use is also subject to ongoing evaluation and monitoring as well – e.g., vulnerability scanning and management, access review, etc.

A data file list will be maintained in Amazon S3 and tracked through Cloudtrail and Cloudwatch. Reporting of data file availability for any file stored in an S3 bucket will be controlled by MGB.

Amazon EC2, Amazon EBS, and Amazon VPC are integrated with AWS CloudTrail, a service that provides a record of actions taken by a user, role, or an AWS service in Amazon EC2, Amazon EBS, and Amazon VPC. CloudTrail captures all API calls for Amazon EC2, Amazon EBS, and Amazon VPC as

events, including calls from the console and from code calls to the APIs. MGB IT/security staff have full access to CloudTrail to ensure that CloudTrail monitoring is available at all times. Amazon CloudWatch Events delivers a near-real-time stream of system events that describe changes in AWS resources. Amazon CloudTrail can log, continuously monitor, and retain account activity related to actions across the MGB AWS infrastructure. CloudTrail provides event history of MGB AWS account activity. This event history simplifies security analysis, resource change tracking, and troubleshooting and complies with requirements to ensure the data file inventory is controlled by MGB.

Backups: Backups are created using industry recognized Cryptographic mechanisms (e.g., 256-bit AES encryption) as appropriate and required. Data are backed up within the MGB network from the MGB Needham data center to the MGB Marlborough data center via replication/mirroring and volume-level snapshots. AWS Backup supports both instance-level backups as Amazon Machine Images (AMIs) and volume-level backups as separate snapshots based on the resource tags. AMIs allow MGB IT and security staff to create backups of all S3 and EC2 instances. This backup approach allows elimination of EC2 instances when access to CMS data files is no longer needed. Use of temporary instances will allow highest security control to be applied regarding for whom and when CMS data files are accessible.

In addition to the safeguards listed above, the Division follows enterprise privacy and information security policies and maintains internally procedures in connection with this project to safeguard the data in connection with this project as appropriate and required including: Physical Security and Environmental Controls for Electronic Information Policy; IT Access Control Standards for Users policy; Safeguarding Fax Copiers Printers Telephone Use and Pagers; Physical Removal and Transport of Protected Health Information and Personal Information policy, etc.

#### **6.8. Quality control**

Senior Programmers and Research Specialists perform QA/QC on raw or common data model converted data via SAS/R/Aetion software. The protocol will be iteratively developed and pre-specified data checks including feasibility counts and balance on baseline covariates will be conducted with outputs reviewed by both MGB and FDA team members. Team members will review code lists to ensure fidelity to intended algorithms.

## 6.9. Study size and feasibility

See appendix 4 and appendix 5 (feasibility, weighting on age, sex, comorbidity score as well as all predefined propensity score variables). Propensity score distribution plots with c-statistics are available in appendix 6. Table 1 showing prevalence of baseline characteristics and standardized differences in distribution are available in appendix 7. Additional diagnostic evaluations, including balance assessments of laboratory and clinical examination test results not included in the propensity score as well as assessment of heart failure-related medication after follow-up, will be conducted to assess potential residual confounding and divergence of treatment over time.

#### 7. Limitation of the methods

As we are using secondary data and the data were not collected for research, some important variables may not be collected or will be measured imperfectly. We have selected validated algorithms when possible and we have created proxies for important variables that are not directly captured in the data to reduce confounding by unmeasured factors. One measurement difference is for the primary outcome, where for the RCT, MACE was defined as stroke, myocardial infarction, and cardiovascular death, whereas in our database study, it is defined as stroke, myocardial infarction, and all cause death.

When comparing results from an RCT to a database study that emulates the design, we assume that the findings from the single RCT are internally valid.

Although we plan to emulate the important features of each RCT as closely as possible in healthcare claims, there may be some elements of RCT design that are not emulable with a database study, which means that the study generating RWE and the RCT will address slightly different clinical questions. For example, in routine clinical practice, adherence to treatment is typically not as high as it is in an RCT with strong measures in place to encourage adherence to the study protocol. This means that there is more discontinuation and short-term medication use in the patients identified in claims databases than trial participants.

Apparent agreement between RCT and database study results could occur if the effects of multiple factors (chance, emulation differences, bias) cancel each other out.

## 8. Protection of human subjects

This study has been approved by the Brigham and Women's Hospital Institutional Review Board.

#### 9. References

- 1. Marso S, Bain S, Consoli A, et al. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. *The New England journal of medicine*. 2016;375(19). doi:10.1056/NEJMoa1607141
- 2. A Long-term, Randomised, Double-blind, Placebo-controlled, Multinational, Multi-centre Trial to Evaluate Cardiovascular and Other Long-term Outcomes With Semaglutide in Subjects With Type 2 Diabetes (SUSTAIN<sup>™</sup> 6 Long-term Outcomes). June 20, 2019. Accessed July 26, 2025. https://clinicaltrials.gov/study/NCT01720446
- 3. News Details. Novo Nordisk. Accessed February 17, 2025. https://www.novonordisk.com/content/nncorp/global/en/news-and-media/news-and-ir-materials/news-details.html
- 4. Green Jennifer B., Bethel M. Angelyn, Armstrong Paul W., et al. Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes. *New England Journal of Medicine*. 2015;373(3):232-242. doi:10.1056/NEJMoa1501352
- 5. Scirica BM, Bhatt DL, Braunwald E, et al. Saxagliptin and Cardiovascular Outcomes in Patients with Type 2 Diabetes Mellitus. *New England Journal of Medicine*. 2013;369(14):1317-1326. doi:10.1056/NEJMoa1307684
- 6. Heart Failure, Saxagliptin, and Diabetes Mellitus: Observations from the SAVOR-TIMI 53 Randomized Trial. doi:10.1161/CIRCULATIONAHA.114.010389
- 7. A Multicenter Observational Study of Incretin-based Drugs and Heart Failure | New England Journal of Medicine. Accessed December 2, 2024. https://www-nejmorg.emedien.ub.uni-muenchen.de/doi/10.1056/NEJMoa1506115
- 8. Risk for Hospitalized Heart Failure Among New Users of Saxagliptin, Sitagliptin, and Other Antihyperglycemic Drugs: A Retrospective Cohort Study: Annals of Internal Medicine: Vol 164, No 11. Accessed December 2, 2024. https://www.acpjournals.org/doi/10.7326/M15-2568

- 9. Patorno E, Gopalakrishnan C, Bartels DB, Brodovicz KG, Liu J, Schneeweiss S. Preferential prescribing and utilization trends of diabetes medications among patients with renal impairment: Emerging role of linagliptin and other dipeptidyl peptidase 4 inhibitors. *Endocrinology, Diabetes & Metabolism*. 2018;1(1):e00005. doi:10.1002/edm2.5
- 10. Gallwitz B. Safety and efficacy of linagliptin in type 2 diabetes patients with common renal and cardiovascular risk factors. *Therapeutic Advances in Endocrinology*. 2013;4(3):95-105. doi:10.1177/2042018813486165
- 11. Packer M, Anker SD, Butler J, et al. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. *N Engl J Med*. 2020;383(15):1413-1424. doi:10.1056/NEJMoa2022190
- 12. McMurray JJV, Solomon SD, Inzucchi SE, et al. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019;381(21):1995-2008. doi:10.1056/NEJMoa1911303
- 13. Solomon SD, McMurray JJV, Claggett B, et al. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. *N Engl J Med*. 2022;387(12):1089-1098. doi:10.1056/NEJMoa2206286
- 14. Anker SD, Butler J, Filippatos G, et al. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. *N Engl J Med*. 2021;385(16):1451-1461. doi:10.1056/NEJMoa2107038
- 15. Mohan V, Saboo B, Khader J, et al. Position of Sulfonylureas in the Current ERA: Review of National and International Guidelines. *Clin Med Insights Endocrinol Diabetes*. 2022;15:11795514221074663. doi:10.1177/11795514221074663
- 16. Schneeweiss, S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. *Pharmacoepidemiology and drug safety*. 2010;19(8). doi:10.1002/pds.1926
- 17. Ray W. Evaluating medication effects outside of clinical trials: new-user designs. American journal of epidemiology. 2003;158(9). doi:10.1093/aje/kwq231
- 18. Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. *Pharmacoepidemiol Drug Saf.* 2010;19(6):596-603. doi:10.1002/pds.1924
- 19. Kiyota Y, Schneeweiss S, Glynn R, Cannuscio C, Avorn J, Solomon D. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. *American heart journal*. 2004;148(1). doi:10.1016/j.ahj.2004.02.013
- 20. Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. *J Clin Epidemiol*. 2011;64(7):749-759. doi:10.1016/j.jclinepi.2010.10.004
- 21. Sun JW, Rogers JR, Her Q, et al. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. *Med Care*. 2017;55(12):1046-1051. doi:10.1097/MLR.0000000000000824
- 22. Kim DH, Schneeweiss S, Glynn RJ, Lipsitz LA, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. *J Gerontol A Biol Sci Med Sci*. 2018;73(7):980-987. doi:10.1093/gerona/glx229
- 23. Wang SV, Schneeweiss S, RCT-DUPLICATE Initiative, et al. Emulation of Randomized Clinical Trials With Nonrandomized Database Analyses: Results of 32 Clinical Trials. *JAMA*. 2023;329(16):1376. doi:10.1001/jama.2023.4221

- 24. Franklin JM, Pawar A, Martin D, et al. Nonrandomized Real-World Evidence to Support Regulatory Decision Making: Process for a Randomized Trial Replication Project. Clin Pharmacol Ther. 2020;107(4):817-826. doi:10.1002/cpt.1633
- 25. Jarosek, S. Death Information in the Research Identifiable Medicare Data | ResDAC. Accessed July 26, 2025. https://resdac.org/articles/death-information-research-identifiable-medicare-data
- 26. Hill M, Rosenwaike I. The Social Security Administration's Death Master File: the completeness of death reporting at older ages. *Social security bulletin*. 2001;64(1). Accessed July 26, 2025. https://pubmed.ncbi.nlm.nih.gov/12428517/
- 27. Olubowale O, Safford M, Brown T, et al. Comparison of Expert Adjudicated Coronary Heart Disease and Cardiovascular Disease Mortality With the National Death Index: Results From the REasons for Geographic And Racial Differences in Stroke (REGARDS) Study. *Journal of the American Heart Association*. 2017;6(5). doi:10.1161/JAHA.116.004966
- 28. Research Data Assistance Center (ResDAC). Accessed July 26, 2025. https://resdac.org/

# 10. Appendices

See accompanying excel files that specify the cohort study.

- 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment
- 2 Code algorithms
  - 2a Exposure
  - 2a Inclusion
  - 2c Exclusion
  - 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- **8 Covariate Algorithm Sources**

### **Appendices**

- 1 Target Trial Framework, Operational Definitions and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate algorithm sources

| SUSTAING | ОРТИМ | MEDICARE | MARKETSCAN | Notes/Questions | Color coding |
|---|---|---|---|---|---|
| Treatment assignment Parallel, randomized (treatment A vs B) double blin (time 0, index date) double-dummy | exclusion criteria) | (first eligible entry to study population) | Non-randomized initiation of treatment A vs B (first eligible entry to study population) | | Good proxy definition |
| | Code type: NDC, generic name<br>Care setting: N/A<br>Diagnosis position: N/A | Code type: NDC, generic name Care setting: N/A Diagnosis position: N/A | Code type: NDC, generic name Care setting: N/A Diagnosis position: N/A | | |
| | Washout window: [-183, -1] Incident with respect to: semaglutide and sitagliptin in any | Washout window: [-183, -1] | Washout window: [-183, -1] Incident with respect to: semaglutide and sitagliptin in any dose | | |
| Semaglutide (once-weekly in drug naïve subjects - | dose or formulation Assessement window: N/A | or formulation Assessement window: N/A | or formulation Assessement window: N/A | Algorithm detail: We defined Semaglutide using | |
| monotherapy) Exposure Two experimental arms: (1.0mg and 0.5mg) | Source of algorithm: drug names linked to NDC Measurement characteristics: N/A Code type: NDC | Source of algorithm: drug names linked to NDC Measurement characteristics: N/A Code type: NDC | Source of algorithm: drug names linked to NDC Measurement characteristics: N/A Code type: NDC | NDC codes for drug brand name Ozempic, route of administration injectable, with doses up to 1mg. | Moderate proxy definition |
| | Care setting: N/A Diagnosis position: N/A | Care setting: N/A<br>Diagnosis position: N/A | Care setting: N/A<br>Diagnosis position: N/A | | |
| | Washout window: [-183, -1] Incident with respect to: semaglutide and sitagliptin in any dose or formulation | Washout window: [-183,-1]<br>Incident with respect to: semaglutide and sitagliptinin any dose<br>or formulation | Washout window: [-183, -1]<br>Incident with respect to: semaglutide and sitagliptin in any dose<br>or formulation | Algorithm detail: We used sitagliptin as an active | |
| | Assessement window: N/A<br>Source of algorithm: drug names linked to NDC | Assessement window: N/A Source of algorithm: drug names linked to NDC | Assessement window: N/A Source of algorithm: drug names linked to NDC | comparator proxy for placebo. We allowed sitagliptin alone or in combination pills with | Poorly measured in database but not |
| Comparator Placebo | Measurement characteristics: Code type: DX Care setting: Inpatient for stroke/MI, any for death | Measurement characteristics: Code type: DX Care setting: Inpatient for stroke/MI, any for death | Measurement characteristics: Code type: DX Care setting: Inpatient for stroke/MI, any for death | metformin only. Algorithm detail: Optum death includes information | critical for the analysis |
| | Diagnosis position: Primary for Stroke, any for MI Washout window: | Diagnosis position: Primary for Stroke, any for MI Washout window: | Diagnosis position: Primary for Stroke, any for MI Washout window: | from the inpatient discharged dead status, social security death master file, and deaths scraped from | |
| | Source of algorithm: PROMISE team Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94%. | Source of algorithm: PROMISE team Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94%. | Source of algorithm: PROMISE team Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94%. | obituaries or other sources. MarketScan includes information from the inpatient discharged dead status up until 2016. | |
| MACE, Defined as Cardiovascular Death, Non-fatal | PPV for ischemic stroke using ICD9 codes was 88% and 95%.<br>Both of the above ICD9 codes were mapped to ICD10, but no | PPV for ischemic stroke using ICD9 codes was 88% and 95%<br>Both of the above ICD9 codes were mapped to ICD10, but no | PPV for ischemic stroke using ICD9 codes was 88% and 95%<br>Both of the above ICD9 codes were mapped to ICD10, but no | Medicare includes information from the inpatient discharged dead status, NDI cause of death, and | Poorly measured and important for the |
| Primary Outcome Myocardial Infarction, or Non-fatal Stroke Follow up start Randomization date | validation study was performed. One day after date of initiation of treatment A vs B Earliest of: Outcome, end of data/study period, 109 weeks, | validation study was performed. One day after date of initiation of treatment A vs B Earliest of: Outcome, end of data/study period, 109 weeks, | validation study was performed. One day after date of initiation of treatment A vs B Earliest of: Outcome, end of data/study period, 109 weeks, | social security death master file. | analysis |
| Time Frame: Time from randomisation up to end of | discontinuation (45 days grace window and risk-window),<br>switch within or between GLP1 and DPP4 class or add | discontinuation (45 days grace window and risk-window), switch within or between GLP1 and DPP4 class or add pramlintide, | discontinuation (45 days grace window and risk-window), switch within or between GLP1 and DPP4 class or add pramlintide, | | |
| Follow up end follow-up (scheduled at week 109) Causal estimand Modified intention-to-treat Effect estimation | pramlintide, disenrollment, nursing home stay On-treatment Cox proportional hazards regression model | disenrollment, nursing home stay On-treatment Cox proportional hazards regression model | disenrollment, nursing home stay On-treatment Cox proportional hazards regression model | | |
| Inclusion criteria | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | | |
| | Assessment window: [-365, 0] Code type: DX Care setting: Any | Assessment window: [-365, 0] Code type: DX Care setting: Any | Assessment window: [-365, 0] Code type: DX Care setting: Any | | |
| | Diagnosis position: Any<br>Source of algorithm: PROMISE team | Diagnosis position: Any<br>Source of algorithm: PROMISE team | Diagnosis position: Any<br>Source of algorithm: PROMISE team | | |
| 1 Type 2 DM | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] | Algorithm detail: Not considered in the main cohort | |
| | Code type: DX<br>Care setting: Any | Code type: DX Care setting: Any | Code type: DX<br>Care setting: Any | due to high missingness of HbA1c measurements. A sensitivity analyses on a subset of the cohort with | |
| 2 HbA1c above or equal to 7.0% at screening | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | HbA1c measurements will be conducted in the<br>cohort from the Optum database, including the last<br>recorded value in the propensity score. | |
| Anti-diabetic drug naïve, or treated with one or two oral antidiabetic drug (OAD | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Algorithm detail: We are implementing this by | |
| treated with human Neutral Protamin Hagedorn (Ni<br>insulin or | Care setting: n/a | Assessment window: [-183, 0] Code type: NDC Care setting: n/a | Assessment window: [-183, 0] Code type: NDC Care setting: n/a | scoring each class of antidiabetic medications as 1.<br>Insulin long acting and/or mixed is scored and all<br>other oral antidiabetic medications including | |
| long-acting insulin analogue or pre-mixed insulin, by types of insulin either alone or in combination with a retwo OADs | oth Diagnosis position: n/a one Source of algorithm: PROMISE team Measurement characteristics: N/A | Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A | Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A | combinations are scored as 1. If patients have score of more than 3 then we exclude them. | |
| 4a or 4b | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | exclude tient. | |
| Age above or equal to 50 years at screening | Assessment window: [0, 0] Code type: n/a Care setting: n/a | Assessment window: [0, 0] Code type: n/a Care setting: n/a | Assessment window: [0, 0] Code type: n/a Care setting: n/a | | |
| and clinical evidence of cardiovascular disease (specified below). | Diagnosis position: n/a<br>Source of algorithm: n/a | Diagnosis position: n/a Source of algorithm: n/a | Diagnosis position: n/a Source of algorithm: n/a | | |
| 4a Established CVD as one of the following: | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | | |
| | Code type: DX<br>Care setting: Any | Code type: DX<br>Care setting: Any | Code type: DX<br>Care setting: Any | | |
| 4a1 prior myocardial infarction | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | | |
| | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0] | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | | |
| | Code type: DX Care setting: Any Diagnosis position: Any | Code type: DX Care setting: Any Diagnosis position: Any | Code type: DX Care setting: Any Diagnosis position: Any | | |
| 4a2 prior stroke or prior transient ischemic attack | Source of algorithm: PROMISE team<br>Measurement characteristics: N/A | Source of algorithm: PROMISE team<br>Measurement characteristics: N/A | Source of algorithm: PROMISE team<br>Measurement characteristics: N/A | | |
| | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0]<br>Code type: DX | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0]<br>Code type: DX | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0]<br>Code type: DX | | |
| | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, Investigator review of | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, Investigator review of | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, Investigator review of | | |
| prior coronary, carotid or peripheral arterial 4a3 revascularization | Source of algorithm: PROMISE team, Investigator review of codes Measurement characteristics: N/A | Source of algorithm: PROMISE team, Investigator review of codes Measurement characteristics: N/A | Source of algorithm: PROMISE team, Investigator review of codes Measurement characteristics: N/A | | |

| | | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: PX | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: PX | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: PX | |
|---|---|---|---|---|---|
| | more than 50% stenosis on angiography or imaging of | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Algorithm detail: Part of this is captured in the above inclusion criteria. We also added peripheral vascular disease and coronary artery disease codes |
| 4a4 | coronary, carotid or lower extremities arteries<br>history of symptomatic coronary heart disease<br>documented by e.g. positive exercise stress test or | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A | to be inclusive. |
| 4a5 | any cardiac imaging or unstable angina with ECG changes asymptomatic cardiac ischemia documented by | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| 4a6 | positive nuclear imaging test or exercise test or stress<br>echo or any cardiac imaging | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| | | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0]<br>Code type: DX<br>Care setting: Any | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0]<br>Code type: DX<br>Care setting: Any | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0]<br>Code type: DX<br>Care setting: Any | Algorithm detail: We defined by using heart failure |
| 4a7 | chronic heart failure New York Heart Association<br>(NYHA) class II-III | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Diagnosis position: Any<br>Source of algorithm: PROMISE team<br>Measurement characteristics: N/A | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | codes (patients with type 4 heart failure are<br>excluded so hopefully that will help with capturing<br>patients with milder heart failur of this class). |
| | Chronic renal impairment, documents by estimated | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | |
| 4a8 | eGFR < 60 ml/min/1.73 m2 per MDRD Aged 60 years or older | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [0,0] | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [0, 0] | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [0, 0] | Algorithm detail: We defined it by CKD 3-4. |
| | (specified below).<br>Subclinical cardiovascular risk factors as one of the | Code type: r/a Care setting: n/a Diagnosis position: n/a Source of algorithm: n/a | Code type: r/a Care setting: n/a Diagnosis position: n/a Source of algorithm: n/a | Code type: n/a Care setting: n/a Diagnosis position: n/a Source of algorithm: n/a | |
| 4b | following: | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX | Algorithm detail: We defined it using the diagnosis |
| 4h1 | persistent microalbuminuria (30–299 mg/g) or | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | code for conditions where proteinuria is present<br>(conditions like nephrotic syndrome) or conditions<br>defining proteinuria (example: isolated proteinuria,<br>bence jones proteinuria). |
| | hypertension and left ventricular hypertrophy by<br>electrocardiogram or imaging<br>left ventricular systolic or diastolic dysfunction by<br>imaging | Can't measure in claims Can't measure in claims | Can't measure in claims Can't measure in claims | Can't measure in claims Can't measure in claims | |
| 403 | maging | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | Applied before/after selection of index date: Before<br>Assessment window: [all available data, 0]<br>Code type: DX<br>Care setting: Any | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | |
| 4b4 | ankle/brachial index less than 0.9 | Diagnosis position: Any Source of algorithm: Investigator review of codes Measurement characteristics: N/A | Diagnosis position: Any Source of algorithm: Investigator review of codes Measurement characteristics: N/A | Diagnosis position: Any Source of algorithm: Investigator review of codes Measurement characteristics: N/A | Algorithm detail: We defined it using the diagnosis code for atherosclerosis of native arteries of extremities with intermittent claudication. |
| Exclusion Criteria | | Applied before/after selection of index date: Before Assessment window: [-365,0] | Applied before/after selection of index date: Before<br>Assessment window: [-365,0] | Applied before/after selection of index date: Before<br>Assessment window: [-365, 0] | |
| | Type 1 diabetes mellitus, Secondary diabetes, | Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Algorithm detail: Secondary diabetes, Gestational |
| 1 | Gestational diabetes | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-183, 0] Code type: NDC Care setting: ://a | Measurement characteristics: N/A<br>Applied before/after selection of findex date: Before<br>Assessment window: [183,0]<br>Code type: NDC<br>Care setting: n/a | Measurement characteristics: N/A<br>Applied before/after selection of index date: Before<br>Assessment window: [-183, 0]<br>Code type: NDC<br>Care setting: n/a | diabetes are the 2 additional criteria added. |
| 2 | Use of glucagon-like peptide-1 (GLP-1) receptor agonist (exendite), insplicitly, or other) or pramlintide within 90 days prior to screening | Diagnosis position: "A Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-183,0] Code type: NDC Care setting: n/a | Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of findex date: Before Assessment window: [-183, 0] Code type: NDC Care setting: n/a | Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before 'after selection of index date: Before Assessment window: [-183, 0] Code type: NDC Care setting: n/a | |
| 3 | Use of any dipeptidyl peptidase 4 (DPP-IV) inhibitor within 30 days prior to screening | Diagnosis position: r/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of findex date: Before Assessment window: [-91,0] Code type: Generic | Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-91, 0] Code type: Generic | Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-91,0] Code type: Generic | |
| 4 | Treatment with insulin other than basal and pre-mixed insulin within 90 days prior to screening - except for short-term use in connection with intercurrent illness | Care setting: n/a Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-91, 0] Code type: D/S | Care setting: n/a Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-91,0] Code type: DX | Care setting: n/a Diagnosis position:n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-91, 0] Code two: DX | |
| 5 | Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent acute complications of diabetes (eg diabetic ketoacidosis) within 90 days prior to screening | | Care setting: n/a Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A | Care setting: n/a Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A | Algorithm detail: We defined it by diagnosis of diabetes ketoacdiosis (DKA) OR Hyper osmolar hypergycemic non-ketotic syndrome (HONK). |

| 7 | History of chronic pancreatitis or idiopathic acute pancreatitis Acute coronary or cerebro-vascular event within 90 days prior to randomisation | Applied before/after selection of index date: Before Assessment window: [-183,0] Code type: DX X Care setting: n/a Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-91,0] Code type: DX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [:183,0] Code tyne: DX Care setting: n/a Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [:91,0] Code tyne: DX Care setting: Inpatient Diagnosis position: Arry Source of algorithm: PROMISE team Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [:183,0] Code tyne: DX Care setting: n/a Diagnosis position: n/a Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [:91,0] Code tyne: DX Care setting: Inpatient Diagnosis position: Arry Source of algorithm: PROMISE team Measurement characteristics: N/A | Algorithm detail: We defined this using diagnosis codes for acute MI, ita, unstable angina, stable angina in inpatients setting. |
|---|---|---|---|---|---|
| ۰ | Currently planned coronary, carotid or peripheral artery revascularisation | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| | Chronic heart failure New York Heart Association<br>(NYHA) class IV | Applied before/after selection of index date: Before Assessment window: [:365,0] Code type: DN, PX Care setting: IP, Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | Applied before/after selection of index date: Before Assessment window: [365, 0] Code type: DX, PX Care setting: IP, Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | Applied before/after selection of index date: Before Assessment window: [365, 0] Code type: DX, PX Care setting: IP, Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | Algorithm detail: We defined this as heart failure codes in inpatient setting with oxygen use code on the same day. |
| | Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma | Assessment window: [all available data, 0] Code type: DX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any | Assessment window: [all available data, 0] Code type: DX Care setting: Inpatient Dlagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any | Assessment window: [all available data, 0] Code type: DX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any | |
| | Personal history of non-familial medullary thyroid | Source of algorithm: Investigator review of codes | Source of algorithm: Investigator review of codes | Source of algorithm: Investigator review of codes | Algorithm detail: Assessment window may not |
| 11 | carcinoma | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A | capture cancer in distant past. |
| 13 | Chronic hemodialysis or chronic peritoneal dialysis End-stage liver disease, defined as the presence of acute or chronic liver disease and recent history of one or more of the following: ascites, encephalopathy, variceal bleeding, bilirubin ≥2.0 mg/dl, albumin level ≤3.5 g/dl, protrombin time ≥4.5 econds prolonged, international normalized ratio ≥1.7 or prior liver transplant A prior solid organ transplant or awaiting solid organ transplant | Diagnosis position: Any Source of algorithm: https://pubmed.ncbi.nlm.nih.gov/22674685/ and https://pubmed.ncbi.nlm.nih.gov/34256144/ Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | Can't measure in claims Applied before/after selection of index date: Before Assessment window: [:365, 0] Code type: DX, PX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [:183, 0] Code type: DX, PX, RX Care setting: Any Diagnosis position: Any Source of algorithm: https://pubmed.ncb.inlm.nih.gov/322674685/ and https://pubmed.ncb.inlm.nih.gov/3226144/ Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | Can't measure in claims Applied before/after selection of index date: Before Assessment window: [:365, 0] Code type: DX, PX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [:183, 0] Code type: DX, PX, RX Care setting: Any Diagnosis position: Any Source of algorithm: https://pubmed.ncb.inlmnih.gov/322674685/ and https://pubmed.ncb.inlmnih.gov/3226144/ Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | Algorithm detail: Was defined using CKOS/ESRD/Dialysis/Renal transplant code. Algorithm detail: According to https://pubmed.ncbi.nlm.nih.gov/22674685/,ESLD inclaims can be defined using Citrohosis + Decompensation event. We used the ICD9/ICD10 codes from the above study and https://pubmed.ncbi.nlm.nih.gov/34256144/, to define the codes required for Citrhosis and Decompensation events. |
| | Diagnosis of malignant neoplasm in the previous 5 | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any | |
| 16 | years (except basal cell skin cancer or squamous cell<br>skin cancer)<br>Any acute condition or exacerbation of chronic<br>condition that would in the investigator's opinion<br>interfere with the initial trial visit schedule and<br>procedures | Source of algorithm: PROMISE team Measurement characteristics: N/A Can't measure in claims | Source of algorithm: PROMISE team Measurement characteristics: N/A Can't measure in claims | Source of algorithm: PROMISE team Measurement characteristics: N/A Can't measure in claims | |
| / | procedures | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| 18 | Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice) Known or suspected hypersensitivity to trial products | Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Can't measure in claims | |
| 20 | or related products Known use of non-prescribed narcotics or illicit drugs Previous participation in this trial. | Can't measure in claims Applied before/fafter selection of index date: Before Assessment window: [-183,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: search of clinical code lists Measurement characteristics: N/A Can't measure in claims | Can't measure in claims Applied before/after selection of index date: Before Assessment window: [-183, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: search of clinical code lists Measurement characteristics: N/A Can't measure in claims | Can't measure in claims Applied before/after selection of index date: Before Assessment window: [:183,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: search of clinical code lists Measurement characteristics: N/A Can't measure in claims | Algorithm detail: Defined as drug dependence or abuse disorders. |
| | Simultaneous participation in any other clinical trial of | Can thicasure inclaims | Can timedatio incidina | Can timeasure in claims | |
| | an investigational agent. Participation in a clinical trial with investigational stent(s) is allowed | Can't measure in claims | Can't measure in claims | Can't measure in claims | |

| Receipt of any investigational medicinal product within 30 days prior to screening (Visit 1) or according 23 to local requirements, if longer Any other factor likely to limit protocol compliance or | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
|---|---|---|---|---|
| reporting of adverse event at the discretion of the | | | | |
| 24 investigator | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | Assessment window: [-365,0] | Assessment window: [-365, 0] | Assessment window: [-365, 0] | |
| | Code type: PX | Code type: PX | Code type: PX | |
| | Care setting: Any | Care setting: Any | Care setting: Any | |
| | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any | |
| Proliferative retinopathy/maculopathy requiring acute | Source of algorithm: LEAD-2 | Source of algorithm: LEAD-2 | Source of algorithm: LEAD-2 | Algorith |
| 25 treatment | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A | injectio |
| | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | Assessment window: [0,0] | Assessment window: [0,0] | Assessment window: [0, 0] | |
| | Code type: n/a | Code type: n/a | Code type: n/a | |
| | Care setting: n/a | Care setting: n/a | Care setting: n/a | |
| | Diagnosis position: n/a | Diagnosis position: n/a | Diagnosis position: n/a | |
| | Source of algorithm: n/a | Source of algorithm: n/a | Source of algorithm: n/a | |
| 26 Age OR Gender Missing | Measurement characteristics: n/a | Measurement characteristics: n/a | Measurement characteristics: n/a | |
| - | | | | |

gorithm detail: Defined it by either Anti-VEGFi ections or Photocoagulation


Antidiabetic medication score Antidi

Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiahetic medication score (sum of component 1-8 Antidiahetic medication score (sum of component 1-8 Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8, Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8, Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8, Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiahetic medication score (sum of component 1-8 Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8, Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiahetic medication score (sum of component 1-8 Antidiabetic medication score (sum of component 1-8, Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8, Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8, Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiahetic medication score (sum of component 1-8 Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8. Antidiabetic medication score (sum of component 1-8,

Antidiabetic medication score (sum of component 1-8.


Heart failure class IV component must overlap with oxygen use component

OXYGEN CONCENTRATOR, MANUFACTURER SPECIFIED MAXIMUM FLOW RATE

Heart failure class IV component must overlap with oxygen use component

Heart failure class IV component must overlap with oxygen use component

Heart failure class IV component must overlap with oxygen use component Heart failure class IV component must overlap with oxygen use component Heart failure class IV component must overlap with oxygen use component Heart failure class IV component must overlap with oxygen use component


End stage liver disease (Cirrhosis + Decompensation event) component


MALIGNANT NEOPLASM OF CONNECTIVE AND SOFT TISSUE OF UNSPECIFIED


ANAPLASTIC LARGE CELL LYMPHOMA, ALK-POSITIVE, LYMPH NODES OF


MATERNAL CARE FOR (SUSPECTED) CENTRAL NERVOUS SYSTEM


MATERNAL CARE FOR ABNORMALITIES OF THE FETAL HEART RATE OR RHYTHM,


PRETERM LABOR SECOND TRIMESTER WITH PRETERM DELIVERYTHIRD


OTHER PSYCHOACTIVE SUBSTANCE USE, UNSPECIFIED WITH PSYCHOACTIVE


All database

Marketscan/Optum database Medicare database Optum database

Marketscan database

### Appendix 3. Flowchart for cohort assembly

| OPTUM (Jan 1, 2018 to Feb 28, 2025) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 95,349,410 |
| Patients meeting cohort entry criteria | | 1,141,594 |
| Excluded due to insufficient enrollment | -387,201(34%) | 754,393 |
| Excluded due to prior use of referent | -191,077 (25%) | 563,316 |
| Excluded due to prior use of exposure | -352,033 (62%) | 211,283 |
| Excluded because patient qualified in >1 exposure category | -26 (<1%) | 211,257 |
| Excluded based on 1 - DM Type 2 | -18169 (9%) | 193.088 |
| Excluded based on 3 - Antidiabetic medication score | -2,078 (1%) | 191,010 |
| Exclude if patient is between 50 and 60 years of age without established CVD | -9,216 (5%) | 181,794 |
| Exclude if patient is greater than or equal to 60 years of age without establised or subclinical CVD | -36,043 (20%) | 145,751 |
| Excluded based on Age ≤49 | -9.205(6%) | 136.546 |
| Excluded based on 1 - Type 1 DM | -2,165 (2%) | 134,381 |
| Excluded based on 1 - Gestational DM | -0 (<1%) | 134.381 |
| Excluded based on 1 - Secondary DM | -1.459 (1%) | 132.922 |
| Excluded based on 2 - Sitagliptin/Semaglutide (all formulation, combinations) | -3.817 (3%) | 129105 |
| Excluded based on 2 - DPP4i, GLP-1 Pramlintide | -6.142 (5%) | 122.963 |
| Excluded based on 4 - Bolus Insulin (including combination) | -2.623 (2%) | 120,340 |
| Excluded based on 5 - Hyperosmolar hyperglycemic nonketotic syndrome (HONK) | -169 (<1%) | 120,1/1 |
| Excluded based on 5 - Diabetic ketoacidosis | -90 (<1%) | 120,081 |
| Excluded based on 6 - History of pancreatitis | -162 (<1%) | 119,919 |
| Excluded based on 7 - Acute coronary/cerebro-vascular event | -675 (<1%) | 119,244 |
| Excluded based on 9 - Heart failure class IV | -183 (<1%) | 119,061 |
| Excluded based on 10 - History of MEN-2 | -2 (<1%) | 119,059 |
| Excluded based on 11 - Personal history of non-familial medullary thyroid carcinoma | -153 (<1%) | 118,906 |
| Excluded based on 13 - End-stage renal disease, dialysis or renal transplant | -429 (<1%) | 118,477 |
| Excluded based on 14 - End stage liver disease (Cirrhosis + Decompensation event) | -68 (<1%) | 118,409 |
| Excluded based on 15 - Organ Transplant | -115 (<1%) | 118,294 |
| Excluded based on 16 - Cancer | -4,611 (4%) | 113,683 |
| Excluded based on 18 - Pregnancy | -3 (<1%) | 113,680 |
| Excluded based on 20 - Drug abuse or dependence | -700 (<1%) | 112,980 |
| Excluded based on 25 - Proliferative retinopathy or maculopathy | -635 (<1%) | 112,345 |
| Excluded based on Age | -4 (<1%) | 112,341 |
| Excluded based on Gender | -0 (<1%) | 112,341 |
| Patients in Exposure Group | | 64,841 |
| Patients in Referent Group | | 47,500 |
| Total Patients | | 112,341 |

| | Excluded Datiente | Remaining Patients |
|---|---|---|
| Patients in dataset | Excluded Fasteria | 126.118.01 |
| Patients meeting cohort entry criteria | | 102294 |
| - cluded due to insufficient enrollment | -215.859 (21%) | 807.08 |
| scluded due to prior use of referent | -235.193 (29%) | 571.89 |
| Excluded due to prior use of exposure | -410.684 (72%) | 161.20 |
| excluded due to prior use or exposure excluded because patient qualified in >1 exposure category | -37 (<1%) | 161,20 |
| Excluded based on 1 - DM Type 2 | -41.877 (26%) | 11929 |
| xcluded based on 3 - Antidiabetic medication score | 1.429 (1%) | 117.86 |
| exclude if patient is between 50 and 60 years of age without established CVD | -19.031(16%) | 9883 |
| Exclude if patient is greater than or equal to 60 years of age without establised or subclinical CVD | -16,771 (17%) | 82.06 |
| Excluded based on Age \$49 | -20,252 (25%) | 61.81 |
| Excluded based on 1-Type I DM | -1.112 (2%) | 60.69 |
| Excluded based on 1 - Type I bit Excluded based on 1 - Gestational DM | -0 (<1%) | 60,69 |
| Excluded based on 1 - Secondary DM | -625 (1%) | 60.07 |
| excluded based on 2 - Sitagliptin/Semaglutide (all formulation combinations) | -2.136 (4%) | 57.93 |
| excluded based on 2 - Straggipting Serragional Community Community (Community Community Communit | -2.538 (4%) | 55.40 |
| excluded based on 4 - Bolus Insulin (including combination) | -624 (1%) | 54,77 |
| xcluded based on 5 - Hyperosmolar hyperglycemic nonketotic syndrome (HUNK) | -76(<1%) | 54,77 |
| scluded based on 5 - Nyperoamous hypergrycemic normalistic ayrunome (norm) | -43(<1%) | 5465 |
| xcluded based on 6 - History of pancreatitis | -56 (<1%) | 54.60 |
| xcluded based on 7 - Acute coronary/cerebro-vascular event | -491 (<1%) | 5411 |
| xcluded based on 9 - Heart failure class IV | -43 (<1%) | 54.06 |
| xcluded based on 10 - History of MEN-2 | -0 (<1%) | 54.06 |
| xcluded based on 11 - Personal history of non-familial medullary thyroid carcinoma | -98(<1%) | 53.96 |
| xcluded based on 13 - End-stage renal disease, dialysis or renal transplant | -148 (<1%) | 53,82 |
| excluded based on 14 - End stage liver disease (Cirrhosis + Decompensation event) | -35(<1%) | 53,78 |
| Excluded based on 15 - Organ Transplant | -39 (<1%) | 53,74 |
| xcluded based on 16 - Cancer | -1,776 (3%) | 51,97 |
| xcluded based on 18 - Pregnancy | -10 (<1%) | 51,96 |
| xcluded based on 20 - Drug abuse or dependence | -127 (<1%) | 51,83 |
| xcluded based on 25 - Proliferative retinopathy or maculopathy | -215 (<1%) | 51,61 |
| xcluded based on Age | -7 (<1%) | 51,61 |
| Excluded based on Gender | -0 (<1%) | 51,61 |
| Patients in Exposure Group | | 26,94 |
| Patients in Referent Group<br>Lotal Patients | | 24,67<br>51.61 |

| MEDICARE (May 13, 2022 to Dec 31, 2020) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 28,874,258 |
| Patients meeting cohort entry criteria | | 963,751 |
| Excluded due to insufficient enrollment | -190.182 (20%) | 773.569 |
| Excluded due to prior use of referent | -541,540 (70%) | 232,029 |
| Excluded due to prior use of exposure | -62.834 (27%) | 169.195 |
| Excluded because patient qualified in >1 exposure category | -18 (<1%) | 169,177 |
| Excluded based on 1 - DM Type 2 | -2.389(1%) | 166,788 |
| Excluded based on 3 - Antidiabetic medication score | -1554 (<1%) | 165.234 |
| Exclude if patient is between 50 and 60 years of age without established CVD | -0 (<1%) | 165.234 |
| Exclude if patient is greater than or equal to 60 years of age without establised or subclinical CVD | -41,096 (25%) | 124,138 |
| Excluded based on Age ≤49 | -0 (<1%) | 124,138 |
| Excluded based on 1 Type I DM | -3.677 (3%) | 120,461 |
| Excluded based on 1 - Gestational DM | -0 (<1%) | 120,461 |
| Excluded based on 1 - Secondary DM | -2.228(2%) | 118.233 |
| Excluded based on 2 - Sitagliptin/Semaglutide (all formulation combinations) | -4.853 (4%) | 113,380 |
| Excluded based on 2 - DPP4i.GLP-1. Pramlintide | -4.796(4%) | 108.584 |
| Excluded based on 4 - Bolus Insulin (including combination) | -1073(<1%) | 107.511 |
| Excluded based on b - Hyperosmolar hyperglycemic nonketotic syndrome (HUNK) | -226 (<1%) | 107,285 |
| Excluded based on 5 - Diabetic ketoacidosis | -100 (<1%) | 107,185 |
| Excluded based on 6 - History of pancreatitis | -234 (<1%) | 106,951 |
| Excluded based on 7 - Acute coronary/cerebro-vascular event | -1,310 (1%) | 105,641 |
| Excluded based on 9 - Heart failure class IV | -0 (<1%) | 105,641 |
| Excluded based on 10 - History of MEN-2 | -0 (<1%) | 105,641 |
| Excluded based on 11 - Personal history of non-familial medullary thyroid carcinoma | -177 (<1%) | 105,464 |
| Excluded based on 13 - End-stage renal disease, dialysis or renal transplant | -781 (<1%) | 104,683 |
| Excluded based on 14 - End stage liver disease (Cirrhosis + Decompensation event) | -111 (<1%) | 104,572 |
| Excluded based on 15 - Organ Transplant | -131 (<1%) | 104,441 |
| Excluded based on 16 - Cancer | -6,464 (6%) | 97,977 |
| Excluded based on 18 - Pregnancy | -10 (<1%) | 97,967 |
| Excluded based on 20 - Drug abuse or dependence | -411 (<1%) | 97,556 |
| Excluded based on 25 - Proliferative retinopathy or maculopathy | ·726 (<1%) | 96,830 |
| Excluded based on Age | -2 (<1%) | 96,828 |
| Excluded based on Gender | -0 (<1%) | 96,828 |
| Patients in Exposure Group | | 13,987 |
| Patients in Referent Group | | 82,841 |
| Total Patients | 1 | 96,828 |

#### Appendix 4.1st Feasibility Assessment

#### Table of Contents

A. Patient characteristics by treatment group

B. Summary Parameters of Study Population
C. Median Follow up Time in Overall Study Population
D. Reasons for Censoring in Overall Study Population

E. Initial Power Assessment

F. Aetion report link G. Review by Principal Investigator

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

OPTUM: Study period from Jan1, 2018 to Feb 28, 2025 MARKETSCAN: Study period from Jan1, 2018 to Dec 31, 2023 MEDICARE: Study period from Jan 1, 2018 to Dec 31, 2020

### A. Patient characteristics by treatment group (follow-up start is 1 days after CED, so few patients and dropped, hence table 1 could include sightly fewer patients than the attrition table)

| Before weighting | | Optum | | | Marketscan | · | | Medicare | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference |
| Number of patients | 47,500 | 64,841 | - (-, -) | 24,670 | 26,942 | - (-, -) | 82,841 | 13,987 | - (-, -) |
| Age | | | | | | | | | |
| mean (sd) | 73.14 (7.49) | 67.89 (7.79) | 5.25 (5.16, 5.34) | 66.59 (10.34) | 60.90 (7.39) | 5.69 (5.53, 5.84) | 76.11 (7.18) | 72.42 (5.20) | 3.68 (3.59, 3.78) |
| _median [IQR] | 73.00 [68.00, 79.00] | 68.00 [63.00, 73.00] | - (-, -) | 64.00 [59.00, 74.00] | 60.00 [55.00, 64.00] | - (-, -) | 75.00 [70.00, 81.00] | 71.00 [68.00, 75.00] | - (-, -) |
| Gender | | | | 50.00, 102.00 | 50.00, 97.00 | - (-, -) | | | |
| Male; n (%) | 21,874 (46.1%) | 29,182 (45.0%) | 1.0% (0.5%, 1.6%) | | | | 37,851 (45.7%) | 6,925 (49.5%) | -3.8% (-4.7%, -2.9%) |
| CCI (365 days) | | | | | | | | | |
| _mean (sd) | 2.92 (2.67) | 2.35 (2.33) | 0.56 (0.53, 0.59) | 1.87 (2.27) | 1.51 (1.90) | 0.36 (0.32, 0.39) | 2.75 (2.65) | 2.46 (2.31) | 0.29 (0.25, 0.33) |
| _median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) |

#### B. Summary Parameters of Overall Study Population (Step 1)

| | Optum | Marketscan | Medicare |
|---|---|---|---|
| Variable | Value | Value | Value |
| Number of patients in full cohort | 112,341 | 51,612 | 96,828 |
| Number of patients dropped as incomplete cases | 0 | 0 | 0 |
| Number of patients that did not begin follow-up | 210 | 80 | 569 |
| Number of patients in analytic cohort | 112,131 | 51,532 | 96,259 |
| Number of events | 2,210.00 | 647.00 | 3,720.00 |
| Number of person-years | 58,115.09 | 27,483.66 | 49,198.40 |
| Number of patients in group: Reference-Sitagliptin | 47,372 | 24,614 | 82,300 |
| Number of patients in group: Exposure - Tirzepatide | 64,759 | 26,918 | 13,959 |
| Risk per 1,000 patients | 19.71 | 12.56 | 38.65 |
| Rate per 1,000 person-years | 38.03 | 23.54 | 75.61 |

### C. Median Follow up Time in Overall Study Population (Step 1)

| | Optum | Marketscan | Medicare |
|---|---|---|---|
| Patient Group | Median Follow-Up Time (Days) [IQR] | Median Follow-Up Time (Days) [IQR] | Median Follow-Up Time (Days) [IQR] |
| Overall Patient Population | 154 [92, 302] | 162 [85, 329] | 146 [73, 313] |

### D. Reasons for Censoring in Overall Study Population (Step 1)

| | Optum | Marketscan | Medicare |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 2,210 (2.0%) | 647 (1.3%) | 3,720 (3.9%) |
| Start of an additional exposure | 1,054 (0.9%) | 689 (1.3%) | 667 (0.7%) |
| End of index exposure | 54,722 (48.8%) | 20,797 (40.4%) | 39,890 (41.4%) |
| Maximum follow-up time | 21,851 (19.5%) | 11,358 (22.0%) | 19,395 (20.1%) |
| Specified date reached | 2,302 (2.1%) | 8,771 (17.0%) | 17,967 (18.7%) |
| End of patient data | O (O.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 22,383 (20.0%) | 6,236 (12.1%) | 3,811 (4.0%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 7,609 (6.8%) | 3,034 (5.9%) | 10,809 (11.2%) |

#### Appendix 5. 2nd Feasibility Assessment

### Table of Contents

A. Median Follow up Time by Treatment Group B. Reasons for Censoring by Treatment Group C. Final Power Assessment D. Aetion report link

E. Review by Principal Investigator

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the formulas from Chow et al. (2008).

#### A. Median Follow Up Time by Treatment Group

| Patient Group | Median Follow-Up | Median Follow-Up | Median Follow-Up |
|---|---|---|---|
| Overall Patient Population | 154 [92, 302] | 162 [85, 329] | 146 [73, 313] |

### B. Reasons for Censoring in Overall Study Population

| | Optum | Marketscan | Medicare |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 2,210 (2.0%) | 647 (1.3%) | 3,720 (3.9%) |
| Start of an additional exposure | 1,054 (0.9%) | 689 (1.3%) | 667 (0.7%) |
| End of index exposure | 54,722 (48.8%) | 20,797 (40.4%) | 39,890 (41.4%) |
| Maximum follow-up time | 21,851 (19.5%) | 11,358 (22.0%) | 19,395 (20.1%) |
| Specified date reached | 2,302 (2.1%) | 8,771 (17.0%) | 17,967 (18.7%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 22,383 (20.0%) | 6,236 (12.1%) | 3,811 (4.0%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 7.609 (6.8%) | 3.034 (5.9%) | 10.809 (11.2%) |

#### C. Power Assessment

| Superiority Analysis | Optum | Marketscan | Medicare |
|---------------------------|--------|------------|----------|
| Number of patients | | | |
| Reference | 47,500 | 24,670 | 82,841 |
| Exposed | 64,841 | 26,942 | 13,987 |
| Risk per 1,000 patients | 19.71 | 12.56 | 38.65 |
| Expected HR | 0.7 | 0.7 | 0.7 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 |
| Number of events expected | 2214 | 648 | 3742 |
| Power | 1.00 | 1.00 | 1.00 |

### D. Aetion report link

Optum Step 1: https://hwh-dope.aetion.com/project/2914/rwrs/139464
Marketscan Step 1: https://hwh-dope.aetion.com/project/2912/rwrs/139472
Medicare Step 1: https://bwh-dope.aetion.com/project/2913/rwrs/139394

## E. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krü | ger | Date reviewed: | July | y 30, 2025 |
|-----------------|----------|-----|----------------|------|------------|

# Appendix 6. Balance Assessment - PS Distribution and C-Statistic

C-statistics unadjusted, OPTUM: 0.886



C-statistics adjusted after overlap weighing on the PS, OPTUM: 0.528



C-statistics unadjusted, MARKETSCAN: 0.878



C-statistics adjusted after overlap weighing on the PS, MARKETSCAN: 0.535



### C-statistics unadjusted, MEDICARE: 0.841



C-statistics adjusted after overlap weighing on the PS, MEDICARE: 0.534



| Appendix 7. Balance Assessment - Table 1 | | | | | | |
|---|---|---|---|---|---|---|
| OPTUM<br>Variable | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference |
| Variable Number of patients Year of Cohort Entry Date | 28,279 | 49,843 | - (-, -) | 13,602 | 13,602 | - (-, -) |
| 2018; n (%) | 4,704 (16.6%) | 44 (0.1%) | 16.5% (16.1%, 17.0%) | 65 (0.5%) | 44 (0.3%) | 0.2% (-0.0%, 0.3%) |
| 2019; n (%)<br>2020; n (%) | 4,855 (17.2%)<br>4,659 (16.5%) | 1,369 (2.7%)<br>2,560 (5.1%) | 14.4% (14.0%, 14.9%)<br>11.3% (10.9%, 11.8%) | 1,227 (9.0%)<br>1,893 (13.9%) | 1,203 (8.8%)<br>1,910 (14.0%) | -0.1% (-1.0%, 0.7%) |
| 2021; n (%)<br>2022; n (%) | 4,231 (15.0%)<br>3,451 (12.2%) | 4,304 (8.6%)<br>7,572 (15.2%) | 6.3% (5.8%, 6.8%)<br>-3.0% (-3.5%, -2.5%) | 2,297 (16.9%)<br>2,504 (18.4%) | 2,388 (17.6%)<br>2,535 (18.6%) | -0.7% (-1.6%, 0.2%)<br>-0.2% (-1.2%, 0.7%) |
| 2023; n (%)<br>2024; n (%) | 3,209 (11.3%)<br>3,159 (11.2%) | 15,621 (31.3%)<br>18,081 (36.3%) | -20.0% (-20.5%, -19.4%)<br>-25.1% (-25.7%, -24.5%) | 2,788 (20.5%)<br>2,817 (20.7%) | 2,745 (20.2%)<br>2,766 (20.3%) | 0.3% (-0.6%, 1.3%) 0.4% (-0.6%, 1.3%) |
| 2025; n (%)<br>Age | 11 (0.0%) | 292 (0.6%) | -0.5% (-0.6%, -0.5%) | 11 (0.1%) | 11 (0.1%) | 0.0% (-0.1%, 0.1%) |
| mean (sd)median [IQR] | 72.34 (7.50)<br>72.00 [68.00, 78.00] | 67.49 (7.76)<br>68.00 [62.00, 73.00] | 4.86 (4.74, 4.97) | 70.56 (7.47)<br>71.00 [67.00, 75.00] | 70.57 (7.43)<br>71.00 [66.00, 76.00] | -0.01 (-0.19, 0.17)<br>- (-, -) |
| min, max Gender (male); n (%) | 50.00, 88.00<br>12,564 (44.4%) | 50.00, 88.00<br>21,624 (43.4%) | - (-, -)<br>10% (0.3%, 1.8%) | 50.00, 88.00<br>5,991 (44.0%) | 50.00, 88.00<br>6,005 (44.1%) | - (-, -)<br>-0.1% (-1.3%, 1.1%) |
| Race (Recategorized)White; n (%) | 12,998 (46.0%) | 24,640 (49.4%) | -3.5% (-4.2%, -2.7%) | 6,563 (48.3%) | 6,583 (48.4%) | -0.1% (-1.3%, 1.0%) |
| Black; n (%)<br>Unknown / Missing; n (%) | 4,762 (16.8%)<br>9,385 (33.2%) | 6,869 (13.8%)<br>17.616 (35.3%) | 3.1% (2.5%, 3.6%)<br>-2.2% (-2.8%, -1.5%) | 2,143 (15.8%)<br>4,585 (33.7%) | 2,152 (15.8%)<br>4,553 (33,5%) | -0.1% (-0.9%, 0.8%)<br>0.2% (-0.9%, 1.4%) |
| Others; n (%) | 1,134 (4.0%) | 718 (1.4%) | 26% (2.3%, 2.8%) | 311 (2.3%) | 314 (2.3%) | -0.0% (-0.4%, 0.3%) |
| Region / State<br>Northest; n (%) | 2,992 (10.6%) | 4,487 (9.0%) | 16% (11%, 2.0%) | 1,409 (10.4%) | 1,359 (10.0%) | 0.4% (-0.4%, 1.1%) |
| Midwest / North central; n (%)<br>South; n (%) | 3,803 (13.4%)<br>16,289 (57.6%) | 9,445 (18.9%)<br>27,747 (55.7%) | -5.5% (-6.0%, -5.0%)<br>1.9% (1.2%, 2.7%) | 2,162 (15.9%)<br>7,790 (57.3%) | 2,185 (16.1%)<br>7,811 (57.4%) | -0.2% (-1.0%, 0.7%)<br>-0.2% (-1.3%, 1.0%) |
| West; n (%)Missing n (%) | 5,182 (18.3%)<br>13 (0.0%) | 8,143 (16.3%)<br>21 (0.0%) | 2.0% (1.4%, 2.5%)<br>0.0% (-0.0%, 0.0%) | 2,238 (16.5%)<br>3 (0.0%) | 2,240 (16.5%)<br>7 (0.1%) | -0.0% (-0.9%, 0.9%)<br>-0.0% (-0.1%, 0.0%) |
| Smoking/Tobacco use; n (%) Weight | 7,220 (25.5%) | 13,895 (27.9%) | -2.3% (-3.0%, -1.7%) | 3,512 (25.8%) | 3,501 (25.7%) | 0.1% (-1.0%, 1.1%) |
| Underweight; n (%)<br>Normal weight; n (%) | 388 (1.4%)<br>2,662 (9.4%) | 63 (0.1%)<br>724 (1.5%) | 1.2% (1.1%, 1.4%)<br>8.0% (7.6%, 8.3%) | 52 (0.4%)<br>570 (4.2%) | 56 (0.4%)<br>553 (4.1%) | -0.0% (-0.2%, 0.1%)<br>0.1% (-0.4%, 0.6%) |
| Overweight; n (%)<br>Class 1 Obesity; n (%) | 6,852 (24.2%)<br>3,959 (14.0%) | 5,293 (10.6%)<br>5,185 (10.4%) | 13.6% (13.0%, 14.2%)<br>3.6% (3.1%, 4.1%) | 2,612 (19.2%)<br>1,848 (13.6%) | 2,646 (19.5%)<br>1.844 (13.6%) | -0.2% (-1.2%, 0.7%)<br>0.0% (-0.8%, 0.9%) |
| Class 2 Obesity; n (%)<br>Class 3 Obesity; n (%) | 1,703 (6.0%)<br>5,460 (19.3%) | 3,415 (6.9%)<br>19,481 (39.1%) | -0.8% (-1.2%, -0.5%)<br>-19.8% (-20.4%, -19.1%) | 892 (6.6%)<br>3,557 (26.2%) | 928 (6.8%)<br>3,554 (26.1%) | -0.3% (-0.9%, 0.3%)<br>0.0% (-1.0%, 1.1%) |
| Unspecified Obesity; n (%) | 7,255 (25.7%) | 15,481 (35.1%)<br>15,682 (31.5%)<br>4,047 (8.1%) | -5.8% (-6.5%, -5.2%)<br>2.8% (2.3%, 3.2%) | 4,071 (29.9%)<br>1.335 (9.8%) | 4,021 (29.6%)<br>1.393 (10.2%) | 0.4% (-0.7%, 1.5%) |
| Diabetic retinopathy; n (%) Diabetic neuropathy; n (%) | 9,795 (34.6%) | 14,480 (29.1%) | 5.6% (4.9%, 6.3%) | 4,474 (32.9%) | 4,536 (33.3%) | -0.5% (-1.6%, 0.7%) |
| Diabetic nephropathy; n (%) Diabetes with other ophthalmic complications; n (%) | 10,091 (35.7%)<br>1,862 (6.6%) | 12,927 (25.9%)<br>2,382 (4.8%) | 9.7% (9.1%, 10.4%)<br>1.8% (1.5%, 2.2%) | 4,260 (31.3%)<br>805 (5.9%) | 4,296 (31.6%)<br>797 (5.9%) | -0.3% (-1.4%, 0.8%)<br>0.1% (-0.5%, 0.6%) |
| Diabetes with peripheral circulatory disorders; n (%) Diabetic foot, n (%) | 5,796 (20.5%)<br>898 (3.2%) | 8,322 (16.7%)<br>1,434 (2.9%) | 3.8% (3.2%, 4.4%)<br>0.3% (0.0%, 0.6%) | 2,579 (19.0%)<br>399 (2.9%) | 2,607 (19.2%)<br>439 (3.2%) | -0.2% (-1.1%, 0.7%)<br>-0.3% (-0.7%, 0.1%) |
| Erectile dysfunction; n (%)<br>Hypoglycemia; n (%) | 1,064 (3.8%)<br>7,495 (26.5%) | 2,471 (5.0%)<br>12,276 (24.6%) | -1.2% (-1.5%, -0.9%)<br>1.9% (1.2%, 2.5%) | 577 (4.2%)<br>3,521 (25.9%) | 578 (4.2%)<br>3,607 (26.5%) | -0.0% (-0.5%, 0.5%)<br>-0.6% (-1.7%, 0.4%) |
| Hyperglycemia/DKA/HONK; n (%)<br>Skin infections; n (%) | 14,525 (51.4%)<br>2,841 (10.0%) | 23,311 (46.8%)<br>5,344 (10.7%) | 4.6% (3.9%, 5.3%)<br>-0.7% (-1.1%, -0.2%) | 6,883 (50.6%)<br>1,368 (10.1%) | 7,018 (51.6%)<br>1,381 (10.2%) | -1.0% (-2.2%, 0.2%)<br>-0.1% (-0.8%, 0.6%) |
| Stable angina; n (%) Unstable angina; n (%) | 1,990 (7.0%)<br>1,001 (3.5%) | 3,737 (7.5%)<br>1,795 (3.6%) | -0.5% (-0.8%, -0.1%)<br>-0.1% (-0.3%, 0.2%) | 975 (7.2%)<br>465 (3.4%) | 966 (7.1%)<br>443 (3.3%) | 0.1% (-0.6%, 0.7%)<br>0.2% (-0.3%, 0.6%) |
| Hypertension; n (%) | 26,616 (94.1%)<br>1.411 (5.0%) | 46,038 (92.4%)<br>1.864 (3.7%) | 18% (1.4%, 2.1%)<br>1.2% (0.9%, 1.6%) | 12,721 (93.5%)<br>568 (4.2%) | 12,714 (93.5%)<br>593 (4.4%) | 0.1% (-0.5%, 0.6%) |
| Hypotension; n (%)<br>Hyperlipidemia; n (%) | 25,165 (89.0%) | 43,970 (88.2%) | 0.8% (0.3%, 1.2%) | 12,081 (88.8%) | 12,150 (89.3%) | -0.5% (-1.3%, 0.2%) |
| Atrial fibrillation; n (%) Cardiac conduction disorder; n (%) | 4,414 (15.6%)<br>2,488 (8.8%) | 7,576 (15.2%)<br>4,036 (8.1%) | 0.4% (-0.1%, 0.9%)<br>0.7% (0.3%, 1.1%) | 2,087 (15.3%)<br>1,121 (8.2%) | 2,008 (14.8%)<br>1,140 (8.4%) | 0.6% (-0.3%, 1.4%)<br>-0.1% (-0.8%, 0.5%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%)<br>Ischemic stroke; n (%) | 614 (2.2%)<br>264 (0.9%) | 1,178 (2.4%)<br>354 (0.7%) | -0.2% (-0.4%, 0.0%)<br>0.2% (0.1%, 0.4%) | 308 (2.3%)<br>110 (0.8%) | 279 (2.1%)<br>114 (0.8%) | 0.2% (-0.1%, 0.6%) |
| PVD diagnosis or surgery; n (%) Other cardiac dysrhythmia; n (%) | 4,767 (16.9%)<br>7,334 (25.9%) | 6,364 (12.8%)<br>13,141 (26.4%) | 4.1% (3.6%, 4.6%)<br>-0.4% (-1.1%, 0.2%) | 2,002 (14.7%)<br>3,459 (25.4%) | 2,031 (14.9%)<br>3,463 (25.5%) | -0.2% (-1.1%, 0.6%)<br>-0.0% (-1.1%, 1.0%) |
| Cardiomyopathy; n (%) Valve disorders; n (%) | 2,291 (8.1%)<br>4,810 (17.0%) | 3,880 (7.8%)<br>7,987 (16.0%) | 0.3% (-0.1%, 0.7%)<br>1.0% (0.4%, 1.5%) | 1,046 (7.7%)<br>2,179 (16.0%) | 1,005 (7.4%)<br>2,180 (16.0%) | 0.3% (-0.3%, 0.9%) |
| Valve replacement; n (%) | 585 (2.1%) | 0.40 (1.00() | | | | |
| | 982 (3.5%) | 940 (1.9%)<br>1.354 (2.7%) | 0.2% (-0.0%, 0.4%) | 274 (2.0%)<br>394 (2.9%) | 286 (2.1%)<br>392 (2.9%) | -0.1% (-0.4%, 0.3%)<br>0.0% (-0.4%, 0.4%) |
| TIA; n (%)<br>Edema; n (%) | | | 0.8% (0.5%, 1.0%)<br>-0.5% (-1.1%, 0.0%) | 394 (2.9%)<br>2,246 (16.5%) | 392 (2.9%)<br>2,200 (16.2%) | 0.0% (-0.4%, 0.4%) |
| TIA: n (%) Edema; n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) | 982 (3.5%)<br>4,621 (16.3%)<br>1,111 (3.9%)<br>1,292 (4.6%) | 1,354 (2.7%)<br>8,407 (16.9%)<br>1,998 (4.0%)<br>2,152 (4.3%) | 0.8% (0.5%, 1.0%)<br>-0.5% (-1.1%, 0.0%)<br>-0.1% (-0.4%, 0.2%)<br>0.3% (-0.1%, 0.6%) | 394 (2.9%)<br>2,246 (16.5%)<br>551 (4.1%)<br>579 (4.3%) | 392 (2.9%)<br>2,200 (16.2%)<br>552 (4.1%)<br>566 (4.2%) | 0.0% (-0.4%, 0.4%)<br>0.3% (-0.5%, 1.2%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.4%, 0.6%) |
| TIA.n (%) Edema; n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable cardioverter defibrillator; n (%) Hyperkalemis, n (%) | 982 (3.5%)<br>4,621 (16.3%)<br>1,111 (3.9%)<br>1,292 (4.6%)<br>128 (0.5%)<br>1,407 (5.0%) | 1.354 (2.7%)<br>8.407 (16.9%)<br>1.998 (4.0%)<br>2.152 (4.3%)<br>186 (0.4%)<br>1.585 (3.2%) | 0.8% (0.5%, 1.0%) -0.5% (-1.1%, 0.0%) -0.1% (-0.4%, 0.2%) 0.3% (-0.1%, 0.6%) 0.1% (-0.0%, 0.2%) 1.8% (1.5%, 2.1%) | 394 (2.9%)<br>2,246 (16.5%)<br>551 (4.1%)<br>579 (4.3%)<br>55 (0.4%)<br>577 (4.2%) | 392 (2.9%)<br>2,200 (16.2%)<br>552 (4.1%)<br>566 (4.2%)<br>50 (0.4%)<br>579 (4.3%) | 0.0% (-0.4%, 0.4%)<br>0.3% (-0.5%, 1.2%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.4%, 0.6%)<br>0.0% (-0.1%, 0.2%)<br>-0.0% (-0.5%, 0.5%) |
| TIA.n (%) Edemia n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Pulmonary hypertension; n (%) (Implantable cardioveter defibrillator, n (%) Hyperkallemia; n (%) Coronary atherosclerosis; n (%) Coronary atherosclerosis; n (%) | 982 (3.5%)<br>4.621 (16.3%)<br>1,111 (3.9%)<br>1,292 (4.6%)<br>128 (0.5%)<br>1,407 (5.0%)<br>10,186 (36.0%)<br>39 (0.1%) | 1.354 (2.7%)<br>8,407 (16.9%)<br>1,998 (4.0%)<br>2,152 (4.3%)<br>186 (0.4%)<br>1,585 (3.2%)<br>18,491 (37.1%)<br>71 (0.1%) | 0.8% (0.5%, 1.0%)<br>-0.5% (-1.1%, 0.0%)<br>-0.1% (-0.4%, 0.2%)<br>0.3% (-0.1%, 0.6%)<br>0.1% (-0.0%, 0.2%)<br>1.8% (1.5%, 2.1%)<br>-1.1% (-1.8%, 0.4%)<br>-0.0% (-0.1%, 0.1%) | 394 (2.9%) 2.246 (16.5%) 551 (4.1%) 579 (4.3%) 55 (0.4%) 577 (4.2%) 4,878 (35.5%) 18 (0.1%) | 392 (2.9%)<br>2,200 (16.2%)<br>552 (4.1%)<br>566 (4.2%)<br>50 (0.4%)<br>579 (4.3%)<br>4,844 (35.5%)<br>21 (0.2%) | 0.0% (-0.4%, 0.4%)<br>0.3% (-0.5%, 1.2%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.4%, 0.6%)<br>0.0% (-0.1%, 0.2%)<br>-0.0% (-0.5%, 0.5%)<br>0.2% (-0.9%, 1.4%)<br>-0.0% (-0.1%, 0.1%) |
| TIA.n (%) Edemax (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Pulmonary hypertension; n (%) Hyperkalemia; n (%) Coronary atherosclerosis; n (%) Coronary atherosclerosis; n (%) Cerebrovascular procedure; n (%) Linsertion of pacemakens; removal of cardiac lead; n (%) | 982 (3.5%)<br>4.621 (16.3%)<br>1.111 (3.9%)<br>1.292 (4.6%)<br>128 (0.5%)<br>1.407 (5.0%)<br>10.186 (36.0%)<br>39 (0.1%)<br>101 (0.4%)<br>2.511 (8.9%) | 1,354 (2.7%) 8,407 (15.9%) 1,998 (4.0%) 2,152 (4.3%) 186 (0.4%) 1,585 (3.2%) 18,491 (37.1%) 71 (0.1%) 117 (0.2%) | 0.8% (0.5%, 1.0%) -0.5% (-1.1%, 0.0%) -0.1% (-0.4%, 0.2%) 0.3% (-0.1%, 0.6%) 0.1% (-0.0%, 0.2%) 1.1% (-1.8%, -0.4%) -0.0% (-0.1%, 0.1%) 0.1% (-0.1%, 0.1%) 0.1% (-0.1%, 0.1%) 0.1% (-0.1%, 0.2%) 2.7% (2.3%, 3.1%) | 394 (29%)<br>2246 (16.5%)<br>551 (4.1%)<br>579 (4.3%)<br>55 (0.4%)<br>577 (4.2%)<br>4.878 (35.9%)<br>18 (0.1%)<br>39 (0.3%)<br>1.031 (7.6%) | 392 (2.9%) 2200 (16.2%) 552 (4.1%) 566 (4.2%) 560 (0.4%) 579 (4.3%) 4844 (35.5%) 21 (0.2%) 42 (0.3%) | 0.0% (-0.4%, 0.4%)<br>0.3% (-0.5%, 0.5%)<br>-0.0% (-0.5%, 0.5%)<br>0.0% (-0.1%, 0.2%)<br>0.0% (-0.5%, 0.5%)<br>0.2% (-0.1%, 0.2%)<br>0.2% (-0.9%, 1.4%)<br>-0.0% (-0.5%, 0.5%)<br>0.2% (-0.9%, 1.4%)<br>0.0% (-0.5%, 0.1%)<br>0.2% (-0.5%, 0.1%) |
| TIA.n (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable cardioverter defibrillator, n (%) Hypersalemia; n (%) Coronary affectselerois; n (%) Cerebrovascular procedure; n (%) Insertion of pacemakers / removal of cardiac lead; n (%) CKD Stage 1-2: n (%) CKD Stage 1-2: n (%) CKD Stage 3-4: n (%) | 982 (3.5%)<br>4.621 (16.3%)<br>1.111 (3.9%)<br>1.292 (4.6%)<br>1.28 (0.5%)<br>1.407 (5.0%)<br>10.186 (36.0%)<br>39 (0.1%)<br>101 (0.4%)<br>2.511 (8.9%)<br>8.496 (30.0%)<br>2.778 (9.8%) | 1,354 (2.7%) 8,407.16.9%) 1.998 (4.0%) 2.152 (4.3%) 1.998 (3.0%) 1.586 (3.2%) 1.849 (3.7%) 7. (0.1%) 11/10.2%) 3.068 (6.2%) 11,499 (23.1%) 3.524 (7.1%) | 0.8% (0.5%, 1.0%) -0.5% (-1.1%, 0.0%) -0.1% (-0.4%, 0.2%) -0.3% (-0.1%, 0.6%) -0.1% (-0.0%, 0.2%) -1.1% (-1.8%, 0.4%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) -0.7% (-0.3%, 3.1%) -7.0% (-0.3%, 7.5%) -2.8% (-2.3%, 3.2%) | 394 (29%) 2.246 (16.5%) 551 (4.1%) 579 (4.3%) 579 (4.3%) 577 (4.2%) 4.878 (35.9%) 18 (0.1%) 39 (0.3%) 1,031 (7.6%) 3,685 (27.1%) 1164 (8.6%) | 392 (29%) 2200 (16 2%) 552 (4 1%) 566 (4 2%) 50 (4 4%) 579 (4 3%) 444 (3 5 5%) 21 (0 2%) 42 (0 3 %) 1,010 (7.4%) 3,704 (27 2%) 1,3704 (27 2%) | 0.0% (-0.4%, 0.4%)<br>0.3% (-0.5%, 1.2%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.4%, 0.6%)<br>0.0% (-0.1%, 0.2%)<br>-0.0% (-0.1%, 0.5%)<br>0.2% (-0.9%, 1.4%)<br>-0.0% (-0.1%, 0.1%)<br>-0.0% (-0.5%, 0.8%)<br>0.2% (-0.5%, 0.8%)<br>0.2% (-0.5%, 0.8%)<br>0.1% (-1.2%, 0.9%) |
| TIA.n (%) Edoma: n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypotrension: n (%) Implemtable cardioverter defibrillator; n (%) Implemtable cardioverter defibrillator; n (%) Lyperialemia; n (%) Ceronary atherosclerosis n (%) | 982 (3.5%) 462 (16.3%) 1.111 (3.9%) 1.292 (4.6%) 128 (0.5%) 1.407 (6.0%) 1.018 (3.6%) 39 (0.1%) 101 (0.4%) 2.511 (8.9%) 2.776 (9.8%) 2.776 (9.8%) 2.776 (9.8%) 2.776 (9.8%) | 1,354 (27%) 8,407.16.9% 1,998 (4.0%) 2,152 (4.3%) 1,598 (3.2%) 1,585 (3.2%) 1,585 (3.2%) 1,585 (3.2%) 1,71 (0.1%) 11/10 (2.2%) 3,058 (6.2%) 3,524 (7.1%) 3,352 (6.7%) 3,352 (6.7%) | 0.8% (0.5% 1.0%)<br>-0.5% (1.1% 0.0%)<br>-0.1% (-0.4% 0.2%)<br>-0.3% (-0.1% 0.6%)<br>-0.3% (-0.1% 0.6%)<br>-0.5% (-0.1% 0.1%)<br>-0.0% (-0.1% 0.1%)<br>-0.0% (-0.1% 0.1%)<br>-0.0% (-0.1% 0.1%)<br>-0.0% (-0.3% 0.2%)<br>-0.0% (-0.3% 0.2%)<br>-0.0% (-0.3% 0.2%)<br>-0.0% (-0.3% 0.2%)<br>-0.0% (-0.3% 0.2%)<br>-0.3% (-0.3% 0.2%)<br>-0.3% (-0 | 394 (29%) 2246 (16.5%) 551 (4.1%) 579 (4.3%) 579 (4.3%) 579 (4.2%) 18 (0.1%) 18 (0.1%) 18 (0.1%) 18 (0.1%) 18 (0.1%) 18 (0.1%) 18 (0.1%) 110 (1.6%) 110 (1.6%) 1117 (1.8%) 1127 (1.8%) | 392 (29%) 2200 (16.2%) 552 (41.5%) 552 (41.5%) 550 (4.4%) 550 (0.4%) 550 (0.4%) 21 (0.2%) 22 (0.2%) 22 (0.2%) 1152 (16.5%) 1152 (16.5%) 1178 (16.7%) | 0.0% (-0.4%, 0.4%)<br>0.3% (-0.5%, 1.2%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.4%, 0.6%)<br>0.1% (-0.4%, 0.6%)<br>0.0% (-0.1%, 0.2%)<br>-0.0% (-0.5%, 0.5%)<br>0.2% (-0.9%, 1.4%)<br>-0.0% (-0.1%, 0.1%)<br>-0.0% (-0.5%, 0.8%)<br>0.2% (-0.5%, 0.8%)<br>0.1% (-0.5%, 0.8%)<br>0.1% (-0.5%, 0.8%)<br>0.1% (-0.5%, 0.8%)<br>0.0% (-0.9%, 1.0%) |
| TIA.n (%) Edeman, n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantatile candioverter defletifistor; n (%) Hypertalemiss; n (%) Coronary attheroscierosis; n (%) Cerebrovascular procedure; n (%) Inselind n (%) activities (%) Cerebrovascular procedure; n (%) Cerebrovascular procedure; n (%) CKI Stage 3-12; n (%) CKI Stage 3-13; n (%) Unspecified CKD; n (%) Acuts kidney high; n (%) | 982(3.5%) 462(16.3%) 1111(3.9%) 1.292(4.6%) 1.292(4.6%) 1.293(6.0%) 1.407(5.0%) 1.407(5.0%) 1.90(1.0%) 1.90(1. | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 185 (0.4%) 185 (0.4%) 184 (1.1%) 17 (0.2%) 3,068 (6.2%) 3,068 (6.2%) 1,499 (2.1%) 3,524 (7.1%) 3,362 (6.7%) | 0.8% (0.5% 1.0%) -0.5% (-1.1% 0.0%) -0.1% (-0.4% 0.2%) -0.3% (-0.1% 0.6%) -0.3% (-0.1% 0.6%) -0.3% (-0.1% 0.6%) -0.5% (-0.5% 0.2%) -1.8% (-1.5% 0.2%) -1.8% (-1.5% 0.2%) -0.0% (-0.1% 0.0%) -0.0% (-0.1% 0.0%) -0.0% (-0.1% 0.3%) -0.0% (-0.5% 0.3%) -0.5% (-0.3% 0.3%) -0.5% (-0.3%) -0.5% (-0.3% 0.3%) - | 394 (29%) 2246 (16.5%) 551 (4.1%) 579 (4.3%) 579 (4.3%) 570 (4.3%) 570 (4.2%) 48.78 (35.9%) 18 (0.1%) 39 (0.3%) 10.331 (7.5%) 3.685 (27.1%) 119 (18.6%) | 392 (29%) 2200 (16.2%) 552 (4.1%) 552 (4.1%) 561 (4.2%) 50 (0.4%) 579 (4.3%) 4,844 (35.6%) 24 (0.2%) 42 (0.3%) 3,704 (27.2%) 1152 (8.5%) | 0.0% (-0.4%, 0.4%) 0.3% (-0.5%, 1.2%) -0.0% (-0.5%, 0.5%) 0.1% (-0.4%, 0.6%) 0.1% (-0.4%, 0.6%) 0.2% (-0.1%, 0.5%) 0.2% (-0.1%, 0.1%) 0.2% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.5%, 0.8%) 0.1% (-0.5%, 0.8%) 0.1% (-0.5%, 0.8%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Palmonary hypertension; n (%) Implantable cardioverter defloritation; n (%) Hypertalemia; n (%) Cononur, atheroscienosis, n (%) Corebovascus personature; n (%) Insertion of pacemakens; / removal of cardiac lead; n (%) CNO Stage 1-2; n (%) CNO Stage 1-2; n (%) Unspecified CNO; n (%) Unspecified CNO; n (%) Hypertensive nephropathy; n (%) Hypertensive nephropathy; n (%) Unsay tract Friedoms; n (%) Gental infections; n (%) Gental infections; n (%) Gental infections; n (%) | 982 (3.5%) 4.621 (6.5%) 1111 (3.9%) 1292 (4.5%) 128 (0.5%) 1407 (5.0%) 10.16 (3.6.0%) 10.10 (4.5%) 10.10 (4.5%) 2.511 (6.9%) 2.511 (6.9%) 2.776 (9.8%) 2.911 (0.3%) 6.296 (2.2.3%) 5.313 (1.8.8%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 185 (0.4%) 185 (0.4%) 185 (1.3%) 18 (4.91(37.1%) 17 (0.2%) 3,068 (6.2%) 3,068 (6.2%) 3,524 (7.1%) 3,524 (7.1%) 8,492 (7.7%) 8,492 (7.7%) 8,492 (7.7%) | 0.8% (0.5% 1.0%) 0.5% (1.1% 0.0%) 0.1% (0.4% 0.2%) 0.1% (0.4% 0.2%) 0.1% (0.00% 0.2%) 0.1% (0.00% 0.2%) 1.1% (1.2% 0.4%) 1.1% (1.5% 0.4%) 0.0% (0.1% 0.0%) 0.1% (0.0% 0.2%) 1.2% (1.2% 0.1%) 0.5% (0.0% 0.2%) 1.3% (1.5% 0.4%) 0.5% (0.2% 0.3%) 1.3% (1.5% 0.4%) 0.5% (0.2% 0.3%) 0.1% (0.0% 0.2%) 1.3% (1.5% 0.5%) 1.3% | 394 (29%) 2246 (16.5%) 551 (4.1%) 579 (4.3%) 579 (4.3%) 577 (4.2%) 48.78 (35.9%) 18 (0.1%) 39 (0.3%) 10.317 (5%) 3.685 (2.71%) 1197 (8.8%) 1273 (19.9%) 273 (19.9%) | 392 (29%) 2200 (16.2%) 552 (4.1%) 566 (4.2%) 501 (4.4%) 501 (4.4%) 501 (4.3%) 4.844 (15.5%) 21 (12.2%) 4.10 (17.4%) 5.704 (17.2%) 1.102 (8.5%) 1.152 (8.5%) 1.152 (8.5%) 2.700 (19.9%) 2.700 (19.9%) 4.75 (15.5%) 4.75 (15.5%) | 0.0% (-0.4%, 0.4%) 0.3% (-0.5%, 1.2%) 0.0% (-0.5%, 0.5%) 0.1% (-0.4%, 0.6%) 0.1% (-0.4%, 0.6%) 0.9% (-0.5%, 0.5%) 0.9% (-0.5%, 0.6%) 0.3% (-0.5%, 0.8%) 0.3% (-0.5%, 0.8%) 0.3% (-0.5%, 0.8%) 0.3% (-0.5%, 0.8%) 0.3% (-0.5%, 0.8%) 0.4% (-0.5%, 0.8%) 0.4% (-0.5%, 0.8%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable cardioverter defibrillator, n (%) Hypertalemin; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Unspecific of pacemakers; / removal of cardiac lead; n (%) COO Stage 1-2; n (%) COO Stage 1-2; n (%) CACUS Edinge 1-2; n (%) Linspecified COCD (%) Acute Active you (%) Hypertensive negativopathy; n (%) Hypertensive negativopathy; n (%) Unitary tack theirotion; n (%) Gential infections; n (%) Gential infections; n (%) COOPD, n (%) Asthman, n (%) | 982 (3.5%) 4.621 (16.3%) 1111 (3.9%) 1292 (4.6%) 128 (0.5%) 1.407 (5.0%) 1.018 (3.6.0%) 39 (0.1%) 39 (0.1%) 39 (0.1%) 39 (0.1%) 3,495 (3.0.0%) 3,495 (3.0.0% | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 185 (0.4%) 18,491 (3.71%) 17 (0.2%) 1,7 (0.5%) 11,40 (2.8%) 1,568 (6.2%) 11,499 (2.31%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 1,420 (2.8%) | 0.8% (0.5% 1.0%) 0.5% (1.1% 0.0%) 0.1% (0.4% 0.2%) 0.1% (0.4% 0.2%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 1.1% (1.2% 0.4%) 0.1% (0.0% 0.2%) 1.1% (1.2% 0.4%) 0.0% (0.1% 0.1%) 0.1% (0.0% 0.2%) 2.7% (2.2% 3.1%) 0.5% (0.0% 0.2%) 2.5% (2.2% 3.2%) 0.5% (0.2% 0.2%) 0.5% (0.2% 0.7%) 0.5% (0.2% 0.7%) 0.5% (0.2% 0.7%) 0.5% (0.2% 0.7%) 0.7% (0.1% 0.2%) 0.7% (0.1% 0.2%) | 394 (29%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (3.5.5%) 18 (0.1%) 19 (0.3%) 10 (0.3%) 10 (0.3%) 1164 (6.6%) 1157 (8.5%) 2,73 (19.9%) 2,73 (19.9%) 4,58 (3.4%) 6,58 (3.4%) 6,58 (3.4%) | 392 (29%) 2200 (16.2%) 552 (4.1%) 552 (4.1%) 550 (0.4%) 550 (0.4%) 550 (0.4%) 550 (0.4%) 21 (0.2%) 22 (0.2%) 12 (0.2%) 12 (0.3%) 13704 (27.2%) 1152 (8.5%) 1157 (8.5%) 170 (1.5%) 270 (1.5%) 270 (1.5%) 270 (1.5%) 270 (1.5%) | 0.0% (1.04%, 0.4%) 0.3% (1.5%), 1.2%) 0.3% (1.5%), 1.2%) 0.0% (1.5%), 0.5%) 0.0% (1.1%, 0.2%) 0.0% (1.1%, 0.2%) 0.0% (1.1%, 0.2%) 0.0% (1.1%, 0.2%) 0.0% (1.0%, 0.5%) 0.0% (1.0%, 0.5%) 0.0% (1.0%, 0.5%) 0.0% (1.0%, 0.5%) 0.0% (1.0%, 0.5%) 0.1% (1.0%, 0.5%) 0.1% (1.0%, 0.5%) 0.1% (1.0%, 0.5%) 0.1% (1.0%, 0.5%) 0.3% (1.1%, 0.0%) 0.3% (1.1%, 0.0%) 0.3% (1.1%, 0.4%) 0.3% (1.1%, 0.5%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable cardioverter defibrillator, n (%) Hypertalemin; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Coronary afferosclerosis; n (%) Unspecified COCD in (%) CACO Stage 1-2; n (%) CACO Stage 1-2; n (%) CACO Stage 1-2; n (%) Linspecified COCD (%) Acute Active you (%) Linspecified COCD (%) Linspecified COCD (%) CACUB Active (%) CACUB Active (%) Coronary afferoscierosis; n (%) Gential infections; n (%) Gential infections; n (%) COPPD, n (%) Asthmus; n (%) Obstructive sleep appea; n (%) Serious bacterial infections; n (%) Obstructive sleep appea; n (%) | 982 (3.5%) 4.621 (16.3%) 1.111 (3.9%) 1.292 (4.6%) 1.28 (0.5%) 1.407 (5.0%) 1.28 (0.5%) 1.407 (5.0%) 1.018 (3.6.0%) 39 (0.1%) 39 (0.1%) 39 (0.1%) 2.778 (9.8%) 3.495 (30.0%) 2.778 (9.8%) 3.495 (30.0%) 3.390 (1.374 (4.9%) 5.055 (17.9%) 3.032 (10.7%) 5.849 (20.7%) 5.849 (20.7%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 18.69 (1.97.1%) 17 (0.5%) 17 (0.2%) 3,668 (6.2%) 11,499 (2.3.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 4,703 (14.7%) 1,420 (2.8%) 8,574 (1.7%) 8,574 (1.7%) 1,420 (2.8%) 8,574 (1.7%) 1,999 (3.7%) 1,999 ( | 0.8% (0.5% 1.0%) 0.5% (1.1% 0.0%) 0.1% (0.4% 0.2%) 0.1% (0.4% 0.2%) 0.1% (0.00% 0.2%) 0.1% (0.00% 0.2%) 0.1% (0.1% 0.0%) 0.5% (0.0% 0.2%) 0.5% (0.2% 0.1%) 0.5% (0.2% 0.7%) | 394 (29%) 2246 f16.5%) 551 (4.1%) 557 (4.1%) 557 (4.3%) 55 (0.4%) 5577 (4.2%) 4.878 (35.5%) 18 (0.1%) 19 (0.2%) 10 (1.0%) 13 (6.5%) 1164 (6.6%) 1197 (8.8%) 273 (19.9%) 458 (3.4%) 655 (5.0%) 2.337 (17.2%) 1644 (12.1%) 3.657 (26.9%) | 392 (29%) 2200 (16.2%) 552 (4.1%) 556 (4.2%) 550 (4.1%) 550 (4.4%) 579 (4.3%) 4.344 (3.5.5%) 4.344 (3.5.5%) 4.210 (3.%) 1.100 (7.4%) 3,704 (27.2%) 1.152 (8.5.%) 1.152 (8.5.%) 2.700 (19.9%) 2.700 (19.9%) 3,734 (7.2%) 1.618 (1.2%) 3,734 (1.2%) 1.618 (1.2%) 3,734 (1.2%) 1.618 (1.2%) 3,697 (27.2%) 3,697 (27.2%) | 0.0% (1.04%, 0.4%) 0.3% (1.5%), 1.2%) 0.3% (1.5%), 1.2%) 0.3% (1.5%), 1.2%) 0.3% (1.5%), 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.2% (1.9%, 1.4%) 0.0% (1.5%, 0.5%) 0.2% (1.9%, 1.4%) 0.0% (1.5%, 0.5%) 0.3% (1.3%, 0.5%) 0.3% (1.3%, 0.5%) 0.3% (1.3%, 0.5%) 0.3% (1.3%, 0.5%) 0.3% (1.3%, 0.5%) 0.3% (1.4%, 0.8%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonany embolism; n (%) Pulmonany hypertension; n (%) Implantable cardioverter defibrillator, n (%) Hypertalemin, n (%) Coronany afferosclerosis, n (%) Coronany afferosclerosis, n (%) Coronany afferosclerosis, n (%) Coronany afferosclerosis, n (%) Coronany afferosclerosis, n (%) Unspecified COCD, n (%) CACO Stage 1-2, n (%) CA | 982 (3.5%) 4.621 (16.3%) 1.111 (3.9%) 1.292 (4.6%) 1.28 (0.5%) 1.407 (5.0%) 1.018 (3.6.0%) 1.018 (3.6.0%) 30 (0.1%) 30 (0.1%) 2.778 (3.6.0%) 3.495 (3.0.0%) 3.312 (18.6%) 3.414 (3.3.9%) 1.274 (4.9%) 5.055 (17.9%) 3.032 (10.7%) 5.849 (20.7%) 5.849 (20.7%) 1.894 (7.0%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 18.69 (1.7%) 17 (0.5%) 17 (0.2%) 3,068 (6.2%) 11,409 (2.3%) 18,491 (2.1%) 18,491 (2.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 1,420 (2.8%) 1,420 (2.8% | 0.8% (0.5% 1.0%) -0.5% (1.1%) -0.1% (0.4%) -0.2%) -0.3% (-0.1%) -0.3% (-0.1%) -0.2%) -0.3% (-0.1%) -0.5% (0.2%) -0.3% (-0.1%) -0.5% (-0.1%) -0.5% (-0.1%) -0.5% (-0.1%) -0.5% (-0.1%) -0.5% (-0.1%) -0.5% (-0.1%) -0.5% (-0.3%) -0 | 394 (29%) 2246 (16.5%) 551 (4.1%) 557 (4.1%) 557 (4.3%) 55 (0.4%) 55 (0.4%) 55 (0.4%) 55 (0.5%) 18 (0.1%) 19 (0.2%) 19 (0.2%) 103 (0.5%) 1164 (2.6%) 1157 (2.8%) 1158 (1.8%) 1159 (1.8%) 1154 (2.6%) 1157 (2.8%) 1154 (2.6%) 1157 (2.8%) 1154 (2.6%) 1157 (2.6%) 1 | 392 (29%) 2200 (16.2%) 552 (4.1%) 556 (4.2%) 550 (4.1%) 550 (4.4%) 570 (4.3%) 4344 (3.5.5%) 421 (2.2%) 421 (2. | 0.0% (1.04%, 0.4%) 0.3% (1.5%), 1.2%) 0.3% (1.5%), 1.2%) 0.3% (1.5%), 1.2%) 0.3% (1.5%), 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.3% (1.3%, 0.5%) |
| TIA.n.(%) Edeman (%) Wenous thromboembolism / Pulmonary embolism; n.(%) Pulmonary hypertensior; n.(%) Implantable cardoverter defibrillator; n.(%) Hyperfallemis; n.(%) Cononary atheroscherosis; n.(%) Cerebrovascular procedure; n.(%) Cerebrovascular procedure; n.(%) Cerebrovascular procedure; n.(%) CKO Stage 3-4; n.(%) CKO Stage 1-2; n.(%) CKO Stage 1-3; n.(%) Acute kidney injury; n.(%) Livaspecified CKD; n.(%) Acute kidney injury; n.(%) Liviasy tract infections; n.(%) CroPt, n.(%) Asthma; n.(%) Obstructive sleep apone; n.(%) Serious bacterial infections; n.(%) Serious bacterial infections; n.(%) Serious bacterial infections; n.(%) MASHMASLD; n.(%) MASHMASLD; n.(%) MASHMASLD; n.(%) Freumonia; n.(%) MASHMASLD; n.(%) | 982 (3.5%) 462 (16.5%) 1111 (3.9%) 1292 (4.6%) 128 (6.5%) 1407 (5.0%) 128 (6.5%) 1407 (5.0%) 130 (10.8%) 131 (10.8%) 131 (10.8%) 131 (10.8%) 132 (10.8%) 133 (10.8%) 134 (10.8%) 135 (10.8%) 135 (10.8%) 137 (4.9%) 137 (4.9%) 138 (4.9%) 139 (10.7%) 139 (10.7%) 139 (10.8%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 2,152 (4.3%) 1,556 (3.2%) 1,569 (3.2%) 1,569 (3.3%) 1,574 (1.2%) 1,574 (1.2%) 1,574 (1.2%) 1,576 (3.3%) 1,574 (1.2%) 1,576 (3.3%) 1,574 (1.2%) 1,576 (3.3%) 1,57 | 0.8% (0.5% 1.0%) -0.5% (1.1%) -0.1% (0.4%, 0.2%) -0.3% (0.4%, 0.2%) -0.3% (0.1%, 0.6%) -0.3% (0.1%, 0.6%) -0.3% (0.1%, 0.6%) -0.3% (0.1%, 0.1%) -0.5% (0.1%, 0.1%) -0.0% (0.1%, 0.1%) -0.0% (0.1%, 0.1%) -0.0% (0.3%, 0.2%) -0.3% (0.3%, 0.2%) -0.3% (0.3%, 0.3%) -0.5% (0.3%, 0.3%) -0.5% (0.3%, 0.3%) -0.5% (0.3%, 0.3%) -0.5% (0.3%, 0.3%) -0.4% (0.7%, 0.3%) -0.4% (0.7%, 0.3%) -0.4% (0.7%, 0.3%) -0.4% (0.7%, 0.1%) -0.4% (0.7%, 0.1%) -0.4% (0.7%, 0.1%) -0.4% (0.1%, 0.1%) -0 | 394 (29%) 2246 10.5%) 551 (4.1%) 551 (4.1%) 579 (4.3%) 55 (0.4%) 577 (4.2%) 18 (0.1%) 19 (3.1%) | 392 (29%) 392 (29%) 552 (41%) 552 (41%) 552 (41%) 550 (04%) 579 (43%) 50 (04%) 579 (43%) 424 (35.6%) 21 (02.8%) 23 (04.8%) 48 (44.8%) 48 (44.8% | 0.0% (-0.4%, 0.4%) -0.0% (-0.4%, 0.4%) -0.0% (-0.5%, 0.5%) -0.3% (-0.5%, 0.3%) -0.3% (-0.3%, 0.5%) -0.3% (-0.3%, 0.5%) -0.3% (-0.4%, 0.5%) |
| TIA.n.(%) Edems. n.(%) Venous thromboembolism / Pulmonary embolism; n.(%) Venous thromboembolism / Pulmonary embolism; n.(%) Pulmonary hypertension; n.(%) Implantable cardoverter defibrillator, n.(%) Hyperhalemia, n.(%) Cerebrovascular procedure; n.(%) Cerebrovascular procedure; n.(%) Cerebrovascular procedure; n.(%) CKO Stage 1-2; n.(%) CKO Stage 1-2; n.(%) CKO Stage 1-4; n.(%) Linspecified CKD; n.(%) Auta kidney injun; n.(%) Livary tract infections; n.(%) Livary tract fineticitions; n.(%) Livaribiasis (fidney and urinary stone); n.(%) CPB; n.(%) Asthma; n.(%) Serious bacterial infections; n.(%) Serious bacterial infections; n.(%) Serious bacterial infections; n.(%) Livar disease; n.(%) MASHMASLD; n.(%) Livar disease; n.(%) Osteoporosis; n.(%) Osteoporosis; n.(%) Osteoporosis; n.(%) Osteoporosis; n.(%) | 982 (3.5%) 4.62 (16.3%) 1.111 (3.9%) 1.292 (4.6%) 1.282 (0.5%) 1.407 (5.0%) 1.28 (0.5%) 1.407 (5.0%) 1.90 (16.4%) 2.511 (8.9%) 8.496 (3.0%) 2.776 (9.8%) 2.781 (9.8%) 2.792 (9.8%) 2.793 (9.8%) 3.312 (18.8%) 3.312 (18.8%) 3.312 (18.8%) 3.312 (18.8%) 3.312 (18.8%) 3.312 (18.8%) 3.312 (18.8%) 4.797 (17.0%) 1.292 (4.6%) 1.294 (6.8%) 1.292 (6.8%) 2.297 (8.8%) 2.297 (8.0%) 9.682 (3.4%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,598 (4.0%) 1,555 (3.2%) 1,557 (3.2%) 1,557 (3.2%) 1,557 (1.3%) 1,524 (7.1%) 1,626 (7.1%) 1,626 (7.1%) 1,627 (7.2%) 1,62 | 0.8% (0.5% 1.0%) 0.5% (1.1%) 0.1% (0.4%, 0.2%) 0.1% (0.4%, 0.2%) 0.3% (4.1%, 0.6%) 0.3% (4.1%, 0.6%) 1.8% (1.1%, 0.6%) 1.8% (1.1%, 0.6%) 1.8% (1.1%, 0.1%) 1.8% (1.1%, 0.1%) 1.8% (1.1%, 0.1%) 1.9% (1.1%, 0.1%) 1 | 394 (29%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 579 (4.3%) 55 (0.4%) 577 (4.2%) 18 (0.1%) | 392 (29%) 392 (29%) 552 (41%) 552 (41%) 556 (42%) 557 (43%) 50 (0.4%) 579 (43%) 370 (42%) 21 (0.2%) 42 (0.3%) 1,000 (7.4%) 3,704 (27.2%) 1,152 (8.5%) 1,152 (8.5%) 1,152 (8.5%) 1,152 (8.5%) 1,152 (8.5%) 1,52 (8.5%) 1,53 (8.5%) 1,54 (8.5%) 1,55 (8. | 0.0% (1.04%, 0.4%) 0.3% (1.05%, 1.2%) 0.3% (1.05%, 1.2%) 0.0% (1.05%, 0.5%) 1.1% (1.04%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.8%) 0.3% (1.1%, 0.5%) 0.3% (1.1%, 0.5%) 0.3% (1.1%, 0.5%) 0.3% (1.1%, 0.5%) 0.3% (1.05%, 0.8%) 0.5% (1.05%, 0.8%) 0.5% (1.05%, 0.8%) 0.5% (1.05%, 0.8%) |
| TIA.n (%) Edems n (%) Venous thromboenbolism / Pulmonary embolism; n (%) Venous thromboenbolism / Pulmonary embolism; n (%) Pulmonary hysiatensism; n (%) Implantable candioverter defibrillator; n (%) Hyperhalemia; n (%) Cerebrovascular procedure; n (%) Cerebrovascular procedure; n (%) Cerebrovascular procedure; n (%) CKO Stage 3-2; n (%) CKO Stage 3-4; n (%) Unspecified CKD; n (%) Acute kidney; hugy, n (%) Hypertensive nephropathy; n (%) Liviany tract infections; n (%) Liviany tract fineticions; n (%) Definition; n (%) Serious bacterial infections; n (%) Serious bacterial infections; n (%) Serious bacterial infections; n (%) Penumonia; n (%) Serious bacterial infections; n (%) Penumonia; n (%) Livian disease; n (%) MASHIMASLD; n (%) Fractures; Falls; n (%) Osteocorbosis; n (%) Depression (%) Depression (%) Dementia; n (%) Dementia; n (%) Dementia; n (%) | 982 (3.5%) 4.621 (6.3%) 1111 (3.9%) 1292 (4.5%) 128 (0.5%) 1407 (5.0%) 128 (0.5%) 1407 (5.0%) 39 (0.1%) 101 (0.4%) 2511 (8.9%) 8.496 (3.0%) 2776 (9.8%) 2511 (8.9%) 8.496 (3.0%) 2781 (8.8%) 2511 (8.9%) 8.496 (3.0%) 1.374 (4.9%) 5.055 (1.7%) 3.032 (0.7%) 5.849 (2.0.7%) 1.292 (4.6%) 1.884 (7.0%) 4.797 (7.0%) 1.292 (4.6%) 1.884 (7.0%) 4.797 (7.0%) 1.292 (6.6%) 2.595 (9.2%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,598 (4.0%) 1,555 (3.2%) 1,552 (3.2%) 1,55 | 0.8% (0.5% 1.0%) 0.5% (1.1%) 0.1% (0.4%, 0.2%) 0.1% (0.4%, 0.2%) 0.1% (0.4%, 0.2%) 0.1% (0.5%, 0.2%) 1.5% (1.5%, 2.1%) 1.5% (1.5%, 2.1%) 1.5% (1.5%, 2.1%) 1.5% (0.5%, 0.2%) 2.7% (2.3%, 3.1%) 2.8% (2.3%, 3.2%) 3.5% (3.1%, 0.7%) 0.4% (0.7%, 0.1%) 0.7% (0.1%, 1.2%) 1.3% (1.5%, 2.5%) | 394 (2.9%) 2246 fl.6.5%) 551 (4.1%) 551 (4.1%) 579 (4.3%) 55 (0.4%) 577 (4.2%) 18 (0.1%) 18 (0.1 | 392 (29%) 392 (29%) 552 (41%) 552 (41%) 556 (42%) 552 (41%) 556 (42%) 50 (0.4%) 579 (43%) 50 (0.4%) 579 (43%) 10 (27%) 110 (27%) 110 (27%) 110 (27%) 1152 (85%) 1152 (85%) 1153 (85%) 1153 (85%) 1154 (85%) 1156 (85%) 1157 (15%) 117 (85%) 117 (85%) 117 (85%) 1075 (75%) | 0.0% (1.04%, 0.4%) 0.0% (1.05%, 0.5%) 0.3% (1.05%, 1.2%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.8%) |
| TIA. n. (%) Edema, n. (%) Venous thromboembolism / Pulmonary embolism; n. (%) Pulmonary hypertension; n. (%) Implantable candioverter defletifistor; n. (%) Implantable candioverter defletifistor; n. (%) Loronary atherosclerosis; n. (%) Coronary atherosclerosis; n. (%) CXI Staps 1-2; n. (%) CXI Staps 1-2; n. (%) CXI Staps 1-2; n. (%) Unspecified CXID; n. (%) Unspecified CXID; n. (%) Hypertensive rephropathy; n. (%) Unspecified CXID; n. (%) Gental infections; n. (%) Unitary tract infections; n. (%) Gental infections; n. (%) Obstructive steep apnex; n. (%) Obstructive steep apnex; n. (%) Pheuronis; n. (%) Destructive; f. (%) MASHMASD; n. (%) MASHMASD; n. (%) Osteoprofisis; n. (%) Osteoprofisis; n. (%) Osteoprofisis; n. (%) Osteoprofisis; n. (%) Osteoprofisis; n. (%) | 982 (3.5%) 4.621 (6.5%) 1111 (3.9%) 129 (4.5%) 129 (4.5%) 128 (0.5%) 1407 (5.0%) 10.186 (3.6.0%) 39 (0.1%) 10.186 (3.6.0%) 39 (0.1%) 10.104%) 2511 (6.9%) 2511 (6.9%) 2511 (6.9%) 39 (0.1%) 10.104%) 2511 (6.9%) 39 (0.1%) 10.104%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,95 | 0.8% (1.5% 1.0%) 0.8% (1.1% 0.0%) 0.1% (1.0 0.0%) 0.2%) 0.2% (1.2%) 0.3% (1.0 0.0%) 0.3% (1.0 0.0% | 394 (2.9%) 394 (2.9%) 551 (4.1%) 551 (4.1%) 551 (4.1%) 55 (0.4%) 577 (4.2%) 4.878 (35.5%) 18 (0.1%) 39 (0.3%) 10.31 (7.5%) | 392 (29%) 392 (29%) 552 (41%) 552 (41%) 556 (42%) 550 (43%) 550 (43%) 550 (43%) 550 (43%) 4,844 (35.6%) 24 (0.2%) 4,240 (3.3%) 1,000 (7.3%) 1,152 (8.5%) 1,152 (8 | 0.0% (1.4%, 0.4%) 0.3% (1.5%), 1.2% 0.3% (1.5%), 1.2% 0.3% (1.5%), 1.2% 0.0% (1.5%, 0.5%) 0.0% (1.5%, 0.5%) 0.0% (1.5%, 0.5%) 0.0% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.3% (1.5%, 0.5%) 0.5% (1.5%, 0.5%) 0.5% (1.5%, 0.5%) 0.5% (1.5%, 0.5%) |
| TIA.n (%) Edems, n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable candioverter defleritation; n (%) Implantable candioverter defleritation; n (%) Lippethalments; n (%) Consulty atherosclerosis; n (%) CXD Staps 3-1; n (%) CXD Staps 3-1; n (%) Unspecified CXD; n (%) Acuta kidney hijv; n (%) Hypertensive nephropathy; n (%) Unspecified CXD; n (%) Gental infections; n (%) Gental infections; n (%) COPE, n (%) Asthmar, n (%) Obstructive sleep apone; n (%) Precurronis; n (%) Precurronis; n (%) Precurronis; n (%) Precurronis; n (%) Osteoporosis; n (%) Demendix, n (%) Demendix, n (%) Demendix, n (%) | 982 (3.5%) 4.621 (6.5%) 1111 (3.9%) 1292 (4.5%) 128 (0.5%) 1407 (5.0%) 10186 (36.0%) 39 (0.1%) 10196 (36.0%) 39 (0.1%) 1010 (0.4%) 39 (0.1%) 1010 (0.4%) 39 (0.1%) 1010 (0.4%) 39 (0.1%) 1010 (0.4%) 39 (0.1%) 1010 (0.4%) 101 | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,95 | 0.8% (0.5% 1.0%) 0.8% (1.1% 0.0%) 0.1% (1.0 0.0%) 0.0% (1.0 0.0%) | 394 (29%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 577 (4.2%) 4.878 (35.5%) 18 (0.1%) 39 (0.3%) 1031 (7.5%) 11031 (7.5%) 11031 (7.5%) 1104 (6.6%) 1197 (8.8%) 4.878 (3.5%) 4.988 (3.5%) 4.988 (3.5%) 4.988 (3.5%) 4.998 (3.5%) | 392 (29%) 2200 (16.2%) 552 (4.1%) 552 (4.1%) 556 (4.2%) 550 (4.3%) 550 (4.3%) 550 (4.3%) 579 (4.3%) 4,844 (3.5.6%) 24 (0.2%) 1,000 (7.3%) 1,100 (7.3%) 1,100 (7.3%) 1,152 (16.5%) 1,152 | 0.0% (1.4%, 0.4%) 0.3% (1.5%), 1.2% 0.3% (1.5%), 1.2% 0.3% (1.5%), 1.2% 0.3% (1.5%), 0.5% 0.5% (1.5%), 0.5% 0.0% (1.5%, 0.5%) 0.0% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.2% (1.5%, 0.5%) 0.3% (1.5%, 0.5%) |
| TIA. n. (%) Edoma; n. (%) Venous thromboembolism / Pulmonary embolism; n. (%) Pulmonary hypertension; n. (%) Implantable candioverter defictifiator, n. (%) Hypertalemia; n. (%) Coronary atherosaction (n. (%) Cerebroviascular procedure; n. (%) Derebroviascular procedure; n. (%) Erestroviascular procedure; n. (%) Erestroviascular procedure; n. (%) CXIS Stage 3-12; n. (%) CXIS Stage 3-14; n. (%) Unspecified CXID: n. (%) CXIS Stage 3-14; n. (%) Unspecified CXID: n. (%) Hypertensive nephropathy; n. (%) Unspecified CXID: n. (%) CVID: n. (%) Gential infections; n. (%) Gential infections; n. (%) Gential infections; n. (%) COPE, n. (%) Asthmur, n. (%) Obstructive sleep apnex; n. (%) Presumonia; n. (%) Distructive sleep apnex; n. (%) Presumonia; n. (%) Distructive sleep apnex; n. (%) Presumonia; n. (%) Obstructive sleep apnex; n. (%) Presumonia; n. (%) Osteoprosis; n. (%) Osteoprosis; n. (%) Osteoprosis; n. (%) Demersion; n. (%) | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 129 (4.5%) 129 (4.5%) 128 (5.5%) 128 (5.5%) 128 (5.5%) 128 (5.5%) 128 (5.5%) 101 (6.4%) 101 (6.5%) 101 (6.5 | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,95 | 0.8% (0.5% 1.0%) 0.3% (1.1% 0.0%) 0.1% (1.0 0.0%) 0.0% (1.0 0. | 394 (29%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (35.9%) 18 (0.1%) 39 (0.3%) 30 (0.5%) 30 | 392 (2.9%) 392 (2.9%) 552 (4.1%) 552 (4.1%) 556 (4.2%) 550 (4.3%) 550 (4.3%) 550 (4.3%) 550 (4.3%) 4,04 (4.2%) 4,0 | 0.0% (1.4%, 0.4%) 0.3% (1.5%), 1.2% 0.0% (1.5%, 0.5%) 0.3% (1.5%, 0.5%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable candioverter deficilitator, n (%) Hyperkalemia, n (%) Coronary atheroscienosis, n (%) Coronary atheroscienosis, n (%) Coronary atheroscienosis, n (%) Coronary atheroscienosis, n (%) Coronary atheroscienosis, n (%) Imsertion of pacternialems / removal of cardiac lead; n (%) CXIS Stage 3-2, n (%) CXIS Stage 3-4, n (%) Unspecified CXID, n (%) CXIS Stage 3-4, n (%) Unspecified CXID, n (%) Evitary tract infections; n (%) Gental infections; n (%) Obstructive sleep apnea, n (%) Serious bacterial infections; n (%) Preumonia; n (%) Distructive sleep apnea, n (%) Serious bacterial infections; n (%) Preumonia; n (%) Distructive sleep apnea, n (%) Distructive | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 129 (4.5%) 129 (4.5%) 128 (5.5%) 128 (5.5%) 128 (5.5%) 128 (5.5%) 128 (5.5%) 101 (6.4%) 101 (6.5%) 101 (6.5 | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 135 (0.4%) 136 (0.5%) 13 (0.5%) 13 (0.5%) 13 (0.5%) 13 (0.5%) 14 (0.5%) 14 (0.5%) 14 (0.5%) 14 (0.5%) 15 (0.5%) 16 (0.5%) 16 (0.5%) 17 (0.5%) 18 (0.5%) 18 (0.5%) 19 (0.5%) | 0.8% (0.5% 1.0%) 0.1% (1.0% 0.0%) 0.1% (1.0% 0.0%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 1.1% (1.2% 0.2%) 1.1% (1.2% 0.2%) 1.1% (1.2% 0.2%) 1.2% (1.2% 0.2%) 1.3% (1.2% 0.2%) | 394 (2.9%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 557 (4.3%) 55 (0.4%) 55 (0.4%) 55 (0.4%) 577 (4.2%) 4.578 (3.5.9%) 18 (0.1%) 39 (0.3%) 1031 (7.6%) 39 (0.3%) 1164 (6.6%) 1167 (6.6%) 1169 (6.6%) 273 (19.9%) 273 (19.9%) 235 (17.2%) 1464 (12.1%) 3.657 (26.9%) 474 (3.5%) 173 (6.4%) 2469 (18.2%) 147 (6.6%) 137 (6.4%) 148 (6.6%) 149 (6.6%) 159 (6.6%) 149 (6.6%) 149 (6.6%) 159 (6.6%) 149 (6.6%) 159 (6.6%) 149 (6.6 | 392 (29%) 392 (29%) 552 (41%) 552 (41%) 556 (42%) 550 (43%) 550 (43%) 550 (43%) 550 (43%) 454 (45.6%) 4,000 (20%) | 0.0% (1.04%, 0.4%) 0.3% (1.05%, 1.2%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.05%) 0.1% (1.05%, 0.05%) 0.1% (1.05%, 0.05%) 0.3% (1.1%, 0.05%) 0.3% (1.0%, 0.05%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertinishor, n (%) Implicitable cardioverter deficitlator, n (%) Implicitable cardioverter deficitlator, n (%) Importinative cardioverter deficitlator, n (%) Dononary afferenceloresis, n (%) Coronary afferenceloresis, n (%) Coronary afferenceloresis, n (%) Insertion of paccemakens / removal of cardiac lead n (%) CXIO Stage 3-2, n (%) CXIO Stage 3-2, n (%) CXIO Stage 3-2, n (%) Unspecified CXIO, n (%) Gental infections; n (%) Gental infections; n (%) Gental infections; n (%) Obstructive sleep apness, n (%) Serious bacterial infections; n (%) Pheumonia; n (%) Distructive sleep apness, n (%) Serious bacterial infections; n (%) Distructive sleep apness; n (%) Distructive sleep apness; n (%) Distructive sleep apness; n (%) Dementia; n (%) Institute of the projectoris; n (%) Anneity, n (%) Reprocessories; n (%) | 982 (3.5%) 4.621 (6.5%) 1111 (3.9%) 1292 (4.6%) 128 (0.5%) 128 (0.5%) 128 (0.5%) 128 (0.5%) 128 (0.5%) 128 (0.5%) 101 (0.4%) 251 (8.9%) 101 (0.4%) 251 (8.9%) 104 (0.4%) 251 (8.9%) 104 (0.5%) 105 (0.5%) 106 (0.5%) 107 (0.5%) 107 (0.5%) 108 (0.5%) 109 (0. | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 185 (0.4%) 185 (0.4%) 18.49 (1.7%) 18.49 (1.7%) 17 (0.2%) 3,068 (6.2%) 18,29 (1.7%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 4,526 (6.3%) 8,452 (7.7%) 1,420 (2.8%) 1, | 0.8% (0.5% 1.0%) 0.1% (1.0% 0.0%) 0.1% (1.0% 0.0%) 0.1% (0.0% 0.2%) 0.2% (0.2% 0.2%) 0.2% (0.2% 0.2%) 0.5% (0.1% 0.0%) 0.5% (0.1% 0.0%) 0.5% (0.1% 0.0%) 0.5% (0.2% 0.2%) 0.5% (0.1% 0.0%) 0.5% (0.0% 0.0%) | 394 (29%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (3.5.9%) 18 (0.1%) 19 (0.2%) 19 (0.2%) 10 (1.1%) 10 (1.1%) 11 | 392 (29%) 392 (29%) 592 (41%) 592 (41%) 595 (41%) 596 (42%) 591 (43%) 591 (43%) 484 (42.65%) 41 (25.65%) 42 (12.75%) 42 (12.75%) 42 (12.75%) 42 (12.75%) 43 (12.75%) 43 (12.75%) 43 (12.75%) 44 (12.75%) 45 (12.75%) 45 (12.75%) 45 (12.75%) 47 (12.75 | 0.0% (1.4%, 0.4%) 0.3% (1.5%), 1.2% 0.3% (1.5%), 1.2% 0.3% (1.5%), 1.2% 0.3% (1.5%), 0.5% 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.3%, 0.5%) 0.0% (1.5%, 0.5%) 0.3% (1.4%, 0.5%) 0.3% (1.5%, 0.5%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertaisation; n (%) Implantable cardioverter deficilitation; n (%) Implantable cardioverter deficilitation; n (%) Dononary afferencelorosis; n (%) Cononary afferencelorosis; n (%) Cononary afferencelorosis; n (%) Cononary afferencelorosis; n (%) Insertion of pacemakens; / removal of cardiac lead; n (%) CXIO Steps 1-2; n (%) CXIO Steps 1-2; n (%) CXIO Steps 1-2; n (%) CXIO Steps 1-2; n (%) Unsepecified CXIO; n (%) CXIO Steps 1-2; n (%) Gental infections; n (%) Gental infections; n (%) University infections; n (%) Districtive sleep apneas; n (%) Serious bacterial infections; n (%) Pheumonia; n (%) Districtive sleep apneas; n (%) Serious bacterial infections; n (%) Pheumonia; n (%) Districtive sleep apneas; n (%) Serious bacterial infections; n (%) Districtive sleep apneas; n (%) Districtive sleep apneas; n (%) Definition or psychosis; n (%) Demonster, n (%) Definition or psychosis; n (%) Demonster, n (%) Definition or psychosis; n (%) Aneity, n (%) Definition or psychosis; n (%) Aneity, n (%) Hyporthyciotism n (%) Universities of (%) Univ | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 1292 (4.6%) 128 (0.5%) 1407 (5.0%) 128 (0.5%) 1407 (5.0%) 10186 (3.6.0%) 101 (0.4%) 2776 (9.8%) 3.495 (3.0.0%) 3.13 (1.8%) 9.44 (3.3.%) 1.174 (4.9%) 5.055 (1.7.9%) 3.032 (0.7.%) 5.812 (0.7%) 1.292 (4.6%) 1.292 (4.6%) 1.292 (4.6%) 1.292 (4.6%) 1.292 (5.6%) 3.012 (3.0.0%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 185 (0.4%) 185 (0.4%) 185 (1.2%) 18 (1.01%) 17 (0.2%) 3,068 (6.2%) 17 (0.2%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 4,525 (7.1%) 8,452 (7.7%) 1,420 (2.8%) 1,420 (2. | 0.8% (0.5% 1.0%) 0.1% (1.0% 0.0%) | 394 (2.9%) 394 (2.9%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.878 (35.9%) 18 (0.3%) 19 (0.2%) 19 (0.2%) 1031 (7.6%) 3.665 (27.7%) 1164 (6.6%) 1197 (8.8%) 4.578 (3.4%) 665 (5.0%) 2.337 (17.2%) 164 (12.1%) 3.657 (2.6.9%) 4.578 (3.8%) 4.58 (3.8%) 5.059 (3.7.2%) | 392 (29%) 392 (29%) 592 (41%) 592 (41%) 595 (41%) 591 (42%) 591 (43%) 591 (43%) 4384 (35%) 421 (23%) 4394 (31%) 4395 (31%) 4395 (31% | 0.0% (1.04%, 0.4%) 0.3% (1.05%, 1.2%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.05%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism (1%) Venous thromboembolism / Pulmonary embolism (1%) Pulmonary hypertension (1%) Implantable cardioverter defibrillator, (1%) Hypertelamin, (1%) Coronary afferencelerosis, (1%) Coronary afferencelerosis, (1%) Coronary afferencelerosis, (1%) Coronary afferencelerosis, (1%) Insertin of pacemakens / removal of cardiac lead; (1%) COS Stage 1.4: (1%) COS Stage 1.4: (1%) COS Stage 1.4: (1%) CACUS Stage 1.4: (1%) CACUS Stage 1.4: (1%) Linspecified COCD (1%) Acute Moley hyper (1%) Hypertensive nephropathy, (1%) Hypertensive nephropathy, (1%) Univary tract Hollow, (1%) COPPD, (1%) Asthmax (1%) Obstructive sleep apnear, (1%) Serious bacteries (1%) Pheumoniar (1%) Distructive sleep apnear, (1%) Freumoniar (1%) Destructive sleep apnear, (1%) Serious bacteries (1%) MASH/MASLD, (1%) Pheumoniar (1%) Destructive (1%) Destructive (1%) Destructive (1%) Destructive (1%) Seep also structives (1%) Seep acredities (1%) Destructive (1%) Seep acredities (1%) Demenda (1%) Seep acredities (1%) Seep ac | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 1292 (4.6%) 128 (0.5%) 1407 (5.0%) 128 (0.5%) 1407 (5.0%) 1018 (3.6.0%) 1010 ( | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 185 (0.4%) 185 (0.4%) 185 (1.2%) 18 (1.01%) 17 (0.2%) 3,068 (6.2%) 18 (1.1%) 17 (0.2%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 1,703 (1.4%) 1,703 (1.4%) 1,703 (1.4%) 1,703 (1.4%) 1,703 (1.4%) 1,705 (1.4%) | 0.8% (0.5% 1.0%) 0.1% (1.0% 0.0%) 0.0% (1.0% 0.0%) 0.0% (1.0% 0.0%) 0.0% (1.0% 0.0%) | 394 (2.9%) 394 (2.9%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.878 (35.9%) 18 (0.3%) 19 (0.2%) 19 (0.2%) 10 (1.0%) 10 (1.0%) 1164 (6.6%) 1167 (6.6%) 1168 (6.6%) 1169 (6.6%) 1164 (1.1%) 1167 (1.1%) 1168 (1.1%) 1169 (1 | 392 (2.9%) 392 (2.9%) 592 (4.1%) 595 (4.1%) 596 (4.2%) 591 (4.3%) 591 (4.3%) 591 (4.3%) 4,344 (4.2%) 4,344 (4 | 0.0% (1.04%, 0.4%) 0.3% (1.05%, 1.2%) 0.3% (1.05%, 1.2%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.05%) 0.3% (1.14%, 0.05%) 0.3% (1.15%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) |
| TIA.1 (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable cardioverter defibrillator, n (%) Hypertelamin; n (%) Coronary afferoactions; n (%) Coronary afferoactions; n (%) Coronary afferoactions; n (%) Coronary afferoactions; n (%) Insertin of pacemakens; / removal of cardiac lead; n (%) COO Stage 1-2; n (%) COO Stage 1-2; n (%) CAO Stage 1-2; n | 982 (3.5%) 46.21 (16.3%) 1111 (3.9%) 1292 (4.6%) 1292 (4.6%) 128 (0.5%) 1407 (5.0%) 1018 (3.6.0%) 1010 (3.6.0%) 10 | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 185 (0.4%) 185 (0.4%) 185 (1.2%) 18 (1.01%) 17 (0.2%) 3,068 (6.2%) 18 (1.2%) 18 (1.1%) 18 ( | 0.8% (0.5% 1.0%) 0.9% (1.0% 0.0%) 0.1% (1.0% 0.0%) 0.5% (1.0% 0.0%) 0.0% (1.0% 0.0%) | 394 (2.9%) 394 (2.9%) 551 (4.1%) 551 (4.1%) 557 (4.3%) 55 (0.4%) 557 (4.2%) 4.878 (3.5.9%) 4.878 (3.5.9%) 4.878 (3.5.9%) 3.685 (27.1%) 1164 (6.6%) 1167 (6.6%) 2.73 (19.9%) 3.685 (27.1%) 1164 (6.6%) 1167 (6.6%) 4.878 (3.5.9%) 4.878 | 392 (2.9%) 392 (2.9%) 552 (4.1%) 552 (4.1%) 556 (4.2%) 550 (4.4%) 579 (4.3%) 501 (4.4%) 579 (4.3%) 4,344 (3.5%) 4,344 (3.1%) 4,344 (3.1 | 0.0% (1.04%, 0.4%) 0.0% (1.04%, 0.4%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.05%) |
| TIA.n. (%) Edomac, n. (%) Venous thromboembolism / Pulmonary embolism; n. (%) Pulmonary hymerisasion; n. (%) Implantable cardioverter defibrillator, n. (%) Hyperkalemia; n. (%) Coronary atherosclerosis; n. (%) CXD Staps 3-2; n. (%) Unspecified CXD; n. (%) Acute kidney hijm; n. (%) Unspecified CXD; n. (%) Acute kidney hijm; n. (%) Unspecified CXD; n. (%) Cyronary through n. (%) Unspecified CXD; n. (%) Gential infections; n. (%) Gential infections; n. (%) Coronary atheroscleros; n. (%) Obstructive alees annex; n. (%) Coronary atheroscleros; n. (%) Presumonias; n. (%) Demonias; n. (%) Demonias; n. (%) Osteoprosis; n. (%) Osteoprosis; n. (%) Osteoprosis; n. (%) Demonias; n. (%) Osteoprosis; n. (%) Osteoprosis | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 1292 (4.6%) 128 (0.5%) 1407 (5.0%) 128 (0.5%) 1407 (5.0%) 1018 (3.6.0%) 1010 ( | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 186 (0.4%) 185 (0.4%) 185 (0.4%) 185 (0.4%) 185 (1.2%) 18 (1.01%) 17 (0.2%) 3,068 (6.2%) 18 (2.1%) 17 (0.2%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 1,703 (1.4%) 1,703 (1.4%) 1,703 (1.4%) 1,703 (1.4%) 1,703 (1.4%) 1,705 (1.4%) | 0.8% (0.5% 1.0%) 0.1% (1.0% 0.0%) 0.0% (1.0% 0.0%) 0.0% (1.0% 0.0%) 0.0% (1.0% 0.0%) | 394 (2.9%) 394 (2.9%) 2246 (16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.878 (35.9%) 18 (0.3%) 19 (0.2%) 19 (0.2%) 10 (1.0%) 10 (1.0%) 1164 (6.6%) 1167 (6.6%) 1168 (6.6%) 1169 (6.6%) 1164 (1.1%) 1167 (1.1%) 1168 (1.1%) 1169 (1 | 392 (2.9%) 392 (2.9%) 592 (4.1%) 595 (4.1%) 596 (4.2%) 591 (4.3%) 591 (4.3%) 591 (4.3%) 4,344 (4.2%) 4,344 (4 | 0.0% (1.04%, 0.4%) 0.3% (1.05%, 1.2%) 0.3% (1.05%, 1.2%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.2% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.05%) 0.3% (1.14%, 0.05%) 0.3% (1.15%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) 0.3% (1.05%, 0.05%) |
| TIA.n (%) Edems, n (%) Venous thromboembolism / Pulmonary embolism; n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable candioverter defletifistor; n (%) Hypertelments; n (%) Coronary atherosclerosis: n (%) Cox O Stapa 3-12; n (%) Cox O Stapa 3-12; n (%) Coronary atherosclerosis: n (%) Precurronis: n (%) Precurronis: n (%) Precurronis: n (%) Osteocorosis: n (%) Osteocorosis: n (%) Demension n (%) Precurronis: n (%) Demension n (%) | 982 (3.5%) 4621 (6.5%) 1111 (3.9%) 1292 (4.5%) 128 (0.5%) 1407 (5.0%) 10186 (36.0%) 39 (0.1%) 10186 (36.0%) 39 (0.1%) 10196 (36.0%) 39 (0.1%) 1010 (0.4%) 2511 (8.9%) 34 (0.1%) 1010 (0.4%) 2511 (8.9%) 34 (0.1%) 1010 (0.4%) 36 (0.0%) 2511 (0.3%) 6,296 (2.2%) 5313 (18.8%) 944 (3.3%) 1274 (4.9%) 5,055 (17.9%) 30,137 (4.6%) 1274 (4.9%) 1592 (6.6%) 1292 (6.6%) 1292 (6.6%) 1292 (6.6%) 1293 (6.6%) 1293 (6.6%) 1294 (6.6%) 1295 (6.6%) 1296 (6.6%) 1296 (6.6%) 1296 (6.6%) 1297 (17.2%) 1297 (17.2%) 1297 (17.2%) 1297 (17.2%) 1297 (17.2%) 1297 (17.2%) 1297 (17.2%) 1298 (17.2%) 1299 (17.2%) 1290 (17.2%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,95 | 0.8% (1.5% 1.0%) 0.8% (1.1% 0.0%) 0.1% (1.0 0.0%) 0.2%) 0.2% (1.2%) 0.3% (1.2%) | 394 (2.9%) 394 (2.9%) 551 (4.1%) 551 (4.1%) 551 (4.1%) 557 (4.3%) 55 (0.4%) 577 (4.2%) 4.878 (35.5%) 18 (0.1%) 18 (0.1%) 19 (1.1%) 19 (1 | 392 (29%) 392 (29%) 552 (41%) 552 (41%) 556 (42%) 552 (41%) 56 (42%) 579 (43%) 4,844 (35.6%) 24 (0.2%) 4,844 (35.6%) 24 (0.2%) 4,844 (35.6%) 1,100 (7.4%) 3,704 (27.2%) 1,152 (8.5%) 1,153 (8.5%) 1,154 (8.5%) 1,154 (8.5%) 1,364 (28.4%) 1,364 ( | 0.0% (1.04%, 0.4%) 0.0% (1.04%, 0.4%) 0.0% (1.05%, 0.5%) 0.1% (1.06%, 0.05%) 0.1% (1.06%, 0.05%) 0.1% (1.06%, 0.05%) 0.1% (1.05%, 0.05%) |
| TIA. n. (%) Edeman, n. (%) Venous thromboembolism / Pulmonary embolism; n. (%) Pulmonary hypertension; n. (%) Implantable candioverter defictifiator, n. (%) Hypertalemia, n. (%) Caronary atherosaction of editoritists, n. (%) Cerebroviascular procedure, n. (%) Deservoviascular procedure, n. (%) Insertion of pacemiaters, 1 (%) Cerebroviascular procedure, n. (%) Insertion of pacemiaters, 1 (%) CKI Stage 3-12, n. (%) CKI Stage 3-12, n. (%) Unspecified CKID, n. (%) Hypertensive nephropathy; n. (%) Hypertensive nephropathy; n. (%) Hypertensive nephropathy; n. (%) Unspecified CKID, n. (%) Gential infections; n. (%) Gential infections; n. (%) Gential infections; n. (%) Gorbon, n. (%) Obstructive sleep apnex; n. (%) Serious bacterial infections; n. (%) Pheumonia; n. (%) Distructive sleep apnex; n. (%) Pheumonia; n. (%) MASHVAASLD n. (%) Pheumonia; n. (%) Osteoprosis; n. (%) Osteoprosis; n. (%) Osteoprosis; n. (%) Demendia; n. (%) Pheumonia; n. (%) Demendia; n. (%) Demendia; n. (%) Demendia; n. (%) Demendia; n. (%) Pheumonia; n. (%) Demendia; n. (%) Coxcomitant use or initiation of Metformix; n. (%) Coxcomitant use or initiation of Metformix; n. (%) | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 129 (4.5%) 128 (0.5%) 140 (3.6%) 128 (0.5%) 140 (3.6%) 128 (0.5%) 140 (1.6%) 101 (6.4%) 101 (6.5%) 101 (6.4%) 101 (6.5%) 101 (6.5 | 1,354 (2.7%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,849 (1.71%) 1,100 (1.0%) 1,10 | 0.8% (1.5% 1.0%) 0.1% (1.0% 0.0%) 0.1% (1.0% 0.0%) 0.1% (1.0% 0.2%) 0.1% (1.0% 0.0%) 0.0% (1.0% 0.0%) | 394 (29%) 2246 fl6.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (3.5.9%) 18 (0.1%) 18 (0.1%) 18 (0.1%) 19 (1.5.9%) 10 (1.5.9%) 110 (1.6.9%) 111 (1.6.9%) 110 (1.6.9%) 111 (1.6.9%) | 392 (2.9%) 392 (2.9%) 592 (4.1%) 595 (4.1%) 596 (4.2%) 591 (4.3%) 591 (4.3%) 591 (4.3%) 4,04 (4.1%) 4, | 0.0% (1.0% 0.4%) 0.4% 0.4% 0.3% 0.3% (1.0% 0.4% 0.4%) 0.0% (1.0% 0.5% 0.5%) 0.0% (1.0% 0.4% 0.6%) 0.0% (1.0% 0.4% 0.6%) 0.0% (1.0% 0.4% 0.6%) 0.0% (1.0% 0.4% 0.6%) 0.0% (1.0% 0.4% 0.6%) 0.0% (1.0% 0.4% 0.4% 0.4% 0.4% 0.4% 0.4% 0.4% 0 |
| TIA. n. (%) Edeman (n.)% Venous thromboembolism / Pulmonary embolism; n. (%) Pulmonary hypertension; n. (%) Implantable candioverter defictifiator, n. (%) Hyperkalemia, n. (%) Conomizer attreascelerosis; n. (%) Conomizer attreascelerosis; n. (%) Conomizer attreascelerosis; n. (%) Cerebrovascelar procedure; n. (%) Implantable candioverter (%) Implantable candioverter (%) Implantable candioverter (%) Implantable candioverter (%) CRIS Stage 3-12, n. (%) CRIS Stage 3-12, n. (%) CRIS Stage 3-14, n. (%) Unspecified CKD; n. (%) Acute kidney hypor, n. (%) Hypertensive nephropathy; n. (%) Hypertensive nephropathy; n. (%) Unspecified CKD; n. (%) Gental infections; n. (%) Gental infections; n. (%) Gental infections; n. (%) Gorbania infections; n. (%) Obstructive sleep apnex; n. (%) Serious bacterial infections; n. (%) Pheumonia; n. (%) Data (%) | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 129 (4.5%) 128 (0.5%) 140 (3.6%) 128 (0.5%) 140 (3.6%) 128 (0.5%) 140 (1.6%) 1016 (3.6%) 101 (0.4%) 101 (0.5%) 101 (0.4%) 101 (0.5%) 101 (0. | 1,354 (2.7%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,849 (1.71%) 1,100 (1.0%) 1,10 | 0.8% (1.5% 1.0%) 0.18% (1.1% 0.0%) 0.19% (1.0% 0.2%) 0.19% (1.0% 0.2%) 0.19% (1.0% 0.2%) 0.19% (1.0% 0.2%) 0.19% (1.0% 0.2%) 1.1% (1.1.8% 0.4%) 0.10% (1.0.1% 0.1%) 0.10% (1.0.2%) 0.2% (1.1% 0.1%) 0.10% (1.0.2%) 0.2% (1.2% 0.2%) 0.2% (1.2% 0.2%) 0.2% (1.2% 0.2%) 0.2% (1.2% 0.2%) 0.5% (1.0.2% 0.2%) 0.5% (1.0.2% 0.2%) 0.5% (1.0.2% 0.0%) 0.0% (1.0.2% 0.0%) | 394 (29%) 2246 fl6.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (3.5.9%) 18 (0.1%) 39 (0.3%) 31 (0.3%) 32 (0.3%) 31 (0.3%) 32 | 392 (2.9%) 392 (2.9%) 592 (4.1%) 592 (4.1%) 595 (4.1%) 596 (4.2%) 591 (4.3%) 591 (4.3%) 4,04 (4.1%) 4, | 0.0% (1.0% 0.4%) 0.4% 0.4%) 0.3% (1.2%) 0.0% (1.0% 0.4%) 0.0% (1.0% 0.5%) 0.5% |
| TIA. n. (%) Edeman (n.)% Venous thromboembolism / Pulmonary embolism (n. (%) Pulmonary hypertension (n. (%) Implantable candioverter defiritietor, n. (%) Implantable candioverter defiritietor, n. (%) Hyperkalemia, n. (%) Conomir attreoscienosis, n. (%) Conomir attreoscienosis, n. (%) Conomir attreoscienosis, n. (%) Insertion of pacternalwers / removal of candiac lead; n. (%) CKB Stage 3-2, n. (%) CKB Stage 3-4, n. (%) Unspecified CKD; n. (%) CKB Stage 3-4, n. (%) Unspecified CKD; n. (%) Hypertensive nephropathy; n. (%) Unspecified CKD; n. (%) Gental infections; n. (%) Gental infections; n. (%) Gental infections; n. (%) Gental infections; n. (%) Obstructive sleep apnex; n. (%) Serious bacterial infections; n. (%) Pheumonia; n. (%) Distructive sleep apnex; n. (%) Pheumonia; n. (%) Distructive sleep apnex; n. (%) Serious bacterial infections; n. (%) Pheumonia; n. (%) Distructive sleep apnex; n. (%) Distructive sleep | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 129 (6.5%) 1128 (6.5%) 129 (6.5%) 128 (6.5%) 128 (6.5%) 128 (6.5%) 128 (6.5%) 128 (6.5%) 101 (6.4%) 101 (6.5%) 101 (6. | 1,354 (2.7%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,849 (1.71%) 1,149 (2.21%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 3,524 (7.1%) 1,429 (2.21%) 1,429 (2.21%) 1,429 (2.21%) 1,429 (2.21%) 1,420 (2.8%) 1,420 (2.1%) | 0.8% (1.5% 1.0%) 0.18% (1.0% 0.0%) 0.19% (1.0% 0.0%) 0.2% (2.3% 3.1%) 0.19% (1.0% 0.0%) 0.2% (2.3% 3.1%) 0.5% (1.0% 0.0%) 0.0% (1.0% 0.0%) 0.1% (1.0% 0.0%) | 394 (2.9%) 394 (2.9%) 551 (4.1%) 551 (4.1%) 557 (4.3%) 55 (0.4%) 557 (4.3%) 55 (0.4%) 55 (0.4%) 577 (4.2%) 4.578 (3.5%) 39 (0.3%) 1031 (7.5%) 39 (0.3%) 1104 (6.6%) 1197 (8.8%) 273 (19.9%) 273 (19.9%) 273 (19.9%) 273 (19.9%) 238 (17.2%) 458 (3.4%) 658 (5.0%) 2387 (17.2%) 144 (12.1%) 3.657 (2.6.9%) 474 (3.5%) 147 (8.6.9%) 148 (8.6.%) 149 (8.6.%) 149 (8.6.%) 149 (8.6.%) 149 (8.6.%) 149 (8.6.%) 149 (8.6.%) 149 (8.6.%) 130 (4.1%) | 392 (29%) 392 (29%) 592 (41%) 552 (41%) 556 (42%) 552 (41%) 56 (42%) 50 (43%) 579 (43%) 434 (42.5%) 434 (42.5%) 441 (23%) 442 (43%) 442 (43%) 442 (43%) 443 (43%) 443 (43%) 444 (43%) 445 (45%) 447 | 0.0% (1.4%, 0.4%) 0.0% (1.5%, 0.5%) |
| TIA. in (%) Edeman (1%) Venous thromboembolism / Pulmonary embolism in (%) Pulmonary hypertension in (%) Implantable cardioverter deficilitator, n (%) Hypertelemia (%) Dononary atherosclerosis, in (%) Dononary atherosclerosis, in (%) Dononary atherosclerosis, in (%) Dononary atherosclerosis, in (%) Dononary atherosclerosis, in (%) Imsertion of paccemakens / removal of cardiac lead in (%) CXIS Stage 3-12, n (%) CXIS Stage 3-12, n (%) CXIS Stage 3-14, n (%) Unspecified CXID, n (%) Acute kidney hypory in (%) Hypertensive nephropathy; n (%) Hypertensive nephropathy; n (%) Unsay fact inflow, and uninary stone); n (%) Gental infections; n (%) Gental infections; n (%) Obstructive sleep apneas; n (%) Serious bacterious infections; n (%) Preumoniar n (%) Data (%) DASHMASID, n (%) Preumoniar n (%) Destroctive sleep apneas; n (%) Destroctive sleep apneas; n (%) Destroctive sleep apneas; n (%) Destroctive n (%) Bland destroctive n (%) Gast top or inflation of submoniar n (%) Concombant use or inflation of submoniar n (%) Concombant use or inflation of submoniar n (%) Past use of Mathory, who in submon in (%) Concombant use or inflation of submoniars; n (%) Past use of the submoniar n (%) Past use of submoniar n (%) | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 129 (3.5%) 1128 (0.5%) 129 (4.6%) 128 (0.5%) 128 (0.5%) 128 (0.5%) 128 (0.5%) 128 (0.5%) 101 (0.4%) 101 (6.4%) 101 (6.5%) 101 (6. | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 185 (0.4%) 185 (0.4%) 185 (0.4%) 185 (0.4%) 185 (1.2%) 18.49 (12.71%) 17 (0.2%) 18.49 (1.2%) 18.49 (1.2%) 18.59 (1.2%) 18.50 (1.2%) | 0.8% (1.5% 1.0%) 0.18% (1.0% 0.0%) 0.19% (1.0% 0.0%) | 394 (2.9%) 394 (2.9%) 2246 f16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (3.5.9%) 18 (0.3%) 19 (0.3%) 19 (0.3%) 19 (0.3%) 19 (0.3%) 19 (0.3%) 1164 (6.5%) 1164 (6.5%) 1167 (6.5%) 1164 (6.5%) 1164 (6.5%) 1164 (6.5%) 1164 (6.5%) 1164 (1.1%) 1165 (1.1%) 1166 (1.1%) 1166 (1. | 392 (29%) 392 (29%) 592 (41%) 566 (42%) 592 (41%) 566 (42%) 591 (43%) 591 (43%) 591 (43%) 484 (42.65%) 24 (23.65%) 25 (23.65%) | 0.0% (1.0% 0.4%) 0.0% (1.0% 0.4%) 0.0% (1.0% 0.5%) 0.0% (1.0% 0.0%) |
| TIA. n. (%) Edeman (n.)% Venous thromboembolism / Pulmonary embolism; n. (%) Palmonary hypertension; n. (%) Implicitable cardioverter deficitator, n. (%) Hypertelemia, n. (%) Dononary afferencelemia, n. (%) Dononary afferencelemia, n. (%) Dononary afferencelemia, n. (%) Dononary afferencelemia, n. (%) Dononary afferencelemia, n. (%) Insertion of pacemilleris, n. (%) Insertion of pacemilleris, n. (%) Insertion of pacemilleris, n. (%) Insertion of pacemilleris, n. (%) Insertion of pacemilleris, n. (%) CXIS Stage 3-12, n. (%) CXIS Stage 3-12, n. (%) CXIS Stage 3-13, n. (%) Insertion of pacemilleris, n. (%) Gental infections; n. (%) Unsertionary of the n. (%) COPP. n. (%) Asthmar n. (%) Obstructive sleeps apneas, n. (%) Serious bacteris n. (%) Pheumonia; n. (%) Dementia, n. (%) Infections; n. (%) Dementia, n. (%) Infections; n. (%) Covicinations of mittalion of Metformix n. (%) Covicinations of mittalion of sulfornylures, n. (%) Past use of Methorium n. (%) Past use of Installation of Justices, n. (%) Past use of Installation of Installation of Justices, n. (%) Past use of Installation of Justices, n. (%) Past use of Sol. T. 2s. n. (%) | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 129 (4.5%) 128 (0.5%) 140 (3.6%) 128 (0.5%) 140 (3.6%) 128 (0.5%) 140 (3.6%) 101 (0.4%) 127 (0.5%) 101 (0.4%) 101 (0.5%) 101 (0.5 | 1,354 (2.7%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,958 (1.0%) 1,958 | 0.8% (0.5% 1.0%) 0.8% (1.1% 0.0%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 0.1% (0.0% 0.2%) 1.1% (1.2% 0.2%) 1.1% (1.2% 0.2%) 1.1% (1.2% 0.2%) 1.2% ( | 394 (29%) 394 (29%) 2246 f16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (35.5%) 39 (0.3%) 39 (0.3%) 39 (0.3%) 31 (0.5%) 39 (0.3%) 31 (0.5%) 39 (0.3%) 31 (0.5%) 39 (0.3%) 31 (0.5%) 31 (0.5%) 32 (0.3%) 33 (0.5%) 34 (0.5%) | 392 (29%) 392 (29%) 392 (29%) 552 (4.1%) 556 (4.2%) 552 (4.1%) 556 (4.2%) 550 (4.3%) 550 (4.3%) 550 (4.3%) 550 (4.3%) 4.844 (3.5.5%) 4.844 (3.5.5%) 4.10 (2.7.4%) 4.20 (3.5.5%) 4.20 (3.5%) 4.20 (3.5% | 0.0% (1.04%, 0.4%) 0.0% (1.05%, 0.5%) 0.3% (1.05%, 0.5%) 0.0% (1.05%, 0.05%) 0.0% (1.05%, 0.05%) 0.05% (1 |
| TIA. n. (%) Edemse, n. (%) Venous thromboembolism / Pulmonary embolism; n. (%) Pulmonary hymerisasion; n. (%) Implantable cardioverter deficitient; n. (%) Hyperkalemist; n. (%) Coronary atherosclerosis; n. (%) Coronary atherosclerosis; n. (%) Coronary atherosclerosis; n. (%) Coronary atherosclerosis; n. (%) Lesebrovascular procedure; n. (%) Insperition of peremitkers; / removal of cardiac lead; n. (%) CXD Staps 3-4; n. (%) Unspecified CXD; n. (%) Acute kidney hijver, n. (%) Hypertensive nephropathy; n. (%) Unspecified CXD; n. (%) Gental infections; n. (%) Gental infections; n. (%) Gental infections; n. (%) COPD; n. (%) Asthmar, n. (%) Othat nuclev sleep anome; n. (%) Presumonias, n. (%) Presumonias, n. (%) Presumonias, n. (%) Presumonias, n. (%) Presumonias, n. (%) Osteoporosis; n. (%) Osteoporosis; n. (%) Osteoporosis; n. (%) Osteoporosis; n. (%) Demensit; n. (%) De | 982 (3.5%) 46.21 (6.5%) 1111 (3.9%) 1292 (4.6%) 128 (0.5%) 1407 (5.0%) 128 (0.5%) 1407 (5.0%) 10186 (3.6.0%) 1010 | 1,354 (2.7%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,958 (4.0%) 1,958 (1.0%) 1,958 | 0.8% (1.5% 1.0%) 0.1% (1.0% 0.0%) 0.0% (1.0% 0.0%) 0.0% ( | 394 (29%) 394 (29%) 2246 f16.5%) 551 (4.1%) 551 (4.1%) 5579 (4.3%) 55 (0.4%) 5577 (4.2%) 4.578 (35.5%) 39 (0.3%) 310 (3.3%) 313 (6.2%) 313 (6.2 | 392 (29%) 392 (29%) 392 (29%) 552 (4.1%) 556 (4.2%) 552 (4.1%) 550 (4.3%) 550 (4.3%) 550 (4.3%) 550 (4.3%) 484 (4.25.5%) 41 (2.25.5%) 42 (2.3%) 43 (2.3%) 43 | 0.0% (1.04%, 0.4%) 0.0% (1.05%, 0.5%) 0.0% (1.05%, 0.05%) |
| TIA.n (%) Edems, n (%) Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable cardioverter defletifish; n (%) Implantable cardioverter defletifish; n (%) Loronary atherosclerosis; n (%) Coronary atherosclerosis; n (%) Coronary atherosclerosis; n (%) Coronary atherosclerosis; n (%) Loronary atherosclerosis; n (%) Coronary atheroscleros; n (%) Gorotal infections; n (%) Unspecified CKD; n (%) Gental infections; n (%) Gental infections; n (%) Unitary tract infections; n (%) Gental infections; n (%) Coronary atherosclerosis; n (%) Obstructive sleep apone; n (%) Presumonis; n (%) Distructive sleep apone; n (%) Presumonis; n (%) Distructive sleep apone; n (%) Presumonis; n (%) Osteoporosis; n (%) Osteoporosis; n (%) Osteoporosis; n (%) Demensit; n (%) Demen | 982 (3.5%) 4621 (8.5%) 1111 (3.9%) 129 (3.5%) 129 (3.5%) 129 (3.5%) 129 (3.5%) 129 (3.5%) 10.186 (3.6.0%) 39 (0.1%) 10.186 (3.6.0%) 39 (0.1%) 10.10 (4.9%) 2511 (8.9%) 2511 (8.9%) 2511 (8.9%) 2511 (8.9%) 2511 (8.9%) 2511 (8.9%) 34 (3.3%) 1374 (4.9%) 353 (2.1%) 353 (2.1%) 353 (2.1%) 353 (2.1%) 354 (2.0%) 354 (2.0%) 355 (2.2%) 357 (2.3%) | 1,354 (2.7%) 8,407 (16.9%) 1,998 (4.0%) 1,998 (4.0%) 1,958 (4.0%) 1,95 | 0.8% (1.5% 1.0%) 0.8% (1.1% 0.0%) 0.1% (1.0 0.0%) 0.2%) 0.2% (1.2%) 0.3% (1.0 0.0%) 0.3% ( | 394 (2.9%) 394 (2.9%) 551 (4.1%) 551 (4.1%) 551 (4.1%) 557 (4.3%) 55 (0.4%) 577 (4.2%) 4.878 (35.5%) 18 (0.1%) 18 (0.1%) 18 (0.1%) 19 (1.0%) 10 (1.0%) 11 (1.0%) | 392 (29%) 392 (29%) 592 (41%) 552 (41%) 556 (42%) 552 (41%) 56 (42%) 579 (43%) 570 (43%) 579 (43%) 4,844 (35.6%) 24 (0.2%) 4,844 (35.6%) 24 (0.2%) 4,844 (35.6%) 1152 (8.5%) 1367 (22.5%) 1367 (22.5%) 1368 (1.5%) 1370 (22.5%) 1370 (22.5%) 1383 (1.3%) 1384 (1.3%) 1384 (1.3%) 1384 (1.3%) 1384 (1.3%) 1385 (1.2%) 1386 (1.2 | 0.0% (1.0.4%, 0.4%) 0.0% (1.0.5%, 0.5%) |

| Digoxin / Digitoxin; n (%) | 516 (1.8%) | 464 (0.9%) | 0.9% (0.7%, 1.1%) | 198 (1.5%) | 177 (1 20/) | 0.2% (-0.1% 0.4%) |
|---|---|---|---|---|---|---|
| Loop diuretics; n (%) | 6,593 (23.3%) | 12,730 (25.5%) | -2.2% (-2.9%, -1.6%) | 3,224 (23.7%) | 177 (1.3%)<br>3,214 (23.6%) | 0.1% (-0.9%, 1.1%) |
| Other diuretics; n (%)<br>Intravenous diuretics; n (%) | 2,393 (8.5%)<br>514 (1.8%) | 5,875 (11.8%)<br>910 (1.8%) | -3.3% (-3.8%, -2.9%)<br>-0.0% (-0.2%, 0.2%) | 1,297 (9.5%)<br>217 (1.6%) | 1,295 (9.5%)<br>216 (1.6%) | 0.0% (-0.7%, 0.7%) |
| Nitrates; n (%) | 2,841 (10.0%) | 4,979 (10.0%) | 0.1% (-0.4%, 0.5%) | 1,332 (9.8%) | 1,314 (9.7%) | 0.1% (-0.6%, 0.8%) |
| Anti-arrhythmics; n (%)<br>Statins; n (%) | 933 (3.3%)<br>23,398 (82.7%) | 1,885 (3.8%)<br>40,844 (81.9%) | -0.5% (-0.8%, -0.2%)<br>0.8% (0.2%, 1.4%) | 477 (3.5%)<br>11,337 (83.3%) | 450 (3.3%)<br>11,337 (83.3%) | 0.2% (-0.2%, 0.6%)<br>0.0% (-0.9%, 0.9%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 3,633 (12.8%) | 7,683 (15.4%) | -2.6% (-3.1%, -2.1%) | 1,951 (14.3%) | 1,967 (14.5%) | -0.1% (-1.0%, 0.7%) |
| Antiplatelet medications; n (%) Oral anticoagulants; n (%) | 4,106 (14.5%)<br>3,966 (14.0%) | 6,992 (14.0%)<br>7,548 (15.1%) | 0.5% (-0.0%, 1.0%)<br>-1.1% (-1.6%, -0.6%) | 1,906 (14.0%)<br>1,985 (14.6%) | 1,808 (13.3%)<br>1,925 (14.2%) | 0.7% (-0.1%, 1.5%)<br>0.4% (-0.4%, 1.3%) |
| COPD/Asthma medications; n (%) | 9,683 (34.2%) | 19,893 (39.9%) | -5.7% (-6.4%, -5.0%) | 4,983 (36.6%) | 5,022 (36.9%) | -0.3% (-1.4%, 0.9%) |
| NSAIDS; n (%) Oral corticosteroids; n (%) | 8,230 (29.1%)<br>5,976 (21.1%) | 16,906 (33.9%)<br>14,125 (28.3%) | -4.8% (-5.5%, -4.1%)<br>-7.2% (-7.8%, -6.6%) | 4,321 (31.8%)<br>3,202 (23.5%) | 4,261 (31.3%)<br>3,152 (23.2%) | 0.4% (-0.7%, 1.6%)<br>0.4% (-0.6%, 1.4%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) Opioids; n (%) | 1,379 (4.9%)<br>8,809 (31.2%) | 1,676 (3.4%)<br>17,708 (35.5%) | 1.5% (1.2%, 1.8%)<br>-4.4% (-5.1%, -3.7%) | 542 (4.0%)<br>4,334 (31.9%) | 536 (3.9%)<br>4,400 (32.3%) | 0.0% (-0.4%, 0.5%) |
| Anti-depressants; n (%) | 9,311 (32.9%) | 21,362 (42.9%) | -9.9% (-10.6%, -9.2%) | 4,950 (36.4%) | 4,959 (36.5%) | -0.1% (-1.2%, 1.1%) |
| Antipsychotics; n (%) Anxiolytics / hypnotics, benzos; n (%) | 1,193 (4.2%)<br>5,399 (19.1%) | 2,421 (4.9%)<br>11.876 (23.8%) | -0.6% (-0.9%, -0.3%)<br>-4.7% (-5.3%, -4.1%) | 590 (4.3%)<br>2,733 (20.1%) | 587 (4.3%)<br>2,694 (19.8%) | 0.0% (-0.5%, 0.5%)<br>0.3% (-0.7%, 1.2%) |
| Dementia medications; n (%) | 1,396 (4.9%) | 819 (1.6%) | 3.3% (3.0%, 3.6%) | 433 (3.2%) | 426 (3.1%) | 0.1% (-0.4%, 0.5%) |
| Urinary tract infections antibiotics; n (%) Laxatives; n (%) | 13,197 (46.7%)<br>1,053 (3.7%) | 24,575 (49.3%)<br>1,870 (3.8%) | -2.6% (-3.4%, -1.9%)<br>-0.0% (-0.3%, 0.3%) | 6,436 (47.3%)<br>454 (3.3%) | 6,456 (47.5%)<br>452 (3.3%) | -0.1% (-1.3%, 1.0%)<br>0.0% (-0.4%, 0.4%) |
| Number of distinct medications | | | 0.01/.0.00.0.70 | 15.01 (6.61) | | 0.04/ 0.00 0.00 |
| mean (sd)median [IQR] | 14.66 (6.48)<br>14.00 [10.00, 18.00] | 15.47 (6.76)<br>15.00 [11.00, 19.00] | -0.81 (-0.90, -0.71)<br>-(-, -) | 14.00 [10.00, 19.00] | 15.05 (6.46)<br>14.00 [10.00, 19.00] | -0.04 (-0.20, 0.11)<br>- (-, -) |
| min, max Number of office visits | 1.00, 57.00 | 1.00, 62.00 | - (-, -) | 1.00, 57.00 | 1.00, 59.00 | - (-, -) |
| mean (sd) | 9.88 (6.83) | 10.81 (7.12) | -0.93 (-1.03, -0.82) | 10.17 (7.01) | 10.22 (6.63) | -0.05 (-0.21, 0.11) |
| median [IQR] | 8.00 [5.00, 13.00]<br>0.00, 99.00 | 9.00 [6.00, 14.00]<br>0.00, 93.00 | - (-, -)<br>- (-, -) | 9.00 [5.00, 14.00]<br>0.00, 93.00 | 9.00 [6.00, 13.00]<br>0.00, 84.00 | - (-, -)<br>- (-, -) |
| Number of endocrinologist visits | | | | | | |
| mean (sd)median [IQR] | 0.30 (1.20)<br>0.00 [0.00, 0.00] | 0.37 (1.24)<br>0.00 [0.00, 0.00] | -0.07 (-0.09, -0.05)<br>-(-, -) | 0.33 (1.34)<br>0.00 [0.00, 0.00] | 0.34 (1.08)<br>0.00 [0.00, 0.00] | -0.01 (-0.04, 0.02)<br>- (-, -) |
| min, max | 0.00, 34.00 | 0.00, 40.00 | - (-, -) | 0.00, 34.00 | 0.00, 23.00 | - (-, -) |
| Number of cardiologist visitsmean (sd) | 2.24 (3.96) | 2.23 (3.87) | 0.01 (-0.05, 0.06) | 216 (3.95) | 2.12 (3.76) | 0.04 (-0.05, 0.13) |
| median [IQR] | 1.00 [0.00, 3.00]<br>0.00, 78.00 | 1.00 [0.00, 3.00]<br>0.00, 85.00 | -(-, -)<br>-(-, -) | 1.00 [0.00, 3.00]<br>0.00, 78.00 | 1.00 [0.00, 3.00]<br>0.00, 83.00 | - (-, -)<br>- (-, -) |
| Number of internal/family medicine visits | | | | | | |
| mean (sd)median [IQR] | 9.21 (9.36)<br>7.00 [4.00, 12.00] | 8.05 (8.56)<br>6.00 [3.00, 10.00] | 116 (1.03, 1.29) | 8.63 (9.11)<br>6.00 (3.00, 11.00) | 8.72 (9.25)<br>6.00 [3.00, 11.00] | -0.09 (-0.31, 0.13)<br>- (-, -) |
| min, max | 0.00,189.00 | 0.00, 219.00 | - (-, -) | 0.00, 154.00 | 0.00, 219.00 | - (-, -)<br>- (-, -) |
| Number of electrocardiograms (ECG/EKG)mean (sd) | 1.30 (1.90) | 1.22 (1.75) | 0.08 (0.05, 0.11) | 123 (1.87) | 1.19 (1.72) | 0.04 (-0.00, 0.08) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max<br>Number of echocardiograms | 0.00, 30.00 | 0.00, 28.00 | -(-, -) | 0.00, 30.00 | 0.00, 26.00 | - (-, -) |
| mean (sd)median [IQR] | 0.38 (0.70) | 0.39 (0.71)<br>0.00 [0.00, 1.00] | -0.01 (-0.02, 0.00) | 0.37 (0.70)<br>0.00 [0.00, 1.00] | 0.37 (0.69)<br>0.00 [0.00, 1.00] | 0.01 (-0.01, 0.02) |
| min, max | 0.00, 9.00 | 0.00,10.00 | - (-, -)<br>- (-, -) | 0.00, 9.00 | 0.00, 8.00 | - (-, -)<br>- (-, -) |
| Out-of-pocket medication cost<br>mean (sd) | 518.72 (663.16) | 606.72 (828.66) | -88.00 (-98.62, -77.39) | 547.44 (736.98) | 546.68 (605.66) | 0.76 (-15.27, 16.79) |
| median [IQR] | 306.90 [125.23, 687.83] | 366.06 [146.95, 800.31] | - (-, -) | 303.46 [127.15, 718.12] | 345.01 [143.55, 743.16] | - (-, -) |
| min, max Unique brand medicines | 0.00, 19,558.36 | 0.00, 51,242.99 | - (-, -) | 0.00, 19,558.36 | 0.00, 10,678.19 | - (-, -) |
| mean (sd) | 14.90 (6.67) | 15.71 (6.95) | -0.80 (-0.90, -0.70) | 15.25 (6.80) | 15.30 (6.65) | -0.05 (-0.21, 0.11) |
| median [IQR]min, max | 14.00 [10.00, 19.00]<br>1.00, 63.00 | 15.00 [11.00, 20.00]<br>1.00, 65.00 | - (-, -)<br>- (-, -) | 14.00 [10.00, 19.00]<br>1.00, 63.00 | 14.00 [11.00, 19.00]<br>1.00, 62.00 | - (-, -)<br>- (-, -) |
| Unique generic medicinesmean (sd) | 14.55 (5.40) | | | | | |
| | | | | 15.01 (6.61) | | -0.04 (-0.20, 0.11) |
| median [IQR] | 14.66 (6.48)<br>14.00 [10.00, 18.00] | 15.47 (6.76)<br>15.00 [11.00, 19.00] | -0.81 (-0.90, -0.71)<br>-(-, -) | 15.01 (6.61)<br>14.00 [10.00, 19.00] | 15.05 (6.46)<br>14.00 [10.00, 19.00] | -0.04 (-0.20, 0.11)<br>- (-, -) |
| median [IQR]min, max | 14.00 [10.00, 18.00]<br>1.00, 57.00 | 15.00 [11.00, 19.00]<br>1.00, 62.00 | - (-, -)<br>- (-, -) | 14.00 [10.00, 19.00]<br>1.00, 57.00 | 14.00 [10.00, 19.00]<br>1.00, 59.00 | |
| _median [IQR]<br>_mir, max<br>Colonoscopy Sigmoidoscopy; n (%)<br>Flu Pneumococcal vaccine; n (%) | 14.00 [10.00, 18.00]<br>1.00, 57.00<br>2,631 (9.3%)<br>11,130 (39.4%) | 15.00 [11.00, 19.00]<br>1.00, 62.00<br>5,709 (11.5%)<br>17,564 (35.2%) | -(-, -)<br>-(-, -)<br>-2.2% (-2.6%, -1.7%)<br>4.1% (3.4%, 4.8%) | 14.00 [10.00, 19.00]<br>1.00, 57.00<br>1.391 (10.2%)<br>5,013 (36.9%) | 14.00 [10.00, 19.00]<br>1.00, 59.00<br>1.402 (10.3%)<br>4,992 (36.7%) | - (-, -)<br>- (-, -)<br>-0.1% (-0.8%, 0.6%)<br>0.2% (-1.0%, 1.3%) |
| _median [IQR]<br>_min, max<br>Colonoscopy Sigmoidoscopy; n (%) | 14.00 [10.00, 18.00]<br>1.00, 57.00<br>2,631 (9.3%) | 15.00 [11.00, 19.00]<br>1.00, 62.00<br>5,709 (11.5%) | - (-, -)<br>- (-, -)<br>-2.2% (-2.6%, -1.7%) | 14.00 [10.00, 19.00]<br>1.00, 57.00<br>1,391 (10.2%) | 14.00 [10.00, 19.00]<br>1.00, 59.00<br>1,402 (10.3%) | - (-, -)<br>- (-, -)<br>-0.1% (-0.8%, 0.6%) |
| Imedian (IQR) Imis max Colonoscopy Sigmoidoscopy; n (%) Fiu Prisumococcal vaccine; n (%) Pga smean n (%) PSA test n (%) FSA test n (%) FSA test n (%) | 14.00 [10.00, 18.00]<br>1.00, 57.00<br>2.631 (9.3%)<br>11,130 (39.4%)<br>937 (3.3%)<br>6,262 (221%)<br>2,515 (8.9%) | 15.00 [11.00, 19.00]<br>1.00, 62.00<br>5.709 (11.5%)<br>17.564 (35.2%)<br>2.659 (5.3%)<br>11.948 (24.0%)<br>2.370 (4.8%) | -(-,-)<br>-(-,-)<br>-2.2% (-2.6%,-1.7%)<br>4.1% (3.4%, 4.8%)<br>-2.0% (-2.3%, -1.7%)<br>-1.8% (-2.4%, -1.2%)<br>4.1% (3.8%, 4.5%) | 14.00 [10.00, 19.00]<br>1.00, 57.00<br>1.391 (10.2%)<br>5.013 (36.9%)<br>530 (3.9%)<br>3,133 (23.0%)<br>914 (6.7%) | 14.00 [10.00, 19.00]<br>1.00, 59.00<br>1.402 [10.3%)<br>4,992 (36.7%)<br>537 (3.9%)<br>3.112 (22.9%)<br>920 (6.8%) | - (-, -)<br>- (-, -)<br>- 0.1% (-0.8%, 0.6%)<br>0.2% (-1.0%, 1.3%)<br>- 0.1% (-0.5%, 0.4%)<br>0.2% (-0.9%, 1.2%)<br>- 0.0% (-0.6%, 0.6%) |
| Imedian (1(R)) Imit; max Colonoscopy Sigmoidoscopy; n (%) Flu Presumeroccal vaccine; n (%) Flu Presumeroccal vaccine; n (%) Pay smean; n (%) Pay smean; n (%) Pasal local thod test; n (%) Bone mineral density tests; n (%) Marmograms; n (%) | 14.00 [10.00,18.00]<br>1.00,57.00<br>2.631 (9.3%)<br>11.130 (3.9.4%)<br>937 (3.3%)<br>6.262 (221%)<br>2.515 (8.9%)<br>2.550 (9.0%)<br>6.299 (22.3%) | 15.00 (11.00, 19.00)<br>1.00, 62.00<br>5.709 (11.5%)<br>17.564 (35.2%)<br>26.59 (5.3%)<br>11.948 (24.0%)<br>2.370 (4.8%)<br>4.838 (9.7%)<br>14.310 (28.7%) | -(, -)<br>-(, -)<br>-(2% (-2.6%, -1.7%)<br>4.1% (3.4%, 4.8%)<br>-2.0% (-2.3%, -1.7%)<br>1.8% (-2.4%, -1.2%)<br>-0.7% (-1.1%, -0.3%)<br>-6.4% (-7.1%, -5.8%) | 14.00 [10.00, 19.00]<br>100, 57.00<br>1,391 [10.2%)<br>5,013 (36.9%)<br>530 (3.9%)<br>3,133 (23.0%)<br>914 (6.7%)<br>1,246 (9.2%)<br>3,420 (25.1%) | 14.00 (10.00, 19.00)<br>1.402 (10.3%)<br>1.492 (36.7%)<br>537 (3.9%)<br>3.112 (22.9%)<br>920 (6.8%)<br>1.240 (9.1%)<br>3.454 (25.4%) | -(, -)<br>-(, -)<br>-0.1% (-0.8%, 0.6%)<br>-0.2% (-1.0%, 1.3%)<br>-0.1% (-0.5%, 0.4%)<br>-0.2% (-0.5%, 0.6%)<br>-0.0% (-0.6%, 0.5%)<br>-0.0% (-0.6%, 0.7%)<br>-0.2% (-1.3%, 0.8%) |
| _median [LQR] _min; max Colomoscopy Sigmoidoscopy; n (%) Flu Preumcoccal vaccine; n (%) Flu Preumcoccal vaccine; n (%) Flu Statis, n (%) PSA test, n (%) Feat occur th blood test, n (%) Bone mineral density tests; n (%) Mammograms; n (%) Mammograms; n (%) Telemedicine; n (%) | 14.00 [10.00, 18.00]<br>1.00, 57.00<br>2,631 (9.3%)<br>11,130 (39.4%)<br>937 (3.3%)<br>6.262 (22.1%)<br>2,515 (8.9%)<br>2,550 (9.0%) | 15.00 [11.00, 19.00]<br>1.00, 62.00<br>5.709 (11.5%)<br>17.564 (35.2%)<br>2.659 (5.3%)<br>11.948 (24.0%)<br>2.370 (4.8%)<br>4.838 (9.7%) | -(-, -)<br>-(-, -)<br>-(-, -)<br>-2.2% (-2.6%, -1.7%)<br>4.1% (3.4%, 4.8%)<br>-2.0% (-2.3%, -1.7%)<br>-1.8% (-2.4%, -1.2%)<br>4.1% (3.8%, 4.5%)<br>-0.7% (-1.1%, -0.3%) | 14.00 [10.00, 19.00]<br>1.00, 57.00<br>1.391 (10.2%)<br>5,013 (36.9%)<br>530 (3.9%)<br>3,133 (23.0%)<br>914 (6.7%)<br>1,246 (9.2%) | 14.00 [10.00, 19.00]<br>100, 59.00<br>1,402 (10.3%)<br>4,992 (36.7%)<br>537 (3.9%)<br>3,112 (22.9%)<br>920 (6.8%)<br>1,240 (9.1%) | - (-, -)<br>- (-, -)<br>- 0.1% (-0.8%, 0.6%)<br>0.2% (-1.0%, 1.3%)<br>-0.1% (-0.5%, 0.4%)<br>0.2% (-0.9%, 1.2%)<br>-0.0% (-0.6%, 0.6%)<br>0.0% (-0.6%, 0.7%) |
| Imedian (IQR) Imit max Colonoscopy Sigmoldoscopy, n (%) Flu Presumcoccal vaccine; n (%) Pag anmean (%) PSA test n (%) FSA test n (%) FSA test n (%) Bone mineral dentity tests; n (%) Marmongams; n (%) Telemedicine; n (%) HBAI c tests Iman (s) | 14.00 [10.00, 18.00]<br>100, 57.00<br>2631 [9.3%]<br>11.130 (39.4%)<br>937 (3.3%)<br>6.262 (22.1%)<br>2515 (8.9%)<br>2550 (9.0%)<br>4,742 (16.8%)<br>245 (1.30) | 15.00 (11.00, 19.00) 1.00, 62.00 5.709 (11.5%) 17.564 (15.2%) 17.564 (15.2%) 18.488 (24.0%) 2.370 (4.8%) 4.838 (9.7%) 12.448 (25.0%) 12.448 (25.0%) | -(, -)<br>-(-, -)<br>-(2.2% (-2.6%, -1.7%)<br>-4.1% (3.4%, 4.8%)<br>-2.0% (-2.3%, -1.7%)<br>-1.8% (-2.4%, -1.2%)<br>-4.1% (3.8%, 4.5%)<br>-0.7% (-1.1%, -0.3%)<br>-6.4% (-7.1%, -5.8%)<br>-8.2% (-8.8%, -7.6%)<br>0.09 (0.07, 0.11) | 14.00 [10.00, 19.00] 1.00, 57.00 1.391 [10.2%) 5.013 (36.9%) 5.013 (3.9%) 31.33 (23.0%) 914 (6.7%) 1.246 (9.2%) 3.070 (22.6%) 2.45 (1.28) | 14-00 [10.00 19.00] 10.0, 59.00 1.402 [10.3%) 4.992 [36.7%) 5.37 [3.9%] 3.112 [22.9%) 9.20 [6.8%] 1.240 [9.1%] 3.454 [25.4%) 3.47 [22.1%) 2.47 (1.36) | (-, -)<br>-(1, -)<br>-(1)% (-0.8%, 0.6%)<br>0.2% (-1.0%, 1.3%)<br>-0.1% (-0.5%, 0.4%)<br>-0.2% (-0.9%, 1.2%)<br>-0.0% (-0.6%, 0.6%)<br>-0.0% (-0.6%, 0.7%)<br>-0.2% (-1.9%, 0.8%)<br>-0.6% (-1.6%, 0.4%)<br>-0.02 (-0.05, 0.02) |
| Imedian (1(R)) Imit; max Coloroscopy Sigmoidoscopy; n (%) Flu Pheumococcal vaccine n (%) Pap amean n (%) Pap amean n (%) Pas tent n (%) Pas t | 14.00 [10.00, 18.00]<br>1.00, 57.00<br>2.631 [9.3%]<br>11.130 (39.4%)<br>9.37 (3.3%)<br>6.262 (22.1%)<br>2.515 (8.9%)<br>6.299 (22.3%)<br>4,742 (16.8%) | 15.00 (11.00, 19.00)<br>1.00, 62.00<br>5.709 (11.5%)<br>17.564 (15.7%)<br>2.659 (5.3%)<br>11.948 (24.0%)<br>2.370 (4.8%)<br>4.838 (9.7%)<br>12.448 (25.0%) | (-, -)<br>-(-, -)<br>-22% (-2.6%, -1.7%)<br>-4.1% (.3.4%, -4.8%)<br>-2.0% (-2.3%, -1.7%)<br>-1.8% (-2.4%, -1.2%)<br>-4.1% (.3.9%, -4.5%)<br>-0.7% (-1.1%, -0.3%)<br>-6.4% (-7.1%, -5.8%)<br>-8.2% (-8.8%, -7.6%) | 14.00 (10.00, 19.00)<br>1.00, 57.00<br>1.391 (10.2%)<br>5.013 (36.9%)<br>5.30 (3.9%)<br>3.133 (23.0%)<br>914 (6.7%)<br>1.246 (9.2%)<br>3.470 (25.1%)<br>3.070 (22.6%) | 14.00 (10.00, 19.00)<br>1.402 (10.3%)<br>1.402 (10.3%)<br>537 (3.9%)<br>537 (3.9%)<br>3.112 (2.2.9%)<br>920 (6.5%)<br>1,240 (9.1%)<br>3,454 (25.4%)<br>3,447 (23.1%) | -(-, -)<br>-(-, -)<br>-(-, -)<br>-(-) -(-) -(-) -(-) -(-)<br>-(-) -(-) -(-) -(-) -(-)<br>-(-) -(-) -(-) -(-) -(-)<br>-(-) -(-) -(-) -(-) -(-) -(-)<br>-(-) -(-) -(-) -(-) -(-) -(-)<br>-(-) -(-) -(-) -(-) -(-) -(-) -(-)<br>-(-) |
| Imedian (10R) min, max Colonaccopy, Sigmoidescopy, n (%) Bith Presumboscopi, n (%) Play smear, n (%) Teal could blood test, n (%) Bone mineral donnity tests, n (%) Marmingamen, n (%) Telemedicine n (%) HibALE tests Limban (td) Limba (max Lijid panels | 14.00 (10.00. 18.00] 100. 57.00 26.31 (3.3%) 11.130 (3.3%) 11.130 (3.3%) 137 (3.3%) 25.51 (3.5%) 25.51 (3.0%) 25.51 (3.0%) 25.51 (3.0%) 4,742 (3.6.5%) 245 (13.0%) 245 (13.0%) 245 (13.0%) 245 (13.0%) 000 (10.0%) | 15.00 (11.00, 15.00) 10.0 6.200 5.709 (11.5%) 17.564 (15.2%) 2.659 (5.3%) 11.946 (24.0%) 2.470 (4.8%) 4.380 (6.7%) 14.310 (28.7%) 12.446 (5.50%) 2.36 (13.2%) 2.36 (13.2%) 2.36 (13.2%) 0.00, 37.00 | 16.3<br>17.3<br>17.5 | 14.00 [10.00, 19.00] 1.00, 57.00 1.391 [10.2%] 5.013 [36.9%] 5.013 [36.9%] 5.013 [32.0%] 911 (6.7%) 1.246 [9.2%] 3.420 (25.1%) 3.420 (25.1%) 3.420 (25.1%) 2.45 (1.28) 2.00 [2.00, 3.00] 0.00, 9.00 | 14.00 [10.00 19.00] 10.00 50.00 14.02 (10.3%) 4.992 (16.7%) 5.37 (3.9%) 3.112 (22.9%) 9.20 (6.6.5%) 1.240 (19.1%) 3.454 (22.4.5%) 3.147 (22.1.5%) 2.47 (13.6) 2.40 (13.6) 0.00 , 37.00 | 1(-, 1) -0.1% (-0.8%, 0.6%) -0.2% (-1.0%, 1.3%) -0.1% (-0.5%, 0.4%) -0.2% (-0.5%, 0.6%) -0.2% (-0.6%, 0.6%) -0.0% (-0.6%, 0.6%) -0.2% (-1.3%, 0.8%) -0.2% (-1.3%, 0.8%) -0.2% (-1.3%, 0.8%) -0.2% (-1.3%, 0.4%) -0.02 (-0.05, 0.02) -1, -1 |
| Imedian (IQR) Imis max Colonoscopy Sigmoldoscopy, n (%) Flu Phatumococcal vaccine; n (%) Plu Shatumococcal vaccine; n (%) PSA test n (%) PSA test n (%) PSA test n (%) Bone mineral density tests; n (%) Mammograms; (%) Telemaclicine; n (%) HbAIc testsmedian (IQR)middian (IQR)mid max | 14.00 (10.00, 18.00)<br>100, 57.00<br>26.31 (9.3%)<br>11.130 (39.4%)<br>9377 (3.3%)<br>6.262 (22.1%)<br>2.515 (8.9 0.9%)<br>6.299 (22.3%)<br>4.742 (16.8%)<br>2.45 (1.30)<br>2.00 (2.00, 3.00) | 15.00 (11.00, 19.00) 1.00, 62.00 5.709 (11.5%) 17564 (15.2%) 2.559 (3.3%) 11.948 (24.0%) 2.270 (4.8%) 4.339 (8.7%) 14.330 (28.7%) 12.448 (25.5%) 12.448 (25.5%) 2.36 (13.2) 2.301 (13.2) | 1-(-, 1<br>-(-, 2)<br>-(-2)% (-2.6%, -1.7%)<br>-(-1.9%, -1.7%) | 14.00 [10.00, 19.00] 1.00, 57.00 1.291 [10.2%] 5.013 (36.9%) 5.013 (36.9%) 3.133 (72.0%) 914 (6.7%) 1.246 (9.2%) 3.420 (25.1%) 3.420 (25.1%) 3.420 (25.1%) 3.420 (25.1%) 3.420 (20.0%) | 14.00 [10.00, 19.00] 10.0, 59.00 14.02 (10.3%) 4.992 (26.7%) 5.77 (3.9%) 5.77 (3.9%) 12.00 (6.5%) 12.00 (3.9%) 12.00 (3.9%) 13.47 (23.1%) 2.47 (13.6%) 2.47 (13.6%) 2.47 (13.6%) | 1(-, 1)<br>-0.1% (-0.8%, 0.6%)<br>0.2% (-1.0%, 1.3%)<br>-0.1% (-0.5%, 0.4%)<br>0.2% (-0.9%, 1.2%)<br>0.0% (-0.6%, 0.6%)<br>0.0% (-0.6%, 0.7%)<br>-0.2% (-1.3%, 0.8%)<br>-0.6% (-1.6%, 0.4%)<br>-0.02 (-0.05, 0.02)<br>-1; -1 |
| Imedian (IQR) Imis, mas; Colonescopy, Sigmoldoscopy, n (%) Flu Presumozoccal vaccine; n (%) Plu Presumozoccal vaccine; n (%) Plus State th (%) PSA test n (%) PSA test n (%) PSA test n (%) PSA test n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HABAIC tests Imean (sd) Imedian (IQR) Init max Lisid panels Imean (sd) Imean | 14:00 [10:00.18:00] 1:00,57:00 2:631 (9.3%) 11:130 [39.4%) 937 (3.3%) 6,262 (221%) 2:5516 (9.9%) 6,299 (223%) 4,742 (16.8%) 2:45 (1.30) 2:00 [2:00.300] 0:00,000 | 15.00 (11.00, 19.00) 10.0 62.00 5.709 (11.5%) 17.564 (15.2%) 26.59 (5.3%) 11.948 (24.0%) 2.370 (4.8%) 4.831 (9.7%) 14.310 (28.7%) 12.448 (25.0%) 2.36 (1.12 2.00 (1.00, 3.00) 0.00, 3.700 | 1-1-3<br>1-5-3<br>2.2% (2.6% - 1.7%)<br>4.1% (3.4% - 4.8%)<br>2.0% (2.3% - 1.7%)<br>1.8% (2.4% - 1.7%)<br>1.8% (2.4% - 1.7%)<br>0.7% (1.1% - 0.3%)<br>6.4% (7.1% - 5.8%)<br>8.2% (3.8% - 7.5%)<br>0.09 (0.07, 0.11)<br>1-1-3<br>1-3<br>1-3<br>1-3<br>1-3<br>1-3<br>1-3<br>1 | 14.00 [10.00, 19.00] 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%] 13.91 [10 | 14.00 [10.00, 19.00] 10.00, 59.00 1.402 (10.3%) 4.592 (13.67%) 5.77 (1.3%) 3.112 (22.9%) 9.20 (16.8%) 1.240 (9.1%) 3.454 (25.4%) 3.447 (23.1%) 2.47 (13.6) 2.00 (12.00, 3.00) 0.00, 37.00 | -(-, -) -(-, - |
| Imedian (IQR) Imit; max Colonoscopy, Sigmoldoscopy; n (%) Flu Presumozoccal vaccine; n (%) Flu Presumozoccal vaccine; n (%) PSA test n (%) FSA test n (%) FS | 14.00 (10.00.18.00] 1.00.57.00 2.631 (9.3%) 1.130 (3.3%) 1.130 (3.34%) 937 (3.3%) 6.262 (2.21%) 2.5516 (9.9%) 6.269 (2.21%) 2.550 (9.9%) 6.299 (2.23%) 4,742 (16.8%) 2.45 (1.30) 1.00.10.00 1.74 (1.21) 2.00 (1.00. 2.00) 0.00, 2.00 3.40 (3.50) | 15.00 [1.00, 19.00] 10.0 6.200 5.709 (11.5%) 17.564 (13.5.2%) 26.595 (2.3%) 11.948 (2.40%) 2.370 (4.8%) 4.838 (9.7%) 4.330 (8.7%) 12.448 (25.0%) 2.36 (1.32 2.001 10.0 3.001 0.00, 37.00 1.69 (1.19) 2.001 (1.00, 2.00) 0.00, 36.00 | 16.3 22% (2.6%, 1.7%) 1.53 (2.6%, 1.7%) 1.53 (2.6%, 1.7%) 1.54 (3.4%, 4.8%) 2.0% (2.3%, 1.7%) 1.8% (2.4%, 1.2%) 1.8% (2.4%, 1.2%) 1.8% (2.4%, 1.2%) 1.8% (3.6%, 4.5%) 0.7% (1.1%, 0.3%) 6.4% (7.1%, 5.6%) 8.2% (3.8%, 7.5%) 1.6% (3.8%, 7.5%) 1.6% (3.6%, 4.7%) 1.6% (3. | 14.00 [10.00, 19.00] 1.00, 57.00 1.391 [10.2%) 5.013 [36.9%) 5.013 [36.9%) 5.013 [36.9%) 3.133 [23.0%) 914 [6.7%) 1.246 [9.2%) 3.420 (25.1%) 3.070 (22.6%) 2.45 (1.28) 2.00 [2.00, 3.00] 0.00, 9.00 172 (1.18) 2.00 [10.0, 2.00] 0.00, 2.00 3.30 (2.52) | 14.00 [10.00. 19.00] 10.00. 59.00 14.02 (10.3%) 4.992 (36.7%) 5.77 (3.9%) 3.112 (22.9%) 12.40 (21.1%) 12.40 (21.1%) 12.41 (21.1%) 12.47 (13.1%) 12.47 (13.1%) 12.47 (13.1%) 17.3 (1.22) 17.3 (1.22) 17.3 (1.22) 17.3 (1.22) 17.3 (1.22) 17.3 (1.23) 17.3 (1.24) 17.3 (1.25) 17.3 (1.25) 17.3 (1.25) 17.3 (1.26) 17.3 (1.26) 17.3 (1.26) 17.3 (1.27) 17.3 (1.28) | -(-, -)<br>-(-, -)<br>-(-) -(-) -(-) -(-) -(-)<br>-(-) -(-) -(-) -(-) -(-) -(-) -(-)<br>-(-) |
| Imedian (IQRI Imris max Colonoscopy Sigmoidoscopy n (%) Flu Pretermococcal vacciner n (%) Flu Pretermococcal vacciner n (%) Flos Ates in (%) FSA test n (%) | 14.00 (10.00, 18.00] 100, 57.00 26.31 (3.3%) 11.310 (3.3%) 13.73 (3.3%) 937 (3.3%) 6, 622 (2.2%) 2,515 (6.9%) 2,550 (9.0%) 6,259 (2.23%) 4,742 (16.5%) 2,45 (1.30) 2,00 (1.00, 3.00) 0,00 (1.00) 1,74 (1.2) 2,00 (1.00, 2.00) 0,00 (2.00) | 15.00 (11.00, 15.00) 10.0 6.200 5.709 (11.5%) 17.564 (13.2%) 2.655 (6.3%) 11.948 (24.0%) 2.370 (48.5%) 12.370 (48.5%) 12.310 (28.7%) 12.418 (25.5%) 12.418 (25.5%) 12.418 (20.0%) 12.418 (20.0%) 10.00, 37.00 16.9 (119) 10.00, 36.00 | 16-3<br>12-98 (2.0% -1.7%)<br>43% (3.4% -8.8%)<br>2.0% (2.2% -1.7%)<br>43% (2.4% -1.7%)<br>43% (2.4% -1.7%)<br>43% (2.4% -1.5% -5.0%)<br>6.2% (4.5% -5.0%)<br>6.2% (4.6% -1.7% -5.0%)<br>6.2% (4.6% -1.7% -5.0%)<br>6.2% (4.6% -1.7% -5.0%)<br>6.2% (4.6% -1.7% -1.7%)<br>6.3% (4.6% -1.7% -1.7%)<br>6.3% (4.6% -1.7% -1.7% -1.7%)<br>6.3% (4.6% -1.7% -1.7% -1.7%)<br>6.3% (4.6% -1.7% | 14.00 [10.00, 19.00] 1.00, 57.00 1.331 [10.2%) 5.013 (36.5%) 5.013 (36.5 | 14.00 [10.00 19.00] 10.00 59.00 14.02 [10.319] 14.02 [10.319] 14.02 [10.319] 13.112 [22.91] 13.112 [22.91] 13.112 [22.91] 13.147 [23.119] 24.71 [13.6] 24.71 [13.6] 20.01 [2.00] 17.01 [12.2] 17.01 [12.2] 17.01 [12.2] | 1() 0.1% (-0.8%, 0.6%) 0.1% (-0.8%, 0.6%) 0.2% (-1.0%, 1.3%) 0.1% (-0.5%, 0.4%) 0.7% (-0.5%, 0.4%) 0.0% (-0.6%, 0.6%) 0.0% (-0.6%, 0.7%) 0.2% (-1.5%, 0.6%) 0.0% (-0.6%, 0.4%) 0.0% (-0.6%, 0.4%) 0.0% (-0.6%, 0.4%) 0.0% (-0.0%, 0.4%) 0.0% (-0.0%, 0.0%) 1() 1() 1() 0.01 (-0.04, 0.02) 1() |
| Imedian (IQR) Imis max Colonoscopy Sigmoidoscopy, n (%) Flu Pretumococcal vaccine; n (%) Plu Pretumococcal vaccine; n (%) PSA test n (%) FSA test n (%) Inclination (%) Inclination (%) Inclination (%) Inclination (IQR) Inclination (IQR | 14-00 [10.00.18.00] 1.00,5700 2631 (9.3%) 11.130 [39.4%) 937(3.3%) 6,262 (221%) 2,5516 (9.9%) 6,299 (221%) 2,451 (1.3%) 4,742 (16.3%) 245 (1.30) 200 [200,300] 0,000,10.00 1.74 (1.21) 200 [10.0,200] 0,000,200 3,40(3.50) 3,40(3.50) 3,40(3.50) 3,40(3.50) 3,60(3.00) | 15.00 [11.00, 19.00] 10.00 62.00 5.709 [11.5%] 17.564 (35.2%) 17.564 (35.2%) 18.948 (24.0%) 2.370 (4.8%) 4.383 (9.7%) 4.381 (9.7%) 12.448 (25.0%) 2.36 (1.32) 2.00 11.00, 3.001 0.00, 3.700 16.9 (11.9) 2.00 [10.0, 2.00] 0.00 3.000 3.17(2.6%) 3.00 (2.00, 4.00) 0.00, 92.00 | 14; 1<br>1; 3<br>22% (2.6%, 1.7%)<br>41% (3.4%, 4.8%)<br>41% (3.4%, 4.6%)<br>1.8% (2.4%, 1.2%)<br>41% (3.8%, 4.5%)<br>0.7% (1.1%, 0.3%)<br>6.4% (7.1%, 5.5%)<br>10.2% (3.8%, 7.6%)<br>0.09 (0.07, 0.11)<br>(1; 4)<br>0.05 (0.03, 0.07)<br>(1; 4)<br>0.23 (0.18, 0.28)<br>(1; 4)<br>0.23 (0.18, 0.28) | 14.00 [10.00, 19.00] 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%) 13.91 [10.2%] 13.91 [10 | 14.00 [10.00 ; 19.00] 10.00 59.00 1.402 [10.3%) 4.592 [13.67%] 5.77 (3.9%) 3.112 [22.9%) 9.201 [6.8%] 1.240 [9.1%) 3.454 [25.4%] 3.47 (23.1%) 2.47 (13.6) 2.001 [20.0, 3.00] 0.00, 37.00 1.73 (1.22) 2.001 [10.20] 0.00 (30.00) 3.30 (2.88) 3.00 [2.00, 4.00] 0.00, 92.00 | -(-, -) -(-, - |
| Imedian (1QR) Imit; max Colonoscopy Sigmoidoscopy; n (%) Flu Presumacoccal vaccine; n (%) Flu Presumacoccal vaccine; n (%) Flu Presumacoccal vaccine; n (%) FSA test n (%) | 14-00 [10.00.18.00] 1.00, 57:00 2.631 (9.3%) 11.130 [39.4%) 937 (3.3%) 6.262 (22.1%) 6.259 (22.1%) 6.259 (22.1%) 4.742 (16.8%) 4.742 (16.8%) 4.742 (16.8%) 1.744 (1.2%) 1.744 | 15.00 [11.00, 19.00] 10.0 62.00 5.709 (11.5%) 17.564 (15.2%) 17.564 (15.2%) 17.564 (15.2%) 11.948 (24.0%) 2.370 (4.8%) 4.838 (9.7%) 14.310 (28.7%) 12.448 (25.0%) 2.36 (13.2) 2.00 (10.0, 3.00) 0.00, 3.700 1.69 (11.9) 2.00 (10.0, 2.00) 0.00, 2.00 0.00, 0.00 0.00 | 16.3 22% (2.6%, 1.7%) 1.53 (2.6%, 1.7%) 1.53 (2.6%, 1.7%) 1.54 (3.4%, 4.8%) 2.0% (2.3%, 1.7%) 1.8% (2.4%, 1.2%) 1.8% (2.4%, 1.2%) 1.8% (2.4%, 1.2%) 1.8% (3.6%, 4.5%) 0.7% (1.1%, 0.3%) 6.4% (7.1%, 5.6%) 8.2% (3.8%, 7.5%) 1.6% (3.8%, 7.5%) 1.6% (3.6%, 4.7%) 1.6% (3. | 14.00 [10.00, 19.00] 13.00 5.700 13.91 [10.2%) 5.013 13.65 9%) 5.013 13.65 9%) 5.013 13.65 9%) 3.133 (23.0%) 914 (6.7%) 1.246 [9.2%) 3.420 (25.1%) 3.070 (22.6%) 2.45 (1.28) 2.00 [2.00, 3.00] 0.00, 9.00 1.72 [118] 2.00 [10.0, 2.00] 0.00, 2.00 | 14.00 [10.00 ; 19.00] 10.00 59.00 1.402 (10.3%) 4.592 (16.5%) 5.77 (1.3%) 3.112 (22.9%) 9.201 (16.8%) 1.240 (9.1%) 3.454 (25.4%) 3.454 (25.4%) 3.47 (23.1%) 2.47 (13.6) 2.00 (2.00, 3.00) 0.00, 37.00 1.73 (1.22) 2.00 [10.00, 2.00] 0.00, 2.00 0.00, 0.00 0.00 | -(-, -)<br>-(-, -)<br>-(-) -(-) -(-) -(-) -(-)<br>-(-) -(-) -(-) -(-) -(-) -(-) -(-)<br>-(-) |
| Imedian (10R) Imit; max Colonocopy Sigmoidescopy; n (%) Pla Phenomococal vaccine n (%) Pap samean n (%) Pap samean n (%) PSA test n (%) PSA t | 14.00 (10.00.18.00] 1.00.57.00 2.631 (3.3%) 1.1320 (3.3%) 1.1320 (3.34%) 337 (3.3%) 337 (3.3%) 6.262 (2.21%) 2.550 (9.9%) 6.269 (2.21%) 2.450 (1.30) 2.00 (2.00, 3.00) 0.00, 1.00 1.74 (1.21) 2.00 (1.00, 2.00) 0.00, 2.00 3.40 (3.50) 3.00 (2.00, 4.00) 0.00, 3.600 0.03 (6.00) | 15.00 [1.00, 19.00] 10.0, 62.00 5.709 (11.5%) 17.564 (13.5%) 2.659 (5.3%) 11.948 (24.0%) 2.2570 (4.5%) 4.838 (9.7%) 14.310 (28.7%) 12.448 (25.0%) 12.448 (25.0%) 12.448 (25.0%) 13.00 (30.0) 0.00 37.00 169 (11.9) 2.001 [0.0, 2.00] 0.00 36.00 317 (2.5%) 300 (20.0, 4.0) 0.00 92.00 0.00 92.00 0.00 92.00 | 16.3<br>2.2% (2.6%, 1.7%)<br>2.1% (2.6%, 1.7%)<br>2.1% (2.4%, 1.2%)<br>2.0% (2.3%, 1.7%)<br>1.8% (2.4%, 1.2%)<br>1.8% (2.4%, 1.2%)<br>1.8% (2.4%, 1.2%)<br>1.9% (2.4%, 1.2%)<br>0.7% (1.1%, 0.3%)<br>6.4% (7.1%, 5.5%)<br>8.2% (8.8%, 7.6%)<br>0.09 (0.07, 0.11)<br>16.3<br>0.05 (0.03, 0.07)<br>16.3<br>0.23 (0.18, 0.28)<br>16.3<br>0.23 (0.18, 0.28)<br>16.3<br>0.01 (0.04, 0.02) | 14.00 [10.00, 19.00] 10.0, 5700 1.391 [10.2%) 5.013 [36.9%) 5.30 [3.59%) 5.30 [3.59%) 5.30 [3.59%) 1.34 [2.2.0%) 914 [6.7%) 1.246 [9.2%] 3.420 [25.1%) 3.070 [2.26%) 2.45 [1.28] 2.00 [2.00, 3.00] 0.00, 9.00 1.77 [1.18] 2.00 [1.00, 2.00] 0.00, 2.00 3.30 [2.52] 3.00 [2.00, 4.00] 0.00, 2.00 0.00, 2.00 | 14.00 10.00 19.00 | -(-, -) -(-) -(-) -(-) -(-) -(-) -(-) -(-) - |
| Imedian (IQRI) Imis max Colonoscopy Sigmoidoscopy; n (%) Fili Phisumoroccal vaccine; n (%) Fili Phisumoroccal vaccine; n (%) Fili Phisumoroccal vaccine; n (%) Fish test n (%) Fish test n (%) Fish test n (%) Fish test n (%) Bone mineral density tests; n (%) Mammagrams; n (%) Telemadicine; n (%) Telemadicin | 14-00 [10.00.18.00] 1.00, 57:00 2.631 (9.3%) 11.130 [39.4%) 937 (3.3%) 6.262 (22.1%) 6.259 (22.1%) 6.259 (22.1%) 4.742 (16.8%) 4.742 (16.8%) 4.742 (16.8%) 1.744 (1.2%) 1.744 | 15.00 11.00, 15.00 10.0, 62.00 5.709 11.519 17564 (15.2%) 2559 (3.3%) 11.948 (24.0%) 2.270 (4.8%) 4.330 (28.7%) 4.330 (28.7%) 1.448 (25.0%) 12.448 (25.0%) 2.36 (1.32) 2.36 (1.32) 2.301 (1.03, 3.00) 3.00 (3.00, 3.00) 3.00 (3.00, 3.00) 3.00 (3.00, 3.00) 3.17 (2.6%) 3.00 (2.00, 4.00) 0.00 (32.00) | 16.3 22% (2.6%, 1.7%) 41% (3.4%, 4.8%) 41% (3.4%, 4.6%) 41% (3.4%, 4.6%) 41% (3.4%, 4.5%) 4.8% (2.4%, 1.7%) 4.8% (2.4%, 1.7%) 4.8% (2.4%, 1.7%) 4.8% (2.4%, 1.7%) 4.9% (3.8%, 4.5%) 0.7% (1.1%, 0.3%) 6.4% (7.1%, 5.8%) 8.2% (8.8%, 7.6%) 0.09 (0.07, 0.11) (6.4) 1.6.4 (7.1%, 5.8%) 8.2% (8.8%, 7.6%) 0.09 (0.07, 0.11) (6.4) 1.6.4 (7.4%, 1.2%) 4.6.4 (7.4%, 1.2% | 14.00 [10.00, 19.00] 13.00 5.700 13.91 [10.2%) 5.013 13.65 9%) 5.013 13.65 9%) 5.013 13.65 9%) 3.133 (23.0%) 914 (6.7%) 1.246 [9.2%) 3.420 (25.1%) 3.070 (22.6%) 2.45 (1.28) 2.00 [2.00, 3.00] 0.00, 9.00 1.72 [118] 2.00 [10.0, 2.00] 0.00, 2.00 | 14.00 [10.00 ; 19.00] 10.00 59.00 1.402 (10.3%) 4.592 (16.5%) 5.77 (1.3%) 3.112 (22.9%) 9.201 (16.8%) 1.240 (9.1%) 3.454 (25.4%) 3.454 (25.4%) 3.47 (23.1%) 2.47 (13.6) 2.00 (2.00, 3.00) 0.00, 37.00 1.73 (1.22) 2.00 [10.00, 2.00] 0.00, 2.00 0.00, 0.00 0.00 | -(-, -) |
| Imedian (IQR) Imis mass Colonescopy Sigmoidoscopy; n (%) Fiu Presumcooccal vaccine; n (%) Fiu Presumcooccal vaccine; n (%) PSA test n (%) FSA test n (%) FSA test n (%) FSA test n (%) Bone mineral density tests; n (%) Manningame; n (%) Telemedicine; n (%) Telemedicin | 14-00 [10.00.18.00] 1.100, 57.00 2.631 (9.3%) 11.130 (3.3%) 11.130 (3.3%) 11.130 (3.3%) 11.130 (3.3%) 11.130 (3.3%) 6.262 (2.21%) 2.550 (9.0%) 6.269 (2.23%) 4.742 (16.5%) 2.45 (1.30) 2.00 [2.00, 3.00] 0.00 [1.00 1.74 (1.21) 2.00 [1.00, 2.00] 0.00, 2.20 0.00, 2.20 0.00, 3.65.00 0.03 (3.65.00 0.00 (3.00) | 15.00 11.00, 19.00 10.00 62.00 5.709 11.5% 17.564 13.5.2% 26.595 (2.3%) 11.948 (2.4.0%) 2.270 (4.8%) 4.381 (9.7%) 4.381 (9.7%) 4.381 (9.7%) 12.448 (2.5.0%) 2.361 13.2 2.001 10.0.3.00 0.00, 37.00 16.9 (1.9) 2.001 10.0.2.00 0.00, 36.00 3.17 (2.6.9) 3.001 (2.0.0.4.00) 0.00, 92.00 0.001 (2.0.0.00) | 14.3 2.2% (2.6%, 1.7%) 2.2% (2.6%, 1.7%) 4.1% (3.4%, 4.8%) 2.0% (2.3%, 1.7%) 3.8% (2.4%, 1.7%) 3.8% (2.4%, 1.7%) 0.7% (1.1%, 0.3%) 6.4% (7.1%, 5.8%) 8.2% (3.8%, 7.6%) 0.09 (0.07, 0.11) 1.0-1 1 | 14.00 10.00 19.00 | 14.00 10.00 19.00 | -(-, -) -(-, - |
| Imedian (IQRI Imit; max Colonscopy Sigmoldoscopy; n (%) Flu Presumozoccal vaccine; n (%) Flu Presumozoccal vaccine; n (%) PSA test n (%) FSA | 14.00 [10.00.18.00] 1.00.57.00 2.631 (9.3%) 1.130 (3.3%) 1.130 (3.3%) 1.130 (3.3%) 937 (3.3%) 937 (3.3%) 937 (3.3%) 937 (3.3%) 947 (3.3%) 1.2550 (9.0%) 1.2550 (9.0%) 1.2550 (9.0%) 1.245 (1.30) 1.200 (1.00.30) 1.74 (1.21) 1.200 (1.00.20) 1.74 (1.21) 1.200 (1.00.20) 1.74 (1.22) 1.200 (1.00.20) 1.74 (1.23) 1.74 (1.24) 1.75 (1.25) 1 | 15.00 [1.00, 15.00] 10.0 6.200 5.709 (11.5%) 17.564 (35.2%) 26.59 (3.3%) 11.948 (24.0%) 2.270 (4.5%) 4.331 (9.7%) 4.331 (9.7%) 4.331 (9.7%) 4.331 (9.7%) 12.448 (25.0%) 2.36 (1.32 2.001 1.00, 3.00) 0.00, 37.00 16.9 (1.19) 2.001 (1.00, 2.00) 0.00, 36.00 3.17 (2.69) 3.00 (2.00, 4.00) 0.00, 92.00 0.00, 77.00 1.21 (1.65) 1.00 (1.00, 0.00) 0.00, 77.00 | 16.3 22% (2.5%, 1.7%) 2.2% (2.5%, 1.7%) 4.1% (3.4%, 4.8%) 2.0% (2.2%, 1.7%) 1.8% (2.4%, 1.7%) 1.8% (2.4%, 1.7%) 0.7% (1.1%, 0.3%) 6.4% (1.7%, 5.8%) 8.2% (3.8%, 7.5%) 0.09 (0.07, 0.11) 4.5 (1.3%, 0.3%) 6.4% (7.7%, 5.8%) 0.09 (0.07, 0.11) 4.5 (1.3%, 0.3%) 6.4% (7.7%, 5.8%) 0.09 (0.07, 0.11) 4.5 (1.3%, 0.3%) 6.5 ( | 14.00 10.00 19.00 | 14.00 10.00 19.00 | -(-, -) -(-, - |
| Imedian (10R) Imit; max Colonoccopy Sigmoidoscopy; n (%) Rip Pheumococcal vaccine n (%) Pap amear, n (%) Pap | 14-00 [10.00.18.00] 1.100, 57.00 2.631 (9.3%) 11.130 [3.9%) 11.130 [3.94%) 937 [3.3%) 6.262 [2.21%) 2.550 (9.9%) 6.299 [2.23%) 4,742 [16.8%) 2.45 (1.30) 2.00 [2.00.300] 0.00 [10.00 1.74 (1.21) 2.00 [10.0.20] 0.00, 2.200 3.40 [3.50) 3.00 [2.00.40] 0.00, 3.66.00 0.23 [2.29] 0.23 [2.29] 0.23 [2.29] 0.00 [3.60.00] 0.00 [3.60.00] 1.32 (2.29) 0.00 [3.60.00] 0.00 [3.60.00] 1.32 (2.28) | 15.00 11.00, 19.00 10.00 62.00 5.709 11.5% 17.564 13.5.2% 26.595 (2.3%) 11.948 (2.4.0%) 2.270 (4.8%) 4.381 (9.7%) 4.381 (9.7%) 4.381 (9.7%) 12.448 (2.5.0%) 2.361 13.2 2.001 10.0.3.00 0.00, 37.00 16.9 (1.9) 2.001 10.0.2.00 0.00, 36.00 3.17 (2.6.9) 3.001 (2.0.0.4.00) 0.00, 92.00 0.001 (2.0.0.00) | 16.3 2.2% (2.5% -1.7%) 1.5.3 2.2% (2.5% -1.7%) 1.1% (3.4% 4.5%) 2.2% (2.5% -1.7%) 1.5% (2.5% -1.7%) 1.5% (2.4% -1.7%) 1.5% (2.4% -1.7%) 1.5% (2.4% -1.7%) 1.5% (2.5% - | 14.00 10.00 19.00 10.0 57.00 1391 10.2% 50.13 26.5% 50.1 | 14.00 10.00 19.00 10.00 59.00 14.02 (10.3%) 14.92 (26.7%) 577 (3.9%) 3.112 (22.9%) 3.112 (22.9%) 3.12 (23.1%) 3.45 (25.4%) 3.45 (25.4%) 3.47 (23.1%) 24.7 (1.36) 20.01 20.03 0.00 0.00 37.00 1.73 (1.22) 20.01 20.03 0.00 3.30 (2.8%) | 1(-, -) 0.1% (-0.8%, 0.6%) 0.2% (-1.0%, 1.3%) 0.2% (-1.0%, 1.3%) 0.2% (-0.0%, 0.4%) 0.2% (-0.9%, 0.4%) 0.2% (-0.9%, 0.6%) 0.0% (-0.6%, 0.6%) 0.0% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) 0.0% (-0.6%, 0.0%) 0.0% (-0.6%, 0.0%) 0.0% (-0.6%, 0.0%) 0.0% (-0.6%, 0.0%) 1(-, -) 0.00 (-0.04, 0.02) 1(-, -) 0.00 (-0.06, 0.06) 1(-, -) 0.00 (-0.06, 0.06) 1(-, -) 1(-, -) 0.00 (-0.05, 0.03) 1(-, -) 1(-, -) 0.01 (-0.05, 0.03) |
| Imedian (191) min, max Colonoccopy Sigmoidoscopy; n (%) Bit Pherumococcal vaccine; n (%) Pip Samear, | 14.00 [10.00.18.00] | 15.00 11.00, 15.00 10.0, 62.00 5.709 11.519 17.564 (15.2%) 25.509 (3.3%) 11.946 (24.0%) 2.770 (4.8%) 4.330 (28.7%) 4.330 (28.7%) 12.448 (25.0%) 2.36 (1.32) 2.36 (1.32) 2.36 (1.32) 2.301 (1.03) 2.36 (1.32) 2.301 (1.03) 2.301 | 16.3 22% (2.6%, 1.7%) 4.1% (3.4%, 4.8%) 2.2% (2.6%, 1.7%) 4.1% (3.4%, 4.8%) 2.0% (2.3%, 1.7%) 4.1% (3.6%, 4.5%) 4.1% (3. | 14.00 10.00 19.00 | 14.00 14.00 19.00 10.00 50.00 14.02 (10.3 %) 4.992 (16.7 %) 537 (13.9 %) 3112 (22.9 %) 920 (6.8 %) 1240 (19.1 %) 3454 (25.4 %) 3454 (25.4 %) 3454 (25.4 %) 3474 (23.1 %) 1274 (19.1 %) 1 | -(-, -) |
| Imedian (IQR) Imit; max Coloroscopy Sigmoidoscopy; n (%) Flu Presumacroccal vaccine; n (%) Flu Presumacroccal vaccine; n (%) PSA test n (%) FSA test n (%) F | 14.00 (10.00.18.00] 1.00.57.00 2.631 (9.3%) 1.130 (13.9%) 1.130 (13.9%) 937 (3.3%) 937 (3.3%) 937 (3.3%) 937 (3.3%) 937 (3.3%) 937 (3.3%) 947 (3.3%) 947 (3.3%) 947 (3.3%) 947 (3.3%) 947 (3.3%) 947 (10.0%) 948 (10.0%) 949 (2.2%) 949 (2.2%) 949 (2.2%) 949 (2.2%) 949 (2.2%) 940 (3.5%) 940 | 15.00 11.00, 15.00 10.06 20.00 5.709 11.15% 17.564 (15.2%) 25.509 (15.3%) 17.564 (15.2%) 25.509 (15.3%) 17.564 (15.2%) 25.70 (4.8%) 4.380 (2.7%) 14.380 (2.7%) 14.380 (2.7%) 14.380 (2.7%) 14.380 (2.7%) 12.448 (2.5%) 12.448 (2.5%) 12.448 (2.5%) 12.448 (2.5%) 12.458 (2.5%) 12.468 (2.5%) 12.469 (2.5%) | 16.3 2.2% (2.5%, 1.7%) 41% (2.6%, 1.7%) 41% (3.4%, 4.2%) 2.2% (2.2%, 1.7%) 41% (3.4%, 4.2%) 42% (2.2%, 1.7%) 1.8% (2.4%, 4.2%) 4.2% (4.4%, 4.2%) 4.2% (4.4%, 4.2%) 4.2% (4.5%, 4.5%) 0.7% (1.1%, 0.3%) 6.4% (7.7%, 5.5%) 8.2% (3.8%, 7.5%) 0.09 (0.07, 0.11) (1.5, 3.2%) (1.5, | 14.00 10.00 19.00 10.0 57.00 1391 10.2% 50.13 26.5% 50.1 | 14.00 10.00 19.00 10.00 50.00 14.02 (10.3 %) 4.992 (36.7 %) 5.77 (3.9 %) 5.77 (3 | 1(-, -) 1(-, -) 1(-) 1(-) 1(-) 1(-) 1(-) 1(-) 1(-) 1( |
| Imedian (IQR) Imit; max Colonoscopy Sigmoidoscopy; n (%) Flu Presumcoccal vaccine; n (%) Flu Presumcoccal vaccine; n (%) Flu Presumcoccal vaccine; n (%) Flu State (1, %) Fiscal occult blood test n (%) Bone mineral density tests; n (%) Marmograms; n (%) Telemedicine; n (%) Telemedicine; n (%) Hablat tests _mean (sd) _min; max Upid panels _mean (sd) _median (IQR) _min; max Coedine tests _mean (sd) _median (IQR) _min; max Upid panels _median (IQR) _min; max _median (IQR) _median (IQR) _median (IQR) | 14.00 [10.00.18.00] 1.00.5700 2.631 (8.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3 4%) 337 (3.3%) 337 (3.3%) 337 (3.3%) 337 (3.3%) 2.550 (9.0%) 2.550 (9.0%) 2.550 (9.0%) 2.550 (9.0%) 2.45 (1.30) 2.00 [2.00, 3.00] 0.00, 1.00 1.74 (1.2) 2.00 [1.00, 2.00] 0.00, 2.00 3.40 (3.50) 3.00 [2.00, 4.00] 0.00, 366.00 0.23 (2.29) 0.00 [0.00, 0.00] 0.00, 366.00 1.32 (2.29) 1.00 [0.00, 0.00] 1.31 (2.73) 3.00 [1.00, 5.00] 2.20, 1.600 0.19 [1.00] 0.19 [1.00] 0.19 [1.00] 0.19 [1.00] 0.19 [1.00] | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 10.00 5.200 15.90 11.500 15.94 12.520 26.529 5.370 11.546 24.050 25.70 14.550 14.310 28.770 14.310 28.770 12.448 25.070 12.448 25.070 12.448 25.070 12.448 25.070 12.448 25.070 13.00 20.00 13.00 1 | 16.3 22% (2.5%, 1.7%) 2.2% (2.5%, 1.7%) 3.1% (2.4%, 1.2%) 4.1% (2.4%, 1.2%) 4.1% (2.4%, 1.2%) 4.1% (3.5%, 4.5%) 0.7% (1.1%, 0.3%) 6.4% (1.2%, 1.5%) 4.1% (3.5%, 4.5%) 0.9% (0.1%, 0.3%) 6.4% (1.7%, 5.5%) 8.2% (3.8%, 7.5%) 0.99 (0.07, 0.11) (1.5) 1.5% (1.5 | 14.00 10.00 19.00 | 14.00 10.00 10.00 10.00 50.00 14.02 (10.3 %) 4.092 (16.7 %) 527 (1.3 %) 527 (1.3 %) 527 (1.3 %) 528 (1.3 %) 527 (1.3 %) 528 (1.3 %) 528 (1.3 %) 529 (1 | -(-, -) -(-, -) -(-) -(-) -(-) -(-) -(-) -(-) -(-) - |
| Imedian (10R) Imit, max Colonoccopy Sigmoidoscopy; n (%) By Pheumoscocal vaccine; n (%) Phy Pheumoscocal vaccine; n (%) Phy Sha text n (%) Phy Sha text n (%) Phy Sha text n (%) Phy Sha text n (%) Bore mineral density tests; n (%) Marrinograms, n (%) Telsimedicine; n (%) HibAla tests _mean (sd) _min; max Uicid panels _mean (sd) _min; max Uicid panels _mean (sd) _min; max White tests _mean (sd) _min; max White tests _mean (sd) _min; max Uicid panels _min; max Uicid panels _min; max Uicid panels _min; max Coedinine tests _mean (sd) _min; max Uicid panels _min; max Coedinine tests _mean (sd) _min; max Uicid panels _min; max Combined (liQR) _min; max Uicid panels _min; max Combined (liQR) _min; max Uicid panels _mean (sd) | 14.00 [10.00.18.00] 1.00.57.00 2.631 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.2550 (3.0%) 1.2550 (3.0%) 1.2550 (3.0%) 1.2550 (3.0%) 1.245 (1.30) 1.200 (1.00, 3.00) 1.00.10.00 1.74 (1.2) 1.200 (1.00, 2.00) 1.00, 2.00 1.340 (3.50) 1.300 (2.00, 4.00) 1.00, 3.600 1.32 (2.2%) 1.00 (1.00, 0.00) 1.32 (2.2%) 1.00 (1.00, 0.00) 1.31 (2.3%) 1.00 (1.00, 5.00) 1.20 (1.00, 5.00) 1.20 (1.00, 5.00) 1.21 (1.00) | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 15.700 11.500 17.564 (15.200 25.520 15.200 25.5 | 16.3 22% (2.6%, 1.7%) 4.1% (2.4%, 1.2%) 4.1% (2.4%, 1.2%) 1.8% (2.6%, 1.2%) 1.8% (2. | 14.00 [10.00, 19.00] 13.00 [10.00, 19.00] 13.00 [10.2%) 13.01 [10.2%] 13.01 [10.2%] 13 | 14.00 [10.00 19.00] 10.00 59.00 14.02 (10.3 %) 4.992 (16.7 %) 5.97 (13.9 | 1(-, -) 1-(-, -) 1-(- |
| Imedian (10R) min, max Debreamcoccus Sigmoidescopy, n (%) Dis Presumcoccus accinen (%) Play smear n (%) Play | 14.00 [10.00.18.00] 1.00.5700 2.631 (8.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3 4%) 337 (3.3%) 337 (3.3%) 337 (3.3%) 337 (3.3%) 2.550 (9.0%) 2.550 (9.0%) 2.550 (9.0%) 2.550 (9.0%) 2.45 (1.30) 2.00 [2.00, 3.00] 0.00, 1.00 1.74 (1.2) 2.00 [1.00, 2.00] 0.00, 2.00 3.40 (3.50) 3.00 [2.00, 4.00] 0.00, 366.00 0.23 (2.29) 0.00 [0.00, 0.00] 0.00, 366.00 1.32 (2.29) 1.00 [0.00, 0.00] 1.31 (2.73) 3.00 [1.00, 5.00] 2.20, 1.600 0.19 [1.00] 0.19 [1.00] 0.19 [1.00] 0.19 [1.00] 0.19 [1.00] | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 10.00 5.200 15.90 11.500 15.94 12.520 26.529 5.370 11.546 24.050 25.70 14.550 14.310 28.770 14.310 28.770 12.448 25.070 12.448 25.070 12.448 25.070 12.448 25.070 12.448 25.070 13.00 20.00 13.00 1 | 16.3 22% (2.5%, 1.7%) 2.2% (2.5%, 1.7%) 3.1% (2.4%, 1.2%) 4.1% (2.4%, 1.2%) 4.1% (2.4%, 1.2%) 4.1% (3.5%, 4.5%) 0.7% (1.1%, 0.3%) 6.4% (1.2%, 1.5%) 4.1% (3.5%, 4.5%) 0.9% (0.1%, 0.3%) 6.4% (1.7%, 5.5%) 8.2% (3.8%, 7.5%) 0.99 (0.07, 0.11) (1.5) 1.5% (1.5 | 14.00 10.00 19.00 | 14.00 10.00 10.00 10.00 50.00 14.02 (10.3 %) 4.092 (16.7 %) 527 (1.3 %) 527 (1.3 %) 527 (1.3 %) 528 (1.3 %) 527 (1.3 %) 528 (1.3 %) 528 (1.3 %) 529 (1 | -(-, -) -(-, -) -(-) -(-) -(-) -(-) -(-) -(-) -(-) - |
| Imedian (IQR) Imit mass Colonoscopy Sigmoldoscopy: n (%) File Presentacoccal vaccine: n (%) File Presentacoccal vaccine: n (%) File Presentacoccal vaccine: n (%) PSA test n (%) FSA test | 14.00 [10.00, 18.00] 100, 57.00 26.31 (3.3%) 11.310 (3.3%) 11.310 (3.3%) 13.73 (3.3%) 6.262 (2.2%) 2.515 (8.9%) 2.550 (9.0%) 6.299 (2.23%) 4.742 (16.8%) 2.49 (1.30) 2.00 (1.00, 1.00) 1.74 (1.2) 2.00 (1.00, 2.00) 1.00 (2.20) 1.00 (3.65 (0.00) 1.00 (3.65 (0.00) 1.00 (3.65 (0.00) 1.32 (2.8) 1.32 (2.8) 1.30 (1.00, 5.00) 1.31 (2.73 3.00 (1.00, 5.00) 1.31 (2.73 3.00 (1.00, 5.00) 1.31 (2.73 3.00 (1.00, 5.00) 1.30 (3.00) 1.30 (3.0 | 15.00 11.00, 15.00 10.06 20.00 10.06 20.00 17.564 13.52% 25.576 13.58% 17.564 13.52% 25.576 13.58% 17.564 13.52% 25.576 13.58% 23.70 14.510 22.7% 17.564 13.52% 23.70 14.510 22.7% 17.564 13.52% 23.70 14.510 22.7% 17.564 13.52% 17.564 13.52% 17.564 13.52% 17.565 13.52% 17.566 13.52% 17 | 16-3 22% (2.6% -1.7%) 41% (3.4% -1.8%) 41% (3.4% -1.8%) 2.0% (2.2% -1.7%) 41% (3.4% -1.8%) 2.0% (2.2% -1.7%) 41% (3.6% -1.8%) 4.1% | 14.00 10.00 19.00 10.0 57.00 1391 10.2% 5013 136 59% 5014 57% 245 128 246 128 247 128 247 128 248 128 249 249 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 240 | 14.00 14.00 19.00 10.00 59.00 14.02 (10.3%) 4.92 (26.7%) 537 (3.9%) 31.12 (2.9%) 590 (6.8%) 1240 (21.1%) 247 (1.36) 248 (1.36) 249 (1.36) 240 (1.36) 240 (1.36) 250 (1.36) 250 (1.36) 260 (1.36) 277 (2.55) 200 (1.06) 200 (1.06) 210 (1.36) 211 (1.36) 220 (1.36) 200 (1.36) 211 (1.36) 220 (1.36) 231 (1.36) 241 (1.36) 252 (1.36) 253 (1.36) 254 (1.36) 255 (1.36) 256 (1.36) 257 (1.36) 258 (1.36) 258 (1.36) 259 (1.36) 250 (1.36) 25 | 1() (1) |
| Imedian (IQR) Imit; max Colonocopy Sigmoidoscopy; n (%) File Presumococcal vaccine n (%) File Presumococcal vaccine n (%) File Presumococcal vaccine n (%) File Presumococcal vaccine n (%) File All Presumococcal vaccine n (%) File All Presumococcal vaccine n (%) File Court blood test n (%) Bone mineral density tests; n (%) Marmogames, 1%) Telemedicine; n (%) Hibbla tests Limean (sd) Limit; max Uicid panels Limean (sd) Limit; max Uicid panels Limean (sd) Limit; max Coestriane tests Limean (sd) Limit; max Uicid panels Limit; max Uicid panels Limit; max Coestriane tests Limean (sd) Limit; max Uicid panels Limit; max Uicid pan | 14-00 [10.00.18.00] 1-00.5700 2-631 (6.3%) 1-100.5700 2-631 (6.3%) 1-120.63 (6 | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 17.564 (15.2%) 25.59 (15.3%) 17.564 (15.2%) 25.59 (15.3%) 11.546 (24.0%) 25.70 (4.5%) 43.30 (25.7%) 13.448 (25.0%) 12.448 (25.0%) 13.70 (15.0%) 13.70 (15 | 16.3 2286 (26%, 1.7%) 4.1% (2.4%, 1.2%) 1.8% (2.6%, 1.2%) 1.8% (2. | 14.00 10.00 19.00 | 14.00 14.00 19.00 10.00 50.00 14.02 (10.3 %) 4.992 (24.5 %) 537 (3.9 %) 537 (3.9 %) 537 (3.9 %) 537 (3.9 %) 537 (3.9 %) 537 (3.9 %) 538 (3 | 1() (1) |
| Imedian (IQR) Imin max Colemacopy Sigmoidescopy; n (%) Fib Pheumococcal vaccine n (%) Fib Real occur Bhod lest n (%) Fib Real occur Bhod lest n (%) Fib Real occur Bhod lest n (%) Telemachine n (%) Hib Alz tests Imedian (IQR) Imin max Upid panels Imedian (IQR) Imin max Upid panels Imedian (IQR) Imin max Ocastine tests Imedian (IQR) Imin max Upid panels Imedian (IQR) Imedian (IQ | 14.00 10.00 18.00 | 15.00 11.00, 15.00 10.00 52.00 10.00 52.00 17.564 (15.2%) 25.59 (15.3%) 17.564 (15.2%) 25.59 (15.3%) 17.564 (15.2%) 25.59 (15.3%) 17.464 (26.3%) 17.464 (26.3%) 17.464 (15.3%) 18.464 (15.3%) 18.464 (15 | 16.3 22% (2.6%, 1.7%) 4.1% (2.4%, 4.2%) 2.2% (2.6%, 1.7%) 4.1% (2.4%, 4.2%) 2.0% (2.3%, 1.7%) 1.8% (2.4%, 4.2%) 2.0% (2.3%, 1.7%) 1.8% (2.4%, 4.5%) 0.7% (1.1%, 0.3.5%) 6.4% (7.1%, 5.5%) 8.2% (8.6%, 7.6%) 0.09 (0.07, 0.11) (1.5, 3.5%) 0.09 (0.07, 0.11) (1.5, 3.5%) 0.05 (0.03, 0.07) (1.5, 3.5%) 0.05 (0.03, | 14.00 10.00 19.00 10.00 57.00 1391 10.2% 50.13 36.5% 50.13 50.5% 50. | 14.00 10.00 10.00 10.00 50.00 10 | 1(-, -) (1-, -) (1-) (1-) (1-) (1-) (1-) (1-) (1-) (1 |
| Imedian (10R) Imit; max Colonoccopy Sigmoidoscopy; n (%) Rh Pheumococcal vaccine n (%) Pap amear n (%) Pap ame | 14-00 [10.00.18.00] 1-00.5700 2-631 (3.3%) 1-1130 (3.3%) 1-1312 (3.3%) 1 | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 17.564 (15.2%) 25.509 (15.3%) 17.564 (15.2%) 25.509 (15.3%) 17.564 (15.2%) 25.509 (15.3%) 17.464 (15.0%) 24.704 (15.0%) 25.704 (15.0%) 25.704 (15.0%) 25.704 (15.0%) 26.704 (15.0%) 26.704 (15.0%) 27.705 | 16-3 2-28-(-26%,-1.7%) 4-38-(-24%,-1.2%) 4-38-(-24%,-1.2%) 1.88-(-24%,-1.2%) 1.88-(- | 14.00 10.00 19.00 10.00 17.00 130 11.02% 15.013 16.5% 15.014 16.5% 15.014 | 14.00 14.00 19.00 14.00 14.00 10.00 14.02 10.03 14.02 10.03 14.02 10.33 14.02 10.03 14.02 10.33 14.02 10.03 14.02 10.03 10.03 10.03 14.03 10.03 10.03 10.03 15.03 10.03 10.03 15.03 10.03 10.03 10.03 15.03 10.03 10.03 10.03 15.03 10.03 10.03 10.03 15.03 10.03 10.03 15.03 10.03 10.03 10.03 15.03 10.03 10.03 10.03 15.03 10.03 10.03 10.03 15.03 10.03 10.03 15.03 10.03 10.03 10.03 10.03 15.03 10.03 10.03 10.03 10.03 15.03 10.03 10.03 10.03 10.03 15.03 10.03 10.03 10.03 10.03 10.03 10.03 15.03 10.03 10.0 | 1(-, -) (1-, -) (1-) (1-) (1-) (1-) (1-) (1-) (1-) (1 |
| Imedian (IQR) Imit max Colonoscopy Sigmoidoscopy: n (%) Fili Pinsemacoccal vaccine: n (%) Fili Pinsemacoccal vaccine: n (%) Fili Pinsemacoccal vaccine: n (%) PSA test n (%) PSA test n (%) PSA test n (%) PSA test n (%) Bone mineral density tests; n (%) Bone mineral density tests; n (%) Marmograms: n (%) HABAC tests Imean (sq) Imit max Usid panels Imedian (IQR) Imit max Usid panels Imean (sq) Imedian (IQR) Imit max Imit max Usid panels Imedian (IQR) Imit max Imit max Imedian (IQR) Imit max Imedian (IQR | 14.00 (10.00. 18.00] 14.00 (10.00. 18.00] 14.00, 57.00 26.31 (6.3%) 14.30 (13.3%) 14.30 (13.3%) 14.30 (13.3%) 14.30 (13.3%) 15.31 (13.3%) | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 10.00 5.200 15.90 11.500 15.94 12.520 2.652 (5.370) 11.948 24.050 2.270 (4.870) 13.310 (2.870) 13.448 (2.570) 13.410 (2.870) 13.448 (2.570) 13.410 (2.870) | 16.3 2.2% (2.5% -1.7%) 2.2% (2.6% -1.7%) 2.2% (2.6% -1.7%) 2.2% (2.6% -1.7%) 2.0% (2.3% -1.3%) 2.0% (2.3% -1.3%) | 14.00 10.00 19.00 | 14.00 10.00 10.00 10.00 50.00 10 | 1(-) 1 (-) 21% (-0.8% 0.5%) 0.2% (-0.0% 1.3%) 0.2% (-0.0% 1.3%) 0.2% (-0.0% 1.3%) 0.2% (-0.0% 1.3%) 0.2% (-0.9% 1.2%) 0.2% (-0.9% 1.2%) 0.0% (-0.5% 0.6%) 0.0% (-0.5% 0.6%) 0.0% (-0.5% 0.0%) 0.0% (-0.5% 0.0%) 0.0% (-0.5% 0.0%) 0.0% (-0.0% 0.0%) 0. |
| Imedian (IQR) Infinity Infinity Infinity Colonoscopy Sigmoidoscopy: n (%) Fili Presembococcal vaccine: n (%) Fili Presembococcal vaccine: n (%) Fili Presembococcal vaccine: n (%) PSA test n (%) Fili Presembococcal Fili Presel occur to bood test: n (%) Bone mineral density tests; n (%) Bone mineral density tests; n (%) Marmograms: n (%) Telemodicine; n (%) HAb1c tests Imedian (IQR) Imin max Upid panels Imedian (IQR) Imin max Upid panels Imedian (IQR) Imin max Upid panels Imedian (IQR) Imin max Upid panels Imedian (IQR) Imin max Upid panels Imedian (IQR) Imin max Upid tests Imedian (IQR) Imin max Upid tests Imedian (IQR) Imin max Upid tests Imedian (IQR) Imin max Upid tests Imedian (IQR) Imin max Imedian (IQR) Imin max Imin max Imedian (IQR) Imin max | 14.00 [10.00.18.00] 1.00.5700 2.631 (6.3%) 1.120 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.2550 (9.0%) 2.2550 (9.0%) 2.2550 (9.0%) 2.45 (1.30) 2.00 [2.00, 3.00] 0.00, 1.00 1.74 (1.2) 2.00 [1.00, 2.00] 0.00, 2.00 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 10.00 5.200 15.90 11.500 15.90 12.500 15.90 13.500 15.90 | 16-3 22% (2.5%, 1.7%) 41% (2.4%, 1.2%) 42% (2.5%, 1.7%) 1.8% (2.4%, 2.5%) 1.8% (2.4%, 1.2%) 1.8% (2.5%, 1.4%) 1.9% (1.5%, 1.2%) 1.9% (1.5% | 14.00 10.00 19.00 | 14.00 14.00 19.00 10.00 50.00 14.02 (10.3 %) 4.992 (16.7 %) 527 (1.3 %) 527 (1 | 1(-, 1) (1-, 1) (1-) (1-) (1-) (1-) (1-) (1-) (1-) (1 |
| Imedian (IQR) Imin max Colonsocopy Sigmoidoscopy; n (%) Elly Pheumococcal vaccine; n (%) Pap armet, n (%) Pa | 14.00 [10.00.18.00] | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 17.564 (15.2%) 25.509 (15.3%) 17.564 (15.2%) 25.509 (15.3%) 17.564 (15.2%) 25.509 (15.3%) 17.644 (15.2%) 25.701 (4.8%) 4.3810 (28.7%) 14.3810 (28.7%) 14.3810 (28.7%) 14.3810 (28.7%) 14.3810 (28.7%) 12.448 (15.0%) 12.448 (15.0%) 12.448 (15.0%) 12.468 (15.0%) 12.468 (15.0%) 12.468 (15.0%) 12.468 (15.0%) 12.469 (15.0%) 13.400 (15.0%) 14.400 (15.0%) 14.400 (15.0%) 15.400 (15.0%) 15.200 (16.3%) 14.200 (15.0%) 14.200 (15.0%) 14.200 (15.0%) 15.200 (15.0%) 15.2 | 16-3 2-28-(-26%,-1.7%) 4-38-(-2.4%,-1.2%) 4-38-(-2.4%,-1.2%) 1.8% (-2.4%,-1.2%) 1.8% (-2.4%,-2.4%) 1.8% (-2.4%) | 14.00 10.00 19.00 10.00 17.00 1391 10.2% 10.0 17.00 1391 10.2% 1301 10.2% 1301 10.2% 1301 1308 1303 1308 1313 123.0% 1246 12.2% 1256 12.2% 1267 12.2% 1268 12.2% | 14.00 14.00 19.00 10.00 50.00 14.02 10.03 14.02 10.03 14.02 10.33 14.02 10.33 14.02 10.33 14.02 10.33 14.03 10.33 14 | 1(-, -) (1, -) ( |
| Imedian (IQR) Imin max Colemacopy Sigmoidoscopy, n (%) Bit Phaumacopy Sigmoidoscopy, n (%) Bit Phaumacopy Sigmoidoscopy, n (%) Pipa amear, n (%) Bone mineral density tests; n (%) Bone mineral density tests; n (%) Marmongame, n (%) HibAct tests _mean (sq) _min, max Luici panels _mean (sq) _min, max Luici panels _mean (sq) _min, max Coatinine tests _mean (sq) _min, max Anthropic pedide tests _mean (sq) _min, max Urine tests _mean (sq) _min max Urine tests _mean (sq) _min max Urine tests _mean (sq) _median (LQR) _min, max Namber of Hospitalizations _mean (sq) _median (LQR) _min, max Number of Hospitalizations _mean (sq) _median (LQR) _min, max Any hospitalizations within polor 91 days; n (%) _mean (sq) _mean (sq) _mean (sq) _mean (sq) _mean (sq) _min, max Any hospitalizations within polor 91 days; n (%) _mean (sq) _median (LQR) _min, max Any hospitalizations within polor 92 days; n (%) _mean (sq) _median (LQR) _min, max Any hospitalizations within polor 92 days; n (%) _mean (sq) _median (LQR) _min, max Any hospitalizations within polor 92 days; n (%) _mean (sq) _median (LQR) _min, max Any hospitalization within polor 92 days; n (%) _mean (sq) _median (LQR) _min, max _min, | 14.00 [10.00. 18.00 | 15.00 11.00, 15.00 10.00 62.00 5.709 11.15% 17.564 (15.2%) 25.509 (3.3%) 19.48 (24.0%) 2.370 (4.8%) 4.330 (28.7%) 14.310 (28.7%) 12.448 (15.5%) 12.458 (13.2) 12.418 (15.5%) 12.418 (15 | 16-3 15-3 22% (2.6%, 1.7%) 43% (3.4%, 4.8%) 2.0% (2.2%, 1.7%) 43% (3.4%, 4.5%) 2.0% (2.3%, 1.7%) 43% (3.6%, 4.5%) 43% (3.6%, 4.6%) 43% (3.6%, 4.6%) 43% (3.6%, 4.6%) 43% (3.6%, 4.6%) 43% (3.6%, 4.8%) 43% (3.5%, | 14.00 10.00 19.00 10.00 17.00 1391 10.2% 10.0 17.00 1391 10.2% 15.013 13.5 % 15.013 15.0 % 15.013 15.0 % 15.014 17.0 % 15.014 17.0 % 15.015 | 14.00 14.00 19.00 14.02 14.00 14.00 14.02 16.00 14.00 14.02 16.00 14.00 16.00 14.02 16.00 16.00 16.00 14.02 16.00 16.00 16.00 14.02 16.00 16.00 16.00 14.00 16.00 16.00 16.00 14.00 16.00 16.00 16.00 14.00 16.00 16.00 16.00 14.00 16.00 16.00 16.00 15.00 16.00 16.00 16.00 15.00 16.00 16.00 16.00 15.00 16.00 16.00 16.00 15.00 16.00 16.00 16.00 15.00 16.00 16.00 15.00 16.00 16.00 15.00 16.00 16.00 15.00 16.00 16.00 16.00 16.00 16.00 16.00 16.00 16.00 16.00 16.00 16.00 | -(-, -) -(-, - |
| Imedian (IQR) Imit, max Colonoscopy Sigmoidoscopy; n (%) Flu Presumcoccal vaccine; n (%) Flu Presumcoccal vaccine; n (%) Flu Presumcoccal vaccine; n (%) Flu State th n (%) FSA test n (%) | 14.00 [10.00.18.00] 1.00.57.00 2.631 (6.3%) 1.120 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.1320 (3.3%) 1.2550 (9.0%) 2.2550 (9.0%) 2.2550 (9.0%) 2.2550 (9.0%) 2.45 (1.30) 2.00 (1.00.3.00] 0.00,10.00 1.74 (1.2) 2.00 [1.00.2.00] 0.00,2.00 0.00,2.00 0.00,2.00 0.00,2.00 0.00,3.60 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 10.00 5.200 15.90 11.90 15.94 12.529 26.529 5.378 11.948 24.059 24.5270 44.859 43.310 28.779 12.448 25.579 12.419 12.001 10.200 10.00 3.00 | 16.3 22% (2.5%, 1.7%) 2.2% (2.5%, 1.7%) 3.2% (2.5%, 1.7%) 1.8% (2.4%, 1.2%) 1.8% (2.5%, 1.4%) 1.8% (2.5%, 1.2%) 1.8% (2.5%, 1.4%) 1.8% (2.5%, 1.4%) 1.8% (2.5%, 1.4%) 1.8% (2.5%, 1.4%) 1.9% (1.4%, 2.4%) 1.9% (1. | 14.00 10.00 19.00 | 14.00 14.00 19.00 10.00 50.00 14.02 10.01 50.00 14.02 10.3 50.00 14.02 10.00 14. | 1(-, -) 1-(-, -) 1-(-, -) 2-(-) 2-(- |
| Imedian (IQR) Imit; max Colonoscopy Sigmoidoscopy; n (%) File Presumococcal vaccine n (%) File Presumococcal vaccine n (%) Pays antean n (%) Pays antean n (%) Pass teat n (%) Pass teat n (%) Pass teat n (%) Pass teat n (%) Telemedicine; n (%) Hablat tests Imedian (IQR) Imit; max Upid panels Imedian (IQR) Imit; max Imit; max Imedian (IQR) Imit; max Imi | 14-00 [10.00 18.00] 14-00 [10.00 18.00] 14-00 [2.50] 16.01 [2.50] 16.01 [2.50] 16.02 [2.50] 16.03 [2.50] 16.04 [2.50] 16.05 [2.50] | 15.00 11.00, 15.00 10.00 52.00 10.00 52.00 17.564 (15.2%) 17.564 (16.2%) 17.565 (16.2%) 17.566 | 16-3 15-3 22% (2.5%, 1.7%) 14% (2.4%, 1.2%) 14% (2.4%, 1.2%) 14% (2.4%, 1.2%) 1.8% (2.6%, 1.2%) 1.8% ( | 14.00 10.00 19.00 10.00 17.00 130 11.02% 10.00 17.00 130 11.02% 130 13.00 131 12.20% 131 131 131 131 131 131 13 | 14.00 10.00 10.00 10.00 50.00 10 | 1() -(1.5) -(1 |
| Imedian (10R) Imit, max Colonocopy Sigmoidoscopy, n (%) Bit Pheumococcal vaccine n (%) Phys Imean n (%) Bone mineral density tests; n (%) Bone mineral density tests; n (%) Bone mineral density tests; n (%) Imean (s) Imean | 14-00 [10.00.18.00] 1-00.5700 2-631 (6.3%) 1-100.5700 2-631 (6.3%) 1-120 (6.3%) 1-1 | 15.00 11.00, 15.00 10.00 5.200 10.00 5.200 10.00 5.200 15.90 11.500 15.94 12.520 2.559 5.370 11.546 2.64.050 2.570 4.650 1.546 2.650 1.546 2.650 1.546 2.650 1.546 2.650 1.546 2.550 1.546 2.550 | 16.3 22% (2.5%, 1.7%) 2.2% (2.5%, 1.7%) 3.2% (2.5%, 1.7%) 1.8% (2.4%, 1.2%) 1.8% (2.5%, 1.2%) 1.9% (1.4%, 2.4%) 1.9% (1.4%, 2.4%) 1.9% (1.4%, 2.4%) 1.9% (1.2%, 1.2%) 1.9% (1. | 14.00 10.00 19.00 | 14.00 10.00 10.00 10.00 50.00 10 | 1(-, -) 1-(-, -) 2-(-) 2 |

| Appendix 7. Balance Assessment - Table 1 | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN<br>Variable | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference |
| Variable Number of patients Year of Cohort Entry Date | 13,885 | 19,713 | - (-, -) | 6,554 | 6,554 | - (-, -) |
| 2018; n (%) | 3,221 (23.2%) | 386 (2.0%) | 21.2% (20.5%, 22.0%) | 358 (5.5%) | 375 (5.7%) | -0.3% (-1.1%, 0.5%) |
| 2019; n (%)<br>2020; n (%) | 3,234 (23.3%)<br>2,537 (18.3%) | 1,408 (7.1%)<br>1,784 (9.0%) | 16.1% (15.4%, 16.9%)<br>9.2% (8.5%, 10.0%) | 1,118 (17.1%)<br>1,253 (19.1%) | 1,137 (17.3%)<br>1,280 (19.5%) | -0.3% (-1.6%, 1.0%)<br>-0.4% (-1.8%, 1.0%) |
| 202!; n (%)<br>2022; n (%) | 2,127 (15.3%)<br>1,536 (11.1%) | 2,762 (14.0%)<br>4,473 (22.7%) | 1.3% (0.5%, 2.1%)<br>-11.6% (-12.4%, -10.8%) | 1,408 (21.5%)<br>1,269 (19.4%) | 1,436 (21.9%)<br>1,237 (18.9%) | -0.4% (-1.9%, 1.0%)<br>0.5% (-0.9%, 1.8%) |
| 2023; n (%)<br>Age | 1,230 (8.9%) | 8,900 (45.1%) | -36.3% (-37.1%, -35.4%) | 1,148 (17.5%) | 1,089 (16.6%) | 0.9% (-0.4%, 2.2%) |
| mean (sd)median [IQR] | 66.06 (10.01)<br>64.00 [59.00, 74.00] | 60.81 (7.34)<br>60.00 [55.00, 64.00] | 5.25 (5.06, 5.45)<br>- (-, -) | 62.75 (8.67)<br>61.00 [56.00, 68.00] | 62.62 (7.95)<br>61.00 [57.00, 67.00] | 0.14 (-0.15, 0.42) |
| min, max<br>Gender (male); n (%) | 50.00, 99.00<br>7,259 (52.3%) | 50.00, 92.00<br>9,487 (48.1%) | - (-, -)<br>4.2% (3.1%, 5.2%) | 50.00, 96.00<br>3,374 (51.5%) | 50.00, 92.00<br>3,382 (51.6%) | - (-, -)<br>-0.1% (-1.8%, 1.6%) |
| Region / StateNortheast; n (%) | 2,643 (19.0%) | 2,773 (14.1%) | 5.0% (4.1%, 5.8%) | 1,146 (17.5%) | 1,130 (17.2%) | 0.2% (-1.1%, 1.6%) |
| Widwest / North central; n (%)<br>South; n (%) | 4,710 (33.9%)<br>5,858 (42.2%) | 4,640 (23.5%)<br>10,836 (55.0%) | 10.4% (9.4%, 11.4%)<br>-12.8% (-13.9%, -11.7%) | 1,739 (26.5%)<br>3,273 (49.9%) | 1,773 (27.1%)<br>3,257 (49.7%) | -0.5% (-2.1%, 1.0%)<br>0.2% (-1.5%, 2.0%) |
| West n (%)<br>Missing.n (%) | 654 (4.7%)<br>20 (0.1%) | 1,451 (7.4%)<br>13 (0.1%) | -2.7% (-3.2%, -2.1%)<br>0.1% (-0.0%, 0.2%) | 392 (6.0%)<br>4 (0.1%) | 390 (6.0%)<br>4 (0.1%) | 0.0% (-0.8%, 0.9%) |
| Smoking / Tobacco use; n (%) Weight | 1,742 (12.5%) | 2,566 (13.0%) | -0.5% (-1.2%, 0.3%) | 836 (12.8%) | 811 (12.4%) | 0.4% (-0.8%, 1.5%) |
| Underweight; n (%) | 91 (0.7%) | 16 (0.1%) | 0.6% (0.4%, 0.7%) | 16 (0.2%) | 13 (0.2%) | 0.0% (-0.1%, 0.2%) |
| Normal weight; n (%)Overweight; n (%) | 727 (5.2%)<br>2,779 (20.0%) | 159 (0.8%)<br>1,825 (9.3%) | 4.4% (4.0%, 4.8%)<br>10.8% (10.0%, 11.5%) | 124 (1.9%)<br>969 (14.8%) | 125 (1.9%)<br>929 (14.2%) | 0.6% (-0.6%, 1.8%) |
| Class 1 Obesity; n (%)<br>Class 2 Obesity; n (%) | 1,802 (13.0%)<br>901 (6.5%) | 1,777 (9.0%)<br>1,295 (6.6%) | 4.0% (3.3%, 4.7%)<br>-0.1% (-0.6%, 0.5%) | 734 (11.2%)<br>449 (6.9%) | 737 (11.2%)<br>456 (7.0%) | -0.0% (-1.1%, 1.1%)<br>-0.1% (-1.0%, 0.8%) |
| Class 3 Obesity; n (%)<br>Unspecified Obesity; n (%) | 2,892 (20.8%)<br>4,693 (33.8%) | 5,208 (26.4%)<br>9,433 (47.9%) | -5.6% (-6.5%, -4.7%)<br>-14.1% (-15.1%, -13.0%) | 1,726 (26.3%)<br>2,536 (38.7%) | 1,779 (27.1%)<br>2,515 (38.4%) | -0.8% (-2.3%, 0.7%)<br>0.3% (-1.4%, 2.0%) |
| Diabetic retinopathy; n (%) Diabetic neuropathy; n (%) | 1,072 (7.7%)<br>3,233 (23.3%) | 1,333 (6.8%)<br>3,909 (19.8%) | 1.0% (0.4%, 1.5%)<br>3.5% (2.6%, 4.4%) | 488 (7.4%)<br>1,405 (21.4%) | 491 (7.5%)<br>1,437 (21.9%) | -0.0% (-1.0%, 0.9%)<br>-0.5% (-1.9%, 0.9%) |
| Diabetic nephropathy; n (%) Diabetes with other opthalmic complications; n (%) | 2,822 (20.3%)<br>326 (2.3%) | 3,123 (15.8%)<br>373 (1.9%) | 4.5% (3.6%, 5.3%)<br>0.5% (0.1%, 0.8%) | 1,163 (17.7%)<br>155 (2.4%) | 1,142 (17.4%)<br>163 (2.5%) | 0.3% (-1.0%, 1.6%) |
| Diabetes with peripheral circulatory disorders; n (%) Diabetic foot n (%) | 1,409 (10.1%)<br>336 (2.4%) | 1,927 (9.8%)<br>392 (2.0%) | 0.4% (-0.3%, 1.0%)<br>0.4% (0.1%, 0.8%) | 628 (9.6%)<br>146 (2.2%) | 640 (9.8%)<br>145 (2.2%) | -0.2% (-1.2%, 0.8%)<br>0.0% (-0.5%, 0.5%) |
| Erectile dysfunction; n (%) Hypoglycemia: n (%) | 569 (4.1%)<br>1.929 (13.9%) | 883 (4.5%)<br>3,306 (16.8%) | -0.4% (-0.8%, 0.1%)<br>-2.9% (-3.7%, -2.1%) | 299 (4.6%)<br>991 (15.1%) | 301 (4.6%)<br>948 (14.5%) | -0.0% (-0.8%, 0.7%)<br>0.7% (-0.6%, 1.9%) |
| Hyperglycemia/DKA/HONK; n (%) Skin infections: n (%) | 6,649 (47.9%)<br>1.379 (9.9%) | 9,433 (47.9%)<br>1983 (10.1%) | -2.5% (-3.7%, -2.1%)<br>0.0% (-1.1%, 1.1%)<br>-0.1% (-0.8%, 0.5%) | 3,225 (49.2%)<br>661 (10.1%) | 3,270 (49.9%)<br>643 (9.8%) | -0.7% (-2.4%, 1.0%)<br>-0.3% (-0.8%, 1.3%) |
| Stable angina; n (%) | 766 (5.5%) | 1,176 (6.0%) | -0.4% (-1.0%, 0.1%) | 661 (10.1%)<br>373 (5.7%)<br>258 (3.9%) | 368 (5.6%) | 0.1% (-0.7%, 0.9%) |
| Unstable angina; n (%)<br>Hypertension; n (%) | 541 (3.9%)<br>12,558 (90.4%) | 757 (3.8%)<br>17,392 (88.2%) | 0.1% (-0.4%, 0.5%)<br>2.2% (1.5%, 2.9%) | 5,858 (89.4%) | 268 (4.1%)<br>5,892 (89.9%) | -0.2% (-0.8%, 0.5%)<br>-0.5% (-1.6%, 0.5%) |
| Hypotension; n (%) Hyperlipidemia; n (%) | 433 (3.1%)<br>11,872 (85.5%) | 467 (2.4%)<br>16,612 (84.3%) | 0.7% (0.4%, 1.1%)<br>1.2% (0.5%, 2.0%) | 169 (2.6%)<br>5,588 (85.3%) | 170 (2.6%)<br>5,594 (85.4%) | -0.0% (-0.6%, 0.5%)<br>-0.1% (-1.3%, 1.1%) |
| Atrial fibrillation; n (%) Cardiac conduction disorder; n (%) | 1,791 (12.9%)<br>824 (5.9%) | 2,136 (10.8%)<br>1,056 (5.4%) | 2.1% (1.4%, 2.8%)<br>0.6% (0.1%, 1.1%) | 709 (10.8%)<br>324 (4.9%) | 693 (10.6%)<br>314 (4.8%) | 0.2% (-0.8%, 1.3%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%)<br>Ischemic stroke; n (%) | 375 (2.7%)<br>246 (1.8%) | 570 (2.9%)<br>241 (1.2%) | -0.2% (-0.6%, 0.2%)<br>0.5% (0.3%, 0.8%) | 184 (2.8%)<br>98 (1.5%) | 201 (3.1%)<br>93 (1.4%) | -0.3% (-0.9%, 0.3%)<br>0.1% (-0.3%, 0.5%) |
| PVD diagnosis or surgery; n (%) Other cardiac dysrhythmia: n (%) | 1,394 (10.0%)<br>3,091 (22.3%) | 1,427 (7.2%)<br>4,370 (22.2%) | 2.8% (2.2%, 3.4%)<br>0.1% (-0.8%, 1.0%) | 547 (8.3%)<br>1.395 (21.3%) | 558 (8.5%)<br>1,368 (20.9%) | -0.2% (-1.1%, 0.8%)<br>0.4% (-1.0%, 1.8%) |
| Cardiomyopathy; n (%)<br>Valve disorders: n (%) | 925 (6.7%)<br>1,847 (13.3%) | 1,239 (6.3%)<br>2,349 (11.9%) | 0.4% (-0.2%, 0.9%)<br>1.4% (0.7%, 2.1%) | 425 (6.5%)<br>806 (12.3%) | 396 (6.0%)<br>805 (12.3%) | 0.4% (-0.4%, 1.3%) |
| Valve replacement; n (%)<br>TIA; n (%) | 211 (1.5%)<br>460 (3.3%) | 220 (1.1%)<br>544 (2.8%) | 0.4% (0.1%, 0.7%)<br>0.6% (0.2%, 0.9%) | 79 (1.2%)<br>194 (3.0%) | 76 (1.2%)<br>196 (3.0%) | 0.0% (-0.3%, 0.4%) |
| Edema; n (%) Venous thromboembolism / Pulmonary embolism; n (%) | 1,574 (11.3%)<br>474 (3.4%) | 2,280 (11.6%)<br>688 (3.5%) | -0.2% (-0.9%, 0.5%)<br>-0.1% (-0.5%, 0.3%) | 716 (10.9%)<br>215 (3.3%) | 734 (11.2%)<br>209 (3.2%) | -0.3% (-1.4%, 0.8%)<br>0.1% (-0.5%, 0.7%) |
| Pulmonary hypertension; n (%) | 381 (2.7%) | 470 (2.4%) | 0.4% (0.0%, 0.7%) | 158 (2.4%) | 160 (2.4%) | -0.0% (-0.6%, 0.5%) |
| Implantable cardioverter defibrillator; n (%)<br>Hyperkalemia; n (%) | 59 (0.4%)<br>372 (2.7%) | 81 (0.4%)<br>364 (1.8%) | 0.0% (-0.1%, 0.2%)<br>0.8% (0.5%, 1.2%) | 23 (0.4%)<br>145 (2.2%) | 22 (0.3%)<br>138 (2.1%) | 0.0% (-0.2%, 0.2%)<br>0.1% (-0.4%, 0.6%) |
| Coronary atherosclerosis; n (%) | 5,027 (36.2%) | 6,651 (33.7%) | 2.5% (1.4%, 3.5%) | 2,221 (33.9%) | 2,229 (34.0%) | -0.1% (-1.8%, 1.5%) |
| Cerebrovascular procedure; n (%) | 19 (0.1%) | 16 (0.1%) | 0.1% (-0.0%, 0.1%) | 7 (0.1%) | 7 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Cerebrovascular procedure; n (%) Insertion of pacemakers / removal of cardiac lead; n (%) CKD stage 1-2; n (%) | 19 (0.1%)<br>30 (0.2%)<br>473 (3.4%) | 16 (0.1%)<br>17 (0.1%)<br>548 (2.8%) | 0.1% (-0.0%, 0.1%)<br>0.1% (0.0%, 0.2%)<br>0.6% (0.2%, 1.0%) | 7 (0.1%)<br>7 (0.1%)<br>193 (2.9%) | 7 (0.1%)<br>7 (0.1%)<br>196 (3.0%) | 0.0% (-0.1%, 0.1%)<br>0.0% (-0.1%, 0.1%)<br>-0.0% (-0.6%, 0.6%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 30 (0.2%) | 16 (0.1%)<br>17 (0.1%) | 0.1% (-0.0%, 0.1%)<br>0.1% (0.0%, 0.2%) | 7 (0.1%)<br>7 (0.1%) | 7 (0.1%)<br>7 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Insertion of accomakers / removal of cardiac lead; n (%) CKD stage 1-2; n (%) CKD stage 3-4; n (%) Unspecified CKD; n (%) Acute kidney intry, n (%) | 30 (0.2%)<br>473 (3.4%)<br>2,235 (16.1%)<br>626 (4.5%)<br>940 (6.8%) | 16 (0.1%)<br>17 (0.1%)<br>548 (2.8%)<br>2,338 (11.9%) | 0.1% (-0.0%, 0.1%)<br>0.1% (0.0%, 0.2%)<br>0.6% (0.2%, 1.0%)<br>4.2% (3.5%, 5.0%) | 7 (0.1%)<br>7 (0.1%)<br>193 (2.9%)<br>907 (13.8%) | 7 (0.1%)<br>7 (0.1%)<br>196 (3.0%)<br>882 (13.5%) | 0.0% (-0.1%, 0.1%)<br>0.0% (-0.1%, 0.1%)<br>-0.0% (-0.6%, 0.6%)<br>0.4% (-0.8%, 1.6%) |
| Insertion of pacemakers / removal of cardiac lead: n (%) CKO stage 1-2; n (%) CKD stage 3-4; n (%) Unspecified CKD; n (%) | 30 (0.2%)<br>473 (3.4%)<br>2,235 (16.1%)<br>626 (4.5%) | 16 (0.1%)<br>17 (0.1%)<br>548 (2.8%)<br>2.338 (11.9%)<br>618 (3.1%)<br>890 (4.5%) | 0.1% (-0.0%, 0.1%)<br>0.1% (0.0%, 0.2%)<br>0.6% (0.2%, 1.0%)<br>4.2% (3.5%, 5.0%)<br>1.4% (0.9%, 1.8%)<br>2.3% (1.7%, 2.8%) | 7 (0.1%)<br>7 (0.1%)<br>193 (2.9%)<br>907 (13.8%)<br>209 (3.2%)<br>328 (5.0%) | 7 (0.1%)<br>7 (0.1%)<br>196 (3.0%)<br>882 (13.5%)<br>220 (3.4%)<br>355 (5.4%) | 0.0% (-0.1%, 0.1%)<br>0.0% (-0.1%, 0.1%)<br>-0.0% (-0.6%, 0.6%)<br>0.4% (-0.8%, 1.6%)<br>-0.2% (-0.8%, 0.5%)<br>-0.4% (-1.2%, 0.4%) |
| Insertion of accimaleus / removal of cardiac lead; n (%) CXD stage 1.2; n (%) CXD stage 1.4; n (%) CXD stage 3.4; n (%) Unespecified CXD; n (%) Accute kidney lyiny; n (%) Hypertensive nephropathy; n (%) Univary tract infections; n (%) Gential infections; n (%) Gential infections; n (%) | 30 (0.2%)<br>473 (3.4%)<br>2235 (16.1%)<br>626 (4.5%)<br>940 (6.8%)<br>1.569 (11.3%)<br>1.599 (13.0%)<br>517 (3.7%)<br>740 (5.3%) | 16 (01%) 17 (01%) 548 (2.8%) 2.338 (11.9%) 618 (3.1%) 890 (4.5%) 1.636 (8.3%) 2.092 (10.6%) 688 (3.5%) 1.033 (5.2%) | 0.1% (-0.0%, 0.1%) 0.1% (0.0%, 0.2%) 0.1% (0.0%, 0.2%) 0.6% (0.2%, 1.0%) 4.2% (3.5%, 5.0%) 1.4% (0.9%, 1.8%) 2.3% (1.7%, 2.8%) 3.0% (2.3%, 3.7%) 2.4% (1.7%, 3.1%) 0.2% (-0.2%, 0.6%) 0.1% (-0.2%, 0.6%) | 7 (0.1%)<br>7 (0.1%)<br>907 (13.8%)<br>907 (13.8%)<br>907 (13.8%)<br>209 (3.2%)<br>328 (5.0%)<br>608 (9.3%)<br>728 (11.1%)<br>267 (4.1%)<br>342 (5.2%) | 7 (0.1%)<br>7 (0.1%)<br>196 (3.0%)<br>882 (13.5%)<br>822 (13.5%)<br>355 (5.4%)<br>557 (9.1%)<br>729 (11.1%)<br>284 (4.3%)<br>357 (5.4%) | 0.0% (-0.1%, 0.1%)<br>0.0% (-0.1%, 0.1%)<br>-0.0% (-0.6%, 0.6%)<br>-0.4% (-0.8%, 1.6%)<br>-0.2% (-0.8%, 0.5%)<br>-0.4% (-0.8%, 0.5%)<br>0.4% (-1.2%, 0.4%)<br>0.2% (-0.8%, 1.2%)<br>-0.0% (-1.1%, 1.1%)<br>-0.3% (-1.0%, 0.4%)<br>-0.2% (-1.0%, 0.6%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD staps 1-2, n (%) CXD staps 2-4; n (%) CXD staps 2-4; n (%) CXD staps 2-4; n (%) LXD pecified CXD; n (%) Accute kidney injury; n (%) Pypertensive neighregathy; n (%) Pypertensive neighregathy; n (%) Userany tract reflections; n (%) Gental infections; n (%) Userany tract reflections; n (%) CXD pecified | 30 (0.2%)<br>473 (3.4%)<br>2235 (16.1%)<br>626 (4.5%)<br>940 (6.8%)<br>1.569 (11.3%)<br>1.809 (12.0%)<br>517 (3.7%)<br>740 (5.3%)<br>1.238 (6.9%) | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 93 (11.9%) 1618 (3.1%) 1636 (4.5%) 1636 (3.3%) 1637 (6.8%) 1033 (5.2%) 1639 (8.4%) 1272 (1.0%) | 0.196 (-0.0%, 0.1%) 0.196 (0.0%, 0.2%) 0.196 (0.0%, 0.2%) 0.5% (0.2%, 1.0%) 4.2% (3.5%, 5.0%) 4.2% (3.5%, 5.0%) 1.4% (0.9%, 1.8%) 2.3% (1.7%, 2.8%) 3.0% (2.3%, 3.7%) 2.4% (1.7%, 3.1%) 0.2% (-0.2%, 0.6%) 0.196 (-0.4%, 0.6%) 2.1% (5.4%, 1.5%) | 7 (0.1%)<br>7 (0.1%)<br>193 (2.9%)<br>907 (13.8%)<br>209 (3.2%)<br>328 (5.0%)<br>608 (9.3%)<br>728 (11.1%)<br>267 (4.1%)<br>342 (5.2%)<br>594 (9.1%)<br>618 (9.4%) | 7(0.1%) 7(0.1%) 196 (3.0%) 882 (13.5%) 882 (13.5%) 355 (5.4%) 355 (5.4%) 557 (13.1%) 229 (11.1%) 244 (4.2%) 357 (5.4%) 557 (9.1%) | 0.0% (-0.1%, 0.1%)<br>0.0% (-0.1%, 0.1%)<br>0.0% (-0.5%, 0.6%)<br>0.4% (-0.8%, 0.5%)<br>0.2% (-0.8%, 0.5%)<br>0.2% (-0.8%, 0.5%)<br>0.2% (-0.8%, 1.2%)<br>0.0% (-1.1%, 1.1%)<br>0.3% (-1.0%, 0.6%)<br>0.2% (-1.0%, 0.6%)<br>0.3% (-1.0%, 0.6%)<br>0.0% (-1.0%, 0.6%)<br>0.0% (-1.0%, 0.6%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD Stape 1.2, n (%) CXD Stape 1.2, n (%) CXD Stape 2.4, n (%) Unspecified CXD, n (%) Accete Active y large, n (%) Pypecified CXD, n (%) Accete Active y large, n (%) Pypecifiensive neight-postby; n (%) Universal tract infections; n (%) Central infections; n (%) Central infections; n (%) Company and principle of the princi | 30 (0.2%) 473 (3.4%) 473 (3.4%) 4235 (16.1%) 626 (4.5%) 940 (6.8%) 1,569 (11.3%) 1,569 (11.3%) 1,569 (11.3%) 1,569 (13.3%) 1,569 (13.3%) 1,569 (13.3%) 1,569 (13.5%) | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 890 (4.5%) 16.36 (3.3%) 2.092 (10.6%) 688 (3.5%) 1.033 (5.2%) 1.033 (5.2%) 1.033 (3.8%) 2.172 (11.0%) 7.533 (3.8.2%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.5% (0.2% 0.2%) 0.5% (0.2% 1.0%) 4.2% (3.5% 5.0%) 4.2% (3.5% 5.0%) 1.3% (3.5% 5.0%) 2.3% (1.7% 2.8%) 2.3% (1.7% 2.8%) 2.4% (1.7% 3.3%) 0.2% (0.2% 0.6%) 0.1% (0.4% 0.5%) 2.2% (1.2% 3.1%) 2.1% (2.8% 3.1%) 2.1% (2.8% 3.1%) 2.1% (2.8% 3.1%) 2.1% (2.8% 3.1%) | 7(0.1%)<br>7(0.1%)<br>193 (2.9%)<br>907 (13.8%)<br>209 (3.2%)<br>328 (5.0%)<br>608 (9.3%)<br>728 (11.1%)<br>267 (4.1%)<br>342 (5.2%)<br>594 (9.1%)<br>618 (9.4%)<br>2.090 (3.15%)<br>2.291 (3.15%) | 7(0.1%) 7(0.1%) 196 (3.0%) 882 (13.5%) 822 (13.5%) 325 (13.6%) 355 (5.4%) 557 (3.4%) 729 (11.1%) 224 (4.2%) 357 (5.4%) 557 (3.7%) 557 (3.7%) 557 (3.7%) 557 (3.7%) 557 (3.7%) | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.5%, 0.6%) 0.4% (-0.8%, 1.6%) 0.2% (-0.8%, 0.5%) 0.2% (-0.8%, 1.2%) 0.2% (-0.1%, 0.1%) 0.2% (-0.1%, 0.1%) 0.3% (-1.0%, 0.4%) 0.3% (-1.0%, 0.6%) 0.0% (-1.0%, 0.6%) 0.0% (-1.0%, 1.0%) 0.3% (-1.0%, 0.4%) 0.3% (-1.3%, 0.7%) 0.2% (-1.8%, 1.4%) 0.2% (-1.8%, 1.4%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD 61sps 1-2, n (%) CXD 61sps 1-2, n (%) CXD 61sps 2-4, n (%) Unspecified CXD, n (%) Accete kidney history, n (%) Pypecifiend CXD, n (%) Accete kidney history, n (%) Pypecifiend (%) Accete kidney history, n (%) Universal tract infections; n (%) Central infections; n (%) Central infections; n (%) Combas ( | 30 (0.2%) 473 (3.4%) 2.236 (16.1%) 6.05 (4.5%) 940 (6.5%) 940 (6.5%) 1569 (1.3%) 1569 (1.3%) 157 (3.7%) 770 (5.5%) 1500 (10.5%) 1500 (10.5%) 3,613 (5.6%) 783 (5.6%) 783 (5.6%) | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 1636 (3.3%) 2.092 (10.6%) 688 (3.5%) 1,033 (5.2%) 1,033 (5.2%) 1,033 (5.2%) 2,172 (11.0%) 7,533 (3.8.2%) 639 (3.2%) 920 (4.7%) 920 (4.7%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.5% (0.2%) 0.5% (0.2%) 1.0%) 1.2% (0.2%) 1.0%) 1.2% (0.1%) 1.5%) 1.2% (0.1%) 1.5%) 2.3% (1.1%) 2.3% (1.1%) 2.3% (1.1%) 2.3% (1.1%) 2.3% (1.1%) 2.3% (1.1%) 2.3% (1.2%) 3.1%) 0.1% (-0.4%) 0.6%) 0.1% (-0.4%) 0.6%) 0.1% (-0.4%) 0.6%) 1.2% (1.2%) 1.12%) 1.5% (1.1%) 2.2% (1.2%) 1.12%) 1.5% (1.1%) 2.0%) 1.12%) 1.5% (1.1%) 0.5%) 1.5% | 7(0.1%) 7(0.1%) 193 (2.9%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 328 (5.0%) 608 (9.3%) 728 (11.1%) 342 (5.2%) 544 (9.1%) 618 (9.4%) 209 (33.1%) 21 (3.4%) 22 (3.4%) 314 (4.8%) 324 (4.9%) | 7(0.1%) 7(0.1%) 196 (3.0%) 882 (13.5%) 220 (2.4%) 355 (5.4%) 557 (9.1%) 729 (111%) 284 (4.3%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 244 (3.6%) 245 (3.6%) 246 (3.6%) 247 (3.6%) | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.6%, 0.6%) 0.0% (-0.8%, 1.6%) 0.2% (-0.8%, 1.5%) 0.2% (-0.8%, 1.5%) 0.2% (-0.1%, 1.2%) 0.0% (-1.1%, 1.1%) 0.3% (-1.0%, 0.6%) 0.3% (-1.0%, 0.6%) 0.2% (-1.0%, 1.0%) 0.2% (-1.0%, 1.0%) 0.2% (-1.8%, 1.4%) 0.2% (-1.8%, 1.4%) 0.2% (-0.8%, 0.4%) 0.2% (-0.8%, 0.4%) |
| Insention of accemakers / removal of cardiac lead; n (%) CXD stage 3-1; n (%) CXD stage 3-4; n (%) Unspecified CXD; n (%) Unspecified CXD; n (%) Hypertensive nephropathy; n (%) Unray fract infections; n (%) Genital infections; n (%) Unray fract infections; n (%) Genital infections; n (%) CXP (XI) CX | 30 (0.2%) 473 (3.4%) 473 (3.4%) 473 (3.4%) 474 (3.4%) 474 (3.4%) 475 (3.4%) 476 (3.5%) 477 (3.5%) 4 | 16 (01%) 17 (0.1%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 518 (3.1%) 890 (4.5%) 16.36 (3.3%) 2.092 (0.6%) 688 (3.5%) 1.033 (5.2%) 1.033 (5.2%) 1.033 (5.2%) 539 (3.2%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.5% 1.1%) 2.3% (1.1% 2.8%) 2.3% (1.1% 2.8%) 2.3% (1.1% 2.8%) 2.3% (2.1% 2.8%) 2.4% (1.1% 3.1%) 0.2% (0.2% 0.6%) 0.1% (0.4% 0.6%) 2.2% (1.2% 3.1%) 1.5% (1.1% 2.0%) 1.5% (0.5% 1.1%) 1.5% (1.1% 2.0%) 1.5% (1.5% 1.5%) 1.2% (2.2% 1.1%) 2.3% (2.2% 1.1%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 328 (5.0%) 328 (1.0%) 329 (1.0%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 344 (4.5%) 344 (4.5%) 344 (4.5%) 344 (4.5%) | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.12.5%) 220 (2.4%) 355 (5.4%) 355 (5.4%) 575 (11%) 729 (11%) 284 (4.3%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 220 (3.6%) 235 (5.0%) 325 (5.0%) 325 (5.0%) 325 (5.0%) 325 (5.0%) 345 (3.5%) 545 (3.3%) | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.5%) 0.4% (-1.2%, 0.4%) 0.2% (-0.8%, 0.5%) 0.4% (-1.2%, 0.4%) 0.3% (-1.3%, 0.1%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.2% (-1.0%, 0.6%) 0.2% (-1.2%, 0.7%) 0.2% (-1.2%, 0.7%) 0.2% (-1.2%, 0.7%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD stage 1.2, n (%) CXD stage 1.2, n (%) CXD stage 2.4, n (%) Unspecified CXD, n (%) Accele kidney highly; n (%) Psyspectree of the property of the | 30 (0.2%) 473 (3.4%) 473 (3.4%) 473 (3.4%) 474 (3.4%) 474 (3.4%) 475 (3.4%) 476 (3.5%) | 16 (01%) 17 (0.1%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 850 (4.5%) 618 (3.1%) 850 (4.5%) 1.033 (5.2%) 1.033 (5.2%) 1.033 (5.2%) 1.033 (5.2%) 639 (3.2%) 920 (4.7%) 639 (3.2%) 920 (4.7%) 1.817 (9.2%) 802 (4.1%) 460 (2.3%) 5,338 (27.1%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.18%) 2.3% (1.7% 2.8%) 0.3% (2.3% 3.7%) 2.4% (1.7% 3.1%) 0.2% (-0.4% 0.6%) 0.1% (-0.4% 0.6%) 0.2% (-0.2% 0.5%) 0.1% (-0.2% 0.5%) 0.1% (-0.2% 0.5%) 0.2% (-0.2% 0.5%) 0.6% (0.2% 0.9%) 0.6% (0.2% 0.9%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 328 (5.0%) 328 (13.8%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 548 (9.4%) 229 (3.4%) 320 (4.4%) 334 (4.5%) 334 (4.5%) 160 (2.4%) 160 (2.4%) | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.12.5%) 220 (3.4%) 355 (5.4%) 355 (5.4%) 575 (11%) 779 (11%) 244 (4.3%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 220 (3.6%) 533 (14.2%) 545 (3.8%) 353 (14.2%) 545 (3.8%) 195 (2.5%) 195 (3.5%) 196 (2.5%) 196 (2.5%) 196 (2.5%) | 0.0% (-0.1%, 0.1%) 0.0% (-1.1%, 0.1%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.2% (-1.0%, 0.6%) 0.2% (-1.0%, 0.6%) 0.2% (-1.0%, 0.6%) 0.2% (-1.2%, 0.1%) 0.2% (-0.5%, 0.6%) 0.2% (-0.6%, 0.6%) |
| Insertion of accimaleus / removal of cardiac lead; n (%) CKD stage 3-2; n (%) CKD stage 3-4; n (%) Unspecified CKD; n (%) Unspecified CKD; n (%) Hypertensive nephropathy; n (%) Hypertensive nephropathy; n (%) Unspecified CKD; n (%) Gential infections; n (%) Unsay fact infections; n (%) Unsay fact infections; n (%) Unsay fact infections; n (%) Gential infections; n (%) Gential infections; n (%) Undithasis (Kdney and uninary stone); n (%) Setious bacterial infections; n (%) Presumonia; n (%) Presumonia; n (%) Unwer desease n (%) MASHMASID n (%) Fractures / Falls; n (%) Fractures / Falls; n (%) | 30 to 2% 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (16.1%) 626 (4.5%) 940 (16.8%) 1.559 (11.3%) 1.559 (11.3%) 1.559 (11.3%) 1.509 (13.0%) 517 (3.7%) 740 (5.3%) 1.506 (10.8%) 1.536 (16.8%) 1.536 (16.8%) 1.538 (16.8%) 1.506 (16.8%) 1.506 (16.8%) 1.507 (16.8%) 1.508 (16.8%) | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 1.636 (8.3%) 2.032 (10.6%) 688 (3.5%) 1.630 (8.4%) 2.172 (10.0%) 639 (3.2%) 920 (4.7%) 2.955 (15.0%) 1.817 (9.2%) 802 (4.1%) 802 (4.1%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 1.4% (0.9% 1.8%) 1.4% (0.9% 1.8%) 1.4% (0.9% 1.8%) 1.0% (1.2% 0.6%) 1.0% (1.2% 0.6%) 1.0% (1.2% 0.6%) 1.0% (1.2% 0.6%) 1.1% (1.2% 0.1%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.2% (2.0% 0.5%) 1.2% (2.0% 0.5%) 1.2% (2.0% 0.5%) 1.2% (2.0% 0.5%) 1.2% (2.0% 0.5%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.3%) 209 (3.3%) 228 (5.0%) 608 (9.3%) 227 (4.1%) 342 (5.2%) 524 (9.1%) 618 (9.4%) 227 (3.4%) 314 (4.8%) 920 (14.0%) 334 (4.6%) 304 (4.6%) | 7(0.1%) 7(0.1%) 196 (3.0%) 882 (13.5%) 20 (3.4%) 355 (5.4%) 597 (9.1%) 797 (111%) 224 (4.2%) 357 (5.4%) 357 (6.4%) 377 (6.4%) 377 (6 | 0.9% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.2% (-0.8%, 0.5%) 0.2% (-0.8%, 0.5%) 0.2% (-0.8%, 1.5%) 0.2% (-0.8%, 1.2%) 0.2% (-0.1%, 1.5%) 0.3% (-1.1%, 0.1%) 0.3% (-1.1%, 0.1%) 0.3% (-1.1%, 0.1%) 0.3% (-1.1%, 0.1%) 0.2% (-1.1%, 0.1%) |
| Insertion of accimaleus / removal of cardiac lead; n (%) CKD stage 3-2; n (%) CKD stage 3-4; n (%) Unspecified CKD; n (%) Acute kidney intry, n (%) Hypertensive nephropathy; n (%) Hypertensive nephropathy; n (%) Unspecified CKD; n (%) Gential infections; n (%) Unsay fact infections; n (%) Unsay fact infections; n (%) Undithasis (Kdone) and uninary stone); n (%) COPD; n (%) Asthmar, n (%) Obstructive sleep apnex; n (%) Precurroniz; n (%) Precurroniz; n (%) Precurroniz; n (%) Fractures / Fallis; n (%) Osteoporosis; n (%) Osteoporosis; n (%) Osteoporosis; n (%) Osteoporosis; n (%) Osteoporosis; n (%) | 30 to 2% 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (16.8%) 1.569 (11.3%) 1.569 (11.3%) 1.569 (11.3%) 1.569 (11.3%) 1.569 (11.3%) 1.57 (3.7%) 740 (5.3%) 1.59 (11.3%) | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 1.636 (8.3%) 2.092 (10.6%) 688 (3.5%) 1.635 (8.2%) 1.635 (8.2%) 1.635 (8.2%) 1.635 (8.2%) 1.636 (8.3%) 2.172 (11.0%) 7.533 (3.8.2%) 6.39 (3.2%) 9.20 (4.7%) 2.955 (15.0%) 1.817 (9.2%) 802 (4.1%) 802 (4.1%) 802 (4.1%) 803 (4.1%) 804 (4.1%) 805 (4.1%) 805 (4.1%) 806 (2.3%) 8,338 (27.1%) 8,338 (27.1%) 8,338 (27.1%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.6% (0.2%) 1.0%) 0.6% (0.2%) 1.0%) 1.4% (0.9%) 1.8%) 1.4% (0.9%) 1.8%) 1.4% (0.9%) 1.8%) 1.4% (0.9%) 1.8% 1.0% (0.2%) 0.6%) 1.0% (0.2%) 0.6%) 1.0% (0.2%) 0.6%) 1.0% (0.2%) 0.6%) 1.2% (1.2%) 1.1%) 1.5% (1.1%) 2.0%) 1.5% (1.1%) 2.0% 1.5% (1.5%) 1.5%) 1.2% (1.2%) 0.5%) 1.2% (1.2%) 1.5%) 1.2% (1.2%) 0.5%) 1.2% (1.2%) 0.5%) 1.3% (1.2%) 0.9%) 1.3% (1.2%) 0.9%) 1.3% (1.2%) 0.9%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 907 (13.8%) 907 (13.8%) 328 (5.0%) 608 (9.3%) 328 (5.0%) 608 (9.3%) 728 (11.1%) 227 (4.1%) 342 (5.2%) 554 (9.1%) 342 (5.2%) 342 (5.2%) 344 (4.8%) 344 (4.8%) 930 (4.6%) 160 (2.4%) 160 (2.4%) | 7(0.1%) 7(0.1%) 196 (3.0%) 882(13.5%) 220 (3.4%) 335(15.4%) 537(19.1%) 729 (11.1%) 224 (4.2%) 357 (5.4%) 358 (5.6%) 333 (14.2%) 345 (5.6%) 333 (14.2%) 345 (3.3%) 1616 (2.4.7%) 1638 (2.4.7%) | 0.9% (-1.1%, 0.1%) 0.0% (-1.1%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-0.8%, 0.5%) 0.2% (-0.8%, 1.5%) 0.2% (-0.8%, 1.5%) 0.2% (-0.8%, 1.2%) 0.3% (-1.1%, 1.1%) 0.3% (-1.1%, 0.1%) 0.3% (-1.3%, 0.7%) 0.3% (-1.3%, 0.7%) 0.2% (-0.8%, 0.4%) 0.2% (-0.8%, 0.4%) 0.2% (-0.4%, 0.1%) 0.2% (-0.4%, 0.1%) 0.2% (-0.4%, 0.1%) 0.2% (-0.4%, 0.1%) 0.2% (-0.4%, 0.1%) 0.3% (-0.4%, 0.1%) |
| Insertion of accomaleus / removal of cardiac lead; n (%) CXD stage 1.2 n (%) CXD stage 1.2 n (%) CXD stage 3.4; n (%) Unespecified CXD; n (%) Acute lichney interpretation of the stage of | 30 to 2% 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (6.5%) 16.0% | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 1.636 (8.3%) 1.636 (8.3%) 1.636 (8.3%) 1.637 (8.3%) 1.639 (8.3%) 1.639 (8.3%) 1.639 (8.3%) 1.650 (8.4%) 1.650 (8.4 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.5% (0.2%) 0.3% (0.2%) 0.5% (0.5%) | 7(0.1%) 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 907 (13.8%) 907 (13.8%) 328 (5.0%) 608 (9.3%) 328 (5.0%) 608 (9.3%) 728 (11.1%) 926 (74.1%) 342 (5.2%) 924 (9.1%) 618 (9.4%) 342 (6.2%) 344 (4.8%) 934 (4.8%) 934 (4.8%) 934 (4.8%) 934 (4.8%) 934 (4.8%) 936 (13.6%) 160 (2.4%) 160 (2.4%) 160 (2.4%) | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 220 (3.4%) 220 (3.4%) 355 (5.4%) 597 (9.1%) 729 (111%) 224 (4.3%) 357 (5.4%) 597 (9.1%) 637 (9.7%) 2,105 (3.21%) 234 (3.6%) 325 (5.0%) 333 (4.2%) 545 (8.3%) 246 (3.3%) 164 (2.5%) 164 (2.5%) 165 (2.4%) 165 (2.4%) | 0.9% (-13%, 0.1%) 0.0% (-13%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.5%) 0.4% (-1.0%, 0.5%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.3% (-1.3%, 0.1%) 0.3% (-1.3%, 0.4%) 0.2% (-1.3%, 0.5%) 0.3% (-1.3%, 0.5%) 0.3% (-1.3%, 0.5%) 0.3% (-1.3%, 0.5%) 0.3% (-1.3%, 1.5%) 0.3% (-1.3%, 1.5%) 0.3% (-1.3%, 1.5%) 0.3% (-1.3%, 1.5%) 0.3% (-1.3%, 1.5%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD stage 1.2, n (%) CXD stage 2.4; n (%) CXD stage 3.4; n (%) Line pecified CXD; n (%) Accute kidney injury, n (%) Hypertensive neightropathy; n (%) Hypertensive neightropathy; n (%) Usinary fract infections; n (%) Gential infections; n (%) CoPto, n (%) Asthmar, n (%) Obstructive sleep apnea; n (%) Serious bacterial infections; n (%) Pneumonia; n (%) MASHMASLD; n (%) Pneumonia; n (%) MASHMASLD; n (%) Determents; n (%) Anexis, n (%) Anexis, n (%) Anexis, n (%) Anexis, n (%) | 30 (0.2%) 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (6.5%) 940 (6.5%) 1.569 (11.3%) 1.569 (11.3%) 1.569 (13.5%) 1.57 (3.7%) 740 (5.3%) 1.509 (10.5%) 1.517 (3.7%) 740 (5.3%) 1.509 (10.5%) 1.517 (3.7%) 740 (5.3%) 1.509 (10.5%) 1.50 | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 549 (2.8%) 890 (4.5%) 16.36 (3.1%) 890 (4.5%) 16.36 (3.9%) 2.092 (0.6%) 688 (3.5%) 1.033 (5.2%) 1.034 (1.7%) 1.055 (1.5%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.5% 1.0%) 1.2% (1.1% 2.8%) 1.3% (0.5% 1.0%) 1.4% (0.5% 1.0%) 1.4% (0.5% 1.0%) 1.4% (0.1% 2.8%) 1.4% (0.1% 2.8%) 1.5% (0.6%) 1.5% (0.4% 0.6%) 1.5% (0.4% 0.6%) 1.5% (0.4% 0.6%) 1.5% (0.5% 1.1%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.5% 1.5%) 1.5% (1.5% | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 907 (13.8%) 907 (13.8%) 328 (5.0%) 608 (9.3%) 728 (11.1%) 328 (5.0%) 608 (9.3%) 728 (11.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 344 (4.8%) 344 (4.8%) 344 (4.8%) 344 (4.8%) 160 (2.4%) | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.13.5%) 220 (2.4%) 355 (5.4%) 355 (5.4%) 557 (9.1%) 357 (5.4%) 557 (9.1%) 198 (4.4.3%) 357 (5.4%) 557 (9.1%) 198 (4.3.5%) 244 (3.6%) 325 (5.0%) 325 (5.0%) 325 (5.0%) 325 (5.0%) 325 (5.0%) 326 (5.0%) 326 (5.0%) 327 (5.4%) 327 (5.4%) 328 (5.4%) 328 (5.4%) 329 (5.4%) 329 (5.4%) 320 (5.4%) 320 (5.4%) 321 (5.5%) 322 (5.4%) 323 (6.2%) 324 (5.5%) 325 (5.5%) 325 (5.5%) 326 (5.5%) 327 (5.5%) 327 (5.5%) 328 (5.5%) 329 (5.5%) | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.2% (-0.8%, 0.5%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.3% (-1.0%, 0.5%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.2% (-1.0%, 0.5%) 0.3% (-0.4%, 1.0%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXO stage 2, 4; n (%) CXO stage 3, 4; n (%) Liva pecified CXCn (%) Accele kidney injury n (%) Hypertensive neighropathy; n (%) Hypertensive neighropathy; n (%) Urrany tract infloredors; n (%) Gential infections; n (%) Gential infections; n (%) CXPD: n (%) Asthma; n (%) CXPD: n (%) Asthma; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Pheumonia; n (%) MASH/MASLD: n (%) Pheumonia; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Distructive sleep apnea; n (%) Demension n (%) Demension n (%) Demension n (%) Demension n (%) Arnein; n (%) Arnein; n (%) Arnein; n (%) Infinium n ( | 30 (0.2%) 473 (3.4%) 2.23 (6.6.1%) 6.26 (4.5%) 9.10 (6.6%) 1.559 (1.3%) 1.559 (1.3%) 1.559 (1.3%) 1.559 (1.3%) 1.510 (1.3% | 16 (01%) 17 (0.1%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 16.36 (3.3%) 2.052 (0.6%) 688 (3.5%) 1.033 (5.2%) 1.034 (5.2%) 1.034 (1.7%) 1.034 (1.7%) 1.034 (1.7%) 1.05 (0.5%) 1.05 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.18%) 2.3% (1.7% 2.8%) 2.3% (1.7% 2.8%) 2.3% (1.7% 2.8%) 0.1% (0.4% 0.6%) 2.4% (1.2% 3.1%) 0.1% (0.4% 0.6%) 2.2% (1.2% 0.6%) 0.1% (0.4% 0.6%) 2.2% (1.2% 0.5%) 0.1% (0.4% 0.6%) 2.2% (1.2% 0.5%) 0.1% (0.0% 0.5%) 1.5% (1.1% 0.5%) 1.5% (1.1% 0.5%) 1.5% (1.1% 0.5%) 1.5% (1.5% 0.5%) 0.5% (0.5% 0.5%) 0.5% (0.5% 0.9%) 1.8% (2.2% (1.0%) 1.3% (2.2% 1.7%) 2.7% (1.5% 0.9%) 1.8% (2.5% 1.0%) 0.7% (0.5% 0.9%) 1.8% (2.5% 1.0%) 0.7% (0.5% 0.9%) 0.7% (0.5% 0.0%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 328 (5.0%) 329 (2.0%) 329 (2.0%) 342 (5.2%) 342 (5.2%) 342 (5.2%) 342 (5.2%) 343 (4.0%) 344 (4.0%) 344 (4.0%) 344 (4.0%) 344 (4.0%) 344 (4.0%) 344 (4.0%) 345 (2.4%) 346 (2.4%) 346 (2.5%) 348 (2.5%) 348 (3.0%) 349 ( | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.12.5%) 220 (3.4%) 355 (5.4%) 355 (5.4%) 355 (7.9%) 357 (5.4%) 357 (5.4%) 357 (5.4%) 357 (3.1%) 197 (3.1%) 198 (4.3.5%) 199 (3.1%) 1 | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.2% (-0.8%, 0.5%) 0.4% (-1.2%, 0.4%) 0.2% (-0.8%, 0.5%) 0.4% (-1.2%, 0.4%) 0.2% (-1.0%, 0.1%) 0.3% (-1.3%, 0.1%) 0.2% (-0.1%, 0.1%) 0.3% (-1.3%, 0.7%) 0.2% (-0.1%, 0.1%) 0.3% (-0.1%, 0.1%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD staps 2,4; n (%) CXD staps 3,4; n (%) CXD staps 2,4; n (%) CXD staps 3,4; n (%) CXD staps 3,4; n (%) CXD staps 3,4; n (%) CXD staps 4,4; | 30 (0.2%) 473 (3.4%) 2.235 (16.1%) 6.26 (4.5%) 9.10 (6.6%) 9.10 (6.6%) 1.565 (1.13%) 1.565 (1.13%) 1.565 (1.13%) 1.565 (1.13%) 1.57 (3.7%) 7.10 (5.3%) 1.506 (1.0.6%) 1.507 (1.0.6%) 1.508 | 16 (01%) 17 (0.1%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 589 (4.5%) 589 (4.5%) 589 (4.5%) 1,033 (5.2%) 1,034 (1.5%) 1,044 (1.5%) 1,044 (1.5% | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.18%) 2.3% (1.1% 2.8%) 1.4% (0.9% 1.18%) 2.3% (1.1% 2.8%) 0.3% (2.3% 3.7%) 2.4% (1.1% 3.1%) 0.2% (-0.2% 0.6%) 0.1% (-0.4% 0.6%) 0.1% (-0.2% 0.5%) 1.2% (-2.5% 1.1%) 1.3% (-2.5% 1.1%) 1. | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 328 (5.0%) 329 (13.8%) 342 (5.2%) 344 (5.2%) 344 (6.3%) 344 (6.3%) 345 (6.3%) 344 (6.3%) 345 (6.3%) 346 (6.3%) 346 (6.3%) 347 (6.3%) 348 (6.3%) 348 (6.3%) 349 (6.3%) 349 (6.3%) 340 | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 198 (3.0%) 198 (2.1.2.5%) 220 (3.4.%) 355 (5.4.%) 355 (5.4.%) 357 (9.1%) 729 (11.1%) 224 (4.3.%) 357 (5.4.%) 557 (9.1.%) 637 (9.1.%) 638 | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.2% (-0.2%, 0.1%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.4% (-1.2%, 0.4%) 0.5% (-1.2%, 0.1%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.2% (-1.2%, 0.4%) 0.2% (-1.2%, 0.5%) 0.2% (-1.2%, 0.5%) 0.2% (-1.4%, 1.0%) 0.2% (-1.2%, 0.5%) 0.2% (-1.4%, 1.0%) 0.2% (-1.2%, 0.5%) 0.3% (-1.4%, 1.0%) 0.3% (-1.4%, 0.5%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD stage 1-2; n (%) CXD stage 1-2; n (%) CXD stage 1-2; n (%) CXD stage 1-2; n (%) CXD stage 2-4; n (%) LYD pecified CXD; n (%) Acute kidney injury, n (%) Hypertensive neighropathy; n (%) Hypertensive neighropathy; n (%) LYD stage 1-2; n (%) Gental infections; n (%) LYD stage 1-2; n (%) | 30 (0.2%) 473 (3.4%) 2.236 (16.1%) 2.237 (16.1%) 2.237 (16.1%) 2.238 (16 | 16 (01%) 17 (01%) 18 (12%) 18 (28%) 18 (28%) 18 (21%) 18 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 2.3% (1.1% 2.8%) 2.3% (1.1% 2.8%) 2.3% (1.1% 2.8%) 2.3% (2.1% 2.8%) 2.4% (0.1% 3.1%) 2.4% (0.1% 3.1%) 2.4% (0.1% 3.1%) 2.4% (0.1% 3.1%) 2.1% (2.2% 0.6%) 0.1% (0.4% 0.6%) 0.1% (0.4% 0.6%) 0.1% (0.4% 0.6%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.2% 0.5%) 1.2% (2.0% 0.5%) 1.2% (2.0% 0.5%) 1.3% (2.5% 1.1%) 1.3% (2.5% 1.1%) 1.3% (2.5% 1.1%) 1.3% (2.5% 1.3%) 1.5% (1.5% 0.9%) 1.5% (2.5% 1.0%) 3.3% (2.9% 3.7%) 0.7% (0.5% 0.9%) 1.5% (2.5% 4.2%) 2.7% (1.3% 3.5%) 0.3% (0.0% 0.5%) 3.3% (2.9% 3.5%) 0.3% (1.9% 0.0%) 0.3% (1.2% 0.0%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 328 (5.0%) 329 (1.0%) 329 (1.0%) 320 ( | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.1.3.5%) 20 (3.4.%) 355 (5.4.%) 357 (5.4%) 357 (5.4%) 357 (5.4%) 357 (5.4%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 220 (3.8.%) 325 (5.0%) 933 (14.2%) 933 (14.2%) 933 (14.2%) 934 (14.2%) 934 (14.2%) 195 (2.4.%) 195 (2.4.%) 195 (2.4.%) 195 (2.4.%) 195 (2.4.%) 196 (2.5.%) 197 (2.5.%) 197 (2.5.%) 197 (2.5.%) 198 (3.3.%) 199 (3.3.%) 199 (3.3.%) 199 (3.3.%) 199 (3.3.%) 199 (3.3.%) | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.2% (-0.8%, 0.5%) 0.4% (-1.2%, 0.4%) 0.2% (-1.2%, 0.5%) 0.2% (-1.4%, 0.5%) 0.3% (-1.6%, 0.5%) 0.3% (-1.6%, 0.5%) 0.3% (-1.6%, 0.5%) 0.3% (-1.6%, 0.5%) 0.3% (-1.6%, 0.5%) 0.3% (-1.5%, 0.6%) |
| Insention of accimalisms / removal of cardiac lead; n (%) CKD stage 3-4; n (%) CKD stage 3-4; n (%) Unspecified CKD; n (%) Unspecified CK | 30 (0.2%) 473 (3.4%) 2.236 (16.1%) 2.237 (16.1%) 2.237 (16.1%) 2.238 (16 | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.2%) 184 (3.2%) 185 (3.3%) 185 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.1% (0.4% 0.6%) 0.1% (-0.4% 0.6%) 0.1% (-0.4% 0.6%) 1.2% (-2.2% 1.1.2%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.3% (-2.0% 0.0%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (12.8%) 209 (3.2%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 344 (4.6%) 160 (2.4%) 160 ( | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.13.5%) 20 (3.4%) 355 (5.4%) 355 (5.4%) 357 (5.4%) 357 (6.4%) 358 (6.4%) 358 (6.4%) 358 (6.4%) 358 (6.4%) 369 | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.0%) 0.3% (-1.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD stage 1-2; n (%) CXD stage 1-2; n (%) CXD stage 1-2; n (%) CXD stage 1-2; n (%) CXD stage 2-4; n (%) LXD specified CXD; n (%) Acute kidney injury, n (%) Hypertensive neight-repairty, n (%) LYD specified CXD; n (%) LYD specified LYD spec | 30 (0.2%) 473 (3.4%) 2.236 (16.1%) 6.256 (4.5%) 940 (6.6%) 940 (6.6%) 1569 (11.3%) 1569 (11.3%) 1569 (11.3%) 157 (3.7%) 740 (5.3%) 1509 (10.6%) 157 (3.7%) 750 (5.3%) 1500 (10.5%) 1500 (10 | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 183 (3.1%) 1850 (4.5%) 1636 (3.3%) 1636 (3.3%) 1636 (3.3%) 1636 (3.3%) 1636 (3.3%) 1637 (3.2%) 1638 (3.5%) 1638 (3.5%) 1638 (3.5%) 1639 (3.2%) 1650 (3.4%) 2.172 (11.0%) 7.533 (38.2%) 639 (3.2%) 920 (4.7%) 2.955 (15.0%) 1817 (9.2%) 920 (4.1%) 460 (2.3%) 3.340 (17.3%) 3.402 (17.3%) 3.402 (17.3%) 3.403 (17.3%) 3.41 (1.7%) 105 (0.5%) 3.24 (1.6%) 3.499 (17.7%) 324 (1.6%) 4.980 (2.3.3%) 3.499 (17.7%) 324 (1.6%) 4.980 (2.3.3%) 3.902 (19.8%) 5 (0.0%) 742 (3.3.8%) 4 99 (0.2%) 11 (0.1%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 1.2% (1.7% 2.6%) 1.4% (0.9% 1.8%) 2.3% (1.7% 2.6%) 0.1% (0.4% 0.6%) 0.1% (0.5% 1.5%) 1.2% (2.2% 1.1%) 1.2% (2.2% 1.1%) 1.2% (2.0% 0.5%) 0.5% (0.5% 0.9%) 0.5% (0.5% 0.9%) 0.5% (0.5% 0.9%) 0.3% (0.2% 0.7%) 0.3% (0.2% 0.7%) 0.3% (0.0% 0.6%) 0.3% (0.0% 0.0%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (12.8%) 209 (3.2%) 328 (5.0%) 342 (5.2%) 344 (4.6%) 160 (2.4%) 160 (2.4%) 160 (2.5%) 160 (2.4%) 160 (3.6%) 160 (2.4%) 160 (3.6%) 160 (2.4%) 172 (2.4%) 183 (2.8%) 183 (2.8%) 183 (2.8%) 183 (2.8%) 183 (2.8%) 183 (2.8%) 183 (2.8%) 184 (2.8%) 185 (2.3%) | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.13.5%) 20 (3.4%) 355 (5.4%) 557 (9.1%) 357 (5.4%) 557 (9.1%) 357 (5.4%) 557 (9.1%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 224 (3.6%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 224 (3.6%) 357 (5.4%) 557 (9.1%) 198 (1.1%) 198 | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.0% (-0.0%, 0.0%) |
| Insertion of accomaleus / removal of cardiac lead; n (%) CXD stage 1.2 n (%) CXD stage 2.4; n (%) Use pecified CXD; n (%) Acute kidney inty; n (%) Use pecified CXD; n (%) Acute kidney inty; n (%) Hypertensive nephropathy; n (%) Usery tract intections; n (%) Gential infections; n (%) Gential infections; n (%) Usery tract intections; n (%) COPD; n (%) Asthmar, n (%) Obstructive sleep apnex; n (%) Serious bacterial infections; n (%) Presumonis; n (%) Distructive sleep apnex; n (%) Asthmar, n (%) Distructive sleep apnex; n (%) Serious bacterial infections; n (%) Presumonis; n (%) Distructive sleep apnex; n (%) MASHMASI, n (%) Fractures; Fallis; n (%) Osteoprosis; n (%) Demorris; n (%) Sleep disorders; n (%) Annierz; n (%) Innierz; n (%) Innierz; n (%) Innierz; n (%) Billiany disease; n (%) Billiany disease; n (%) Billiany disease; n (%) Bowel obstruction; n (%) | 30 (0.2%) 473 (3.4%) 2.236 (16.1%) 6.256 (4.5%) 940 (6.6%) 940 (6.6%) 940 (6.6%) 1.5650 (11.3%) 1.5650 (11.3%) 1.5650 (11.3%) 1.576 (11.3%) 1.577 (11.3%) 1. | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.1%) 183 (3.2%) 184 (3.2%) 185 (3.3%) 185 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.2% (1.1% 2.6%) 1.1% (0.4% 0.6%) 0.1% (-0.4% 0.6%) 0.1% (-0.4% 0.6%) 1.2% (-2.2% 1.1.2%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.5% (1.1% 2.0%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.3% (-2.0% 0.0%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (12.8%) 209 (3.2%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 342 (5.2%) 524 (3.1%) 344 (4.6%) 160 (2.4%) 304 (4.6%) 160 (2.4%) 160 (2.4%) 160 (2.5%) 160 (2.4%) 160 (2.4%) 160 (2.5%) 161 (3.5%) 162 (2.4%) 163 (6.5%) 164 (6.5%) 165 (2.4%) 165 ( | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.13.5%) 20 (3.4%) 355 (5.4%) 355 (5.4%) 357 (5.4%) 357 (6.4%) 358 (6.4%) 358 (6.4%) 358 (6.4%) 358 (6.4%) 369 | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.0%) 0.3% (-1.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) |
| Insention of accomalies is removal of cardiac lead; n (%) CXD stage 12, et (%) CXD stage 12, et (%) CXD stage 3.4; n (%) Unespecified CXD; n (%) Acute lichny injury n (%) Hypertensive nephropathy; n (%) Hypertensive nephropathy; n (%) Univary tract infections; n (%) Gential infections; n (%) Gential infections; n (%) Univary tract infections; n (%) Gential infections; n (%) Gential infections; n (%) Gential infections; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Preumonia; n (%) Distructive sleep apnea; n (%) Fractures / Falls; n (%) Distructive sleep apnea; n (%) Fractures / Falls; n (%) Distructive sleep apnea; n (%) Fractures / Falls; n (%) Demonstratifis; n (%) Sleep disorders; n (%) Annelin; n (%) Influenz; n (%) Influenz; n (%) Influenz; n (%) Billiany deesse; n (%) Bi | 30 (0.2%) 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (6.5%) 940 (6.5%) 1.669 (11.3%) 1.669 (11.3%) 1.669 (11.3%) 1.669 (11.3%) 1.670 | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 1636 (8.3%) 890 (4.5%) 1636 (8.3%) 1637 (8.3%) 1638 (8.3%) 1633 (5.2%) 1639 (3.2%) 1640 (1.3%) 1650 (5.5%) 1650 (3.3%) 1650 ( | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.1% (0.4%) 0.6% (0.2%) 0.1% (0.4%) 0.6% (0.2%) 0.1% (0.4%) 0.6% (0.2%) 0.5% (0.2%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 208 (5.0%) 608 (9.3%) 728 (11.1%) 608 (9.3%) 728 (11.1%) 342 (5.2%) 554 (9.1%) 618 (9.4%) 519 (9.1%) 618 (9.4%) 519 (9.1%) 519 | 7(0.1%) 7(0.1%) 196 (3.0%) 186 (3.0%) 188 (2.13.5%) 20 (3.4%) 325 (3.4%) 325 (3.4%) 325 (3.4%) 325 (3.4%) 327 (3.2%) 327 (3.2%) 327 (3.2%) 327 (3.2%) 327 (3.2%) 327 (3.2%) 327 (3.2%) 328 (4.2%) 328 (4.2%) 328 (4.2%) 328 (4.2%) 328 (4.2%) 329 (4.2%) 329 (4.2%) 329 (3.2%) 329 (3.2%) 329 (3.2%) 320 (3.2%) 330 (3.2%) | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.5%) 0.4% (-1.1%, 1.0%) 0.0% (-1.0%, 0.1%) 0.3% (-1.0%, 0.5%) 0.0% (-0.0%, 0.5%) 0.0% (-0.0%, 0.5%) 0.0% (-0.0%, 0.5%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) |
| Insertion of accomales removal of cardiac lead; n (%) CXD stage 1.4; n (%) CXD stage 3.4; n (%) Livespecified CXD; n (%) Accute kidney injury; n (%) Hypertensive nephropathy; n (%) Hypertensive nephropathy; n (%) Livrary tract infections; n (%) Gential infections; n (%) Gential infections; n (%) CXPD; n (%) Asthmar (%) Obstructive sleep apnex; n (%) Serious bacterial infections; n (%) Pasumonia; n (%) MASHMASILD; n (%) Pasumonia; n (%) Distructive sleep apnex; n (%) Serious bacterial infections; n (%) Destroposis; n (%) Distructive sleep apnex; n (%) Demension; n (%) Demension; n (%) Demension; n (%) Demension; n (%) Annex; n (%) Infinienz; n (%) Infinienz; n (%) Infinienz; n (%) Infinienz; n (%) Billing disease; n (%) Pancreatitis; n (%) Destroposis; n (%) Destroposis; n (%) Destroposis; n (%) Distructive sleep apnex; n (%) Distructive sleep apnex; n (%) Distructive sleep apnex; n (%) Distructive sleep apnex; n (%) Distructive sleep apnex; n (%) Destroposis; n (%) Destropo | 30 (0.2%) 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (6.5%) 940 (6.5%) 1.569 (11.3%) 1.569 (11.3%) 1.569 (11.3%) 1.57 (3.7%) 740 (5.3%) 1.500 (10.5%) 1.517 (3.7%) 740 (5.3%) 1.500 (10.5%) 1.517 (3.7%) 740 (5.3%) 1.510 (10.5%) 1.510 (10.5%) 1.510 (10.5%) 1.511 (3.1%) 1.510 (10.5%) 1.510 | 16 (01%) 17 (0.1%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 163 (3.1%) 890 (4.5%) 163 (3.1%) 163 (6.3%) 163 (6.3%) 163 (6.3%) 163 (6.3%) 1033 (6.2%) 1033 (6.2%) 1033 (6.2%) 1033 (6.2%) 1033 (6.2%) 11850 (8.4%) 2172 (11.0%) 7.533 (8.2%) 639 (3.2%) 920 (4.7%) 295 (15.0%) 1817 (9.2%) 802 (4.1%) 460 (2.3%) 5.338 (27.1%) 3.402 (17.3%) 3.402 (17.3%) 3.402 (17.3%) 3.44 (1.7%) 105 (0.5%) 3.24 (1.6%) 3.24 (1.6%) 3.24 (1.6%) 4.980 (2.5.3%) 3.29 (1.6%) 4.980 (2.5.3%) 5.915 (3.0.0%) 3.24 (1.6%) 4.980 (2.5.3%) 3.49 (17.7%) 324 (1.6%) 4.980 (2.5.3%) 4.9 (0.2%) 11 (0.1%) 41 (0.2%) 11 (0.1%) 41 (0.2%) 117 (0.6%) | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.1% (0.4%) 0.6% (0.2%) 0.1% (0.4%) 0.6% (0.2%) 0.1% (0.4%) 0.6% (0.2%) 0.5% (0.2%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 208 (5.0%) 608 (9.3%) 728 (11.1%) 228 (5.0%) 608 (9.3%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (6.2%) 343 (4.6%) 360 (2.4%) 364 (6.6%) 360 (2.4%) 365 (2.4%) 366 (2.4%) 367 (6.2%) 368 (6.2%) 368 (6.2%) 368 (6.2%) 369 | 7(0.1%) 7(0.1%) 196 (3.0%) 186 (3.0%) 188 (2.13.5%) 220 (3.4%) 325 (5.4%) 597 (9.1%) 597 (9.1%) 294 (4.3.7%) 325 (5.4%) 327 (5.4%) 328 (4.2%) 328 (4.2%) 328 (4.2%) 328 (4.2%) 328 (4.2%) 328 (4.2%) 329 (4.2%) 329 (4.2%) 320 (6.2%) 320 (6.2%) 330 (6.2%) 340 (6.2%) 350 (6.2%) 3 | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.5%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXO stage 2, 4; n (%) CXO stage 3, 4; n (%) Livespecified CXCn (%) Accele kidney injury n (%) Hypertensive neighropathy; n (%) Hypertensive neighropathy; n (%) Livrary tract infections; n (%) Gential infections; n (%) Gential infections; n (%) CXPD; n (%) Asthma; n (%) CXPD; n (%) Asthma; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Pheumonia; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Pheumonia; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Distructive sleep apnea; n (%) D | 30 (0.2%) 473 (3.4%) 2235 (16.1%) 2235 (16.1%) 2235 (16.1%) 2235 (16.1%) 2245 (16.1%) 225 (16.1%) 225 (16.1%) 225 (16.1%) 225 (16.1%) 225 (16.1%) 227 (16.1%) 228 (16.1%) 228 (16.1%) 229 (16.1%) 239 (16.1%) 249 | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 1636 (8.3%) 1636 (8.3%) 1636 (8.3%) 1636 (8.3%) 1650 (8.4%) 1650 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.14% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.4%) 1.6% (0.2%) 1.5% (0.1%) 1.5% (0.4%) (1.6%) 1.5% (0.4%) (1.6%) 1.5% (0.4%) (1.6%) 1.5% (0.4%) (1.6%) 1.5% (0.4%) (1.5%) | 7(0.1%) 7(0.1%) 193 (2.9%) 997 (13.8%) 209 (3.2%) 209 (3.2%) 228 (5.0%) 608 (9.3%) 228 (5.0%) 608 (9.3%) 227 (4.1%) 226 (1.1%) 247 (4.1%) 247 (4.1%) 248 (4.1%) 249 (4.1%) 240 (4.1%) 241 (4.6%) 160 (2.4%) 160 (2.5%) 160 ( | 7(0.15%) 7(0.15%) 196 (3.05%) 196 (3.05%) 196 (3.05%) 196 (3.05%) 197 (3.15%) | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.1%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.5%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXO stage 2, 4; n (%) CXO stage 3, 4; n (%) Livespecified CXCn (%) Accele kidney injury n (%) Hypertensive neighropathy; n (%) Hypertensive neighropathy; n (%) Hypertensive neighropathy; n (%) Livraly tract riflorious; n (%) Gential infections; n (%) Distructive sleep apnea; n (%) Senious bacterial infections; n (%) Pheumonit; n (%) Distructive sleep apnea; n (%) Gential infections; n (%) Distructive sleep apnea; n (%) Gential infections; n (%) Distructive sleep apnea; n (%) Demential n (%) D | 30 (0.2%) 473 (3.4%) 2.23 (6.6.1%) 2.23 (6.6.1%) 2.25 (6.5%) 9.01 (6.5%) 9.01 (6.5%) 1.565 (1.3%) 1.565 (1.3%) 1.565 (1.3%) 1.565 (1.3%) 1.565 (1.3%) 1.565 (1.3%) 1.566 (1.3%) 1.567 (1.3%) 1.567 (1.3%) 1.57 (1.3 | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 890 (4.5%) 1636 (3.8%) 1636 (3.8%) 1636 (3.8%) 1639 (3.8%) 1650 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 2.3% (1.1% 2.6%) 2.3% (1.1% 2.6%) 2.3% (1.1% 2.6%) 0.1% (-0.4% 0.6%) 0.1% (-0.5% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.3% (-2.5% 1.0%) 1.3% (-2.5% 1.0%) 0.5% (-0.5% 0.9%) 1.5% (-2.5% 1.0%) 0.3% (-0.1% 0.0%) 0.3% (-0.2% 0.0%) 0.3% (-0.5% 0.2%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 328 (5.0%) 608 (9.3%) 728 (111%) 226 (7.41%) 342 (5.2%) 554 (9.1%) 618 (9.4%) 220 (13.9%) 134 (4.6%) 134 (4.6%) 134 (4.6%) 135 (1.6%) 136 (1.6%) 136 (1.6%) 136 (1.6%) 136 (1.6%) 137 (1.6%) 137 (1.6%) 138 (1.6%) 139 (1.6%) 140 (1.6%) 150 (1.6%) 15 | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.13.5%) 20 (3.4.%) 355 (5.4.%) 357 (5.4.%) 357 (5.4.%) 357 (5.4.%) 357 (5.4.%) 357 (5.4.%) 357 (5.4.%) 357 (3.1.%) 368 (3.1.%) 368 (3.1.%) 368 (3.1.%) 369 (3.1.%) 370 ( | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.2%, 0.1%) 0.0% (-0.2%, 0.1%) 0.0% (-0.2%, 0.1%) 0.0% (-0.2%, 0.1%) 0.0% (-0.2%, 0.1%) |
| Insention of accernaleus; removal of cardiac lead; n (%) CXO stage 12, 4; n (%) CXO stage 2, 4; n (%) Linspecified CXCn (%) Acute Xidew; ripary; n (%) Hyperferentive neightropathy; n (%) Hyperferentive neightropathy; n (%) Univary tract reflections; n (%) Gental infections; n (%) Gental infections; n (%) Univary tract reflections; n (%) Gental infections; n (%) COPD; n (%) Asthma; n (%) Obstructive sleep apnea; n (%) Serious bacterial infections; n (%) Phoeumonia; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Phoeumonia; n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Phoeumonia; n (%) Distructive sleep apnea; n (%) Depression; n (%) Distructive sleep apnea; n (%) Depression; n (%) Depress | 30 (0.2%) 473 (3.4%) 2.235 (1.6.1%) 6.26 (4.5%) 9.40 (6.6.6%) 9.40 (6.6.6%) 1.565 (1.1.3%) 1.565 (1.1.3%) 1.565 (1.1.3%) 1.565 (1.1.3%) 1.565 (1.1.3%) 1.565 (1.1.3%) 1.565 (1.1.3%) 1.566 (1.1.3%) 1.567 | 16 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 18 (3.1%) 890 (4.5%) 16 (3.1%) 890 (4.5%) 16 (3.5%) 18 (3.5%) 19 (3.5%) 19 (3.5%) 10 (3.5%) 10 (3.5%) 10 (3.5%) 11 (0.1%) 11 (0.0.5%) 11 (0.1%) 11 (0.0.5%) 11 (0.0.5%) 11 (0.0.5%) 11 (0.0.5%) 11 (0.0.5%) 11 (0.0.5%) 11 (0.0.5%) 12 (3.5%) 13 (3.5%) 13 (3.5%) 14 (3.5%) 15 (3.5%) 16 (3.5%) 17 (3.5%) 18 (3.5 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 2.3% (1.1% 2.6%) 2.3% (1.1% 2.6%) 2.3% (1.1% 2.6%) 0.1% (-0.4% 0.6%) 0.1% (-0.5% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.2% (-2.0% 0.5%) 1.3% (-2.0% 0.5%) 1.3% (-2.0% 0.5%) 0.5% (-0.5% 0.5%) 0.5% (-0.5% 0.5%) 0.3% (-0.0% 0.6%) 0.3% (-0.2% 0.7%) 0.3% (-0.2% 0.7%) 0.3% (-0.2% 0.7%) 0.3% (-0.2% 0.0%) 0.3% (-0.5% 0.0%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (12.8%) 209 (3.2%) 209 (3.2%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 328 (5.0%) 342 (5.2%) 342 (6.2%) 342 (6.2%) 344 (4.6%) 344 ( | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.13.5%) 20 (3.4%) 355 (5.4%) 357 (5.4%) 357 (5.4%) 357 (5.4%) 357 (5.4%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 2106 (3.2.1%) 234 (3.3.%) 325 (5.0%) 933 (14.2%) 525 (6.3.%) 193 (14.2%) 525 (6.3.%) 193 (14.2%) 195 (6.3.%) 195 (6.4.%) 195 (6.4.%) 195 (6.4.%) 196 (6.4.%) 196 (6.4.%) 196 (6.4.%) 196 (6.4.%) 197 (1.4.%) 197 (1.4.%) 1 | 0.0% (-1.1%, 0.1%) 0.0% (-1.1%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.0% (-0.0%, 0.0%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXD stage 1-2; n (%) CXD stage 1-3; n (%) CXD stage 2-4; n (%) CXD stage 2-4; n (%) Liva pecified CXD, n (%) Acute kidney injury, n (%) Hypertensive nephropathy, n (%) Hypertensive nephropathy, n (%) Hypertensive nephropathy, n (%) Liva pecified CXD, n (%) Gential infections; n (%) Distructive sleep apnea; n (%) Distructive sleep apnea; n (%) Distructive sleep apnea; n (%) Distructive sleep apnea; n (%) Demential n ( | 30 (0.2%) 473 (3.4%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.336 (1.6.1%) 2.337 (1.6.2%) 2.338 (1.6.2%) 2.348 (1.6.2%) 2.349 (1.6.2%) | 16 (01%) 17 (01%) 18 (12%) 548 (2.8%) 548 (2.8%) 18 (3.1%) 19 (3.1%) 19 (3.1 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 0.6% (0.2% 1.0%) 1.4% (0.9% 1.8%) 1.2% (1.1% 2.6%) 1.4% (0.9% 1.8%) 1.2% (1.1% 2.6%) 1.4% (0.9% 1.8%) 1.2% (1.1% 2.6%) 0.1% (0.4% 0.6%) 0.1% (0.4% 0.6%) 0.1% (0.4% 0.6%) 1.2% (1.2% 1.1%) 1.5% (1.1% 2.0%) 1.2% (1.2% 1.1%) 1.5% (1.1% 2.0%) 1.2% (2.0% 0.5%) 1.2% (2.0% 0.0%) 1.2% | 7(0.1%) 7(0.1%) 7(0.1%) 193 (2.9%) 907 (12.8%) 209 (3.2%) 328 (5.0%) 608 (9.3%) 328 (5.0%) 608 (9.3%) 728 (111%) 328 (5.0%) 608 (9.3%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (6.2%) 344 (4.6%) 160 (2.4%) 304 (4.6%) 160 (2.4%) 160 (3.4%) 160 (3.4 | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (3.1%) 20 (3.4%) 355 (5.4%) 557 (9.1%) 355 (5.4%) 557 (9.1%) 357 (5.4%) 557 (9.1%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 220 (3.2%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 224 (3.6%) 357 (5.4%) 557 (9.1%) 637 (9.7%) 224 (3.6%) 357 (5.4%) 557 (9.1%) 537 (9.7%) 235 (5.0%) 933 (14.2%) 545 (8.2%) 106 (24.7%) 10.59 (15.5%) 106 (24.7%) 10.81 (6.5%) 108 (16.5%) 108 (16.5%) 108 (16.5%) 108 (16.5%) 109 (16.5%) 109 (16.5%) 100 ( | 0.0% (-1.1%, 0.1%) 0.0% (-1.1%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.0% (-0.0%, 0.0%) |
| Insertion of accemakers / removal of cardiac lead; n (%) CXO staps 1-2; n (%) CXO staps 2-4; n (%) CXO staps 2-4; n (%) Lyo pecified CXO; n (%) Acute kidney injury, n (%) Hypertensive nephropathy; n (%) Hypertensive nephropathy; n (%) Lyo pecified CXO; n (%) Cottal state infections; n (%) Gental infections; n (%) Gental infections; n (%) Cottal state (%) Past use of Metions in (%) Cottal state | 30 (0.2%) 473 (3.4%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.236 (1.6.1%) 2.237 (1.6.2%) 2.237 (1.6.2%) 2.237 (1.6.2%) 2.238 (2.2%) 2.239 (2.2%) 2.249 (2.2%) 2.249 (2.2%) 2.259 (2.2%) 2.2714 (2.2%) 2.291 (2.2%) 2.291 (2.2%) 2.292 (2.2%) 2.293 (2.2%) 2.291 (2.2%) 2. | 16 (01%) 17 (01%) 18 (12%) 548 (2.8%) 548 (2.8%) 16 (3.1%) 17 (3.1%) 18 (3.1%) 18 (3.1%) 18 (3.1%) 18 (3.1%) 19 (3.1 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.1% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.1%) 1.4% (0.1%) 1.4% (0.1%) 1.4% (0.1%) 1.4% (0.1%) 1.5% (1.1%) 1.5% (1 | 7(0.1%) 7(0.1%) 7(0.1%) 193 (2.9%) 907 (12.8%) 209 (3.2%) 209 (3.2%) 328 (5.0%) 608 (9.3%) 728 (11.1%) 226 (7.41%) 342 (5.2%) 544 (9.1%) 344 (4.8%) 920 (14.0%) 531 (6.1%) 160 (2.4%) 160 ( | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 197 (3.0%) 198 (3.0%) 198 (3.0%) 198 (3.0%) 198 (4.0%) 198 (4 | 0.0% (-1.1%, 0.1%) 0.0% (-1.1%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 1.6%) 0.2% (-1.0%, 1.6%) 0.2% (-1.0%, 1.2%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.0%) |
| Insertion of accernaleus; removal of cardiac lead; n (%) CKO stags 1-2; n (%) CKO stags 3-4; n (%) Liva pecified CKD n (%) Acute Addrey ripary, n (%) Hypertensive negativepathy, n (%) Hypertensive negativepathy, n (%) Hypertensive negativepathy, n (%) Usivary tract Helections; n (%) Gential infections; n (%) Gential infections; n (%) Usivary tract Helections; n (%) Gential infections; n (%) Usivary tract Helections; n (%) Gential infections; n (%) COPP. n (%) Asthmax, n (%) Obstructive sleep apnea; n (%) Serious bacterial infections; n (%) Pneumonia; n (%) Distructive sleep apnea; n (%) Finature (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Pneumonia; n (%) Distructive (%) Distructive (%) Distructive (%) Distructive (%) Degression n (%) | 30 (0.2%) 473 (3.4%) 473 (3.4%) 2.236 (16.1%) 2.236 (16.1%) 2.236 (16.1%) 3.165 (11.3%) 1.565 (11.3%) 1.565 (11.3%) 1.565 (11.3%) 1.57 (3.7%) 3.17 (3.7%) 3.161 (2.6%) 3.17 (3.7%) 3.161 (2.6%) 4.236 (3.9%) 3.161 (2.6%) 4.236 (3.9%) 3.161 (2.6%) 4.25 (3.6%) 1.21 (3.1%) 4.25 (3.6%) 4.27 (3.2%) 4.27 (3.2%) 4.27 (3.2%) 4.27 (3.2%) 4.28 (3.2%) 4.29 (0.81) 4.29 (3.2%) 4. | 16 (01%) 17 (01%) 18 (12%) 548 (2.8%) 548 (2.8%) 16 (3.1%) 17 (3.1%) 18 (3.1%) 18 (3.1%) 18 (3.1%) 19 (3.1 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.1% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.9%) 1.4% (0.1%) 1.4% (0.1%) 1.4% (0.1%) 1.4% (0.1%) 1.4% (0.1%) 1.4% (0.1%) 1.5% (1.1%) 1.5% (1 | 7(0.1%) 7(0.1%) 7(0.1%) 193 (2.9%) 907 (12.8%) 209 (3.2%) 328 (5.0%) 508 (9.3%) 328 (5.0%) 508 (9.3%) 728 (111%) 328 (5.0%) 508 (9.3%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 342 (5.2%) 534 (9.1%) 344 (4.8%) 920 (14.0%) 531 (6.1%) 100 (2.4%) 100 (2.5%) | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 197 (3.1%) 197 (3.1%) 198 (3 | 0.0% (-1.1%, 0.1%) 0.0% (-1.1%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 1.6%) 0.2% (-1.0%, 1.6%) 0.2% (-1.0%, 1.2%) 0.0% (-1.1%, 1.1%) 0.0% (-1.1%, 1.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.1%, 1.1%) 0.2% (-1.1%, 0.1%) 0.2% (-1.1%, 0.1%) 0.3% (-1.1%, 0.1%) |
| Insertion of accernakers; removal of cardiac lead; n (%) CKO stags 1-4; n (%) CKO stags 3-4; n (%) Liva pecified CKD n (%) Acute bidney injury, n (%) Liva pecified CKD n (%) Acute bidney injury, n (%) Liva pecified CKD n (%) Acute bidney injury, n (%) Liva pecified CKD n (%) Acute bidney injury, n (%) Liva pecified CKD n (%) Acute bidney injury, n (%) Liva pecified CKD n (%) Gental infections; n (%) Gental infections; n (%) Gental infections; n (%) COPD: n (%) COPD: n (%) Asthmax n (%) Distructive sleep apnea; n (%) Serious bacterial infections; n (%) Pneumonia; n (%) Distructive sleep apnea; n (%) Finature infections; n (%) Distructive sleep apnea; n (%) Finature infections; n (%) Distructive sleep apnea; n (%) Distructive sleep apnea; n (%) Distructive sleep apnea; n (%) Distructive sleep apnea; n (%) Distructive sleep apnea; n (%) Decreasis n (%) Distruction n (%) Decreasis n (%) | 30 (0.2%) 473 (3.4%) 473 (3.4%) 2.235 (16.1%) 2.235 (16.1%) 2.235 (16.1%) 2.235 (16.1%) 2.235 (16.1%) 2.245 (16.1%) 2.245 (16.1%) 2.247 (16.2%) 2.247 (16.2%) 2.247 (16.2%) 2.248 (16.2%) 2.248 (2.2%) 2.248 (16.2%) 2.249 (16.2%) 2.259 (16.2%) 2.269 (16.2%) 2.270 (16.2%) 2.290 (16.2%) 2.290 (16.2%) 2.290 (16.2%) 2.290 (16.2%) 2.291 (16.2%) | 16 (01%) 17 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 680 (3.1%) 690 (4.8%) 1.636 (8.3%) 1.636 (8.3%) 1.636 (8.3%) 1.637 (8.3%) 1.637 (8.3%) 1.638 (8.3%) 1.638 (8.3%) 1.638 (8.3%) 1.638 (8.3%) 1.639 (3.2%) 1.649 (3.2%) 1.659 (3.3%) 1.6 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.1%) 0.5% (0.0% 0.1%) 0.5% (0.0% 0.2%) 0.5% (0.0% 0.1%) 0.5% (0.0% 0.1%) 0.5% (0.0% 0.1%) 0.5% (0.0% 1.5%) 0.5% (0.0% 0.1%) 0.0% (0.0% 0.0%) 0.0% (0.0% 0.0%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 208 (5.0%) 608 (9.3%) 728 (11.1%) 608 (9.3%) 728 (11.1%) 342 (5.2%) 544 (9.1%) 344 (4.6%) 180 (2.4%) 344 (4.6%) 180 (2.4%) 344 (4.6%) 180 (2.4%) 140 (3.6%) 180 (2.4%) 140 (3.6%) 180 (2.4%) 180 | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 198 (2.0%) 20 (3.4%) 20 (3.4%) 20 (3.4%) 357 (5.4%) 557 (0.1%) 557 (0.1%) 357 (5.4%) 557 (0.1%) 358 (5.4%) 368 (3.5%) 369 (3.5%) 370 (3.5%) 370 (3.5%) 370 (3.5%) 381 (5.5%) | 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.1%, 0.1%) 0.0% (-0.0%, 0.1%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) 0.2% (-0.0%, 1.0%) 0.2% (-0.0%, 1.0%) 0.2% (-0.0%, 1.0%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.2% (-1.0%, 0.0%) 0.3% (-1.0%, 0.0%) 0.0% (-0.0%, 0.0%) |
| Insention of accomakers; removal of cardiac lead; n (%) CXO stage 1-2; n (%) CXO stage 2-4; n (%) Unspecified CXD: n (%) Acute kidney inyn n (%) Hypertensive nisphropathy; n (%) Hypertensive nisphropathy; n (%) Hypertensive nisphropathy; n (%) Gental infections; n (%) Districtive sleep apnea; n (%) Gental infections; n (%) Districtive sleep apnea; n (%) Gental infections; n (%) Districtive sleep apnea; n (%) Gental infections; n (%) Districtive sleep apnea; n (%) Demendration (%) Districtive sleep appear (%) Districtive sleep appear (%) Districtive sleep appear (%) Demendration (%) Demend | 30 (0.2%) 473 (3.4%) 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (6.6%) 1.669 (11.3%) 1.669 (11.3%) 1.669 (11.3%) 1.669 (11.3%) 1.670 | 16 (01%) 17 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 680 (3.1%) 680 (3.5%) 1.636 (8.3%) 688 (3.5%) 1.636 (8.3%) 1.637 (8.3%) 1.637 (8.3%) 1.638 (8.3%) 1.638 (8.3%) 1.638 (8.3%) 1.638 (8.3%) 1.639 (3.2%) 1.649 (3.2%) 1.659 (3.3%) 1.659 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.5% (0.2%) 0.14% (0.9%) 0.14% (0.9%) 0.14% (0.6%) 0.14% (0.6%) 0.15% (0.4%) 0.15% (0.4%) 0.15% (0.4%) 0.15% (0.4%) 0.15% (0.15%) 0.25% (0.15%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (1.1%) 608 (9.3%) 728 (1.1%) 608 (9.3%) 728 (1.1%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 344 (4.8%) 920 (14.0%) 334 (4.8%) 920 (14.0%) 334 (4.8%) 105 (12.4%) 11.03 (15.5%) 11.03 (15.5%) 11.03 (15.5%) 11.03 (16.5%) 11.03 (16.5%) 11.07 (14.1%) 11 | 7(0.1%) 7(0.1%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 196 (3.0%) 197 (3.1%) 197 (3 | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.3%, 0.7%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.0% (-0.0%, 0.0%) 0.0% (-0.0%, 0.0%) |
| Insention of accomakers / removal of cardiac lead; n (%) CXO stage 1-2 (%) CXO stage 2-4; n (%) Linspecified CXC n (%) Acute kidney inyn n (%) Hypertensive nisphropathy n (%) Hypertensive nisphropathy n (%) Hypertensive nisphropathy n (%) Gental infections; n (%) District we sleep apnea; n (%) District we sleep (%) District we sleep apnea; n (%) District we sleep (%) District we sleep (%) District we sleep (%) Demender (%) District we sleep (%) District we sleep (%) District we sleep (%) District we sleep (%) District we sleep (%) Demender (%) Demender (%) Demender (%) Demender (%) Demender (%) District we sleep (%) Dis | 30 (0.2%) 473 (3.4%) 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (6.6%) 1569 (11.3%) 1569 (11.3%) 1569 (11.3%) 1576 (1.3%) 1576 (1.3%) 1576 (1.3%) 1576 (1.3%) 1500 (1.0.5%) 1576 (1.3%) 1500 (1.0.5%) 1576 | 16 (01%) 17 (01%) 17 (01%) 548 (2.8%) 548 (2.8%) 548 (2.8%) 618 (3.1%) 689 (3.4%) 618 (3.1%) 689 (3.5%) 1.636 (8.3%) 1.636 (8.3%) 1.637 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.6% (0.2%) 0.14% (0.9%) 0.14% (0.9%) 0.14% (0.9%) 0.14% (0.4%) 0.14% (0.6%) 0.15% (0.4%) 0.15% (0.4%) 0.15% (0.4%) 0.15% (0.4%) 0.15% (0.15%) 0. | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (1.1%) 608 (9.3%) 728 (1.1%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 342 (5.2%) 544 (9.1%) 344 (4.8%) 920 (14.0%) 531 (8.1%) 304 (4.6%) 105 (2.4%) 14.0%) 304 (4.6%) 105 (2.4%) 14.0%) 133 (18.5%) 105 (2.2%) 14.0% 133 (1.5%) 156 (2.2%) 147 (2.2%) 148 (3.3%) 137 (12.1%) 137 (12.1%) 138 (1.3%) 139 (1.3%) 139 (1.3%) 130 (0.9%) 147 (2.2%) 148 (0.7%) 149 (0.3%) 149 (0.3%) 140 (0.3%) 140 (0.3%) 140 (0.3%) 140 (0.3%) 141 (0.5%) 141 (0.5%) 142 (0.2%) 143 (0.5%) 144 (0.5%) 145 (0.7%) 147 (0.5%) 147 (0.2%) 148 (0.7%) 149 (0.3%) 149 (0.3%) 140 (0.3%) 141 (0.5%) 141 (0.5%) 142 (0.2%) 143 (0.5%) 144 (0.5%) 145 (0.7%) 144 (0.5%) 147 (2.2.5%) | 7(0.15%) 7(0.15%) 136 (3.0%) 136 (3.0%) 136 (3.0%) 136 (3.0%) 136 (3.0%) 137 (3.4%) 135 (3.2%) 135 (3.2%) 135 (3.2%) 135 (3.2%) 136 (3.2%) 136 (3.2%) 136 (3.2%) 136 (3.2%) 136 (3.2%) 137 (3.2%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 139 (3.3%) 130 | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.3%, 0.7%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.1%) 0.3% (-1.0%, 0.5%) 0.2% (-1.0%, 0.5%) 0.2% (-1.0%, 0.5%) 0.3% (-1.0%, 0.5%) 0.0% (-0.3%, 0.1%) 0.0% (-0.3%, 0.1%) 0.0% (-0.3%, 0.1%) 0.0% (-0.3%, 0.1%) 0.0% (-0.3%, 0.1%) 0.0% (-0.3%, 0.3%) 0.0% (-1.0%, 0.5%) 0.0% (-1.0%, 0.5%) 0.0% (-1.0%, 0.5%) 0.0% (-1.0%, 0.5%) 0.0% (-1.0%, 0.1%) |
| Insention of accernaleurs / removal of cardiac lead; n (%) CXO stage 1-2, n (%) CXO stage 2-4; n (%) Linspecified CXCn (%) Acute Motive y injury; n (%) Hyperbrender neight property n (%) Hyperbrender neight property n (%) Unsay tract infections; n (%) Gential infections; n (%) | 30 (0.2%) 473 (3.4%) 473 (3.4%) 2235 (16.1%) 626 (4.5%) 940 (6.6%) 1.665 (11.3%) 1.665 (11.3%) 1.665 (11.3%) 1.665 (11.3%) 1.665 (11.3%) 1.675 | 16 (01%) 17 (01%) 15 (01%) 15 (10%) 15 (10%) 15 (10%) 15 (10%) 16 (3.1%) 17 (3.1%) 18 | 0.1% (-0.0% 0.1%) 0.1% (0.0% 0.2%) 0.6% (0.2%) 0.1% (0.4%) 0.1% (0.4%) 0.1% (0.4%) 0.1% (0.4%) 0.1% (0.4%) 0.5% (0.2%) 0.3% (0.2%) | 7(0.1%) 7(0.1%) 193 (2.9%) 907 (13.8%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (3.2%) 209 (1.3%) 608 (9.3%) 728 (11.1%) 228 (1.1%) 342 (5.2%) 342 (5.2%) 344 (9.1%) 342 (5.2%) 344 (4.8%) 920 (14.0%) 334 (4.6%) 105 (2.4%) 116 (2.4%) 116 (2.4%) 116 (2.4%) 116 (2.4%) 116 (2.4%) 116 (2.4%) 117 (1.1%) 118 (1.1%) 118 (1.1%) 119 | 7(0.15%) 7(0.15%) 136 (3.0%) 136 (3.0%) 136 (3.0%) 136 (3.0%) 136 (3.0%) 137 (3.4%) 135 (3.2%) 135 (3.2%) 135 (3.2%) 135 (3.2%) 136 (3.2%) 136 (3.2%) 136 (3.2%) 136 (3.2%) 136 (3.2%) 137 (3.2%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 138 (3.3%) 139 (3.3%) 130 | 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.0% (-1.0%, 0.1%) 0.2% (-1.0%, 0.1%) 0.3% (-1.0%, 0.5%) 0.3% (-1.0%, 0.0%) |

| DOCKO : 1.12 | Interior 400 | 2422 45 000 | 0.50/ / 1.30/ 0.30/) | 1 000 #5 000 | 070 (54 00/) | 0.40/ / 0.00/ 3.50/ |
|---|---|---|---|---|---|---|
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) Antirelatelet medications: n (%) | 2,142 (15.4%)<br>2,581 (18.6%) | 3,133 (15.9%) | -0.5% (-1.3%, 0.3%) | 1,002 (15.3%)<br>1 188 (18.1%) | 978 (14.9%)<br>1156 (17.6%) | 0.4% (-0.9%, 1.6%) |
| Oral anticoagulants; n (%) | 1,869 (13.5%) | 2,458 (12.5%) | 1.0% (0.3%, 1.7%) | 795 (12.1%) | 802 (12.2%) | -0.1% (-1.2%, 1.0%) |
| COPD/Asthma medications; n (%) | 4,461 (32.1%) | 7,363 (37.4%) | -5.2% (-6.3%, -4.2%) | 2,215 (33.8%) | 2,186 (33.4%) | 0.4% (-1.2%, 2.1%) |
| NSAIDS; n (%) | 4,244 (30.6%)<br>3.227 (23.2%) | 6,989 (35.5%)<br>5.786 (29.4%) | -4.9% (-5.9%, -3.9%)<br>-6.1% (-7.1%, -5.2%) | 2,181 (33.3%) | 2,134 (32.6%) | 0.7% (-0.9%, 2.3%)<br>-0.8% (-2.3%, 0.7%) |
| Oral corticosteroids; n (%) Osteoporosis agents (incl. bisphosphonates); n (%) | 3,227 (23.2%) | 361 (1.8%) | 0.5% (0.2%, 0.9%) | 1,593 (24.3%) | 1,646 (25.1%)<br>131 (2.0%) | 0.0% (-0.5%, 0.7%) |
| Opioids; n (%) | 4,072 (29.3%) | 6,236 (31.6%) | -2.3% (-3.3%, -1.3%) | 1,965 (30.0%) | 1,960 (29.9%) | 0.1% (-1.5%, 1.7%) |
| Anti-depressants; n (%) | 4,110 (29.6%) | 7,613 (38.6%) | -9.0% (-10.0%, -8.0%) | 2,159 (32.9%) | 2,203 (33.6%) | -0.7% (-2.3%, 1.0%) |
| Antipsychotics; n (%) | 400 (2.9%)<br>2,457 (17.7%) | 621 (3.2%) | -0.3% (-0.6%, 0.1%)<br>-5.2% (-6.0%, -4.3%) | 185 (2.8%) | 191 (2.9%) | -0.1% (-0.7%, 0.5%)<br>-0.2% (-1.6%, 1.2%) |
| Anxiolytics / hypnotics, benzos; n (%) Dementia medications; n (%) | 352 (2.5%) | 4,509 (22.9%)<br>130 (0.7%) | 1.9% (1.6%, 2.2%) | 1,313 (20.0%)<br>72 (1.1%) | 1,325 (20.2%)<br>68 (1.0%) | 0.1% (-0.3%, 0.4%) |
| Urinary tract infections antibiotics; n (%) | 6,415 (46.2%) | 9,522 (48.3%) | -2.1% (-3.2%, -1.0%) | 3,017 (46.0%) | 2,989 (45.6%) | 0.4% (-1.3%, 2.1%) |
| Laxatives; n (%) | 441 (3.2%) | 669 (3.4%) | -0.2% (-0.6%, 0.2%) | 208 (3.2%) | 193 (2.9%) | 0.2% (-0.4%, 0.8%) |
| Number of distinct medications<br>mean (sd) | 13.49 (6.23) | 14.90 (6.66) | -1.40 (-1.54, -1.26) | 14.03 (6.60) | 14.05 (6.12) | -0.01 (-0.23, 0.20) |
| median [IQR] | 13.00 [9.00, 17.00] | 14.00 [10.00, 19.00] | - (-, -) | 13.00 [9.00, 18.00] | 13.00 [10.00, 17.00] | - (-, -) |
| min, max | 1.00, 65.00 | 1.00, 61.00 | - (-, -) | 1.00, 65.00 | 100,46.00 | - (-, -) |
| Number of office visits | | | | | | |
| mean (sd)median [IQR] | 9.50 (6.68)<br>8.00 [5.00, 13.00] | 10.33 (6.91)<br>9.00 [6.00, 13.00] | -0.84 (-0.98, -0.69)<br>- (-, -) | 9.74 (6.69)<br>8.00 [5.00, 13.00] | 9.78 (6.42)<br>8.00 [5.00, 13.00] | -0.04 (-0.26, 0.19)<br>- (-, -) |
| min, max | 0.00, 185.00 | 0.00, 75.00 | - (-, -) | 0.00, 94.00 | 0.00, 57.00 | - (-, -) |
| Number of endocrinologist visits | | | | | | |
| mean(sd) | 0.29 (1.08) | 0.45 (1.29) | -0.16 (-0.18, -0.13) | 0.37 (1.31) | 0.39 (1.06) | -0.02 (-0.06, 0.02) |
| median (IQR)min, max | 0.00 [0.00, 0.00]<br>0.00, 34.00 | 0.00 [0.00, 0.00] | - (-, -)<br>- (-, -) | 0.00 [0.00, 0.00]<br>0.00, 34.00 | 0.00 [0.00, 0.00] | - (-, -)<br>- (-, -) |
| Number of cardiologist visits | 0.00, 54.00 | 0.00, 50.00 | 157 | 0.00, 54.00 | 0.00, 11.00 | - (5.7) |
| mean (sd) | 1.90 (3.46) | 1.91 (3.51) | -0.01 (-0.08, 0.07) | 1.85 (3.42) | 187 (3.39) | -0.02 (-0.13, 0.10) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 3.00] | - (-, -) |
| min, max Number of internal/family medicine visits | 0.00, 70.00 | 0.00, 85.00 | - (-, -) | 0.00, 70.00 | 0.00, 85.00 | - (-, -) |
| mean (sd) | 6.70 (7.59) | 5.61 (6.01) | 1.09 (0.94, 1.24) | 5.89 (6.11) | 5.99 (6.17) | -0.10 (-0.31, 0.11) |
| median [IQR] | 5.00 [3.00, 8.00] | 4.00 [2.00, 7.00] | - (-, -) | 4.00 [2.00, 8.00] | 5.00 [2.00, 8.00] | - (-, -) |
| min, max | 0.00, 114.00 | 0.00, 178.00 | - (-, -) | 0.00, 86.00 | 0.00, 101.00 | - (-, -) |
| Number of Electrocardiograms (ECG/EKG)mean (sd) | 1.34 (2.36) | 1.24 (1.76) | 0.11 (0.06, 0.15) | 1.22 (1.69) | 125 (1.77) | -0.03 (-0.09, 0.03) |
| mean (sd)median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | -(-, -) |
| min, max | 0.00,173.00 | 0.00, 45.00 | - (-, -) | 0.00, 27.00 | 0.00, 35.00 | - (-, -) |
| Number of Echocardiograms | | | | | | |
| mean (sd) | 0.43 (0.83) | 0.42 (0.80)<br>0.00 [0.00, 1.00] | 0.02 (0.00, 0.04) | 0.41 (0.79) | 0.41 (0.78) | 0.01 (-0.02, 0.03) |
| median [1QR]min, max | 0.00 [0.00, 1.00] | 0.00 (0.00, 1.00) | - (-, -)<br>- (-, -) | 0.00 [0.00, 100] | 0.00 [0.00, 1.00] | - (-, -)<br>- (-, -) |
| Out-of-pocket medication cost | | | 177 | | | |
| mean (sd) | 441.60 (588.87) | 542.89 (792.22) | -101.29 (-116.06, -86.52) | 478.72 (702.85) | 482.74 (553.45) | -4.02 (-25.68, 17.64) |
| median [IQR]min, max | 300.00 [143.32, 565.83]<br>-4 490 96, 21 723 25 | 344.91 [144.90, 700.00]<br>-3,255.71, 26,458.73 | - (-, -)<br>- (-, -) | 308.63 [134.98, 619.28]<br>-4 490 96, 21 723 25 | 328.46 [150.00, 634.00]<br>-3 255 71 9 193 18 | - (-, -)<br>- (-, -) |
| min, max Unique brand medicines | -4,490.96, 21,723.25 | -3,255./1, 26,458./3 | - (-, -) | -4,490.96, 21,723.25 | -3,255.71, 9,193.18 | - (-, -) |
| mean (sd) | 13.76 (6.43) | 15.16 (6.84) | -1.39 (-1.54, -1.25) | 14.29 (6.80) | 14.30 (6.29) | -0.01 (-0.23, 0.22) |
| median [IQR] | 13.00 [9.00, 17.00] | 14.00 [10.00, 19.00] | - (-, -) | 13.00 [10.00, 18.00] | 13.00 [10.00, 18.00] | - (-, -) |
| min, max | 1.00, 69.00 | 1.00, 65.00 | - (-, -) | 1.00, 69.00 | 1.00, 49.00 | - (-, -) |
| Unique generic medicines | 13 49 (6 23) | 14 90 (6 66) | -140 (-154 -126) | 14 03 (6 60) | 14 05 (6 12) | -0.01 (-0.23, 0.20) |
| median [IQR] | 13.00 [9.00, 17.00] | 14.00 [10.00, 19.00] | -(-, -) | 13.00 [9.00, 18.00] | 13.00 [10.00, 17.00] | - (-, -) |
| min, max | 1.00, 65.00 | 1.00, 61.00 | - (-, -) | 1.00, 65.00 | 100,46.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%)<br>Flu Pneumococcal vaccine; n (%) | 1,526 (11.0%) | 2,474 (12.6%) | -1.6% (-2.3%, -0.9%) | 731 (11.2%) | 728 (11.1%) | 0.0% (-1.0%, 1.1%) |
| | | | | 2 227 (2 4 10/) | 3.3C3 (3.4 E0/) | 0.40/ ( 3.00/ 1.30/) |
| | 5,128 (36.9%)<br>840 (6.0%) | 6,183 (31.4%)<br>1.831 (9.3%) | 5.6% (4.5%, 6.6%)<br>-3.2% (-3.8%, -2.7%) | 2,237 (34.1%)<br>495 (7.6%) | 2,262 (34.5%)<br>504 (7.7%) | -0.4% (-2.0%, 1.3%)<br>-0.1% (-1.1%, 0.8%) |
| Pap smear; n (%) PSA test n (%) | 840 (6.0%)<br>3,456 (24.9%) | 1,831 (9.3%)<br>5,034 (25.5%) | -3.2% (-3.8%, -2.7%)<br>-0.6% (-1.6%, 0.3%) | 495 (7.6%)<br>1,721 (26.3%) | 504 (7.7%)<br>1,771 (27.0%) | -0.1% (-1.1%, 0.8%)<br>-0.8% (-2.3%, 0.8%) |
| Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) | 840 (6.0%)<br>3,456 (24.9%)<br>923 (6.6%) | 1,831 (9.3%)<br>5,034 (25.5%)<br>897 (4.6%) | -3.2% (-3.8%, -2.7%)<br>-0.6% (-1.6%, 0.3%)<br>2.1% (1.6%, 2.6%) | 495 (7.6%)<br>1,721 (26.3%)<br>366 (5.6%) | 504 (7.7%)<br>1,771 (27.0%)<br>371 (5.7%) | -0.1% (-1.1%, 0.8%)<br>-0.8% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%) |
| Pap smear, n (%) PSA test, n (%) Feal occult blood test: n (%) Bone mineral density tests; n (%) | 840 (6.0%)<br>3,456 (24.9%)<br>923 (6.6%)<br>621 (4.5%) | 1,831 (9.3%)<br>5,034 (25.5%)<br>897 (4.6%)<br>1,057 (5.4%) | -3.2% (-3.8%, -2.7%)<br>-0.6% (-1.6%, 0.3%)<br>2.1% (1.6%, 2.6%)<br>-0.9% (-1.4%, -0.4%) | 495 (7.6%)<br>1,721 (26.3%)<br>366 (5.6%)<br>330 (5.0%) | 504 (7.7%)<br>1,771 (27.0%)<br>371 (5.7%)<br>317 (4.8%) | -0.1% (-1.1%, 0.8%)<br>-0.8% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%) |
| Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) | 840 (6.0%)<br>3,456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2,651 (19.1%) | 1,831 (9.3%)<br>5,034 (25.5%)<br>897 (4.6%)<br>1,057 (5.4%)<br>5,323 (27.0%) | -3.2% (-3.8%, -2.7%)<br>-0.6% (-1.6%, 0.3%)<br>2.1% (1.6%, 2.6%)<br>-0.9% (-1.4%, -0.4%)<br>-7.9% (-8.8%, -7.0%) | 495 (7.6%)<br>1,721 (26.3%)<br>366 (5.6%)<br>330 (5.0%)<br>1,516 (23.1%) | 504 (7.7%)<br>1,771 (27.0%)<br>371 (5.7%)<br>317 (4.8%)<br>1,494 (22.8%) | -0.1% (-11%, 0.8%)<br>-0.8% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%)<br>0.3% (-11%, 1.8%) |
| Pap smear n (%) PSA test n (%) Fiscal occult blood test n (%) Fiscal occult blood test n (%) Bone mineral density tests; n (%) Mammagama; (%) (%) Mammagama; (%) | 840 (6.0%)<br>3.456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2.651 (19.1%)<br>2.300 (16.6%) | 1,831 (9.3%)<br>5,034 (25.5%)<br>897 (4.6%)<br>1,057 (5.4%)<br>5,323 (27.0%)<br>6,395 (32.4%) | -3.2% (-3.8%, -2.7%)<br>-0.6% (-1.6%, 0.3%)<br>2.1% (1.6%, 2.6%)<br>-0.9% (-1.4%, -0.4%)<br>-7.9% (-8.8%, -7.0%)<br>-15.9% (-16.8%, -15.0%) | 495 (7.6%)<br>1.721 (26.3%)<br>366 (5.6%)<br>330 (5.0%)<br>1.516 (23.1%)<br>1.634 (24.9%) | 504 (7.7%)<br>1,771 (27.0%)<br>371 (5.7%)<br>317 (4.8%)<br>1,494 (22.8%)<br>1,665 (25.4%) | -0.1% (-1.1%, 0.8%)<br>-0.8% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%)<br>0.3% (-1.1%, 1.8%)<br>-0.5% (-2.0%, 1.0%) |
| Pap smear n (%) PSA test n (%) FSA t | 940 (6.0%)<br>3,456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2651 (19.1%)<br>2,300 (16.6%) | 1.831 (9.3%)<br>5.034 (25.5%)<br>897 (4.6%)<br>1.057 (5.4%)<br>5.323 (27.0%)<br>6.395 (32.4%) | 3.2% (-3.8%, -2.7%)<br>0.6% (-1.6%, 0.3%)<br>21% (1.6%, 2.6%)<br>-0.9% (-1.4%, -0.4%)<br>7.9% (-8.8%, -7.0%)<br>15.9% (-16.8%, -15.0%)<br>-0.12 (-0.16, -0.09) | 495 (7.6%)<br>1,721 (26.3%)<br>366 (5.6%)<br>330 (5.0%)<br>1,516 (23.1%)<br>1,634 (24.9%) | 504 (7.7%)<br>1,771 (27.0%)<br>371 (5.7%)<br>317 (4.8%)<br>1,494 (22.8%)<br>1,665 (25.4%) | -0.1% (-1.1%, 0.8%)<br>-0.3% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%)<br>0.3% (-1.1%, 1.8%)<br>-0.5% (-2.0%, 1.0%)<br>-0.00 (-0.05, 0.05) |
| Pap smearn (%) PSA fest n (%) Fecal occult Blood fest n (%) Bone mineral density feets; n (%) Mammagams; n (%) Telemedicine; n (%) HEALC feetsmean (sd)median (lQR) | 840 (6.0%)<br>3.456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2651 (191%)<br>2300 (16.6%)<br>209 (1.62)<br>200 (1.02) | 1831 (9.3%)<br>5.034 (25.5%)<br>897 (4.6%)<br>1.057 (5.4%)<br>5.323 (27.0%)<br>6.395 (32.4%)<br>221 (1.49)<br>220 (1.00, 3.00) | 3.2% (-3.8%, -2.7%)<br>0.6% (-1.6%, 0.3%)<br>2.1% (1.6%, 2.6%)<br>0.9% (-1.4%, -0.4%)<br>-7.9% (-8.8%, -7.0%)<br>45.9% (-16.8%, -15.0%)<br>-0.12 (-0.16, -0.09)<br>-(-, -) | 495 (7.6%)<br>1,721 (26.3%)<br>366 (5.6%)<br>330 (5.0%)<br>1,516 (23.1%)<br>1,634 (24.9%)<br>2,24 (1,51)<br>2,00 (1,00,3.00) | 504 (7.7%)<br>1,771 (2.7%)<br>371 (5.7%)<br>317 (4.8%)<br>1,494 (2.2.%)<br>1,665 (25.4%)<br>224 (1.62)<br>200 (1.00, 3.00) | 0.1% (-1.1%, 0.8%) 0.5% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) -0.5% (-2.0%, 1.0%) -0.00 (-0.05, 0.05) |
| Pap smear n (%) PSA test n (%) FSA t | 940 (6.0%)<br>3,456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2651 (19.1%)<br>2,300 (16.6%) | 1.831 (9.3%)<br>5.034 (25.5%)<br>897 (4.6%)<br>1.057 (5.4%)<br>5.323 (27.0%)<br>6.395 (32.4%) | 3.2% (-3.8%, -2.7%)<br>0.6% (-1.6%, 0.3%)<br>21% (1.6%, 2.6%)<br>-0.9% (-1.4%, -0.4%)<br>7.9% (-8.8%, -7.0%)<br>15.9% (-16.8%, -15.0%)<br>-0.12 (-0.16, -0.09) | 495 (7.6%)<br>1,721 (26.3%)<br>366 (5.6%)<br>330 (5.0%)<br>1,516 (23.1%)<br>1,634 (24.9%) | 504 (7.7%)<br>1,771 (27.0%)<br>371 (5.7%)<br>317 (4.8%)<br>1,494 (22.8%)<br>1,665 (25.4%) | -0.1% (-1.1%, 0.8%)<br>-0.3% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%)<br>0.3% (-1.1%, 1.8%)<br>-0.5% (-2.0%, 1.0%)<br>-0.00 (-0.05, 0.05) |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammagams; (%) Telemedicine; n (%) HabAIC tests maan (sd)median IQR min max iman (sd)men (sd) | 840 (6.0%)<br>3.456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2.651 (9.1%)<br>2.300 (16.6%)<br>2.09 (1.6.2)<br>2.00 (1.00, 3.00)<br>0.00, 55.00 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 897 (4.6%) 1057 (5.4%) 5.232 (27.0%) 6.395 (32.4%) 220 (1.49) 220 (1.09) 0.00, 40.00 | 3.2% (-3.8%, -2.7%) -0.6% (-1.6%, 0.3%) -2.1% (1.6%, 0.2%) -0.9% (-1.4%, -0.4%) -7.9% (-8.8%, -7.0%) -15.9% (-16.8%, -15.0%) -0.12 (-0.16, -0.09) -(, -) -(, -) -(, -) -0.12 (-0.15, -0.09) | 495 (7.5%)<br>1,721 (26.3%)<br>366 (5.6%)<br>330 (5.0%)<br>1,516 (23.1%)<br>1,634 (24.9%)<br>2,00 (1.00, 3.00)<br>0,00, 33.00<br>1,61 (1.29) | 504 (7.7%)<br>1771 (27.0%)<br>371 (5.7%)<br>317 (4.8%)<br>1494 (22.8%)<br>1665 (25.4%)<br>2244 (16.2<br>200110.0, 3.00)<br>0.00, 40.00 | -0.1% (-1.1%, 0.8%)<br>-0.8% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%)<br>-0.2% (-0.6%, 1.0%)<br>-0.3% (-1.1%, 1.8%)<br>-0.5% (-2.0%, 1.0%)<br>-0.00 (-0.05, 0.05)<br>-(; -)<br>-(; -)<br>-0.02 (-0.05, 0.03) |
| Pap smearn (%) PSA test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammograms, n (%) Mammograms, n (%) Telemeticine n (%) HALIC testsmean (sd)median (lpti]min, max Lipid panets | 840 (6.0%)<br>3.456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2.651 (19.1%)<br>2.300 (16.6%)<br>2.09 (1.62)<br>2.00 (1.03.300)<br>0.00.55.00 | 1,831 (9.3%) 5,034 (25.5%) 897 (4.6%) 1057 (5.4%) 5,322 (27.0%) 6,355 (32.4%) 2,00 (100,3.00) 0,00,40,00 | 3.2% (-3.8%, 2.7%) -0.6% (-1.6%, 0.3%) -2.1% (1.6%, 2.6%) -0.9% (-1.4%, -0.4%) -7.9% (-3.8%, -7.0%) -15.9% (-1.6, -0.09) -(-, -) -0.12 (-0.15, -0.09) -(-, -) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 330 (5.0%) 1.516 (23.1%) 1.634 (24.9%) 2.24 (1.51) 2.00 (1.00, 3.00) 0.00, 3.30 0 1.61 (1.29) 1.00 (1.00, 2.00) | 504 (77%)<br>1771 (27%)<br>371 (57%)<br>371 (57%)<br>371 (45%)<br>1,494 (228%)<br>1,494 (228%)<br>1,665 (25.4%)<br>2,244 (16.2)<br>2,201 (10.0,3.00)<br>0.00,40.00<br>163 (13.4)<br>100 (10.0,2.00) | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) -0.00 (-0.06, 0.05) -(-, -) -(-, -) -0.02 (-0.06, 0.03) -(-, -) |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests, n (%) Mammograms, n (%) Telemedicine, n (%) Telemedicine, n (%) HAAKC tests Lmean (sd) Lmedian (ligR) Lmin, max Upid panels Lmean (sg) Lmean (sg) Lmean (sg) Lmean (sg) | 840 (6.0%)<br>3.456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2.651 (9.1%)<br>2.300 (16.6%)<br>2.09 (1.6.2)<br>2.00 (1.00, 3.00)<br>0.00, 55.00 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 897 (4.6%) 1057 (5.4%) 5.232 (27.0%) 6.395 (32.4%) 220 (1.49) 220 (1.09) 0.00, 40.00 | 3.2% (-3.8%, -2.7%) -0.6% (-1.6%, 0.3%) -2.1% (1.6%, 0.2%) -0.9% (-1.4%, -0.4%) -7.9% (-8.8%, -7.0%) -15.9% (-16.8%, -15.0%) -0.12 (-0.16, -0.09) -(, -) -(, -) -(, -) -0.12 (-0.15, -0.09) | 495 (7.5%)<br>1,721 (26.3%)<br>366 (5.6%)<br>330 (5.0%)<br>1,516 (23.1%)<br>1,634 (24.9%)<br>2,00 (1.00, 3.00)<br>0,00, 33.00<br>1,61 (1.29) | 504 (7.7%)<br>1771 (27.0%)<br>371 (5.7%)<br>317 (4.8%)<br>1494 (22.8%)<br>1665 (25.4%)<br>2244 (16.2<br>200110.0, 3.00)<br>0.00, 40.00 | -0.1% (-1.1%, 0.8%)<br>-0.8% (-2.3%, 0.8%)<br>-0.1% (-0.9%, 0.7%)<br>-0.2% (-0.6%, 1.0%)<br>-0.3% (-1.1%, 1.8%)<br>-0.5% (-2.0%, 1.0%)<br>-0.00 (-0.05, 0.05)<br>-(; -)<br>-(; -)<br>-0.02 (-0.05, 0.03) |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammagams; (%) Telemedicine; n (%) HabAIC tests maan (sd)median IQR min max iman (sd)men (sd) | 840 (6.0%)<br>3.456 (24.9%)<br>923 (6.6%)<br>621 (4.5%)<br>2.651 (19.1%)<br>2.300 (16.6%)<br>2.09 (1.62)<br>2.00 (1.03.300)<br>0.00.55.00 | 1,831 (9.3%) 5,034 (25.5%) 897 (4.6%) 1057 (5.4%) 5,322 (27.0%) 6,355 (32.4%) 2,00 (100,3.00) 0,00,40,00 | 3.2% (-3.8%, 2.7%) -0.6% (-1.6%, 0.3%) -2.1% (1.6%, 2.6%) -0.9% (-1.4%, -0.4%) -7.9% (-3.8%, -7.0%) -15.9% (-1.6, -0.09) -(-, -) -0.12 (-0.15, -0.09) -(-, -) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 330 (5.0%) 1.516 (23.1%) 1.634 (24.9%) 2.24 (1.51) 2.00 (1.00, 3.00) 0.00, 3.30 0 1.61 (1.29) 1.00 (1.00, 2.00) | 504 (77%)<br>1771 (27%)<br>371 (57%)<br>371 (57%)<br>371 (45%)<br>1,494 (228%)<br>1,494 (228%)<br>1,665 (25.4%)<br>2,244 (16.2)<br>2,201 (10.0,3.00)<br>0.00,40.00<br>163 (13.4)<br>100 (10.0,2.00) | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) -0.00 (-0.06, 0.05) -(-, -) -(-, -) -0.02 (-0.06, 0.03) -(-, -) |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammagamar, n (%) Telemedicine; n (%) Telemedicine; n (%) HabAIC tests Lmean (sd) Lmedan IIQR Limit max Lipid panels Limean (sd) Lmedan IIQR Limit max Creatinine tests Lmean (sd) Lmedan IIQR Lmini max Creatinine tests Lmean (sd) Lmedan IIQR | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 2.651 (19.1%) 2.851 (19.1%) 2.300 (16.6%) 2.001 (16.2) 2.001 (16.2) 2.001 (10.0, 3.00) 0.00, 55.00 15.0 (1.38) 1.001 (1.00, 2.00) 0.00, 9.00 0.00 (0.00, 0.00) | 1,831 (9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.395 (22.4%) 2.20 (100.3.00) 0.00, 40.00 162 (12.7) 100 (1.00, 2.00) 0.00, 3.00 0.00, 0.00 0.00, 0.00 0.00, 0.00 0.00, 0.00 0.00, 0.00 0.00, 0.00 0.00, 0.00 | 3.2% (-3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.9% (1.0%, 2.6%) -0.9% (1.4%, 0.4%) -7.9% (8.8%, -7.0%) -15.9% (8.8%, -7.0%) -15.9% (1.6.6.%, 15.0%) -0.12 (-0.16, -0.09) -(c) | 495 (7.6%) 1,721 (26.3%) 366 (5.6%) 360 (5.6%) 330 (5.0%) 1,516 (2.3.1%) 1,634 (24.9%) 200 (1.00. 3.00) 0,00. 3.3.00 1,51 (1.29) 1,00 (1.00. 2.00) 0,00 (1.00. 0.00) 0,00 (1.00. 0.00) | 504 (7.7%)<br>1771 (27.0%)<br>371 (5.7%)<br>371 (5.7%)<br>371 (4.5%)<br>1,655 (25.4%)<br>1,655 (25.4%)<br>2,001 (100, 3.00)<br>0,00, 40.00<br>1,63 (13.4)<br>1,001 (100, 2.00)<br>0,00, 3.00<br>0,00 (3.00)<br>0,00 (3.00)<br>0,00 (0,00)<br>0,00 (0,00) | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.9%) 0.5% (-2.0%, 1.0%) -0.00 (-0.05, 0.05) -11 -11 -11 -0.02 (-0.06, 0.03) -11 - |
| Pap smear n (%) Fecal occult blood test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Marmorgams; n (%) Telemedicine; n (%) HABAC tests _mean (sd) _meit n nax _upid n nax _median (QR _min; nax _upid n nax _median (QR _min; nax _median (QR _min; nax _median (QR _min; nax _median (QR _min; nax _median (QR _min; nax | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 622 (4.5%) 2230 (1.6.5%) 2230 (1.6.5%) 2209 (1.6.2) 2209 (1.6.2) 2201 (1.0.3.30) 0.00.55.00 150 (1.38) 100 (1.0.2.00) 0.00, 45.00 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 897 (4.6%) 1.057 (5.4%) 5.252 (27.0%) 6.395 (32.4%) 220 (1.49) 220 (1.49) 220 (1.00, 3.00) 0.00, 40.00 152(127) 100 (10.0, 2.00) 0.00, 34.00 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.6%, -2.6%) -0.9% (1.6, -2.6%) -0.12 (0.16, -0.09) -(-, -) -(-, -) -0.12 (0.15, -0.09) -(-, -) | 495 (7.6%) 1.771 (26.3%) 366 (5.6%) 330 (5.0%) 1.56 (23.1%) 1.56 (23.1%) 1.56 (24.5%) 2.24 (1.51) 2.20 (1.00, 3.00) 0.00, 33.00 1.61 (1.29) 1.00 (1.00, 2.00) 0.00, 19.00 0.06 (0.38) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 317 (4.8%) 1454 (22.8%) 1665 (25.4%) 224 (162) 2201 (103.300) 0.00, 40.00 153 (1.34) 1.00 (10.0, 2.00) 0.00, 34.00 | 0.1% (-1.1%, 0.8%) 0.3% (-2.3% 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.6%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.05) -(-, -) |
| Pap smear n (%) Fiscal occult blood test n (%) Fiscal occult blood test n (%) Fiscal occult blood test n (%) Bone mineral density tests; n (%) Marmograms; (%) Fiscandicine; n (%) HabAIC tests Limean (sd) Limean | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 821 (4.5%) 923 (6.0%) 2651 (19.1%) 2651 (19.1%) 269 (1.62) 200 (1.6.0%) 209 (1.62) 200 (1.0.0, 3.00) 000, 55.00 150 (1.38) 100 (1.00, 2.00) 000, 49.40) 000 (9.0.0, 0.00) 000 (1.0.0, 0.00) | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.323 (27.0%) 6.224%) 2.201.00, 3.00) 0.00, 40.00 1.621 (127) 1.621 (127) 1.601 (100, 2.00) 0.00, 40.00 0.05 (0.39) 0.001 (0.00, 0.00) 0.00, 23.00 | 3.2% (-3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -7.9% (8.8%, -7.0%) -15.9% (1.6.5%, 15.0%) -0.12 (0.16, -0.09) -(c) | 495 (7.6%) 1,721 (26.3%) 366 (5.6%) 360 (5.6%) 330 (5.0%) 1,516 (2.3.1%) 1,536 (2.3.1%) 1,536 (2.3.1%) 1,534 (24.9%) 2,24 (1.51) 2,001(.00, 3.00) 0,00, 3.3.00 1,516 (1.29) 1,517 (1.20) 1,518 (1.20) 1, | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (6.7%) 1394 (22.5%) 1494 (23.5%) 1494 (23.5%) 14 | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.9%) 0.5% (-2.0%, 1.0%) 0.00 (-0.05, 0.05) -(1) - |
| Pap smear n (%) Fecal occult blood test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Marmorgams; n (%) Telemedicine; n (%) HABAC tests _mean (sd) _meit n nax _upid n nax _median (QR _min; nax _upid n nax _median (QR _min; nax _median (QR _min; nax _median (QR _min; nax _median (QR _min; nax _median (QR _min; nax | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 621 (4.5%) 923 (6.0%) 2651 (19.1%) 2651 (19.1%) 2650 (19.1%) 200 (16.6%) 209 (1.62) 200 (10.0 3.00) 000. 55.00 1001 (10.0 2.00) 000. 49.00 008 (0.48) 000 (0.00, 0.00) 000 (0.00, 0.00) 0018 (0.97) | 1,831(9,3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5,323 (27.0%) 6,335 (22.4%) 2,27 (4.4%) 2,001 (0.0, 0.00) 0,00, 40.00 1,00, 40 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.6%, -2.6%) -0.9% (1.6, -2.6%) -0.12 (0.16, -0.09) -(-, -) -(-, -) -0.12 (0.15, -0.09) -(-, -) | 495 (7.6%) 1,721 (26.3%) 366 (5.6%) 369 (5.6%) 330 (5.0%) 1,516 (2.3.1%) 1,534 (24.9%) 2,24 (1.51) 2,001 (0.0.3.00) 0,00,33.00 1,00 (1.0.0.2.00) 0,00 (1.0.0.2.00) 0,00 (1.0.0.00) 0,00 (1.0.0.00) 0,19 (1.0.00) | 504 (77%) 1771 (27%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1394 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (23.5%) 1494 (2 | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.9%) 0.5% (-2.0%, 1.0%) -0.00 (-0.05, 0.05) -11 -11 -11 -0.02 (-0.06, 0.03) -11 - |
| Pap smearn (%) PSA fest In (%) Fecal occult Blood set in (%) Bone mineral density teets; in (%) Marrinogams; n (%) Marrinogams; n (%) Telemedicine n (%) HEALC teetsmean (sd)median (IQR]min, max Upid panelsmean (sd)median (IQR]min, max Condition (S)median (IQR]min, max Respectively Respectivel | 840 (6.0%) 3.456 (24.9%) 923 (6.6%) 621 (4.5%) 621 (4.5%) 622 (4.5%) 623 (1.6%) 623 (1.6%) 624 (1.6%) 625 (1.6%) 626 (1.6%) 626 (1.6%) 626 (1.6%) 627 (1.6%) 628 (1.6%) 628 (1.6%) 629 (1.6%) 620 (1.6 | 1831(9.3%) 5.034 (25.5%) 897 (4.6%) 1.057 (5.4%) 5.232 (27.0%) 6.399 (3.24%) 5.232 (27.0%) 6.399 (3.24%) 2.21 (1.4%) 2.20 (1.0%) 0.00, 40.00 162 (1.27) 100 (1.0%) 100 (1.0%) 0.00, 40.00 0.05 (0.39) 0.00 (0.0%) 0.00, 23.00 0.00, 23.00 0.00, 23.00 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, 2.6%) -2.1% (1.6%, 2.6%) -2.1% (1.6%, 2.6%) -7.9% (-8.8%, -7.0%) -15.9% (-1.6.%, -0.4%) -0.12 (-0.15, -0.09) -(-), -1 -(-) -0.12 (-0.15, -0.09) -(-) -(-) -0.12 (-0.15, -0.09) -(-) -(-) -0.3 (-0.05, -0.01) | 495 (7.6%) 1.771 (26.3%) 366 (5.6%) 320 (5.0%) 1.516 (23.1%) 1.534 (24.5%) 1.534 (24.5 | 504 (77%) 1771 (27%) 371 (57%) 371 (57%) 371 (57%) 371 (48%) 1494 (22.8%) 1494 (22. | 0.1% (-1.1%, 0.8%) 0.1% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.05) -(c, -) -(c, - |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests n (%) Mammograms; n (%) Telemedicine; n (%) Telemedicine; n (%) HABAE tests Lmean (sd) Lmedan (lQR) Lmin, max Upid panels Lmean (sd) Lmedan (lQR) Lmin max Ceatinine tests Lmean (sd) Lmean (sd) Lmean (lQR) Lmin max Veratione tests Lmean (sd) Lmean (sd) Lmean (lQR) Lmin max Veratione tests Lmean (sd) Lmean (sd) Lmean (sd) Lmean (sd) Lmean (sd) Lmean (sd) Lmean (sd) Lmin max Veratione tests Lmean (sd) Lmin max Veratione tests Lmean (sd) Lmin max Veratione tests Lmean (sd) Lmin max Veratione tests | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 621 (4.5%) 923 (6.0%) 2651 (19.1%) 2651 (19.1%) 2650 (19.1%) 200 (16.5) 200 (16.5) 200 (16.5) 200 (16.0) 200 (16.0) 000, 55.00 000 (10.0) | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5,232 (27.0%) 6,395 (32.4%) 220 (1.49) 220 (1.49) 220 (1.00, 3.00) 0.00, 40.00 162 (1.27) 100 (1.00, 2.00) 0.00, 34.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00, 22 (0.97) 0.00 (0.00, 0.00) 0.00 (2.00) | 3.2% (3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -7.9% (8.8%, 7.0%) -1.5.9% (1.6.5%, 1.5.0%) -0.12(-0.15, -0.09) -(c) | 495 (7.6%) 1,721 (26.3%) 366 (5.6%) 369 (5.6%) 330 (5.0%) 1,516 (23.1%) 1,536 (23.1%) 1,536 (23.1%) 1,534 (24.9%) 2,24 (1.51) 2,001 (0.0, 3.00) 0,00, 3.3.00 1,516 (2.1%) 1,516 (1.2%) 1,51 | 504 (77%) 1771 (27%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1394 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (23.5%) 1494 (2 | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.9%) 0.3% (-1.1%, 1.9%) 0.00 (-0.05, 0.05) -(, -) - |
| Pap smearn (%) PSA fest In (%) Fecal occult Blood set in (%) Bone mineral density teets; in (%) Marrinogams; n (%) Marrinogams; n (%) Telemedicine n (%) HEALC teetsmean (sd)median (IQR]min, max Upid panelsmean (sd)median (IQR]min, max Condition (S)median (IQR]min, max Respectively Respectivel | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 621 (4.5%) 923 (6.0%) 2651 (19.1%) 2651 (19.1%) 2650 (19.1%) 200 (16.6%) 209 (1.62) 200 (10.0 3.00) 000. 55.00 1001 (10.0 2.00) 000. 49.00 008 (0.48) 000 (0.00, 0.00) 000 (0.00, 0.00) 0018 (0.97) | 1,831(9,3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5,323 (27.0%) 6,335 (22.4%) 2,27 (4.4%) 2,001 (0.0, 0.00) 0,00, 40.00 1,00, 40 | 3.2% (-3.8%, -2.7%) -0.5% (1.6%, 2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -1.5% (1.6%, 2.6%) -0.9% (1.6%, 2.6%) -0.9% (1.6%, 1.5.0%) -0.12 (-0.15, -0.09) -1.5, -1.5 | 495 (7.6%) 1,721 (26.3%) 366 (5.6%) 369 (5.6%) 330 (5.0%) 1,516 (2.3.1%) 1,534 (24.9%) 2,24 (1.51) 2,001 (0.0.3.00) 0,00,33.00 1,00 (1.0.0.2.00) 0,00 (1.0.0.2.00) 0,00 (1.0.0.00) 0,00 (1.0.0.00) 0,19 (1.0.00) | 504 (77%) 1771 (27%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1394 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (23.5%) 1494 (2 | 0.1% (-1.1%, 0.8%) 0.8% (-2.3% 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.9%) 0.3% (-1.1%, 1.9%) 0.00 (-0.05, 0.05) (-1.1%, 1.9%) 0.00 (-0.05, 0.05) (-1.1%, 1.9%) 0.00 (-0.05, 0.05) (-1.1%, 1.9%) 0.00 (-0.05, 0.05) (-1.1%, 1.9%) 0.00 (-0.05, 0.05) (-1.1%, 1.9%) (-1. |
| Pap smearn (%) PSA fest In (%) Fecal occult Blood fest in (%) Bone mineral density feets; in (%) Manningams; in (%) "median (light) "min, max Upid panels "mean (sd) "min, max Creatifine tests "mean (sd) "min, max Nathuretic peptide feets "mean (sd) "min, max Varientic feets "mean (sd) "min, max Unim max Urin max Urin max Urin tests "mean (sd) "min, max Urin max Urin tests "mean (sd) "min, max Urin tests "mean (sd) "min, max Urin tests "mean (sd) "min, max Urin tests "mean (sd) | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 250 (16.6%) 250 (16.6%) 250 (16.6%) 250 (16.6%) 250 (16.5%) 150 (1.38) 100 (1.00, 2.00) 0.00, 45.00 0.03 (0.48) 0.00 (1.00, 0.00) 0.00, 59.00 | 1,831 (9.3%) 5,034 (25.5%) 897 (4.6%) 10.57 (5.4%) 5,221 (27.0%) 6,395 (32.4%) 5,323 (27.0%) 6,395 (32.4%) 220 (1.0%) 0,00,40,00 10.00 (1.0%) | 3.2% (3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -7.9% (8.8%, 7.0%) -1.5.9% (1.6.5%, 1.5.0%) -0.12(-0.15, -0.09) -(c) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 366 (5.6%) 360 (5.6%) 1.516 (23.1%) 1.516 (23.1%) 1.516 (23.1%) 1.534 (24.5%) 1.634 (24.5%) | 504 (77%) 1771 (27%) 371 (57%) 371 (57%) 371 (57%) 371 (57%) 371 (48%) 1,494 (228%) 1,494 (248%) | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.8%) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.5% (-2.0% 1.0%) 0.00 (-0.06, 0.05) -(c, -) |
| Pap smear n (%) Fecal occult blood test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Marmorgams; n (%) Telemedicine; n (%) HABAC tests Lman (sd) Lmedan (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedan (lQR) Lmin; nax Ceatimin tests Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax | 840 (6.0%) 3.456 (24.9%) 923 (6.6%) 621 (4.5%) 621 (4.5%) 2.300 (1.6.0%) 2.300 (1.6.0%) 2.300 (1.6.0%) 2.300 (1.6.0%) 1.50 (1.3.0%) 1.50 (1.3. | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 1057 (5.4%) 5.232 (27.0%) 6.399 (32.4%) 221 (1.49) 220 (1.09) 0.00, 40.00 152 (127) 100 (1.00, 2.00) 0.00, 40.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00, 0.00 0.00, | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.6%, -2.6%) -0.9% (1.6%, -0.6%) -0.9% (1.6%, -0.6%) -0.12 (-0.15, -0.09) -(-, -) | 495 (7.6%) 1.771 (26.3%) 365 (5.6%) 336 (5.6%) 336 (5.6%) 330 (5.0%) 1.516 (23.1%) 1.534 (24.9%) 2.24 (1.51) 2.201 (1.00, 3.00) 0.00, 3.00 1.51 (1.29) 1.001 (1.00, 2.00) 0.00 (1.30) 0.00 (1.00) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (7.1%) 371 (7.4.8%) 1655 (25.4%) 1655 (25.4%) 1655 (25.4%) 1655 (25.4%) 1650 (25.4%) 1651 (25.4%) | 0.1% (-1.1%, 0.8%) 0.3% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.2% (-0.6%, 1.0%) 0.2% (-0.6%, 1.0%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.05) -(-, 2) -(-, 3) -(-, 2) -(-, 3) -(-, 3 |
| Pap smear n (%) PSA test n (%) Fecal occult bload test n (%) Bone mineral density tests; n (%) Mammograms; n (%) "min max Upid panels "man (sd) "min max Upim tests "man (sd) "min max Üm tests "medan (lQR] | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.0%) 2001 (10.0 3.00) 0.00, 55.00 150 (13.8) 150 (13.8) 0.08 (0.48) 0.00 (10.0, 0.00) 0.00, 19.00 110 (19.7) 100 (10.0, 2.00) 110 (1.97) 100 (1.90, 2.00) 200, 25.00 | 1,831(9,3%) 5,034 (25.5%) 897 (4.6%) 1057 (5.4%) 5,322 (27.0%) 5,322 (27.0%) 5,325 (32.4%) 2,001 (10.3.00) 0,00 (40.00) 162 (12.7) 100 (10.0.200) 0,00,34.00 0,00 (30.0.00) 0,00 (30.0.00) 0,00 (30.0.00) 0,00 (30.0.00) 1,00 (10.0.00) | 3.2% (3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -7.9% (8.8%, 7.0%) -1.5.9% (1.6.5%, 1.5.0%) -0.12(-0.15, -0.09) -(c) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 360 (5.6%) 360 (5.6%) 1.516 (23.1%) 1.516 (23.1%) 1.516 (23.1%) 1.524 (1.51) 1.524 (1.51) 1.534 (24.9%) 1.536 (23.1%) 1.536 (23.1%) 1.536 (23.1%) 1.536 (23.1%) 1.536 (23.1%) 1.537 (2.00) 1.500 (1.00, 3.00) 1.73 (2.00) 1.73 (2.00) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (4.5%) 1374 (5.7%) 1374 (5.7%) 1494 (22.8%) 1665 (22.4%) 1665 (22.4%) 1665 (22.4%) 1663 (13.4%) 163 (13.4%) 163 (13.4%) 163 (13.4%) 160 (10.0, 2.00) 174 (2.00) | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.8%) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.5% (-2.0% 1.0%) 0.00 (-0.06 0.05) -1;,-3 -1 |
| Pap smear n (%) Fecal occult blood test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Marmorgams; n (%) Telemedicine; n (%) HABAC tests Lman (sd) Lmedan (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedan (lQR) Lmin; nax Ceatimin tests Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax Lipid panels Lmean (sd) Lmedin (lQR) Lmin; nax | 840 (6.0%) 3.456 (24.9%) 923 (6.6%) 621 (4.5%) 621 (4.5%) 2.300 (1.6.0%) 2.300 (1.6.0%) 2.300 (1.6.0%) 2.300 (1.6.0%) 1.50 (1.3.0%) 1.50 (1.3. | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 1057 (5.4%) 5.232 (27.0%) 6.399 (32.4%) 221 (1.49) 220 (1.09) 0.00, 40.00 152 (127) 100 (1.00, 2.00) 0.00, 40.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00, 0.00 0.00, | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.6%, -2.6%) -0.9% (1.6%, -0.6%) -0.9% (1.6%, -0.6%) -0.12 (-0.15, -0.09) -(-, -) | 495 (7.6%) 1.771 (26.3%) 365 (5.6%) 336 (5.6%) 336 (5.6%) 330 (5.0%) 1.516 (23.1%) 1.534 (24.9%) 2.24 (1.51) 2.201 (1.00, 3.00) 0.00, 3.00 1.51 (1.29) 1.001 (1.00, 2.00) 0.00 (1.30) 0.00 (1.00) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (7.1%) 371 (7.4.8%) 1655 (25.4%) 1655 (25.4%) 1655 (25.4%) 1655 (25.4%) 1650 (25.4%) 1651 (25.4%) | 0.1% (-1.1%, 0.8%) 0.3% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.05) -(;-) |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Marmingams; n (%) Telemédicine n (%) HabAlC tests _mean (sd) _median ID(R] _min, max | 840 (6.0%) 3.456 (24.9%) 923 (6.6%) 621 (4.5%) 621 (4.5%) 2.300 (1.6.2%) 2.300 (1.6.2%) 2.300 (1.6.2%) 2.300 (1.0.3 300) 0.00, 55.00 1.50 (1.38) 1.001 (1.0.2 2.00) 0.00 (1.0.48) 0.00 (1.0.0.0 0.00) 0.00 (1.0.0 0.00) | 1831(9.3%) 5334(25.5%) 887(4.6%) 1057(5.4%) 5.523(27.0%) | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -1.8% (1.6%, -2.6%) -1.9% (1.4%, -0.4%) -7.9% (4.8%, -7.6%) -1.9% (1.6.%, -7.6%) -1.9% (1.6.%, -7.6%) -1.9% (1.6.%, -1.6.%) -1.9% (1.6.%, | 495 (7.6%) 1.771 (26.3%) 365 (5.6%) 360 (5.6%) 360 (5.6%) 1.616 (23.1%) 1.616 (23.1%) 1.634 (24.9%) | 504 (77%) 1771 (27%) 371 (57%) 371 (57%) 371 (57%) 371 (57%) 371 (48%) 1494 (22.8%) 1494 (23.8%) 1494 (24.8%) | 0.1% (-1.1%, 0.8%) 0.3% (-2.3% 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.05) -(c, -) |
| Pas smearn (%) Post a test n (%) Fecal occult bload test n (%) Fecal occult bload test n (%) Mammograms; n (%) Mammogram | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.0%) 2300 (16.0% | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.395 (22.4%) 5.323 (27.0%) 6.395 (22.4%) 200 (100, 3.00) 0.00, 40.00 162 (12.7) 100 (100, 2.00) 0.00, 34.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00, 23.00 0.01 (0.00, 0.00) 0.00, 42.00 106 (1.82 0.00 (1.00, 1.00) 0.00, 53.00 165 (1.82 0.00 (1.00, 1.00) 0.00, 53.00 165 (1.95) 166 (1.95) 166 (1.95) | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -7.9% (1.8%, -0.4%) -7.9% (1.8%, -7.0%) -15.9% (1.6.5%, -1.5.0%) -0.12 (-0.15, -0.09) -(-, -) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 360 (5.6%) 330 (5.0%) 1.516 (23.1%) 1.634 (24.9%) 2.24 (1.51) 2.00 (1.00, 3.00) 0.00, 33.00 1.61 (1.29) 1.61 (1.29) 0.00 (1.00, 2.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (2.00 (2.00 0.00 (2.00 ( | 504 (77%) 1771 (270%) 371 (57%) 371 (57%) 371 (57%) 371 (57%) 371 (47%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (24.8%) 1494 (24.8% | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) -1.00 (-0.06, 0.05) -1.00 (-0.06, 0.05) -1.00 (-0.06, 0.03) -1.00 (-0.06, 0.03) -1.00 (-0.06, 0.03) -1.00 (-0.06, 0.03) -1.00 (-0.07, 0.06) -1.00 (-0.07, 0.06) -1.00 (-0.07, 0.06) -1.00 (-0.07, 0.06) -1.00 (-0.08, 0.06) -1.00 (-0.08, 0.06) -1.00 (-0.09, 0.09) |
| Pap smearn (%) Fiscal occult Blood set n (%) Fiscal occult Blood set n (%) Bone mineral density tests; n (%) Marrinogams; n (%) Telemedicine; n (%) Telemedicine; n (%) HAAC testsmeal n (sd)median (IQR)min, max Upid panelsmeal n (sd)median (IQR)min, max Contine testsmean (sd)median (IQR)min, max Nathuretic peptide testsmean (sd)median (IQR)min, max Unin max Combined (IQR)min, max Combined (IQR)min, max Combined (IQR)min, max Combined comobility scoremean(sd)median (IQR)min, max Combined comobility scoremean(sd)median (IQR)min, max Combined comobility scoremean(sd)median (IQR)min, maxmean(sd)median (IQR)min, max | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 2260 (1.6.6%) 2200 (1.6.0%) 2200 (1.0.0 (1.0.0%) 200 (1.0.0 (1.0.0%) 150 (1.3.8) 100 (1.0.0 (1.0.0 (1.0.0%) 0.00 (1.0.0 (1.0.0 (1.0.0%) 0.00 (1.0.0 (1.0 | 1831(9.3%) 5.034 (25.5%) 897 (4.6%) 1.057 (5.4%) 5.232 (27.0%) 6.399 (32.4%) 5.232 (27.0%) 6.399 (32.4%) 182 (12.7) 100 (100.2.00) 0.00, 40.00 0.55 (3.2%) 0.00 (3.0%) | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -1.2% (1.6%, -2.6%) -1.2% (1.6%, -2.6%) -1.5% (1.6%, -2.6%) -1.5% (1.6%, -3.6%) -1.5% | 495 (7.6%) 1.771 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (23.1%) | 504 (77%) 1771 (27%) 371 (57%) 371 (57%) 371 (57%) 371 (57%) 371 (48%) 1494 (228%) 1494 (248%) 1494 (2 | 0.1% (-1.1%, 0.8%) 0.1% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.05) -(c, -) |
| Pas smearn (%) Post a test n (%) Fecal occult bload test n (%) Fecal occult bload test n (%) Mammograms; n (%) Mammogram | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.0%) 2300 (16.0% | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.395 (22.4%) 5.323 (27.0%) 6.395 (22.4%) 200 (100, 3.00) 0.00, 40.00 162 (12.7) 100 (100, 2.00) 0.00, 34.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00, 23.00 0.01 (0.00, 0.00) 0.00, 42.00 106 (1.82 0.00 (1.00, 1.00) 0.00, 53.00 165 (1.82 0.00 (1.00, 1.00) 0.00, 53.00 165 (1.95) 166 (1.95) 166 (1.95) | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -7.9% (1.8%, -0.4%) -7.9% (1.8%, -7.0%) -15.9% (1.6.5%, -1.5.0%) -0.12 (-0.15, -0.09) -(-, -) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 360 (5.6%) 330 (5.0%) 1.516 (23.1%) 1.634 (24.9%) 2.24 (1.51) 2.00 (1.00, 3.00) 0.00, 33.00 1.61 (1.29) 1.61 (1.29) 0.00 (1.00, 2.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (2.00 (2.00 0.00 (2.00 ( | 504 (77%) 1771 (270%) 371 (57%) 371 (57%) 371 (57%) 371 (57%) 371 (47%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (22.8%) 1494 (24.8%) 1494 (24.8% | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.8%) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.5% (-2.0% 1.0%) 1.6, -1.1% 1.8%) 0.00 (-0.06, 0.05) 1.6, -1 1.6, - |
| Pap smear n (%) PSA test n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Morningarins; n (%) Mammograms; n (%) HeALC testsmean (sd)min max Upid panelsmeal n (pidmin max Upid panelsmeal n (pidmin max Condition testsmeal n (pidmin max Maturetic poptide testsmeal n (pidmin, max Upid panelsmin max Combined condition (pidmin, max Upid panelsmin max Upid panels | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 923 (6.6%) 250 (14.5%) 250 (10.0%) 250 (10.0%) 200 (10.0 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.395 (22.4%) 200 1100, 3.001 0.00, 40.00 162 (12.7) 100 (1.00, 2.00) 0.00, 3.00 0.00, 40.00 0.00 (2.00, 0.00) 0.00, 3.00 0.00 (2.00, 0.00) 0.00, 3.00 0.00 (2.00, 0.00) 0.00, 3.00 0.00 (2.00, 0.00) 106 (1.82 0.00 (1.00, 0.00) 106 (1.82 0.00 (1.00, 0.00) 107 (1.00) 108 (1.00) 109 (1.00) | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -1.2% (1.6%, -2.6%) -1.2% (1.6%, -2.6%) -1.5% (1.6%, -2.6%) -1.5% (1.6%, -3.6%) -1.5% | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.524 (24.9%) 2.24 (1.51) 2.001(1.00, 3.00) 0.00, 3.3.00 1.61 (1.29) 1.001(1.00, 2.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (2.00) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (6.7%) 1,655 (25.4%) 1,655 ( | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.03) -(-, -) |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Manningams; n (%) Manningams; n (%) Telemeticine n (%) HabAC tests _media (sd) _media (sd) _min max Upid panels _mean (sd) _man (sd) _min max Continue tests _mean (sd) _min max Upid panels _min max Combined (sd) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _median (lQR) _min max Upid panels _median (lQR) _median (lQR) _min max Upid panels _median (lQR) | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 2250 (16.6%) 2200 (16.0%) 2200 (16.0%) 2200 (10.0%) 200 (10.0%) 150 (13.8) 100 (10.0%) 100 ( | 1,831(9,3%) 5,034 (25.5%) 897 (4.6%) 10.57 (5.4%) 5,221 (27.0%) 6,399 (32.4%) 220 (1.4%) 162 (12.77) 100 (10.0,200) 0.00, 34.00 105 (0.38) 0.001 (0.00,000) 0.00, 23.00 106 (1.82) 0.001 (0.00,000) 106 (1.82) 0.001 (0.00,000) 106 (1.82) 0.001 (0.00,000) 105 (1.38) 0.001 (0.00,000) 106 (1.83) 106 (1.83) 107 (1.84) 108 (1.85) 109 (1 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.6%, -0.4%) -0.12 (0.15, -0.09) -(-, -) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 366 (5.6%) 367 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.5 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (4.8%) 1,494 (22.8%) 1,494 (23.8%) 1,49 | 0.1% (.11% 0.8%) 0.8% (.23% 0.89) 0.1% (.0.9% 0.87) 0.1% (.0.9% 0.7%) 0.2% (.0.6% 1.0%) 0.3% (.1.1% 1.8%) 0.5% (.2.0% 1.0%) 0.00 (-0.06, 0.05) 1(c.) |
| Pap smear n (%) PSA test n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Mormorgrams; n (%) Mormorgrams; n (%) Mormorgrams; n (%) HeALC tests | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 821 (4.5%) 923 (6.6%) 263 (19.1%) 265 (19.1%) 265 (19.1%) 260 (16.0%) 200 (16.0 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.395 (22.4%) 2.00 (100.3.00) 0.00, 40.00 160 (100.2.00) 0.00, 3.00 0.00 (20.0.00) 0.00 (20.0.00) 0.00 (20.0.00) 0.00 (20.0.00) 0.00 (20.0.00) 106 (18.2 0.00 (100.0.00) 106 (18.3 0.00 (100.0.00) 106 (100.0.00) 106 (100.0.00) 106 (100.0.00) 106 (100.0.00) 106 (100.0.00) 106 (100.0.00) 106 (100.0.00) | 3.2% (3.8%, 2.7%) 0.6% (1.6%, 2.6%) 0.6% (1.6%, 2.6%) 0.9% (1.4%, 0.4%) 7.9% (8.8%, 7.0%) 15.9% (16.6%, 1.50%) 0.12 (0.16, 0.0%) 16.9 0.12 (0.16, 0.0%) 16.9 0.02 (0.01, 0.0%) 16.9 0.03 (0.05, 0.01) 16.9 0.04 (0.00, 0.08) 16.9 0.37 (0.33, 0.42) 16.9 0.01 (0.01, 0.01) 16.9 0.10 (0.01, 0.01) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (2.3.1%) 1.511 (2.3.1%) 1.511 (2.3.1 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1,655 (25.4%) 1,655 (25.4%) 2,001 (100, 3.00) 0,00, 40.00 0,00, 40.00 1,63 (13.4) 1,001 (100, 2.00) 0,00, 34.00 0,00 (100, 3.00) 0,00 (100, 3.00) 0,00 (100, 3.00) 0,00 (100, 3.00) 1,00 (10 | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.89) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.5% (-2.0% 1.0%) 0.00 (-0.06 0.05) 1.(-1) 1. |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Manningams; n (%) Manningams; n (%) Telemeticine n (%) HabAC tests _media (sd) _media (sd) _min max Upid panels _mean (sd) _man (sd) _min max Continue tests _mean (sd) _min max Upid panels _min max Combined (sd) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _min max Upid panels _median (lQR) _median (lQR) _min max Upid panels _median (lQR) _median (lQR) _min max Upid panels _median (lQR) | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 2250 (16.6%) 2200 (16.0%) 2200 (16.0%) 2200 (10.0%) 200 (10.0%) 150 (13.8) 100 (10.0%) 100 ( | 1,831(9,3%) 5,034 (25.5%) 897 (4.6%) 10.57 (5.4%) 5,221 (27.0%) 6,399 (32.4%) 220 (1.4%) 162 (12.77) 100 (10.0,200) 0.00, 34.00 105 (0.38) 0.001 (0.00,000) 0.00, 23.00 106 (1.82) 0.001 (0.00,000) 106 (1.82) 0.001 (0.00,000) 106 (1.82) 0.001 (0.00,000) 105 (1.38) 0.001 (0.00,000) 106 (1.83) 106 (1.83) 107 (1.84) 108 (1.85) 109 (1 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.6%, -0.4%) -0.12 (0.15, -0.09) -(-, -) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 366 (5.6%) 367 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.5 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (4.8%) 1,494 (22.8%) 1,494 (23.8%) 1,49 | 0.1% (.11% 0.8%) 0.8% (.23% 0.89) 0.1% (.0.9% 0.87) 0.1% (.0.9% 0.7%) 0.2% (.0.6% 1.0%) 0.3% (.1.1% 1.8%) 0.5% (.2.0% 1.0%) 0.00 (-0.06, 0.05) 1(c.) |
| Pap smear n (%) Fecal occult blood lest n (%) Fecal occult blood lest n (%) Bone mineral density tests; n (%) Mammograms, n (%) Telemekine n (%) HabALC testsmedian [DR]min, max Lipid panelsmedian [DR]min, max Lipid panelsmedian [DR]min, max Constitute testsmedian [DR]min, max Lipid panelsmedian [DR]min, max Lipid panelsmedian [DR]min, maxmedian [DR]min, maxmin, max _ | 840 (6.0%) 3456 (24.9%) 923 (6.5%) 621 (4.5%) 2250 (16.6%) 2200 (16.6%) 2200 (16.6%) 2200 (16.0%) 200 | 1831(9.3%) 5034(25.5%) 897(4.6%) 1057(5.4%) 5.323 (27.0%) 6.395 (32.4%) 5.323 (27.0%) 6.395 (32.4%) 9.201(10.9.3.00) 0.00.40.00 162 (12.7) 100 (10.0.2.00) 0.00,34.00 0.05 (0.39) 0.00 (0.00,0.00) 0.00 (32.00) 0.00 (30.00) 0.00 (30.00) 106 (1.82) 0.00 (0.00) 106 (1.83) 109 (1.84) 109 (1.85) 109 (1.8 | 3.2% (-3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -0.9% (1.4%, 0.4%) -0.9% (1.4%, 0.4%) -0.9% (1.6%, 0.4%) -0.12 (0.15, 0.0%) -0.13 (0.15, 0.0%) -0.14 (0.00, 0.0%) -0.15 (0.15, | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 366 (5.6%) 367 (5.6%) 1.516 (23.1%) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (4.7%) 1.494 (22.8%) 1.49 | 0.1% (.11% 0.8%) 0.8% (.23% 0.89) 0.1% (.0.9% 0.87) 0.1% (.0.9% 0.7%) 0.2% (.0.6% 0.7%) 0.3% (.11% 1.8%) 0.5% (.20% 1.0%) 0.00 (.0.06, 0.05) 1(c, 1) 1(c, 2) 1(c, 3) 1 |
| Pap smear n (%) Pecal accult blood test n (%) Pecal accult blood test n (%) Pecal accult blood test n (%) Pecal accult blood test n (%) Bone minard lassify last is; n (%) Marmorgams; n (%) HeA1C tests | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 923 (6.0%) 924 (6.0%) 925 (14.5%) 926 (14.5%) 926 (14.5%) 926 (14.5%) 927 (14.5%) 928 (14.5%) 929 (14.5%) 929 (14.5%) 920 (14.5 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.323 (27.0%) 6.323 (27.0%) 6.00 (100.3.00) 0.00, 40.00 160 (100.3.00) 0.00 (100.0.00) | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -7.9% (1.8, -0.4%) -7.9% (1.8, -0.4%) -7.9% (1.6, -0.4%) -1.5% (1. | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.516 (25.1%) 1.516 (25.7%) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1394 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (23.6%) 1495 (23.6%) 1495 (23.6%) 1495 (23.6%) 1496 (23 | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.89) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.3% (-1.1% 1.8%) 0.00 (-0.05, 0.05) (-1.1 |
| Pap smear n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammograms, n (%) Telemekione n (%) HabALC tests Lmoan (sd) Lmodan (JoR] Lmin max Llyipid panels Lmean (sd) Lmean (sd) Lmodan (JoR] Lmin max Llyipid panels Lmean (sd) Lmodan (JoR] Lmin max Llyipid panels Lmean (sd) Lmodan (JoR] Lmin max Llyipid panels Lmodan (JoR] Lmin max Llyipid panels Lmodan (JoR) Lmodan (JoR) Lmin max Llyipid Llyipid (JoR) Lmodan (JoR) Lmin max Llyipid (JoR) Lmodan (JoR) Lmod | 840 (6.0%) 3456 (24.9%) 923 (6.5%) 621 (4.5%) 923 (6.5%) 621 (4.5%) 250 (1.6.5%) 25 | 1831(9.3%) 50.34 (25.5%) 897 (4.6%) 1057 (5.4%) 5.322 (27.0%) 6.395 (32.4%) 5.322 (27.0%) 6.395 (32.4%) 22 (0.10) 0.00, 40.00 162 (12.7) 100 (10.0, 2.00) 0.00, 34.00 0.00 (20.0, 0.00) 0.00, 34.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00 (20.0, 0.00) 0.00 (20.0, 0.00) 106 (18.2) 0.00 (0.00, 0.00) 0.00, 30.00 106 (18.2) 0.00 (0.00, 0.00) 0.00, 30.00 0.00, 30.0 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.9% (1.4%, -0.4%) -0.12 (-0.16, -0.09) -(-), -(- | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 366 (5.6%) 367 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.517 (20.1%) 1.5 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (6.7%) 371 (6.7%) 371 (6.7%) 1.094 (22.2%) 1.094 (2.2%) 1.094 (2.2% | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) 0.5% (-2.0%, 1.0%) 0.00 (-0.06, 0.05) -1c, -1 -1c, - |
| Pap smear n (%) Pecal accult blood test n (%) Pecal accult blood test n (%) Pecal accult blood test n (%) Pecal accult blood test n (%) Bone minard lassify last is; n (%) Marmorgams; n (%) HeA1C tests | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 923 (6.0%) 924 (6.0%) 925 (14.5%) 926 (14.5%) 926 (14.5%) 926 (14.5%) 927 (14.5%) 928 (14.5%) 929 (14.5%) 929 (14.5%) 920 (14.5 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.395 (23.4%) 2011.00.3.001 0.00, 40.000 122 (1.4%) 2011.00.3.001 0.00, 40.00 105 (0.3%) 0.00, 40.00 105 (0.3%) 0.00, 40.00 105 (0.3%) 105 (0.3% | 3.2% (-3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -7.9% (8.8%, 7.0%) -1.5 9% (1.6.5%, 1.5.0%) - | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.516 (25.7%) | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1394 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (22.5%) 1494 (23.5%) 1494 (23 | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.89) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.3% (-1.1% 1.8%) 0.00 (-0.05, 0.05) (-1.1 |
| Pap smear n (%) Fecal occult Blood set n (%) Fecal occult Blood set n (%) Bone mineral density tests; n (%) Marmingams; n (%) Telemoticine n (%) HabAlC testsmean (sd)median [IQR]min, max Upid panelsmean (sd)men (sd)men (sd)men (sd)min (sd)min (sd)min (sd)min (sd)min (sd)min (sd)min (sd)men (sd)min (naxmen (sd)min (naxmen (sd)min (sd) | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 923 (6.0%) 923 (6.0%) 924 (6.0%) 925 (14.5%) 926 (14.5%) 926 (14.5%) 929 (1.62) 920 (1 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.335 (32.4%) 2.27 (1.4%) 2.001 (1.0%) 2.001 (1. | 3.2% (3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -7.9% (8.8%, 7.0%) -1.5.9% (1.6.5%, 1.5.0%) -0.12 (0.15, 0.09) -() | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.517 (20.1%) 1.518 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1394 (22.8%) 1494 (22.8%) 1201 (10.3.00) 10.00, 40.00 10.00, 50.00 10.00, | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.89) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.3% (-1.1% 1.8%) 0.0 (-0.05, 0.05) (-1.1 |
| Pas mean n (%) Fecal occult Mond lest n (%) Fecal occult Mond lest n (%) Fecal occult Mond lest n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemekcine n n (%) HebALC tests | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 923 (6.6%) 621 (4.5%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.0%) 23 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 532 (27.0%) 6.395 (22.4%) 5.323 (27.0%) 6.395 (22.4%) 200 (100, 3.00) 0.00, 40.00 162 (12.7) 100 (100, 2.00) 0.03, 40.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00 (20.0, 0.00) 0.01 (0.00, 0.00) 0.00 (20.0, 0.00) 106 (1.82 0.00 (1.00, 0.00) 0.00, 3.00 106 (1.82 0.00 (1.00, 1.00) 0.00, 3.00 106 (1.82 0.00 (1.00, 1.00) 0.00, 3.00 0.00, | 3.2% (-3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -0.9% (1.4%, 0.4%) -0.9% (1.4%, 0.4%) -0.12 (-0.15, -0.09) -(-), -(- | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 336 (5.6%) 336 (5.6%) 336 (5.6%) 330 (5.0%) 1.516 (23.1%) 1.634 (24.9%) 224 (1.51) 200 (1.00, 3.00) 0.00, 33.00 1.61 (12.9) 1.00 (1.00, 2.00) 0.00, 33.00 1.61 (12.9) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (2.00, 0.00) 0.00 (2.00 1.11 (1.75) 1.00 (1.00, 2.00) 1.173 (2.02) 1.00 (1.00, 3.00) 0.01 (1.00, 3.00) 0.05 (0.38) 0.05 (0.38) 0.00 (0.00) 0. | 504 (77%) 1771 (27%) 371 (57%) 371 (57%) 371 (57%) 371 (57%) 371 (47%) 371 (47%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (26.4%) 1,665 (13.4%) 1,665 | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.8%) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.5% (-2.0% 1.0%) 0.5% (-2.0% 1.0%) 0.00 (-0.06 0.05) 1(-) 1(-) 1(-) 1(-) 1(-) 1(-) 1(-) 1(- |
| Pap smear n (%) Fiscal social thood set n (%) Fiscal social thood set n (%) Bone mineral density teets; n (%) Marrinogams; n (%) Telemedicine n (%) HabAC teetsmeal (sd)median [IQR]min, max Upid panelsmeal (sd)median [IQR]min, max Contine testsmean (sd)median [IQR]min, max Nathuretic peptide testsmean (sd)median [IQR]min, max Contine testsmean (sd)median [IQR]min, max Contine testsmean (sd)median [IQR]min, max Contine testsmean (sd)median [IQR]min, max Urine testsmean (sd)median [IQR]min, max Contine controlled (sd)median [IQR]min, max Martinetic peptide testsmean (sd)median [IQR]min, max Martinetic peptide testsmean (sd)median [IQR]min, max Martinetic peptide testsmean (sd)median [IQR]min, max Martinetic peptide (sd)median [IQR]min, max Martinetic peptide (sd)median [IQR]min, max Martinetic peptide (sd)median [IQR]min, max Martinetic peptide (sd)median [IQR]min, max Martinetic peptide (sd)min pask Martinetic peptid | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 923 (6.0%) 923 (6.0%) 924 (6.0%) 925 (14.5%) 926 (14.5%) 926 (14.5%) 929 (1.62) 920 (1 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5.323 (27.0%) 6.395 (23.4%) 2.20 (1.0%) 2.2 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -1.2% (1.6%, 2.6%) -1.5% (1.6%, | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.516 (23.1%) 1.516 (23.1%) 1.516 (23.1%) 1.524 (24.9%) 2.24 (1.51) 2.001 (0.0, 3.00) 0.00, 3.3.00 1.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (2.00) 1.11 (1.75) 1.00 (1.00, 3.00) 1.00 (2.00, 2.00) 1.00 (2.00, 2.00) 1.00 (2.00, 2.00) 1.00 (2.00, 0.00) 0.00 (2.00) 1.00 (2.00, 0.00) 0.00 (2.00) 1.73 (2.02) 1.00 (1.00, 3.00) 1.76 (2.5, 7.7) 0.00 (1.00, 0.00) 0.00 (2.700) 1.78 (1.1%) 1.79 (1.1%) 1.79 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 1394 (22.8%) 1494 (22.8%) 1201 (10.3.00) 10.00, 40.00 10.00, 50.00 10.00, | 0.1% (-1.1%, 0.8%) 0.3% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 0.1%) 0.3% (-1.1%, 1.8%) 0.3% (-1.1%, 1.8%) 0.00 (-0.05, 0.05) (-1, 1, 1 |
| Pas mean n (%) Fecal occult Mond lest n (%) Fecal occult Mond lest n (%) Fecal occult Mond lest n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemekcine n n (%) HebALC tests | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 923 (6.6%) 621 (4.5%) 2300 (16.6%) 2300 (16.6%) 2300 (16.6%) 2300 (16.0%) 2300 (16.0%) 2300 (16.0%) 2300 (16.0%) 2300 (16.0%) 2300 (16.0%) 2300 (16.0%) 2400 (16.0%) 2410 (16.0%) 24 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 532 (27.0%) 6.395 (22.4%) 5.323 (27.0%) 6.395 (22.4%) 200 (100, 3.00) 0.00, 40.00 162 (12.7) 100 (100, 2.00) 0.03, 40.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00 (20.0, 0.00) 0.01 (0.00, 0.00) 0.00 (20.0, 0.00) 106 (1.82 0.00 (1.00, 0.00) 0.00, 3.00 106 (1.82 0.00 (1.00, 1.00) 0.00, 3.00 106 (1.82 0.00 (1.00, 1.00) 0.00, 3.00 0.00, | 3.2% (-3.8%, 2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -0.9% (1.4%, 0.4%) -0.9% (1.4%, 0.4%) -1.5% (1.6, 0.5%) -1.5% (1.6, 0.5%) -1.5% ( | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 3361 (5.6%) 3361 (5.6%) 3361 (5.6%) 1.516 (23.1%) 1.634 (24.9%) 2.24 (1.51) 2.001 (1.00, 3.00) 0.00, 33.00 1.61 (1.29) 1.61 (1.29) 0.00 (1.00, 3.00) 0.00 (1.00, 3.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (2.00, 0.00) 0.00 (2.00, 0.00) 1.11 (1.75) 1.00 (1.00, 2.00) 1.00 (1.00, 3.00) | 504 (77%) 1771 (27%) 371 (57%) 371 (57%) 371 (57%) 371 (57%) 371 (47%) 371 (47%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (25.4%) 1,665 (26.4%) 1,665 (13.4%) 1,665 | 0.1% (-1.1%, 0.8%) 0.3% (-2.3%, 1.0%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 0.7%) 0.5% (-2.0%, 1.0%) 0.5% (-2.0%, 1.0%) 1.0, 0.00 (-0.06, 0.05) 1.0, |
| Pap smear n (%) Fecal occult Mond lest n (%) Fecal occult Mond lest n (%) Fecal occult Mond lest n (%) Monremorganics n (%) Mammogramics n (%) Mam | 840 (6.0%) 3456 (24.9%) 923 (6.0%) 923 (6.0%) 923 (6.0%) 924 (6.0%) 925 (14.5%) 926 (14.5%) 926 (14.5%) 929 (1.62) 920 (1 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 532 (27.0%) 6.395 (22.4%) 5.323 (27.0%) 6.395 (22.4%) 200 (100, 3.00) 0.00, 40.00 162 (12.77) 100 (100, 2.00) 0.00, 34.00 0.05 (0.39) 0.00 (0.00, 0.00) 0.00 (3.00, 0.00) 0.00 (20.0, 0.00) 0.00 (20.0, 0.00) 105 (18.2 0.00 (10.0, 0.00) 105 (18.2 0.00 (10.0, 0.00) 0.00 (20.0, 0.00) | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, 2.6%) -0.6% (1.6%, 2.6%) -1.2% (1.6%, 2.6%) -1.5% (1.6%, | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 369 (5.6%) 369 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.516 (23.1%) 1.516 (23.1%) 1.516 (23.1%) 1.524 (24.9%) 2.24 (1.51) 2.001 (0.0, 3.00) 0.00, 3.3.00 1.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (2.00) 1.11 (1.75) 1.00 (1.00, 3.00) 1.00 (2.00, 2.00) 1.00 (2.00, 2.00) 1.00 (2.00, 2.00) 1.00 (2.00, 0.00) 0.00 (2.00) 1.00 (2.00, 0.00) 0.00 (2.00) 1.73 (2.02) 1.00 (1.00, 3.00) 1.76 (2.5, 7.7) 0.00 (1.00, 0.00) 0.00 (2.700) 1.78 (1.1%) 1.79 (1.1%) 1.79 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (6.7%) 371 (6.7%) 371 (6.7%) 1.695 (22.4%) | 0.1% (-1.1% 0.8%) 0.8% (-2.3% 0.89) 0.1% (-0.9% 0.7%) 0.2% (-0.6% 1.0%) 0.3% (-1.1% 1.8%) 0.3% (-1.1% 1.8%) 0.00 (-0.05 0.05) (-1.1% 1.1%) (-1.1% 1.1%) 0.00 (-0.05 0.05) (-1.1% 0.5%) 0.05% (-1.2% 0.5%) 0.3% (-0.7% 0.5%) 0.3% (-0.0% 0.5%) |
| Pap smear n (%) Fecal occult blood lest n (%) Fecal occult blood lest n (%) Fecal occult blood lest n (%) Bone mineral density teets; n (%) Mammograms; n (%) Telemedicine n (%) HabAlC feetsmedian [IQR]min, max Upid panelsmedian [IQR]min, max Upid panelsmedian [IQR]min, max Construction lestsmedian [IQR]min, max Construction lestsmedian [IQR]min, max Viment lestsmedian [IQR]min, max Construction lestsmedian [IQR]min, max Viment lestsmedian [IQR]min, max Construction lestsmedian [IQR]min, max Viment lests lestsmedian [IQR]min, max Viment lests les | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 923 (6.6%) 621 (4.5%) 250 (1.6.6%) 250 (1.6.6%) 250 (1.6.6%) 250 (1.6.6%) 150 (1.38) 100 (1.00, 2.00) 0.00, 55.00 150 (1.38) 100 (1.00, 2.00) 0.00, 49.00 0.00 (1.00, 2.00) 0.00, 59.00 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 110 (1.97) 110 (1.98) 110 (1. | 1331(9.3%) 1331(9.3%) 13034(25.5%) 13074(5.6%) 13074(6.6%) 13074(6 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -1.9% (1.4%, -0.4%) -1.9% (1.4%, -0.4%) -1.9% (1.6%, -0.6%) -1.9% | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 366 (5.6%) 367 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.5179 (23.1%) 1.517 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (6.7%) 371 (6.7%) 371 (6.7%) 371 (6.7%) 1.494 (22.8%) 1.494 (22.8%) 1.494 (22.8%) 1.494 (22.8%) 1.665 (22.4%) 1.63 (13.4%) 1.60 (1.00, 2.00) 1.63 (13.4%) 1.60 (1.00, 2.00) 1.63 (13.4%) 1.60 (1.00, 2.00) 1.74 (2.02) 1.74 (2.02) 1.75 (2.8.5%) 1.75 (2.8.5%) 1.795 (28.5%) 1.799 (11.5%) | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 0.7%) 0.3% (-1.1%, 1.9%) 0.5% (-1.1%, 1.9%) 0.5% (-1.1%, 1.9%) 0.00 (-0.06, 0.05) -(-, -) -(-, - |
| Pap smear n (%) Fecal occult stood test n (%) Fecal occult stood test n (%) Fecal occult stood test n (%) Fecal occult stood test n (%) Mammograms; n (%) Ma | 840 (6.0%) 3456 (24.9%) 923 (6.5%) 621 (4.5%) 923 (6.5%) 621 (4.5%) 2.651 (19.1%) 2.300 (16.6%) 2.300 (16.6%) 2.300 (16.6%) 2.301 (16.6%) 2.30 | 1831(9.3%) 5034 (25.5%) 897 (4.6%) 1057 (5.4%) 5323 (27.0%) 6.395 (22.4%) 5323 (27.0%) 6.395 (22.4%) 200 (100, 3.00) 0.00, 40.00 160 (100, 2.00) 0.00, 40.00 160 (100, 2.00) 0.00, 3.00 0.00 (100, 0.00) 0.00, 3.00 0.00 (100, 0.00) 0.00, 23.00 0.01 (100, 0.00) 0.00, 23.00 0.01 (100, 0.00) 0.00, 23.00 0.01 (100, 0.00) 0.00, 23.00 0.01 (100, 0.00) 0.00, 3.00 0.00 (100, 0.00) 0.00, 3.00 0.00 (100, 0.00) 0.00, 3.00 0.00 (100, 0.00) 0.00, 3.00 0.00 (100, 3.00) 0.00 (10 | 3.2% (3.8%, 2.7%) 0.6% (1.6%, 2.6%) 0.6% (1.6%, 2.6%) 0.9% (1.4%, 0.4%) 7.9% (8.8%, 7.0%) 15.9% (16.5%, 1.50%) 0.12 (0.16, 0.0%) 16.9% (1.0%, 0.0%) 17.9% (1.0%, 0.0%) | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 3361 (5.6%) 3361 (5.6%) 3361 (5.6%) 1.516 (23.1%) 1.524 (1.4.3%) 1.524 (1.4.3%) 1.524 (1.4.3%) 1.524 (1.4.3%) 1.524 (1.5.3%) 1.525 (1.5.3%) 1.526 (1.5.3%) 1.527 (1.5 | 504 (7.7%) 1771 (270%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (6.7%) 371 (6.7%) 1.655 (25.4%) 1.655 (25.4%) 1.655 (25.4%) 1.601 (100, 3.00) 1.00, 40.00 1.00, 50.00 1.00, 50.50 1. | 0.1% (-1.1%, 0.8%) 0.3% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 0.7%) 0.3% (-1.1%, 1.8%) 0.5% (-2.0%, 1.0%) 0.5% (-2.0%, 1.0%) 1.6, -1 1 |
| Pap smear n (%) Fecal socult blood lest n (%) Fecal socult blood lest n (%) Bloom mineral density tests; n (%) Mammogams, n (%) Mammogams, n (%) Telemedicine n (%) Hald Clests _median [DR] _min max Upid panels _median [DR] _min max Upid panels _median [DR] _min max Creatinine tests _median [DR] _min max Utime tests _median [DR] _min max Utime tests _median [DR] _median [DR] _median [DR] _min max Creatinine d (min max) _median [DR] _min max Creatinine d (min max) _median [DR] _min max _median [DR] _min max _min max _median [DR] _min max _min | 840 (6.0%) 3456 (24.9%) 923 (6.6%) 621 (4.5%) 923 (6.6%) 621 (4.5%) 250 (1.6.6%) 250 (1.6.6%) 250 (1.6.6%) 250 (1.6.6%) 150 (1.38) 100 (1.00, 2.00) 0.00, 55.00 150 (1.38) 100 (1.00, 2.00) 0.00, 49.00 0.00 (1.00, 2.00) 0.00, 59.00 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 100 (1.00, 2.00) 110 (1.97) 110 (1.97) 110 (1.98) 110 (1. | 1331(9.3%) 1331(9.3%) 13034(25.5%) 13074(5.6%) 13074(6.6%) 13074(6 | 3.2% (-3.8%, -2.7%) -0.6% (1.6%, -2.6%) -0.6% (1.6%, -2.6%) -0.9% (1.4%, -0.4%) -1.9% (1.4%, -0.4%) -1.9% (1.4%, -0.4%) -1.9% (1.6%, -0.6%) -1.9% | 495 (7.6%) 1.721 (26.3%) 366 (5.6%) 366 (5.6%) 367 (5.6%) 369 (5.6%) 1.516 (23.1%) 1.5179 (23.1%) 1.517 | 504 (7.7%) 1771 (27.0%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (5.7%) 371 (6.7%) 371 (6.7%) 371 (6.7%) 371 (6.7%) 1.494 (22.8%) 1.494 (22.8%) 1.494 (22.8%) 1.494 (22.8%) 1.665 (22.4%) 1.63 (13.4%) 1.60 (1.00, 2.00) 1.63 (13.4%) 1.60 (1.00, 2.00) 1.63 (13.4%) 1.60 (1.00, 2.00) 1.74 (2.02) 1.74 (2.02) 1.75 (2.8.5%) 1.75 (2.8.5%) 1.795 (28.5%) 1.799 (11.5%) | 0.1% (-1.1%, 0.8%) 0.8% (-2.3%, 0.8%) 0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 0.7%) 0.3% (-1.1%, 1.9%) 0.5% (-1.1%, 1.9%) 0.5% (-1.1%, 1.9%) 0.00 (-0.06, 0.05) -(-, -) -(-, - |

| Appendix 7. Balance Assessment - Table 1 | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE<br>Variable | Potomog CitE " | Evangum Com-shill-1111 | Difference | Professore City attack | Exposure Commentation 1 11 | Difference - |
| Vanable Number of patients | Reference: Sitagliptin<br>38,610 | Exposure: Semaglutide injection 7,980 | - (-, -) | Reference: Sitagliptin<br>6,877 | Exposure: Semaglutide injection<br>6,877 | - (-, -) |
| Year of Cohort Entry Date2018; n (%) | 13,930 (36.1%) | 571 (7.2%) | 28.9% (28.2%, 29.7%) | 562 (8.2%) | 566 (8.2%) | -0.1% (-1.0%, 0.9%) |
| 2019; n (%)<br>2020; n (%) | 13,697 (35.5%)<br>10,983 (28.4%) | 3,028 (37.9%)<br>4,381 (54.9%) | -2.5% (-3.6%, -1.3%)<br>-26.5% (-27.6%, -25.3%) | 2,764 (40.2%)<br>3,551 (51.6%) | 2,727 (39.7%)<br>3,584 (52.1%) | 0.5% (-11%, 2.2%) |
| Age<br>mean (sd) | 75.45 (6.86) | 72.12 (4.96) | 3.33 (3.20, 3.46) | 72.48 (5.37) | 72.41 (5.05) | 0.07 (-0.11, 0.24) |
| median [IQR]min, max | 74.00 [70.00, 80.00]<br>65.00, 106.00 | 71.00 [68.00, 75.00]<br>65.00, 96.00 | - (-, -)<br>- (-, -) | 71.00 [68.00, 76.00]<br>65.00, 99.00 | 72.00 [68.00, 75.00]<br>65.00, 96.00 | - (-, -)<br>- (- a) |
| Gender (male); n (%) | 16,946 (43.9%) | 3,846 (48.2%) | -4.3% (-5.5%, -3.1%) | 3,252 (47.3%) | 3,281 (47.7%) | -0.4% (-21%, 1.3%) |
| Race (Recategorized)White; n (%) | 29,995 (77.7%) | 6,706 (84.0%) | -6.3% (-7.3%, -5.4%) | 5,762 (83.8%) | 5,737 (83.4%) | 0.4% (-0.9%, 1.6%) |
| Other; n (%)<br>Black; n (%) | 2,757 (7.1%)<br>4,419 (11.4%) | 327 (4.1%)<br>664 (8.3%) | 3.0% (2.5%, 3.6%)<br>3.1% (2.4%, 3.8%) | 304 (4.4%)<br>581 (8.4%) | 302 (4.4%)<br>598 (8.7%) | 0.0% (-0.7%, 0.7%)<br>-0.2% (-1.2%, 0.7%) |
| Unknown / Missing; n (%)<br>Region / State | 1,439 (3.7%) | 283 (3.5%) | 0.2% (-0.3%, 0.6%) | 230 (3.3%) | 240 (3.5%) | -0.1% (-0.8%, 0.5%) |
| Northest; n (%) Midwest / North central: n (%) | 7,473 (19.4%)<br>8,005 (20.7%) | 1,264 (15.8%)<br>1,845 (23.1%) | 3.5% (2.6%, 4.4%) | 1,092 (15.9%) | 1,092 (15.9%) | 0.0% (-1.2%, 1.2%) |
| South; n (%)<br>West; n (%) | 17,616 (45.6%)<br>5,443 (14.1%) | 3,851 (48.3%)<br>1,016 (12.7%) | -2.6% (-3.8%, -1.4%)<br>1.4% (0.5%, 2.2%) | 3,342 (48.6%)<br>869 (12.6%) | 3,327 (48.4%)<br>894 (13.0%) | 0.2% (-1.5%, 1.9%)<br>-0.4% (-1.5%, 0.8%) |
| Missing n (%) | 73 (0.2%) | 4 (0.1%) | 0.1% (0.1%, 0.2%) | 4 (0.1%) | 4 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Smoking / Tobacco use; n (%) Weight | 10,680 (27.7%) | 2,235 (28.0%) | -0.3% (-1.4%, 0.7%) | 1,929 (28.1%) | 1,934 (28.1%) | -0.1% (-1.6%, 1.4%) |
| Underweight; n (%)<br>Normal weight; n (%) | 810 (2.1%)<br>3,876 (10.0%) | 32 (0.4%)<br>235 (2.9%) | 1.7% (1.5%, 1.9%)<br>7.1% (6.6%, 7.6%) | 25 (0.4%)<br>219 (3.2%) | 32 (0.5%)<br>232 (3.4%) | -0.1% (-0.3%, 0.1%)<br>-0.2% (-0.8%, 0.4%) |
| Overweight; n (%)<br>Class 1 Obesity: n (%) | 12,521 (32.4%)<br>3.034 (7.9%) | 1,769 (22.2%)<br>599 (7.5%) | 10.3% (9.2%, 11.3%)<br>0.4% (-0.3%, 1.0%) | 1,675 (24.4%)<br>595 (8.7%) | 1,657 (24.1%)<br>542 (7.9%) | 0.3% (-1.2%, 1.7%) |
| Class 2 Obesity; n (%)<br>Class 3 Obesity; n (%) | 1,429 (3.7%)<br>5,921 (15.3%) | 403 (5.1%)<br>2,126 (26.6%) | -1.3% (-1.9%, -0.8%)<br>-11.3% (-12.3%, -10.3%) | 333 (4.8%)<br>1,711 (24.9%) | 339 (4.9%)<br>1,698 (24.7%) | -0.1% (-0.8%, 0.6%)<br>0.2% (-1.3%, 1.6%) |
| | 11,019 (28.5%)<br>3,745 (9.7%) | 2,816 (35.3%)<br>996 (12.5%) | -6.7% (-7.9%, -5.6%)<br>-2.8% (-3.6%, -2.0%) | 2,319 (33.7%)<br>816 (11.9%) | 2,377 (34.6%)<br>793 (11.5%) | -0.8% (-2.4%, 0.8%)<br>0.3% (-0.8%, 1.4%) |
| Diabetic neuropathy; n (%) | 10,973 (28.4%) | 2,696 (33.8%) | -5.4% (-6.5%, -4.2%) | 2,259 (32.8%) | 2,230 (32.4%) | 0.4% (-1.2%, 2.0%) |
| Diabetic nephropathy; n (%) Diabetes with other opthalmic complications; n (%) | 11,209 (29.0%)<br>1,013 (2.6%) | 2,403 (30.1%)<br>206 (2.6%) | -1.1% (-2.2%, 0.0%)<br>0.0% (-0.3%, 0.4%) | 2,043 (29.7%)<br>185 (2.7%) | 2,000 (29.1%)<br>173 (2.5%) | 0.6% (-0.9%, 2.2%) |
| Diabetes with peripheral circulatory disorders; n (%) Diabetic foot; n (%) | 4,680 (12.1%)<br>1,372 (3.6%) | 1,074 (13.5%)<br>259 (3.2%) | -1.3% (-2.2%, -0.5%)<br>0.3% (-0.1%, 0.7%) | 914 (13.3%)<br>235 (3.4%) | 879 (12.8%)<br>208 (3.0%) | 0.5% (-0.6%, 1.6%) |
| Erectile dysfunction; n (%)<br>Hypoglycemia; n (%) | 566 (1.5%)<br>4.937 (12.8%) | 185 (2.3%)<br>1,091 (13.7%) | -0.9% (-1.2%, -0.5%)<br>-0.9% (-1.7%, -0.1%) | 158 (2.3%)<br>897 (13.0%) | 147 (2.1%)<br>894 (13.0%) | 0.2% (-0.3%, 0.7%) |
| Hyperglycemia / DKA / HONK; n (%) Skin infections: n (%) | 17,806 (46.1%)<br>4,516 (11.7%) | 4.461 (55.9%)<br>950 (11.9%) | -9.8% (-11.0%, -8.6%)<br>-0.2% (-1.0%, 0.6%) | 3,662 (53.2%)<br>803 (11.7%) | 3,656 (53.2%)<br>791 (11.5%) | 0.1% (-1.6%, 1.8%) |
| Stable angina; n (%) | 2,328 (6.0%) | 632 (7.9%) | -1.9% (-2.5%, -1.2%) | 504 (7.3%) | 511 (7.4%) | -0.1% (-1.0%, 0.8%) |
| Unstable angina; n (%)<br>Hypertension; n (%) | 1,629 (4.2%)<br>34,600 (89.6%) | 414 (5.2%)<br>7,109 (89.1%) | -1.0% (-1.5%, -0.4%)<br>0.5% (-0.2%, 1.3%) | 345 (5.0%)<br>6,134 (89.2%) | 337 (4.9%)<br>6,117 (88.9%) | 0.1% (-0.6%, 0.9%) |
| Hypotension; n (%) Hyperlipidemia; n (%) | 2,368 (6.1%)<br>29,388 (76.1%) | 372 (4.7%)<br>6,207 (77.8%) | 1.5% (0.9%, 2.0%)<br>-1.7% (-2.7%, -0.7%) | 329 (4.8%)<br>5,308 (77.2%) | 331 (4.8%)<br>5,303 (77.1%) | -0.0% (-0.8%, 0.7%)<br>0.1% (-1.3%, 1.5%) |
| Atrial fibrillation; n (%) Cardiac conduction disorder; n (%) | 8,887 (23.0%)<br>3.952 (10.2%) | 1,662 (20.8%)<br>711 (8.9%) | 2.2% (1.2%, 3.2%)<br>1.3% (0.6%, 2.0%) | 1,454 (21.1%)<br>582 (8.5%) | 1,437 (20.9%)<br>624 (9.1%) | 0.2% (-11%, 1.6%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 1,209 (3.1%)<br>860 (2.2%) | 368 (4.6%)<br>127 (1.6%) | -1.5% (-2.0%, -1.0%)<br>0.6% (0.3% 1.0%) | 278 (4.0%)<br>116 (1.7%) | 287 (4.2%)<br>110 (1.6%) | -0.1% (-0.8%, 0.5%)<br>0.1% (-0.4%, 0.5%) |
| PVD diagnosis or surgery; n (%) | 4,988 (12.9%) | 906 (11.4%) | 1.6% (0.8%, 2.3%) | 810 (11.8%) | 775 (11.3%) | 0.5% (-0.6%, 1.6%) |
| Other cardiac dysrhythmia; n (%) Cardiomyopathy; n (%) | 11,191 (29.0%)<br>3,287 (8.5%) | 2,053 (25.7%)<br>676 (8.5%) | 3.3% (2.2%, 4.3%)<br>0.0% (-0.6%, 0.7%) | 1,767 (25.7%)<br>560 (8.1%) | 1,784 (25.9%)<br>562 (8.2%) | -0.2% (-1.7%, 1.2%)<br>-0.0% (-1.0%, 0.9%) |
| Valve disorders; n (%) Valve replacement; n (%) | 7,167 (18.6%)<br>1,157 (3.0%) | 1,290 (16.2%)<br>235 (2.9%) | 2.4% (1.5%, 3.3%)<br>0.1% (-0.4%, 0.5%) | 1,099 (16.0%)<br>194 (2.8%) | 1,120 (16.3%)<br>205 (3.0%) | -0.3% (-1.5%, 0.9%)<br>-0.2% (-0.7%, 0.4%) |
| TIA; n (%)<br>Edema: n (%) | 1,496 (3.9%)<br>6.118 (15.8%) | 204 (2.6%)<br>1.269 (15.9%) | 1.3% (0.9%, 1.7%) | 181 (2.6%)<br>1.099 (16.0%) | 185 (2.7%)<br>1.066 (15.5%) | -0.1% (-0.6%, 0.5%)<br>0.5% (-0.8%, 1.7%) |
| Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) | 1,758 (4.6%)<br>1,953 (5.1%) | 326 (4.1%)<br>349 (4.4%) | 0.5% (-0.0%, 1.0%) | 285 (4.1%)<br>285 (4.1%) | 273 (4.0%)<br>292 (4.2%) | 0.2% (-0.5%, 0.8%) |
| Implantable cardioverter defibrillator; n (%) | 283 (0.7%) | 55 (0.7%)<br>131 (1.6%) | 0.0% (-0.2%, 0.3%) | 42 (0.6%) | 44 (0.6%) | -0.0% (-0.3%, 0.2%) |
| Hyperkalemia; n (%) Coronary atherosclerosis; n (%) | 887 (2.3%)<br>16,767 (43.4%) | 3,616 (45.3%) | 0.7% (0.3%, 1.0%)<br>-1.9% (-3.1%, -0.7%) | 115 (1.7%)<br>3,057 (44.5%) | 110 (1.6%)<br>3,067 (44.6%) | 0.1% (-0.4%, 0.5%)<br>-0.1% (-1.8%, 1.5%) |
| Cerebrovascular procedure; n (%)<br>Insertion of pacemakers / removal of cardiac lead; n (%) | 126 (0.3%)<br>238 (0.6%) | 27 (0.3%)<br>39 (0.5%) | -0.0% (-0.2%, 0.1%)<br>0.1% (-0.1%, 0.3%) | 25 (0.4%)<br>35 (0.5%) | 24 (0.3%)<br>31 (0.5%) | 0.0% (-0.2%, 0.2%) |
| CKD stage 1-2; n (%) CKD stage 3-4; n (%) | 1,530 (4.0%)<br>9,602 (24.9%) | 317 (4.0%)<br>2,096 (26.3%) | -0.0% (-0.5%, 0.5%)<br>-1.4% (-2.5%, -0.3%) | 277 (4.0%)<br>1,754 (25.5%) | 268 (3.9%)<br>1,758 (25.6%) | 0.1% (-0.5%, 0.8%)<br>-0.1% (-1.5%, 1.4%) |
| Unspecified CKD; n (%) Acute kidney injury: n (%) | 4,258 (11.0%)<br>5,487 (14.2%) | 809 (10.1%)<br>845 (10.6%) | 0.9% (0.2%, 1.6%)<br>3.6% (2.9%, 4.4%) | 694 (10.1%)<br>747 (10.9%) | 681 (9.9%)<br>733 (10.7%) | 0.2% (-0.8%, 1.2%) |
| Hypertensive nephropathy; n (%) Urinary tract infections: n (%) | 8,274 (21.4%)<br>9,285 (24.0%) | 1,649 (20.7%)<br>1.493 (18.7%) | 0.8% (-0.2%, 1.8%)<br>5.3% (4.4%, 6.3%) | 1,392 (20.2%) | 1,392 (20.2%)<br>1.316 (19.1%) | 0.0% (-1.3%, 1.3%) |
| Genital infections; n (%) | 1,085 (2.8%) | 221 (2.8%)<br>429 (5.4%) | 0.0% (-0.4%, 0.4%) | 210 (3.1%)<br>347 (5.0%) | 192 (2.8%) | 0.3% (-0.3%, 0.8%) |
| Urolithiasis (Kidney and urinary stone); n (%) COPD; n (%) | 1,997 (5.2%)<br>7,568 (19.6%) | 1,489 (18.7%) | -0.2% (-0.8%, 0.3%)<br>0.9% (-0.0%, 1.9%) | 1,288 (18.7%) | 370 (5.4%)<br>1,286 (18.7%) | 0.0% (-1.3%, 1.3%) |
| Asthma; n (%) Obstructive sleep apnea; n (%) | 3,741 (9.7%)<br>7,779 (20.1%) | 880 (11.0%)<br>2,602 (32.6%) | -1.3% (-2.1%, -0.6%)<br>-12.5% (-13.6%, -11.3%) | 763 (11.1%)<br>2,050 (29.8%) | 737 (10.7%)<br>2,089 (30.4%) | 0.4% (-0.7%, 1.4%)<br>-0.6% (-2.1%, 1.0%) |
| Serious bacterial infections; n (%) Pneumonia; n (%) | 3,058 (7.9%)<br>3,643 (9.4%) | 401 (5.0%)<br>570 (7.1%) | 2.9% (2.3%, 3.5%)<br>2.3% (1.6%, 2.9%) | 379 (5.5%)<br>510 (7.4%) | 358 (5.2%)<br>500 (7.3%) | 0.3% (-0.5%, 1.1%) 0.1% (-0.7%, 1.0%) |
| Liver disease; n (%) MASH/MASI D n (%) | 3,915 (10.1%)<br>1,656 (4.3%) | 905 (11.3%)<br>473 (5.9%) | -1.2% (-2.0%, -0.4%)<br>-1.6% (-2.2%, -1.1%) | 739 (10.7%)<br>363 (5.3%) | 753 (10.9%)<br>382 (5.6%) | -0.2% (-1.3%, 0.9%)<br>-0.3% (-1.0%, 0.5%) |
| Fractures / Falls; n (%) | 2,008 (5.2%) | 317 (4.0%)<br>499 (6.3%) | 1.2% (0.7%, 1.7%) | 280 (4.1%)<br>442 (6.4%) | 273 (4.0%)<br>445 (6.5%) | 0.1% (-0.6%, 0.8%) |
| Osteoarthritis; n (%) | 13,310 (34.5%) | 2,848 (35.7%) | -1.2% (-2.4%, -0.1%) | 2,445 (35.6%) | 2,470 (35.9%) | -0.4% (-2.0%, 1.3%) |
| Depression; n (%) Dementia; n (%) | 7,295 (18.9%)<br>4,587 (11.9%) | 1,608 (20.2%)<br>440 (5.5%) | -1.3% (-2.2%, -0.3%)<br>6.4% (5.8%, 7.0%) | 1,385 (20.1%)<br>418 (6.1%) | 1,362 (19.8%)<br>400 (5.8%) | 0.3% (-1.0%, 1.7%) 0.3% (-0.5%, 1.1%) |
| Delinium or psychosis; n (%) Anxiety; n (%) | 1,145 (3.0%)<br>5,786 (15.0%) | 108 (1.4%)<br>1,192 (14.9%) | 1.6% (1.3%, 1.9%)<br>0.0% (-0.8%, 0.9%) | 118 (1.7%)<br>1,034 (15.0%) | 95 (1.4%)<br>1,041 (15.1%) | 0.3% (-0.1%, 0.8%)<br>-0.1% (-1.3%, 1.1%) |
| Sleep disorders; n (%)<br>Anemia; n (%) | 13,350 (34.6%)<br>11.829 (30.6%) | 2,785 (34.9%) 2,022 (25.3%) | -0.3% (-1.5%, 0.8%)<br>5.3% (4.2%, 6.4%) | 2,400 (34.9%)<br>1,786 (26.0%) | 2,387 (34.7%)<br>1.769 (25.7%) | 0.2% (-1.4%, 1.8%) |
| Influenza; n (%)<br>COVID: n (%) | 1,098 (2.8%)<br>220 (0.6%) | 173 (2.2%)<br>57 (0.7%) | 0.7% (0.3%, 1.0%) | 164 (2.4%)<br>57 (0.8%) | 156 (2.3%)<br>51 (0.7%) | 0.1% (-0.4%, 0.6%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 10,684 (27.7%)<br>8.886 (23.0%) | 2,333 (29.2%) | -1.6% (-2.7%, -0.5%) | 1,993 (29.0%)<br>1,674 (24.3%) | 1,964 (28.6%) | 0.4% (-1.1%, 1.9%) |
| Hypothyroidism; n (%) Nephrotic syndrome; n (%) | 3 (0.0%) | 1,923 (24.1%)<br>0 (0.0%) | -1.1% (-2.1%, -0.0%)<br>0.0% (-0.0%, 0.0%) | 0 (0.0%) | 1,621 (23.6%)<br>0 (0.0%) | 0.8% (-0.7%, 2.2%) |
| Urinary incontinence; n (%) Biliary disease; n (%) | 2,592 (6.7%)<br>164 (0.4%) | 477 (6.0%)<br>15 (0.2%) | 0.7% (0.2%, 1.3%)<br>0.2% (0.1%, 0.4%) | 441 (6.4%)<br>14 (0.2%) | 410 (6.0%)<br>12 (0.2%) | 0.5% (-0.4%, 1.3%) |
| Pancreatitis; n (%) Bowel obstruction; n (%) | 31 (0.1%)<br>106 (0.3%) | 5 (0.1%)<br>18 (0.2%) | 0.0% (-0.1%, 0.1%)<br>0.0% (-0.1%, 0.2%) | 7 (0.1%)<br>12 (0.2%) | 5 (0.1%)<br>11 (0.2%) | 0.0% (-0.1%, 0.1%) |
| Gastroparesis; n (%) Number of antidiabetic druzs on CED | 281 (0.7%) | 55 (0.7%) | 0.0% (-0.2%, 0.2%) | 47 (0.7%) | 49 (0.7%) | -0.0% (-0.3%, 0.3%) |
| mean (sd)mean (IOR) | 2.11 (0.80)<br>2.00 (2.00, 3.00) | 2.23 (0.86)<br>2.00 (2.00, 3.00) | -0.12 (-0.14, -0.10)<br>- (-, -) | 2.21 (0.84) | 2.20 (0.86)<br>2.00 (2.00, 3.00) | 0.01 (-0.02, 0.04) |
| min, max | 1.00, 5.00 | 1.00, 4.00 | - (-, -) | 1.00, 4.00 | 1.00, 4.00 | - (-, -) |
| Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) | 21,268 (55.1%)<br>4,941 (12.8%) | 3,806 (47.7%)<br>2,728 (34.2%) | 7.4% (6.2%, 8.6%)<br>-21.4% (-22.5%, -20.3%) | 3,428 (49.8%)<br>1,962 (28.5%) | 3,432 (49.9%)<br>1,926 (28.0%) | -0.1% (-1.7%, 1.6%)<br>0.5% (-1.0%, 2.0%) |
| Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2i; n (%) | 12,535 (32.5%)<br>1,892 (4.9%) | 1,882 (23.6%)<br>915 (11.5%) | 8.9% (7.8%, 9.9%)<br>-6.6% (-7.3%, -5.8%) | 1,771 (25.8%)<br>716 (10.4%) | 1,768 (25.7%)<br>696 (10.1%) | 0.0% (-1.4%, 1.5%) |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin: n (%) | 2,197 (5.7%)<br>24,716 (64,0%) | 478 (6.0%)<br>5.054 (63.3%) | -0.3% (-0.9%, 0.3%)<br>0.7% (-0.5%, 1.8%) | 428 (6.2%)<br>4.449 (64.7%) | 415 (6.0%)<br>4.431 (64.4%) | 0.2% (-0.6%, 1.0%) |
| Past use of Insulins; n (%) | 7,259 (18.8%)<br>15,926 (41.2%) | 3,636 (45.6%)<br>2,654 (33.3%) | -26.8% (-27.9%, -25.6%)<br>8.0% (6.8%, 9.1%) | 2,683 (39.0%)<br>2.447 (35.6%) | 2,639 (38.4%)<br>2,433 (35.4%) | 0.6% (-1.0%, 2.3%) |
| Past use of Sulfonylureas; n (%) Past use of SGLT-2l; n (%) | 2,973 (7.7%) | 1,401 (17.6%) | -9.9% (-10.7%, -9.0%) | 1,064 (15.5%) | 1,059 (15.4%) | 0.1% (-1.1%, 1.3%) |
| Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) | 3,320 (8.6%)<br>28,677 (74.3%) | 770 (9.6%)<br>6,133 (76.9%) | -11% (-1.8%, -0.3%)<br>-2.6% (-3.6%, -1.6%) | 694 (10.1%)<br>5,308 (77.2%) | 660 (9.6%)<br>5,273 (76.7%) | 0.5% (-0.5%, 1.5%) |
| ARNI; n (%)<br>Thiazides; n (%) | 508 (1.3%)<br>12,173 (31.5%) | 151 (1.9%)<br>2,732 (34.2%) | -0.6% (-0.9%, -0.2%)<br>-2.7% (-3.9%, -1.6%) | 112 (1.6%)<br>2,298 (33.4%) | 123 (1.8%)<br>2,334 (33.9%) | -0.2% (-0.6%, 0.3%)<br>-0.5% (-2.1%, 1.1%) |
| Beta-blockers; n (%) Calcium channel blockers; n (%) | 24,199 (62.7%)<br>15,650 (40.5%) | 5,126 (64.2%)<br>3,011 (37.7%) | -1.6% (-2.7%, -0.4%)<br>2.8% (1.6%, 4.0%) | 4,359 (63.4%)<br>2,622 (38.1%) | 4,357 (63.4%)<br>2,625 (38.2%) | 0.0% (-1.6%, 1.7%) |
| Digoxin / Digitoxin; n (%) Loop diuretics; n (%) | 1,378 (3.6%)<br>12,958 (33.6%) | 214 (2.7%)<br>2.913 (36.5%) | 0.9% (0.5%, 1.3%) | 176 (2.6%)<br>2.406 (35.0%) | 181 (2.6%)<br>2.438 (35.5%) | -0.1% (-0.6%, 0.5%)<br>-0.5% (-2.1%, 1.1%) |
| Other diuretics; n (%) | 4,021 (10.4%) | 1,061 (13.3%) | -2.9% (-3.7%, -2.1%) | 836 (12.2%) | 842 (12.2%) | -0.1% (-1.2%, 1.0%) |
| Intravenous diuretics; n (%) Nitrates; n (%) | 1,157 (3.0%)<br>5,598 (14.5%) | 224 (2.8%)<br>1,280 (16.0%) | 0.2% (-0.2%, 0.6%)<br>-1.5% (-2.4%, -0.7%) | 181 (2.6%)<br>1,075 (15.6%) | 187 (2.7%)<br>1,059 (15.4%) | -0.1% (-0.6%, 0.5%)<br>0.2% (-1.0%, 1.5%) |
| Anti-arrhythmics; n (%) Statins; n (%) | 1,995 (5.2%)<br>30,909 (80.1%) | 384 (4.8%)<br>6,649 (83.3%) | 0.4% (-0.2%, 0.9%)<br>-3.3% (-4.2%, -2.3%) | 324 (4.7%)<br>5,668 (82.4%) | 327 (4.8%)<br>5,693 (82.8%) | -0.0% (-0.8%, 0.7%)<br>-0.4% (-1.6%, 0.9%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 5,321 (13.8%) | 1,326 (16.6%) | -2.8% (-3.7%, -1.9%) | 1,089 (15.8%) | 1,087 (15.8%) | 0.0% (-1.2%, 1.3%) |

| A F. L. L. L. F. E. (97) | 7 400 40 000 | 4 004 (00 40) | 0.70/ / 4.70/ 0.00/) | 4.000 (00.40) | 1.0.10.110.000 | 0.50/ / 0.00/ 4.00/ |
|---|---|---|---|---|---|---|
| Antiplatelet medications; n (%) Oral anticoagulants; n (%) | 7,466 (19.3%)<br>8,073 (20.9%) | 1,601 (20.1%)<br>1,608 (20.2%) | -0.7% (-1.7%, 0.2%)<br>0.8% (-0.2%, 1.7%) | 1,380 (20.1%)<br>1,418 (20.6%) | 1,349 (19.6%)<br>1,388 (20.2%) | 0.5% (-0.9%, 1.8%)<br>0.4% (-0.9%, 1.8%) |
| COPD/Asthma medications; n (%) NSAIDS: n (%) | 13,671 (35.4%)<br>10 567 (27.4%) | 3,068 (38.4%)<br>2,282 (28.6%) | -3.0% (-4.2%, -1.9%)<br>-1.2% (-2.3% -0.1%) | 2,631 (38.3%)<br>1 998 (29.1%) | 2,595 (37.7%)<br>1,960 (28.5%) | 0.5% (-11%, 2.2%) |
| Oral corticosteroids; n (%) | 8,875 (23.0%) | 1,939 (24.3%) | -1.3% (-2.3%, -0.3%) | 1,719 (25.0%) | 1,664 (24.2%) | 0.8% (-0.7%, 2.3%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) Opioids; n (%) | 1,831 (4.7%)<br>13,628 (35.3%) | 302 (3.8%)<br>3,124 (39.1%) | 1.0% (0.5%, 1.4%)<br>-3.9% (-5.0%, -2.7%) | 267 (3.9%)<br>2,656 (38.6%) | 268 (3.9%)<br>2,651 (38.5%) | -0.0% (-0.7%, 0.6%)<br>0.1% (-1.6%, 1.7%) |
| Anti-depressants; n (%) | 14,016 (36.3%) | 3,395 (42.5%) | -6.2% (-7.4%, -5.0%) | 2,889 (42.0%) | 2,836 (41.2%) | 0.8% (-0.9%, 2.4%) |
| Antipsychotics; n (%) | 1,887 (4.9%)<br>8,242 (21.3%) | 306 (3.8%)<br>1,747 (21.9%) | 1.1% (0.6%, 1.5%)<br>-0.5% (-1.5%, 0.5%) | 272 (4.0%)<br>1,558 (22.7%) | 266 (3.9%)<br>1,499 (21.8%) | 0.1% (-0.6%, 0.7%)<br>0.9% (-0.5%, 2.3%) |
| Anxiolytics/hypnotics, benzos; n (%) Dementia medications; n (%) | 2,660 (6.9%) | 288 (3.6%) | 3.3% (2.8%, 3.8%) | 272 (4.0%) | 257 (3.7%) | 0.2% (-0.4%, 0.9%) |
| Urinary tract infections antibiotics; n (%) | 20,605 (53.4%)<br>2,065 (5.3%) | 4,429 (55.5%)<br>297 (3.7%) | -21% (-3.3%, -0.9%)<br>1.6% (1.1%, 2.1%) | 3,802 (55.3%)<br>279 (4.1%) | 3,783 (55.0%)<br>250 (3.6%) | 0.3% (-1.4%, 2.0%) 0.4% (-0.2%, 1.1%) |
| Laxatives; n (%) Number of distinct medications | 2,065 (5.3%) | 297 (3.7%) | 16% (1.1%, 2.1%) | 2/9 (4.1%) | 250 (3.6%) | 0.4% (-0.2%, 1.1%) |
| mean (sd) | 14.57 (6.59) | 15.97 (6.61) | -1.40 (-1.56, -1.24) | 15.81 (6.77) | 15.59 (6.50) | 0.22 (-0.00, 0.44) |
| median [IQR]min, max | 14.00 [10.00, 18.00]<br>1.00, 57.00 | 15.00 [11.00, 20.00]<br>1.00, 55.00 | - (-, -)<br>- (-, -) | 15.00 [11.00, 20.00]<br>1.00, 53.00 | 15.00 [11.00, 19.00]<br>1.00, 55.00 | - (-, -)<br>- (-, -) |
| Number of office visits | | | | | | |
| mean (sd)median [IQR] | 11.74 (7.88)<br>10.00 [6.00, 16.00] | 13.40 (8.24)<br>12.00 [8.00.18.00] | -1.66 (-1.86, -1.46)<br>- (-, -) | 13.06 (8.54)<br>11.00 (7.00, 17.00) | 13.02 (7.86)<br>12.00 (7.00.17.00) | 0.04 (-0.23, 0.32) |
| min, max | 0.00,132.00 | 0.00,145.00 | -(-, -) | 0.00, 109.00 | 0.00, 61.00 | - (-, -) |
| Number of endocrinologist visitsmean (sd) | 0.38 (1.25) | 0.89 (1.97) | -0.51 (-0.55, -0.46) | 0.68 (1.80) | 0.70 (1.63) | -0.02 (-0.08, 0.04) |
| | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max Number of cardiologist visits | 0.00, 50.00 | 0.00, 45.00 | - (-, -) | 0.00, 28.00 | 0.00, 28.00 | - (-, -) |
| mean (sd) | 2.53 (3.92) | 2.36 (3.75) | 0.16 (0.07, 0.25) | 2.31 (3.62) | 2.35 (3.79) | -0.04 (-0.17, 0.08) |
| median [IQR]min, max | 1.00 [0.00, 3.00]<br>0.00, 102.00 | 1.00 [0.00, 3.00]<br>0.00, 62.00 | - (-, -)<br>- (-, -) | 1.00 [0.00, 3.00]<br>0.00, 51.00 | 1.00 [0.00, 3.00]<br>0.00, 62.00 | - (-, -)<br>- (-, -) |
| Number of internal/family medicine visits | 0.00, 102.00 | 0.00, 02.00 | | 0.00, 51.00 | 0.00, 02.00 | -(5-) |
| mean (sd) | 7.35 (7.53) | 6.41 (6.39) | 0.94 (0.79, 1.10) | 6.50 (6.72) | 6.48 (6.43) | 0.02 (-0.20, 0.24) |
| median [IQR]min, max | 5.00 [3.00, 10.00]<br>0.00, 142.00 | 5.00 [2.00, 9.00]<br>0.00, 84.00 | - (-, -)<br>- (-, -) | 5.00 [2.00, 9.00]<br>0.00, 88.00 | 5.00 [2.00, 9.00]<br>0.00, 84.00 | - (-, -)<br>- (-, -) |
| Number of Electrocardiograms (ECG/EKG) | 181(2.37) | 1.62(216) | 0.19 (0.13, 0.24) | 1.60 (210) | 1.62 (2.16) | -0.02 (-0.09, 0.05) |
| mean (sd)median (IQR) | 1.81 (2.37)<br>1.00 [0.00, 2.00] | 1.62 (216)<br>1.00 [0.00, 2.00] | 0.19 (0.13, 0.24) | 1.60 (2.10)<br>1.00 [0.00, 2.00] | 1.62 (2.16)<br>1.00 [0.00, 2.00] | -0.02 (-0.09, 0.05)<br>- (-, -) |
| min, max | 0.00, 87.00 | 0.00, 37.00 | -(-,-) | 0.00, 28.00 | 0.00, 37.00 | -(-,-) |
| Number of Echocardiogramsmean (sd) | 0.57 (0.89) | 0.52 (0.84) | 0.05 (0.03, 0.07) | 0.51 (0.83) | 0.51 (0.84) | -0.00 (-0.03, 0.03) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max Out-of-pocket medication cost | 0.00, 19.00 | 0.00, 11.00 | - (-, -) | 0.00, 8.00 | 0.00, 11.00 | - (-, -) |
| mean (sd) | 659.81 (798.91) | 1,034.73 (1,112.54) | -374.92 (-400.60, -349.24) | 938.92 (1,041.14) | 930.77 (941.27) | 8.14 (-25.03, 41.32) |
| median [IQR]min, max | 424.63 [103.10, 920.09]<br>0.00, 24,114.58 | 747.50 [228.42, 1,505.11]<br>0.00, 42,223.98 | - (-, -)<br>- (-, -) | 689.81 [197.80, 1,337.36]<br>0.00, 20,956.74 | 684.78 [204.44, 1,328.67]<br>0.00, 23,893.53 | - (-, -)<br>- (-, -) |
| Unique brand medicines | 0.00, 24,114.58 | 0.00, 42,223.98 | - (-, -) | 0.00, 20,956.74 | 0.00, 23,893.53 | - (-, -) |
| mean (sd) | 14.86 (6.81) | 16.33 (6.85)<br>15.00 (12.00.20.00) | -1.47 (-1.63, -1.30) | 16.16 (7.03)<br>15.00 (11.00.20.00) | 15.93 (6.74) | 0.23 (0.00, 0.46) |
| median [IQR]min, max | 1.00, 66.00 | 1.00, 57.00 | - (-, -)<br>- (-, -) | 1.00, 54.00 | 1.00, 57.00 | - (-, -)<br>- (-, -) |
| Unique generic medicines | | | | | | |
| mean (sd)median [IQR] | 14.57 (6.59)<br>14.00 [10.00, 18.00] | 15.97 (6.61)<br>15.00 [11.00, 20.00] | -140 (-1.56, -1.24)<br>- (-, -) | 15.81 (6.77)<br>15.00 [11.00, 20.00] | 15.59 (6.50)<br>15.00 (11.00, 19.00) | 0.22 (-0.00, 0.44) |
| min, max | 1.00, 57.00 | 1.00, 55.00 | - (-, -) | 1.00, 53.00 | 1.00, 55.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%)<br>Flu Pneumococcal vaccine: n (%) | 3,665 (9.5%)<br>4,138 (10.7%) | 869 (10.9%)<br>794 (9.9%) | -1.4% (-2.1%, -0.6%)<br>0.8% (0.0%, 1.5%) | 721 (10.5%)<br>686 (10.0%) | 729 (10.6%)<br>678 (9.9%) | -0.1% (-1.2%, 0.9%)<br>0.1% (-0.9%, 1.1%) |
| Pap smear, n (%) | 1,289 (3.3%) | 349 (4.4%) | -1.0% (-1.5%, -0.5%) | 290 (4.2%) | 304 (4.4%) | -0.2% (-0.9%, 0.5%) |
| PSA test; n (%) Fecal occult blood test; n (%) | 7,758 (20.1%)<br>2,836 (7.3%) | 1,899 (23.8%)<br>475 (6.0%) | -3.7% (-4.7%, -2.7%)<br>1.4% (0.8%, 2.0%) | 1,604 (23.3%)<br>409 (5.9%) | 1,615 (23.5%)<br>436 (6.3%) | -0.2% (-1.6%, 1.3%)<br>-0.4% (-1.2%, 0.4%) |
| Bone mineral density tests; n (%) | 3,152 (8.2%) | 731 (9.2%) | -1.0% (-1.7%, -0.3%) | 621 (9.0%) | 633 (9.2%) | -0.2% (-1.2%, 0.8%) |
| Mammograms; n (%) Telemedicine: n (%) | 6,892 (17.9%)<br>3.075 (8.0%) | 1,808 (22.7%)<br>1.390 (17.4%) | -4.8% (-5.8%, -3.8%)<br>-9.5% (-10.3%, -8.6%) | 1,489 (21.7%)<br>1,048 (15.2%) | 1,515 (22.0%)<br>1.099 (16.0%) | -0.4% (-1.8%, 1.0%)<br>-0.7% (-2.0%, 0.5%) |
| HbA1C tests | 3,073 (6.0%) | 1,390 (17.470) | -9.5% (-10.5%, -6.6%) | 1,048 (15.2%) | 1,099 (16.0%) | -0.776 (-2.076, 0.576) |
| mean (sd) | 2.69 (2.62) | 2.94 (2.04)<br>3.00 (2.00, 4.00) | -0.26 (-0.31, -0.20) | 2.89 (2.86) | 2.89 (2.01)<br>3.00 (2.00, 4.00) | -0.00 (-0.09, 0.08) |
| median [IQR]min, max | 3.00 [2.00, 3.00]<br>0.00, 194.00 | 0.00,65.00 | - (-, -)<br>- (-, -) | 3.00 [2.00, 4.00]<br>0.00, 112.00 | 0.00,65.00 | - (-, -)<br>- (-, -) |
| Lipid panels | | | | | | |
| mean (sd)median [IQR] | 1.85 (2.27)<br>2.00 [1.00, 3.00] | 1.95 (1.74)<br>2.00 [1.00, 3.00] | -0.11 (-0.15, -0.06)<br>- (-, -) | 1.93 (214)<br>2.00 [1.00, 3.00] | 1.93 (1.70)<br>2.00 [1.00, 3.00] | -0.01 (-0.07, 0.06)<br>- (-, -) |
| min, max | 0.00, 194.00 | 0.00, 35.00 | - (-, -) | 0.00, 112.00 | 0.00, 35.00 | - (-, -) |
| Creatinine testsmean (sd) | 0.11 (0.78) | 0.10 (0.51) | 0.02 (0.01, 0.03) | 0.09 (0.49) | 0.10 (0.52) | -0.01 (-0.02, 0.01) |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | |
| min, max | 0.00, 59.00 | 0.00, 14.00 | - (-, -) | | | - (-, -) |
| Natriuretic peptide testsmean (sd) | | | -15-7 | 0.00, 17.00 | 0.00,14.00 | -(-,-) |
| | 0.43 (2.12) | 0.41 (1.75) | 0.02 (-0.03, 0.06) | 0.00, 17.00 | 0.40 (1.75) | |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.02 (-0.03, 0.06) | 0.39 (1.31)<br>0.00 [0.00, 0.00] | 0.40 (1.75)<br>0.00 [0.00, 0.00] | -(-, -)<br>-0.01(-0.06, 0.04)<br>-(-, -) |
| median [IQR] | | | 0.02 (-0.03, 0.06) | 0.39 (1.31) | 0.40 (1.75) | -(-, -)<br>-0.01 (-0.06, 0.04) |
| _median [IQR] _min, max _urine tests _mean (sd) | 0.00 [0.00, 0.00]<br>0.00, 193.00<br>1.76 (3.02) | 0.00 [0.00, 0.00]<br>0.00, 84.00<br>1.61 (2.81) | 0.02 (-0.03, 0.06)<br>-(-, -)<br>-(-, -)<br>0.15 (0.08, 0.22) | 0.39 (1.31)<br>0.00 [0.00, 0.00]<br>0.00, 42.00 | 0.40 (1.75)<br>0.00 [0.00, 0.00]<br>0.00, 84.00<br>1.63 (2.90) | -(-,-)<br>-0.01 (-0.06, 0.04)<br>-(-,-)<br>-(-,-)<br>0.01 (-0.08, 0.11) |
| median (IQR)<br>min, max<br>Urine tests | 0.00 [0.00, 0.00]<br>0.00, 193.00 | 0.00 [0.00, 0.00]<br>0.00, 84.00 | 0.02 (-0.03, 0.06)<br>-(-,-)<br>-(-,-)<br>0.15 (0.08, 0.22)<br>-(-,-) | 0.39 (1.31)<br>0.00 [0.00, 0.00]<br>0.00, 42.00 | 0.40 (L75)<br>0.00 [0.00, 0.00]<br>0.00, 84.00 | -(-,-)<br>-0.01(-0.06, 0.04)<br>-(-,-)<br>-(-,-)<br>0.01(-0.08, 0.11)<br>-(-,-) |
| .medan (ICR) .min, max Urine tests Urine tests .mean (edmedan (ICR) .min, max Combined comorbidity score | 0.00 [0.00, 0.00]<br>0.00, 193.00<br>1.76 (3.02)<br>1.00 [0.00, 2.00]<br>0.00, 193.00 | 0.00 [0.00, 0.00]<br>0.00, 84.00<br>1.61 [2.81]<br>1.00 [0.00, 2.00]<br>0.00, 83.00 | 0.02 (-0.03, 0.06)<br>-(-,-)<br>-(-,-)<br>-(1,-)<br>0.15 (0.08, 0.22)<br>-(-,-) | 0.39 (1.31)<br>0.00 (0.00, 0.00)<br>0.00, 42.00<br>164 (2.55)<br>1.00 (0.00, 2.00)<br>0.00, 43.00 | 0.40 (1.75)<br>0.00 (0.00, 0.00)<br>0.00, 84.00<br>1.63 (2.90)<br>1.00 (0.00, 2.00)<br>0.00, 83.00 | -(·, -)<br>-0.01(-0.06, 0.04)<br>-(·, -)<br>-(·, -)<br>-(·, -)<br>-(·, -) |
| _median (IQR) _mix_max _mean_(sd _mean_(sd _median_(IQR) _mix_max _mean_(sd _mean_(sd _median_(IQR) _mix_max _mean_(sd | 0.00 [0.00, 0.00]<br>0.00, 193.00<br>1.76 (3.02)<br>1.00 [0.00, 2.00]<br>0.00, 193.00<br>3.12 (2.81) | 0.00 [0.00, 0.00]<br>0.00, 84.00<br>1.61 [2.81]<br>1.00 [0.00, 2.00]<br>0.00, 83.00<br>2.83 (2.45) | 0.02 (-0.03, 0.06)<br>-(-,-)<br>-(-,-)<br>0.15 (0.08, 0.22)<br>-(-,-) | 0.39 (1.31)<br>0.00 (0.00, 0.00)<br>0.00, 42.00<br>164 (2.55)<br>1.00 (0.00, 2.00)<br>0.00, 43.00<br>2.83 (2.52) | 0.40 (1.75)<br>0.00 (0.00, 0.00)<br>0.00, 84.00<br>1.63 (2.90)<br>1.00 (0.00, 2.00)<br>0.00, 83.00<br>2.80 (2.47) | -(-,-)<br>-0.01(-0.06, 0.04)<br>-(-,-)<br>-(-,-)<br>0.01(-0.08, 0.11)<br>-(-,-) |
| medan (IQR)mic, max Unre testsmean (edmean (edmic, max Combined combridity scoremean (sd)mean (sd)mean (sd) | 0.00 [0.00, 0.00]<br>0.00, 193.00<br>1.76 (3.02)<br>1.00 [0.00, 2.00]<br>0.00, 193.00 | 0.00 [0.00, 0.00]<br>0.00, 84.00<br>1.61 [2.81]<br>1.00 [0.00, 2.00]<br>0.00, 83.00 | 0.02 (-0.03, 0.06)<br>-(-,-)<br>-(-,-)<br>-(1,-)<br>0.15 (0.08, 0.22)<br>-(-,-) | 0.39 (1.31)<br>0.00 (0.00, 0.00)<br>0.00, 42.00<br>164 (2.55)<br>1.00 (0.00, 2.00)<br>0.00, 43.00 | 0.40 (1.75)<br>0.00 (0.00, 0.00)<br>0.00, 84.00<br>1.63 (2.90)<br>1.00 (0.00, 2.00)<br>0.00, 83.00 | -(·, -)<br>-0.01(-0.06, 0.04)<br>-(·, -)<br>-(·, -)<br>-(·, -)<br>-(·, -) |
| .medan (IGR) .min max Urine tests .mean (sid .mean(sid | 0.00 (0.00, 0.00)<br>0.00, 193.00<br>1.76 (3.02)<br>1.00 (0.00, 2.00)<br>0.00, 193.00<br>3.12 (2.81)<br>3.00 (1.00, 5.00)<br>-2.00, 17.00 | 0.00 (0.00, 0.00)<br>0.00, 84.00<br>161(2.81)<br>1.00 (0.00, 2.00)<br>0.00, 83.00<br>2.80 (2.45)<br>2.80 (2.00, 4.00)<br>1.00, 14.00 | 0.02(+0.03, 0.06)<br>1(-1)<br>1(-1)<br>1(-1)<br>1(-1)<br>1(-1)<br>1(-1)<br>1(-2) | 0.39 (1.31)<br>0.00 (0.00, 0.00]<br>0.00, 42.00<br>164 (2.55)<br>100 (10.00, 2.00]<br>0.00, 43.00<br>283 (2.52)<br>200 (1.00, 4.00)<br>-1.00, 15.00 | 0.40 (1.75)<br>0.00 (0.00, 0.00)<br>0.00, 84.00<br>1.60 (1.00, 2.00)<br>1.00 (1.00, 2.00)<br>0.00, 83.00<br>2.80 (2.47)<br>2.00 (1.00, 4.00)<br>1.00, 14.00 | -(-,-) -0.01 (-0.06, 0.04) -(-,-) |
| medan (IQR)mic, max Unre testsmean (edmean (edmic, max Combined combridity scoremean (sd)mean (sd)mean (sd) | 0.00 (0.00 0.00)<br>0.00, 193.00<br>1.76 (3.02<br>1.00 (0.00 2.00)<br>0.00, 193.00<br>3.12 (2.81)<br>3.00 (1.00, 5.00)<br>2.200, 17.00<br>0.23 (0.08)<br>0.21 (0.17, 0.27) | 0.00(0.00,0.09) 0.00,84.00 1.61(2.81) 1.00(0.00,2.00) 0.00,83.00 2.83 (2.45) 2.90(1.00,4.00) 1.90,14.00 0.22 (0.06) 0.22 (0.06) | 0.02 (-0.03, 0.06)<br>-(-)<br>-(-)<br>-(-)<br>0.15 (0.08, 0.22)<br>-(-)<br>-(-)<br>-(-)<br>-(-)<br>-(-) | 0.39 (1.31)<br>0.00 (0.00, 0.00)<br>0.00, 42:00<br>164 (2.55)<br>1.00 (0.00, 2.00)<br>0.00, 43:00<br>2.83 (2.52)<br>2.00 (1.00, 4.00)<br>1.00 (15:00)<br>0.22 (0.07)<br>0.22 (0.07) | 0.40 (1.75) 0.00 (0.00, 0.00) 0.00, 84.00 1.63 (2.90) 1.00 (1.00, 2.00) 0.00, 83.00 2.80 (2.47) 2.00 (1.00, 4.00) 1.00 (1.400) 0.22 (0.07) 0.22 (0.07) | -(·,-) -0.01 (-0.06, 0.04) -(·,-) |
| medan (ICR)min, max Universetsmean (cldmean (cldmean (cldmin, max Combined comorbidity scoremean (cldmin, max Praithy Scoremean (cldmin, max Praithy Scoremean (cldmin, max Praithy Score | 0.00 [0.00, 0.00]<br>0.00, 193.00<br>1.76 (3.02)<br>1.00 [0.00, 2.00]<br>0.00, 193.00<br>3.12 (2.81)<br>3.00 [1.00, 5.00]<br>-2.00, 17.00<br>0.23 (0.08) | 0.00[0.00.00]<br>0.00,84.00<br>161(28)<br>100[0.00,2.00]<br>0.00,83.00<br>2.831(245)<br>2.00[1.00,4.00]<br>1.00,14.00<br>0.22(0.06) | 0.02 (-0.03, 0.06) -1(-1) | 0.39 ft.33)<br>0.00 [0.00, 0.00]<br>0.00, 42.00<br>164 (2.55)<br>160 (2.00)<br>0.00, 43.00<br>283 [2.52]<br>200 [1.00, 4.00]<br>1.00, 15.00<br>0.22 (0.07) | 0.40 (1.75)<br>0.00 (0.00, 0.00)<br>0.00, 84.00<br>1.63 (2.90)<br>1.63 (2.90)<br>1.60 (2.90)<br>0.00, 83.00<br>2.80 (2.47)<br>2.00 (1.00, 4.00)<br>1.00, 14.00<br>0.22 (0.07) | -(·,·) -0.01 (-0.06, 0.04) -(·,·) |
| medan (IQR)min, max Urine testsmean (sidmean (sidmedan (IQR)min, max Combined comorbidity scoremean (sidmean (sidmean (sidmean (sidmean (sidmean (sidmin, max Finity Scoremean (sid | 0.00 (0.00 0.00)<br>0.00, 193.00<br>1.76 (3.02<br>1.00 (0.00 2.00)<br>0.00, 193.00<br>3.12 (2.81)<br>3.00 (1.00, 5.00)<br>2.200, 17.00<br>0.23 (0.08)<br>0.21 (0.17, 0.27) | 0.00(0.00,0.09) 0.00(84.00) 1.61(2.81) 1.00(0.00,2.00) 0.00,83.00 2.83 (24.5) 2.83 (24.5) 2.90(1.00,4.00) 1.90,14.00 0.22 (0.06) 0.22 (0.06) 0.22 (0.06) | 0.02 (-0.03, 0.06)<br>16-1<br>16-1<br>16-1<br>16-1<br>16-1<br>16-1<br>16-1<br>16-2<br>16-3 | 0.39 ft.331<br>0.00 [0.00, 0.00]<br>0.00, 42:00<br>164 (2.55)<br>164 (2.55)<br>100 [0.00, 2.00]<br>0.00, 43:00<br>283 (2.52)<br>2001 [0.04, 4.00]<br>1.00, 15:00<br>0.22 [0.07, 0.25]<br>0.07, 0.65<br>0.39 (0.83) | 0.40 (1.75) 0.00 (0.00, 0.00) 0.00, 84.00 1.63 (2.90) 1.00 (1.00, 2.00) 0.00, 83.00 2.80 (2.47) 2.00 (1.00, 4.00) 1.00 (1.400) 0.22 (0.07) 0.22 (0.07) | -(·,·) 0.01(-0.06, 0.04) -(·,·) -(·,·) 0.01(-0.08, 0.11) -(·,·) 0.03(-0.06, 0.11) -(·,·) -(·,·) 0.00(-0.00, 0.00) |
| medan (ICR)min max Urine testsmean (sdmean (sdmedan (IOR)mean (sdmedan (IOR)medan (IOR)medan (IOR)medan (sdmedan (sdmedan (sd)medan (sd)medan (sd)medan (sd)medan (sd)mean (sdmean (sd)mean (sd) | 0.00 [0.00 a.00] 0.00 [1300 1.76 [3.02) 1.00 [0.00 2.00] 0.00 [33.00 3.12 [2.81] 3.00 [1.00 5.00] 2.00 [17.00 0.23 [0.08] 0.21 [0.17, 0.27] 0.07, 0.69 | 0.00(0.00,00) 0.00(0.00,00) 1.6(1.28) 1.00(1.00,2.00) 0.00,6.30.00 0.00,6.30.00 1.00,1.00 | 0.02 (-0.03, 0.06) (-1) (-1) (-1) (-1) (-1) (-1) (-1) (-1 | 0.39 (1.31) 0.00 (0.00 0.00) 0.00, 42.00 1.64 (7.25) 1.00 (1.00 0.20) 0.00, 43.00 0.00, 43.00 0.00, 43.00 0.00, 43.00 0.00, 43.00 0.00, 43.00 0.00, 43.00 0.22 (0.07) 0.22 (0.07) 0.22 (0.07) 0.25 (0.05) 0.39 (0.83) 0.00 (0.00, 1.00) | 0.40 (1.75) 0.00 (0.00, 0.00) 0.00, 84.00 1.63 (2.90) 1.00 (0.00, 2.00) 0.00, 63.00 2.80 (2.47) 2.00 (1.00, 4.00) 1.00, 14.00 1.00, 14.00 0.22 (0.07) 0.22 (0.07) 0.23 (0.07, 0.25) 0.07, 0.63 0.39 (0.83) 0.000 (0.00, 1.00) | -(c, -) -(0.01 (-0.06, 0.04) -(c, -) |
| .medan (ICR) .min, max bine tests .mean (et al., mean (et al., mean (et al., mean) .medan (ICR) .min, max Combined comorbidity score .mean (et al., min, max Faith Score .mean (et al., min, max Faith Score .mean (et al., min, max Incedan (ICR) .min, max Incedan (ICR) .min, max Incedan (ICR) .min, max Incedan (ICR) .min, max Incedan (ICR) .min, max | 0.00 (0.00 0.00) 0.00, 193.00 1.76 (3.02) 1.00 (0.00, 2.00) 0.00, 193.00 3.12 (2.81) 3.00 (1.00, 5.00) 2.00, 17.00 0.21 (0.17, 0.27) 0.07, 0.59 | 0.0010.00.000<br>0.00,84.00<br>1.65(28)<br>1.65(28)<br>1.0010.00,2.00<br>0.00,83.00<br>2.83(245)<br>2.0011.00.4.00<br>1.00,14.00<br>0.22(0.10,0.4.00<br>0.22(0.17,0.25)<br>0.07,0.63 | 0.02 (-0.03, 0.06) -(-,-) | 0.39 ft.331<br>0.00 [0.00, 0.00]<br>0.00, 42:00<br>164 (2.55)<br>164 (2.55)<br>100 [0.00, 2.00]<br>0.00, 43:00<br>283 (2.52)<br>2001 [0.04, 4.00]<br>1.00, 15:00<br>0.22 [0.07, 0.25]<br>0.07, 0.65<br>0.39 (0.83) | 0.40 (1.75) 0.00 (0.00 0.00) 0.00, 84.00 163 (2.90) 100 (0.00, 2.00) 0.00, 83.00 2.80 (2.47) 2.00 (1.00 0.00) 1.00 (1.40.00) 0.22 (0.07) 0.22 (0.07) 0.22 (0.07) 0.25 (0.07) 0.39 (0.83) | -(c-) -(0.01 (-0.05, 0.04) -(c-) -(c |
| .medan (ICR) .mena (IcR) .mena | 0.00 (0.00 0.00) 1.00,193.00 1.00,193.00 1.00 (1.00,0.20) | 0.0010.00.000<br>0.00,84.00<br>1.0010.00,2.001<br>0.00,83.00<br>2.83 (245)<br>2.83 (245)<br>2.0011.00,4.001<br>1.00,14.00<br>0.22 (1.06)<br>0.22 (1.06)<br>0.22 (1.07,0.25]<br>0.07,0.63<br>0.38 (0.82)<br>0.0010.00 | 0.02 (-0.03, 0.06) -1(-1) -1(- | 0.39 ft.31)<br>0.00 (0.00, 0.00)<br>0.00, 42:00<br>164 (2.55)<br>160 (0.00, 2.00)<br>0.00, 43:00<br>2.83 (2.52)<br>2.001 (0.0, 4.00)<br>1.00 (15:00)<br>0.22 (0.07, 0.05)<br>0.27 (0.07, 0.05)<br>0.39 (0.83)<br>0.00 (0.00, 1.00)<br>0.00, 0.00 | 0.40 (1.75) 0.00 (1.00.0.00) 0.00, 84.00 163 (2.90) 163 (2.90) 160 (1.00, 2.00) 0.00, 83.00 280 (2.47) 200 (1.00, 4.00) 1.00, 14.00 0.22 (0.07) 0.22 (0.07, 0.55) 0.07, 0.63 0.39 (0.83) 0.00 (1.00, 1.00) 0.00, 1.00 | -(c) -(001(008,004) -(c) -(c) -(c) -(c) -(c) -(c) -(c) -(c |
| medan (ICR)mix max Urine testsmean (sdmean (sdmean (sdmean (sdmean (sd)mean (sd) | 0.00 [0.00 a.00] 0.001 [33.00 1.76 [3.02 1.001 [0.00 2.00] 0.001 [33.00 3.12 [2.81] 3.00 [1.00 5.00] 2.00 [17.00 0.23 [0.08] 0.24 [0.17, 0.27] 0.07, 0.69 0.77 [1.08] 0.00 [0.00, 1.00] 0.00 [8.00 5.234 [1.3.6%] 9,784 [25.3%] | 0.0010.00.000 1.000,84.00 1.61(28) 1.61(28) 1.0010.00.2001 0.00,83.00 2.83(245) 2.0011.00.4.001 1.00.1400 0.22(0.06) 0.21(0.17,0.25] 0.07,0.63 0.38(0.82) 0.0010.00.1.00] 0.0010.00 | 0.02 (-0.03, 0.06) (-) (- | 0.39 (1.31) 0.00 (0.00. 0.00) 1.00 (1.00. 0.00) 1.00 (1.25) 1.00 (1.00. 0.20) 0.00 (1.3.00) 1.00 (1.00. 0.00) 1.00 (1.00 (1.00) 1.00 (1.00 | 0.40 (1.75) 0.00 (0.00, 0.00) 1.63 (2.90) 1.00 (0.00, 2.00) 1.00 (0.00, 2.00) 0.00, 63.00 2.80 (2.47) 2.00 (1.00, 4.00) 1.00 (1.00, 4.00) 1.00 (1.00, 4.00) 1.00 (1.00, 6.00) 0.22 (0.07) 0.22 (0.07) 0.22 (0.07) 0.33 0.39 (0.83) 0.39 (0.83) 0.00 (0.00, 1.00) 0.00 (1.00) 1.518 (2.21%) | -(c-) -(01)(-006, 0.04) -(c-) |
| .medan (IQR) .min, max Usine tests .mean (udmedan (IQR) .metan (IQR | 0.00 [0.00 a.00] 0.00 [130 0.0] 176 [3 02) 1.00 [0.00 2.00] 0.00 [130 0.0] 3.12 [2.81] 3.00 [1.00 5.00] 2.00 [17.00 0.23 [0.08] 0.23 [0.17, 0.27] 0.07, 0.69 0.57 [1.08] 0.00 [0.00, 1.00] 0.00 [1.00] | 0.0010.00.000 1.000.84.00 1.61(28) 1.0010.00.200 1.00,83.00 2.83(2.45) 2.0011.00.4.00 1.00.14.00 1.00.10.00 1.00.10.00 1.00.10.00 1.00.10.00 1.00.10.00 1.762(22).99 1.762(22).99 1.762(22).99 | 0.02 (-0.03, 0.06) (-) (- | 0.39 (1.31) 0.00 (0.00.00) 0.00 (2.00) 1.64 (2.55) 1.00 (1.00.0.20) 1.00 (1.30.0) 2.31 (2.52) 2.00 (1.00.0.40) 1.00 (1.50.0) 2.21 (0.07) 2 | 0.40 (1.75) 0.00 (0.00, 0.00) 0.00 (0.00) 1.63 (2.90) 1.00 (0.00, 2.00) 0.00, 83.00 2.80 (2.47) 2.00 (1.00, 4.00) 1.00 (1.00, 4.00) 1.00 (1.00, 4.00) 1.00 (1.00, 6.30) 0.22 (0.07) 0.22 (0.07) 0.22 (0.07, 0.53) 0.39 (0.83) 0.39 (0.83) 0.00 (0.00, 1.00) 0.00 (1.00) 1.518 (2.21%) 5.115 (74.4%) 1.1188 (1.74%) | -(c-) -(00)(-006, 0.04) -(c-) -(00)(-006, 0.04) -(c-) |
| medan (IQR)mix max bine tests bine testsmean (sdmedan (sd)mix max combined comorbidity scoremean (sd)medan (IQR)mix max Fally Scoremean (sd)medan (IQR)mix max Fally Scoremean (sd)medan (IQR)mix max Any hosplatizationsmean (sd)medan (IQR)mix max Any hosplatization within prior 91 days; n (%) Any hosplatization within prior 92-385 days; n (%) Aumber of hosplatization within prior 92-385 days; n (%) Aumber of hosplatization within prior 92-385 days; n (%) Aumber of hosplatization within prior 92-385 days; n (%) Aumber of hosplatization (0, 1, 2 or more)+2 n (%)+2 n (%) | 0.00 (0.00 0.00) 0.00 (193.00 1.76 (3.02) 1.00 (0.00, 2.00) 0.00 (193.00 3.12 (2.81) 3.12 (2.81) 3.12 (2.81) 3.12 (2.81) 3.12 (3.00) 0.00 (1.00, 5.00) 2.00 (1.70, 0.00) 0.23 (0.08) 0.23 (0.08) 0.27 (1.08) 0.07 (1.08) 0.00 (1.00, 1.00) | 0.0010.00.009 0.00,84.00 1.01,84.00 1.02,84.00 1.03,84.00 1.04,84.00 1.05,84.00 1.05,84. | 0.02 (-0.03, 0.06) 1-(-) | 0.39 (1.31) 0.00 (0.00, 0.00) 0.00, 42.00 164 (12.55) 164 (12.55) 160 (10.00, 2.00) 0.00, 43.00 2.83 (2.52) 2.00 (10.0, 4.00) 4.00, 15.00 0.22 (0.07) 0.22 (0.07) 0.22 (0.07) 0.29 (0.07) 0.40 (1.50) 0.40 (1.50) 0.50 (1.50) | 0.40 (1.75) 0.00 (0.00, 0.00) 0.00, 84.00 1.63 (2.90) 1.63 (2.90) 1.63 (2.90) 1.63 (2.90) 1.63 (2.90) 1.63 (2.90) 1.63 (2.90) 1.60 (1.90) | 16-3 |
| .medan (IQR) .min, max Unne tests Unne tests Unne tests Unne tests Unne tests Unne tests .mean (IQR) .min, max .medan (IQR) .min, max .medan (IQR) .min, max .medan (IQR) .min, max .medan (IQR) .min, max .medan (IQR) .min, max .mean (IQR) .min, max .mean (IQR) .min, max .mean (IQR) .min, max .mean (IQR) .min, max .medan (IQR) .min, max .mean (IQR) .min, max .min, | 0.00 (0.00, 0.00) 0.00, 193.00 1.76 (3.02) 1.00 (0.00, 2.00) 0.00, 193.00 3.12 (2.81) 3.00 (1.00, 5.00) 2.00, 1.700 0.23 (0.08) 0.21 (0.17, 0.07) 0.07, 0.69 0.67 (1.08) 0.00 (1.00, 1.00) 0.00 | 0.0010.00.009 0.00,84.00 1.01,84.00 1.02,811 1.0010.00,2.001 0.00,83.00 2.83 (245) 2.83 (245) 2.83 (245) 2.9011.00,4.001 1.00,14.00 2.21 (0.06) 0.22 (0.06) 0.22 (0.06) 0.22 (0.07,0.28) 0.07,0.63 0.38 (0.82) 0.0010.00 (1.00) 0.00,10.00 1.762 (221%) 1.762 (221%) 1.952 (724%) 1.95 | 0.02 (-0.03, 0.06) 1(-)-1 1(-) | 0.39 (1.31) 0.00 (0.00, 0.00) 0.00, 42.00 164 (12.55) 164 (12.55) 160 (10.00, 2.00) 0.00, 43.00 2.83 (2.52) 2.83 (2.52) 2.00 (10.0, 4.00) 1.00, 15.00 0.22 (0.07) 0.22 (0.07) 0.22 (0.07) 0.23 (0.05) 0.39 (0.83) 0.00 (0.00, 1.00) 1.50 (0.00, 9.00) 4.60 (1.50) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.53 (1.21%) 1.56 (74.2%) 1.219 (1.21%) 1.56 (1.21%) 1.56 (1.21%) 1.56 (1.21%) 1.57 (1.21%) 1.58 (1.21%) 1.58 (1.21%) 1.59 ( | 0.40 (1.75) 0.00 (1.00, 0.00) 0.00, 84.00 1.63 (2.90) 1.60 (1.00, 2.00) 1.60 (1.00, | 16-3 O01(-006,004) 16-3 O01(-008,011) 16-3 O03(-006,011) 16-3 O03(-006,011) 16-3 O00(-000,000) 16-3 O00 |
| .medan (ICR) .min. max Usine tests .mean (ICR) .mean ( | 0.00 [0.00 a.00] 0.00 [1300 ] 176 [3 02] 1.00 [0.00 2.00] 0.00 [1300 ] 3.12 [28] 3.00 [1.00 5.00] 2.00 [17.00 2.00 [17.00 0.22 [0.08] 0.22 [0.17, 0.27] 0.07, 0.69 0.00 [0.00, 1.00] 0.00 [18.00 0.22 [0.18.00] 0.00 [18.00 0.22 [0.18.00] 0.00 [18.00 0.00 [18.00 0.00 [18.00 0.00 [18.00 0.00 [18.00 0.00 [18.00 0.00 [18.00] 0.00 [18.00 0.00 [18.00 0.00 [18.00 0.00 [18.00] 0.00 [18.00 0.00 [18.00] 0 | 0.0010.00.000 1.000.84.00 1.61(281) 1.0010.00.2001 0.008.300 0.08.300 0.08.312.45 2.0011.00.4.001 1.00.14.00 1.00.10.00 1.00.10.00 1.00.10.00 1.00.10.00 1.00.10.00 1.00.10.00 1.762(221.99) | 0.02 (-0.03, 0.06) (-7) (-7) (-7) (-7) (-7) (-7) (-7) (-7 | 0.39 (1.31) 0.00 (0.00, 0.00) 1.64 (1.255) 1.00 (1.00, 2.00) 1.00, 4.200 1.00, 4.300 2.83 (2.52) 2.00 (1.00, 4.00) 1.00 | 0.40 (1.75) 0.00 (0.00, 0.00) 1.63 (2.90) 1.63 (2.90) 1.00 (0.00, 2.00) 1.00 (0.00, 2.00) 2.80 (2.47) 2.00 (1.00, 4.00) 1.00 (1.00, 4.00) | -(-) |
| medan (IQR)mixmax Usine testsmean (tidmest indmedan (IQR)mixmaxmedan (IQR)mixmaxmedan (IQR)medan (IQR)mixmaxmedan (IQR)mix maxmedan (IQR)mix maxmix max | 0.00 (0.00, 0.00) 0.00, 193.00 1.76 (3.02) 1.00 (0.00, 2.00) 0.00, 193.00 3.12 (2.81) 3.00 (1.00, 5.00) 2.00, 1.700 0.23 (0.08) 0.21 (0.17, 0.07) 0.07, 0.69 0.67 (1.08) 0.00 (1.00, 1.00) 0.00 | 0.0010.00.009 0.00,84.00 1.01,84.00 1.02,811 1.0010.00,2.001 0.00,83.00 2.83 (245) 2.83 (245) 2.83 (245) 2.9011.00,4.001 1.00,14.00 2.21 (0.06) 0.22 (0.06) 0.22 (0.06) 0.22 (0.07,0.28) 0.07,0.63 0.38 (0.82) 0.0010.00 (1.00) 0.00,10.00 1.762 (221%) 1.762 (221%) 1.952 (724%) 1.95 | 0.02 (-0.03, 0.06) 1(-)-1 1(-) | 0.39 (1.31) 0.00 (0.00, 0.00) 0.00, 42.00 164 (12.55) 164 (12.55) 160 (10.00, 2.00) 0.00, 43.00 2.83 (2.52) 2.83 (2.52) 2.00 (10.0, 4.00) 1.00, 15.00 0.22 (0.07) 0.22 (0.07) 0.22 (0.07) 0.23 (0.05) 0.39 (0.83) 0.00 (0.00, 1.00) 1.50 (0.00, 9.00) 4.60 (1.50) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.52 (1.21%) 1.53 (1.21%) 1.56 (74.2%) 1.219 (1.21%) 1.56 (1.21%) 1.56 (1.21%) 1.56 (1.21%) 1.57 (1.21%) 1.58 (1.21%) 1.58 (1.21%) 1.59 ( | 0.40 (1.75) 0.00 (1.00, 0.00) 0.00, 84.00 1.63 (2.90) 1.60 (1.00, 2.00) 1.60 (1.00, | 16-3 O01(-006,004) 16-3 O01(-008,011) 16-3 O03(-006,011) 16-3 O03(-006,011) 16-3 O00(-000,000) 16-3 O00 |
| .medan (IQR) .min, max Ubre tests .mean (sdd .mean (sdd .medan (IQR) .mix max .medan (IQR) .mix max .medan (IQR) .mean (sdd .mean (s | 0.00 (0.00, 0.00) 1.76 (3.02) 1.00 (0.00, 2.00) 1.00 (0.00, 1.00) | 0.0010.00.009 0.000.84.00 1.61.281 1.0010.00,2.001 0.00,83.00 0.00,93.00 0.00 | 0.02 (-0.03, 0.06) 1(-1) | 0.39 (1.31) 0.00 (0.00, 0.00) 0.00, 42:00 1.64 (2.55) 1.00 (1.00, 2.00) 0.00, 43:00 2.83 (2.55) 1.00 (1.00, 2.00) 0.00, 43:00 2.83 (2.52) 2.83 (2.52) 2.83 (2.52) 0.07 (0.55) 0.07 (0.55) 0.07 (0.55) 0.07 (0.55) 0.08 (0.00, 1.00) 0.09 (0.00, 1.00) 0.09 (0.00, 1.00) 1.523 (2.21%) 1.523 (2.21%) 1.523 (2.21%) 1.523 (2.21%) 1.524 (2.21%) 1.525 (2.00%) 1.526 (2.00%) 1.526 (2.00%) 1.527 (2.21%) 1.527 (2.21%) 1.528 (2.21%) 1.528 (2.21%) 1.528 (2.21%) 1.529 (2.21%) 1.52 | 0.40 (1.75) 0.00 (0.00, 0.00) 0.00, 84.00 1.63 (2.90) 1.60 (1.00, 2.00) 1.60 (1.00, | 16-3 O01(-0.06.04) 16-3 O11(-0.08.01) 16-3 O01(-0.08.01) 16-3 O03(-0.06.01) 16-3 O03(-0.06.01) 16-3 O00(-0.00.00) O00(-0.00.00) 16-3 O00(-0.00.00) O00(-0.00) O00 |
| .medan (IQR) .min, max Usine tests .mean (ud .medan (IQR) | 0.00 (0.00, 0.00) 1.76 (3.02) 1.76 (3.02) 1.00 (0.00, 2.00) 1.00 (0.00, 2.00) 3.12 (2.81) 3.00 (1.00, 5.00) 2.00 (1.70, 0.00) 2.00 (1.70, 0.00) 2.00 (1.70, 0.00) 2.00 (1.70, 0.00) 0.00 (1.00, | 0.0010.00.000 1.000.84.00 1.61(281) 1.0010.00.2001 0.000.2001 0.000.2000 0.000.2001 0.0000000000 | 0.02 (-0.03, 0.06) (-1, 1) (-1 | 0.39 (1.31) 0.00 (0.00, 0.00) 1.64 (2.55) 1.00 (1.00, 2.00) 1.00 (2.00) 2.00 ( | 0.40 (1.75) 0.00 (0.00, 0.00) 1.63 (2.90) 1.63 (2.90) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 3.00) 1.60 (1.00, | 16-3 301(406,004) 10-1(-006,011) 16-3 16-3 001(-006,011) 16-3 16-3 003(-006,011) 16-3 16-3 000(-000,000) 16-3 16-3 000(-000,000) 000(-000,000) |
| .medan (ICR) .menan (ICR) .mena | 0.00 (0.00, 0.00) 0.00 (1.30 0.00) 1.76 (3.02) 1.00 (0.00, 2.00) 1.00 (0.00, 2.00) 3.12 (2.81) 3.00 (1.00, 5.00) 2.00 (1.70 0.00) 2.00 (1.70 0.00) 2.00 (1.70 0.00) 2.00 (1.70 0.00) 0.00 (1.00 0 | 0.0010.00.000 1.000.0000 1.000.0000 1.000.000 | 0.02 (-0.03, 0.06) (1-7) | 0.39 (1.31) 0.00 (0.00, 0.00) 1.64 (2.55) 1.00 (1.00, 2.00) 1.64 (2.55) 1.00 (1.00, 2.00) 0.00, 4.30 (1.00) 2.83 (2.52) 2.00 (1.00, 4.00) 1.00 (1.50 (1.00) 2.21 (0.77, 0.25) 0.07, 0.65 0.22 (0.77, 0.25) 0.07, 0.65 0.39 (0.83) 0.00 (0.00, 1.00) 0.00, 9.00 1.52 (2.21 (1.00) 1.52 (2.2 | 0.40 (1.75) 0.00 (0.00, 0.00) 1.63 (2.90) 1.63 (2.90) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 3.00) 1.60 (1.00, | 16-3 301 (0.05, 0.04) 16-3 |
| .medan (ICR) .min, max Urine tests .mean (sid .min, max .mean (sid .min, max .mean (sid .mean (sid .min (sid . | 0.00 (0.00, 0.00) 1.76 (3.02) 1.76 (3.02) 1.00 (0.00, 2.00) 1.00 (0.00, 2.00) 3.12 (2.81) 3.00 (1.00, 5.00) 2.00 (1.70, 0.00) 2.00 (1.70, 0.00) 2.00 (1.70, 0.00) 2.00 (1.70, 0.00) 0.00 (1.00, | 0.0010.00.000 1.000.84.00 1.61(281) 1.0010.00.2001 0.000.2001 0.000.2000 0.000.2001 0.0000000000 | 0.02 (-0.03, 0.06) (-1, 1) (-1 | 0.39 (1.31) 0.00 (0.00, 0.00) 1.64 (2.55) 1.00 (1.00, 2.00) 1.00 (2.00) 2.00 ( | 0.40 (1.75) 0.00 (0.00, 0.00) 1.63 (2.90) 1.63 (2.90) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 2.00) 1.60 (1.00, 3.00) 1.60 (1.00, | 16-3 1001 (0.05, 0.04) 16-3 |

### Variable name

Age Gender Race

Region

Dual status/Low income subsidy

Smoking / Tobacco use

Underweight Normal weight, if BMI is 20.0-24.9

Overweight, if BMI is 25.0 to 29.9

Class 1 (low-risk) obesity, if BMI is 30.0 to 34.9 Class 2 (moderate-risk) obesity, if BMI is 35.0 to 39.9

Unspecified obesity Diabetic retinopathy Diabetic neuropathy Diabetic nephropathy

Diabetes with other opthalmic complications

Diabetes with peripheral circulatory disorders

Diabetic foot Erectile dysfuntion Hypoglycemia

Hyperglycemia/DKA/HONK

Skin infections Stable angina Unstable angina Hypertension Hypotension

Hvperlipidemia Atrial fibrillation

Acute myocardial infarction Old myocardial infarction

Cardiac conduction disorder

Previous cardiac procedure (CABG, PTCA, Stent)

Ischemic stroke

PVD diagnosis or surgery

Other cardiac dysrhythmia

Heart failure

# Algorithm sources

If region not available, from State, https://www2.census.gov/geo/pdfs/maps-data/maps/reference/us regdiv.pdf https://www.cms.gov/medicare-medicaid-coordination/medicare-and-medicaid-coordination/medicare-

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015,

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Class 3 (high-risk) obesity if BMI is equal to or greater than Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/.

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/.

https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus,

Investigator review of codes based on: (modified codes) https://pubmed.ncbi.nlm.nih.gov/36102675/

Investigator review of codes based on: the paper then used ICD9/ICD10 website to expand it,

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

Investigator review of codes based on:

Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/

DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/, https://pubmed.ncbi.nlm.nih.gov/38262528/

HONK:

Investigator review of codes based on: https://pubmed.ncbi.nlm.nib.gov/34953068/, ICD9 to ICD10 conversion

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/. Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/. Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC8064679/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/31933524/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc 31381 DS8.pdf,

https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf,

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes, https://www.icd10data.com/

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc 31381 DS8.pdf, https://www.health.nv.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf.

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Acute heart failure

Microalbuminuria/proteinuria

Cardiomyopathy

Valve disorders

Valve replacement

TIA

Edema

Venous thromboembolism/ pulmonary embolsim

Pulmonary hypertension

Implantable cardioverter defibrillator

Hyperkalemia

Coronary atherosclerosis

Cerebrovascular procedure

Insertion of pacemakers / removal of cardiac lead

CKD stage 1-2

CKD stage 3-4

**Unspecified CKD** 

Acute kidney injury

Hypertensive nephropathy

Urinary tract infections

Genital infections

Urolithiasis (kidney or urinary stones)

COPD

Asthma

Obstructive sleep apnea

Serious bacterial infections

Pneumonia

Liver disease

MASH/MASLD

Fractures / Falls

Osteoporosis

Osteoarthritis

Depression

Dementia

Delirium or psychosis

Anxiety

Sleep disorder

Anemia

Influenza

COVID-19

Hyperthyroidism and other thyroid gland disorders

Hypothyroidism

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

https://pubmed.ncbi.nlm.nih.gov/38440888/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC875199/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC875199/, https://www.ncbi.nlm.ni

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://www.cms.gov/medicare-coverage-

 $Investigator\ review\ of\ codes\ based\ on: \underline{https://www.sciencedirect.com/science/article/pii/S2666572723000251}$ 

Investigator review of codes

 $Modified\ codes\ based\ on\ eligibility\ criteria, here\ we\ implement\ any\ care\ setting, any\ diagnosis\ position$ 

https://pmc.ncbi.nlm.nih.gov/articles/PMC4399109/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC10251803/

Investigator review of codes, <a href="https://www.icd10data.com/">https://www.icd10data.com/</a>

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC2978782/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC5888226/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637,

https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e29ab67-7a7d-4621-

Investigator reviewed code based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC7558992/#app1-antibiotics-09-

Investigator reviewed codes based on: https://pubmed.ncbi.nlm.nih.gov/30207042/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC7793999/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/,

https://pubmed.ncbi.nlm.nih.gov/29921683/, https://pubmed.ncbi.nlm.nih.gov/17346615/,

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder sir wp002.

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/32300995/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/.

Modified CCW algorithm

https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms

https://pubmed.ncbi.nlm.nih.gov/35043165/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/

https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-and-diagnostic-

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38556924/

https://pubmed.ncbi.nlm.nih.gov/34913208/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/

Investigator review of codes based on: https://www.cms.gov/icd10m/version37-fullcode-

Investigator review of codes based on: https://pmc.ncbi.nlm.nib.gov/articles/PMC10478599/

Nephrotic syndrome Urinary incontinence

Biliary disease

Pancreatitis

Bowel obstruction Gastroparesis

Number of antidiabetic drugs on CED

Concomitant use or initiation of metformin Concomitant use or initiation of insulin

Concomitant use or initiation of sulfonylureas

Concomitant use or initiation of SGLT2i

Concomitant use or initiation of other glucose-lowering dru

Past use of metformin Past use of insulin Past use of sulfonylureas Past use of SGLT2i

Past use of other glucose-lowering drugs

ACEi / ARB

ARNI Thiazides Beta-Blockers

Calcium channel blockers

Digoxin/Digitoxin Loop diuretics Other diuretics Intravenous diuretics

**Nitrates** 

Anti-arrhythmics

Statins

PCSK9 inhibitors and other lipid-lowering drugs

Antiplatelet agents
Oral anticoagulants

COPD/Asthma medication

**NSAIDs** 

Oral corticosteroids

Osteoporosis agents (incl. bisphosphonates)

Opioids

Anti-depressants Antipsychotics

Anxiolytics/hypnotics, benzodiazepines

Medication for dementia

Urinary tract infections antibiotics

Laxatives

Number of distinct medications, median (igr), mean (sd)

Number of office visits median (iqr), mean (sd)

Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637,

Investigator review of codes based on: <a href="https://pubmed.ncbi.nlm.nih.gov/38527324/">https://pubmed.ncbi.nlm.nih.gov/38527324/</a> Investigator review of codes based on: <a href="https://pubmed.ncbi.nlm.nih.gov/37796527/">https://pubmed.ncbi.nlm.nih.gov/38527324/</a> Investigator review of codes based on: <a href="https://pubmed.ncbi.nlm.nih.gov/37796527/">https://pubmed.ncbi.nlm.nih.gov/38527324/</a> Investigator review of codes based on: <a href="https://pubmed.ncbi.nlm.nih.gov/37796527/">https://pubmed.ncbi.nlm.nih.gov/37796527/</a>.

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/36222554/,

Investigator review of codes based on: <a href="https://pubmed.ncbi.nlm.nih.gov/36798959/">https://pubmed.ncbi.nlm.nih.gov/36798959/</a>,

Investigator review of codes: <a href="https://pubmed.ncbi.nlm.nih.gov/34624355/">https://pubmed.ncbi.nlm.nih.gov/34624355/</a>

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/

 $Investigator\ review\ of\ codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/www.ncbi.nlm.nih.gov/books/nbw.nih.gov/books/NBK513225/www.ncbi.nlm.nih.gov/books/nbw.nih.gov/book$ 

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/

ru Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/,

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/

 $Investigator\ review\ of\ codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/nlm.nih.g$ 

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/,

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/linestigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/linestigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/linestigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/linestigator review of codes, https://www.n

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK507904/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK556025/, Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using

Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health-Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health-

Investigator review of codes. https://www.drugs.com. https://www.ncbi.nlm.nih.gov/books/NBK537062/

Investigator review of codes, https://www.drugs.com,

Investigator review of codes, https://www.copdfoundation.org/Learn-More/I-am-a-Person-with-

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK547742/

Investigator review of codes, https://www.drugs.com, https://www.aaaai.org/tools-for-the-public/drug-guide/oral-

Investigator review of codes based on: https://www.drugs.com,

Investigator review of codes, https://www.drugs.com,

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK538182/

Investigator review of codes, https://www.drugs.com

Investigator review of codes, https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-

Investigator review of codes based on: https://www.drugs.com.

https://pubmed.ncbi.nlm.nih.gov/35790044/

Investigator review of codes, https://www.drugs.com

N/A

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-

Number of endocrinologist visits, median (igr), mean (sd)

Number of cardiologist visits, median (igr), mean (sd)

Number of electrocardiograms, median (igr), mean (sd) Number of echocardiograms, median (igr), mean (sd) Pharmacy out-of-pocket cost, median (igr), mean (sd)

Unique brand medications Unique generic medications

Ratio of unique brand to generic medications

Colonoscopy/Sigmoidoscopy

Flu vaccine / Pneumococcal vaccine

Pap smear test PSA test

Fecal occult blood test

Bone mineral density tests

Mammograms

Telemedicine

Number of HbA1c tests, median (igr), mean (sd) Number of lipid panels, median (igr), mean (sd) Number of creatinine tests, median (igr), mean (sd)

Number of natriuretic peptide tests, median (igr), mean (sd) Investigator review of codes Number of urine tests, median (igr), mean (sd)

HbA1c Glucose Creatinine Systolic blood pressure

Heart rate BMI eGFR LDL HDL N/A

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Number of internal medicine/family medicine visits, mediar Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-

https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleId=57326,

https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/, https://www.aapc.com/codes/codinghttps://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/, https://pubmed.ncbi.nlm.nih.gov/34778785/,

N/A

Investigator review of codes. https://www.drugs.com Investigator review of codes, https://www.drugs.com Investigator review of codes, https://www.drugs.com

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytichttps://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder sir wp002,https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleId=54767&DocID=A54767. https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder sir wp002,https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleId=54767&DocID=A54767

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder sir wp002.https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleId=54767&DocID=A54767

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytichttps://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

Investigator review of codes

N/A

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002.https://www.cms.gov/medicare-coverage-

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/.

https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-fact-sheet,

https://pubmed.ncbi.nlm.nih.gov/34953068/ https://pubmed.ncbi.nlm.nih.gov/34953068/ https://pubmed.ncbi.nlm.nih.gov/34953068/

Investigator review of codes

N/A N/A N/A N/A N/A N/A

N/A N/A Total cholesterol N/A
Triglycerides N/A
Combined comorbidity score A combine

Combined comorbidity score A combined comorbidity score predicted mortality in elderly patients better than existing scores, Frailty score

Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index,

Number of any hospitalization, median (iqr), mean (sd)

Any hospitalization within prior 90 days; n (%)

Any hospitalization within prior 91-365 days; n (%)

0,1,>1 hospitalizations (any)

N/A

Hospitalization for heart failure; n (%)

N/A

Different in all 3 databases and measure already created in all 3 as well;

ED visit (Medicare): Revenue center codes: 0450, 0451, 0452, 0456, 0459, 0981; Place of service: 23

ED visit (Optum): Place of service: 23

Calendar year N/A